Dabigatran versus Warfarin in Patients with Atrial Fibrillation (RELY trial)

**DUPLICATE-RELY** 

May 26, 2021

NCT04593043

#### 1. RCT Details

#### 1.1 Title

Dabigatran versus Warfarin in Patients with Atrial Fibrillation (RELY trial)

#### 1.2 Intended aim(s)

To compare the risk of stroke or systemic embolism in atrial fibrillation (AF) patients with dabigatran versus warfarin use.

### 1.3 Primary endpoint for replication

The primary outcome of the study was stroke and systemic embolism.

#### 1.3.1 Required power for primary endpoint and noninferiority margin (if applicable)

Assuming a 2-year recruitment period and at least 1 year of follow-up and a primary event rate of 1.6% per year, it was determined that at least 15,000 patients would be needed to achieve a minimum of 450 events. The study would have approximately 84% power to conclude noninferiority of dabigatran over warfarin at alpha of 0.025 (1-sided) level.

#### 1.4 Secondary endpoint for replication (assay sensitivity) and RCT finding

Major bleeding; RR = 0.93 (95% CI 0.81-1.07)

### 1.5 Trial estimate

RR = 0.66 (95% CI 0.53-0.82) comparing 150mg dabigatran vs warfarin (Connolly et al., 2009)

#### 2. Person responsible for implementation of replication in Aetion

Hemin Lee, MD, MPH and Ajinkya Pawar, PhD implemented the study design in the Aetion Evidence Platform. They are not responsible for the validity of the design and analytic choices. All implementation steps are recorded and the implementation history is archived in the platform.

#### 3. Data Source(s)

United/Optum, MarketScan, Medicare

### 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expedited review.

Figure 1.

Design Diagram – RE-LY TRIAL REPLICATION



#### 5. Cohort Identification

#### 5.1 Cohort Summary

This study will involve a new user, parallel group, propensity score-matched, retrospective cohort study design comparing dabigatran (150mg) to warfarin users. The patients will be required to have continuous enrollment during a baseline period of 180 days before initiation of dabigatran or warfarin (index date). We will restrict the analyses to patients with a diagnosis of AF with risk factors for stroke or systemic embolism in the 12 months prior to drug initiation.

#### 5.2 Important steps for cohort formation

New users (defined as no use in 180 days prior to index date) of an exposure and a comparator drug will be identified.

#### 5.2.1 Eligible cohort entry dates

Market availability of dabigatran in the U.S. for non-valvular atrial fibrillation started on October 19, 2010

- For Medicare: October 19, 2010 December 31, 2017 (end of available data)
- For Marketscan: October 19, 2010 December 31, 2018 (end of available data)
- For Optum: October 19, 2010 December 31, 2019 (end of available data)

#### 5.2.2 Specify <u>inclusion/exclusion</u> criteria for cohort entry and define the index date

Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.

#### 5.3 Flowchart of the study cohort assembly

For dabigatran 150mg vs. warfarin

| | Optum | | Truven | | Medicare | |
|---|---|---|---|---|---|---|
| | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining Patients |
| All patients | | 77,673,639 | | 200,203,908 | | 6,886,908 |
| Did not meet cohort entry criteria | 76,847,731 | 825,908 | 199,014,982 | 1,188,926 | -2,335,930 | 4,550,978 |

| Excluded due to insufficient enrollment | -80,642 | 745,266 | -107,905 | 1,081,021 | -1,565,261 | 2,985,717 |
|---|---|---|---|---|---|---|
| Excluded due to prior use of referent | -564,968 | 180,298 | -751,832 | 329,189 | -2,241,426 | 744,291 |
| Excluded due to prior use of exposure | -44,640 | 135,658 | -71,891 | 257,298 | -196,688 | 547,603 |
| Excluded because patient qualified in >1 exposure category | -5 | 135,653 | -9 | 257,289 | -24 | 547,579 |
| Excluded based on Dabigatran (dose other than 150mg) | -306 | 135,347 | -534 | 256,755 | -2,557 | 545,022 |
| Excluded based on Age | 0 | 135,347 | 0 | 256,755 | -162 | 544,860 |
| Excluded based on Gender | 0 | 135,347 | 0 | 256,755 | 0 | 544,860 |
| Excluded based on Inclusion 1a or 1b or 1 c - Atrial fibrillation | -71,189 | 64,158 | -135,349 | 121,406 | -220,602 | 324,258 |
| Excluded based on Inclusion 2a-2e History of Stroke, TIA, Systemic embolism / EF<40% / NYHA 2 or higher / Age >75 / Age 65+RF | -11,313 | 52,845 | -17,737 | 103,669 | -24,940 | 299,318 |
| Excluded based on Inclusion 3 - Age >= 18 | -1 | 52,844 | -1 | 103,668 | 0 | 299,318 |
| Excluded based on Exclusion 1 - History of heart valve disorders | -17,688 | 35,156 | -5,687 | 97,981 | -94,948 | 204,370 |
| Excluded based on Exclusion 2a - Severe/disabling stroke | -576 | 34,580 | -1,111 | 96,870 | -3,090 | 201,280 |
| Excluded based on Exclusion 2b - Any stroke | -960 | 33,620 | -1,391 | 95,479 | -3,948 | 197,332 |
| Excluded based on Exclusion 3a - Major Surgery | -1,091 | 32,529 | -2,526 | 92,953 | -6,491 | 190,841 |
| Excluded based on Exclusion 3c - Intracranial hemorrhage - Inpatient | -51 | 32,478 | -331 | 92,622 | -595 | 190,246 |
| Excluded based on Exclusion 3d - Gastrointestinal hemorrhage | -4,848 | 27,630 | -1,601 | 91,021 | -5,353 | 184,893 |
| Excluded based on Exclusion 3e - Symptomatic or endoscopically documented gastroduodenal ulcer disease | -121 | 27,509 | -714 | 90,307 | -3,148 | 181,745 |
| Excluded based on Exclusion 3f - Hemorrhagic disorder or bleeding diathesis | -257 | 27,252 | -756 | 89,551 | -1,787 | 179,958 |
| Excluded based on Exclusion 3i - Uncontrolled hypertension | -51 | 27,201 | -400 | 89,151 | -804 | 179,154 |

| Excluded based on Exclusion 7 - Severe renal impairment | -1,301 | 25,900 | -4,674 | 84,477 | -12,016 | 167,138 |
|---|---|---|---|---|---|---|
| Excluded based on Exclusion 8 & 9 - Active infective endocarditis and liver disease | -36 | 25,864 | -255 | 84,222 | -616 | 166,522 |
| Excluded based on Exclusion 10 & 11 - Pregnancy & Anemia and Thrombocytopenia | -191 | 25,673 | -1,229 | 82,993 | -2,798 | 163,724 |
| Excluded based on Exclusion 14 - Alcohol abuse or dependence | -28 | 25,645 | -103 | 82,890 | -138 | 163,586 |
| Excluded based on Exclusion 14 - Drug abuse or dependence | -22 | 25,623 | -47 | 82,843 | -111 | 163,475 |
| Excluded based on Exclusion 14 - CCI (180 days) | -7 | 25,616 | -47 | 82,796 | -1,939 | 161,536 |
| Final cohort | | 25,616 | | 82,796 | | 161,536 |

<sup>\*</sup> Medicare database includes all patients using a novel oral anticoagulant and a subset of patients using warfarin during 2011-2017.

#### 6. Variables

### 6.1 Exposure-related variables:

#### Study drug:

The study exposure of interest is initiation of dabigatran. Initiation will be defined by no use of dabigatran or a comparator in the prior 6 months before treatment initiation (washout period).

### Comparator agents-

- Initiators of dabigatran (150mg) will be compared to initiators of
  - o Warfarin

#### 6.2 Covariates:

- Age
- Sex
- Combined Comorbidity Index (CCI), measured over the baseline covariate assessment period, defined as 180 days prior to and including index date

Covariates listed above represent only a small subset of covariates that will ultimately be controlled for in the design and analysis. We use the covariates above only for initial feasibility analyses to judge whether there is likely to be sufficient overlap between treatment groups to proceed with the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and the initial power assessment and are listed in Table 1 (**Appendix B**).

### 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Primary Effectiveness outcomes of interest: (definitions provided in **Appendix A**):

- Primary Outcome: Stroke (hemorrhagic, ischemic) and systemic embolism
- Secondary outcomes: Individual components
  - o Hospital admission for stroke (principal diagnosis position)
  - o Hospital admission for systemic embolism (principal diagnosis position)

Control outcomes of interest (control outcomes only serve to assess aspects of study validity but are not further interpreted):

1. Major bleeding

#### 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analyses will be conducted with treatment defined as the index drug on the day of cohort entry. Because adherence in the real-world databases is expected to be much worse than in the trial, the AT analysis is the **primary** analysis, as it targets the relative hazard of outcomes on treatment.

For the AT analyses, the follow-up will start the day after initiation of apixaban and comparator and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest, unless otherwise specified for selected outcomes,
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,

- Nursing home admission
  - Nursing home admissions are considered a censoring event because the data sources utilized typically provide little to no data on a patient, particularly on drug utilization, after admission. We will utilize this as an exclusion reason for cohorts for the same reason.
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (dabigatran and comparator) plus a defined grace period (i.e., 10 days after the end of the last prescription's days' supply in main analyses).
- The date of augmentation or switching from exposure to comparator or vice versa or augmentation/switching to any other NOAC (e.g. switching from dabigatran or warfarin to apixaban would be a censoring event);
  - o A dosage change on the index treatment does not fulfill this criterion
  - o An added treatment that is not part of the exposure or comparator group does not fulfill this criterion
- Dispensing of a fibrinolytic agent

For the intention-to-treat (ITT) analyses, the censoring based on the augmentation/switching and treatment discontinuation will be replaced with a maximum allowed follow-up time of 365 days.

### 7. Initial Feasibility Analysis

### Action report name:

For dabigatran vs. warfarin

Optum- https://bwh-dope.aetion.com/projects/details/707/results/59579/result/0

Marketscan- https://bwh-dope.aetion.com/projects/details/708/results/59601/result/0

Medicare- https://bwh-dope.aetion.com/projects/details/709/results/59602/result/0

Date conducted: 10/5/20 (Medicare 10/6/20)

Complete Action feasibility analysis using age, sex, and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome. No measures of association will be computed nor will incidence rates stratified by treatment group.

- Report patient characteristics by treatment group
- Report summary parameters of study population
- Report median follow-up time by treatment group
- Report reasons for censoring in the overall study population

#### 8. Initial Power Assessment

#### Action report name:

For dabigatran vs. warfarin

Optum- <a href="https://bwh-dope.aetion.com/projects/details/707/results/53772/result/0">https://bwh-dope.aetion.com/projects/details/707/results/53772/result/0</a>

Marketscan- https://bwh-dope.aetion.com/projects/details/708/results/53771/result/0

Medicare- https://bwh-dope.aetion.com/projects/details/709/results/53770/result/0

Date conducted: 05/11/2020

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 3 covariates: age, sex, and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

• Stop analyses until feasibility and power are reviewed by primary investigators and FDA. Reviewers evaluate the results of the analyses described above in Sections 7 and 8, including numbers of patients, patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates of outcomes and study power. These parameters are re-evaluated and reported in the subsequent sections, after incorporating feedback and refining the protocol.

• Stop analyses until feasibility and power are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 6/3/20 |
|-------------------------|------------------|----------------|---------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 6/30/20 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

#### 9. Balance Assessment

#### Aetion report links:

Optum: https://bwh-dope.aetion.com/projects/details/707/results/59580/result/0
Marketscan: https://bwh-dope.aetion.com/projects/details/708/results/59603/result/0
Medicare: https://bwh-dope.aetion.com/projects/details/709/results/59604/result/0

Date conducted: 10/5/20 (Medicare 10/6/20)

After review of initial feasibility and power analyses, complete creation of the remaining covariates (see Table 1 below for list of covariates). Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates (excluding laboratory values, which are missing in some patients).

• Provide plot of PS distributions stratified by treatment group.

Note- Please refer to Appendix B.

• Report covariate balance after matching.

Note- For Table 1, please refer to **Appendix B**.

• Report reasons for censoring by treatment group.

| | Overall | Referent | Exposure |
|---|---|---|---|
| Dummy Outcome | 0 (0.00%) | 0 (0.00%) | 0 (0.00%) |
| Death | 657 (0.84%) | 369 (0.94%) | 288 (0.74%) |
| Start of an additional exposure | 2,760 (3.53%) | 1,189 (3.04%) | 1,571 (4.02%) |
| End of index exposure | 62,039 (79.39%) | 31,190 (79.83%) | 30,849 (78.96%) |
| Specified date reached (Dec 17/Dec 18/Dec 19) | 2,483 (3.18%) | 1,281 (3.28%) | 1,202 (3.08%) |
| End of patient enrollment | 4,128 (5.28%) | 1,938 (4.96%) | 2,190 (5.61%) |
| Switch to other NOACs (for censoring) + nursing home admission | 6,073 (7.77%) | 3,103 (7.94%) | 2,970 (7.60%) |

• Report follow-up time by treatment group.

| Median Follow-Up Time (Days) [IQR] | | | |
|---|---|---|---|
| Patient Group Optum Truven Medicare | | | |
| Overall Patient Population | 98 [38-191] | 98 [38-193] | 98 [38-202] |

Effectiveness research with Real World Data to support FDA's regulatory decision making

| Referent | 98 [43-192] | 98 [43-178] | 98 [42-196] |
|----------|-------------|-------------|-------------|
| Exposure | 98 [38-190] | 98 [38-220] | 98 [38-211] |

• Report overall risk of the primary outcome.

| | Optum | Marketscan | Medicare | Pooled |
|-------------------------|-------|------------|----------|--------|
| Risk per 1,000 patients | 4.57 | 5.20 | 6.04 | 5.64 |

#### 10. Final Power Assessment

#### Date conducted:

- Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9. All other parameters in the table should be the same as in Section 8. If the study is to be implemented in more than one database, copy and paste excel sheet to report power for each database separately and for the pooled analysis that uses data from all databases together. Power calculations are based on the formulas from Chow et al. (2008).
  - For dabigatran 150mg vs. warfarin
  - o Pooled

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | 78,140 | Number of patients matched | 78,140 |
| Reference | 39,070 | Reference | 39,070 |
| Exposed | 39,070 | Exposed | 39,070 |
| Risk per 1,000 patients | 5.64 | Risk per 1,000 patients | 5.64 |
| Desired HR from RCT | 0.66 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.46 |
| Number of events expected | 440.7096 | Number of events expected | 440.7096 |
| Power | 0.991836251 | Power | 0.977906369 |

### o Optum

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | 5,580 | Number of patients matched | 5,580 |
| Reference | 2,790 | Reference | 2,790 |
| Exposed | 2,790 | Exposed | 2,790 |
| Risk per 1,000 patients | 4.57 | Risk per 1,000 patients | 4.57 |
| Desired HR from RCT | 0.66 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.46 |
| Number of events expected | 25.5006 | Number of events expected | 25.5006 |
| Power | 0.182503488 | Power | 0.157581463 |

## o MarketScan

| t | | · | |
|---|---|---|---|
| Superiority Analysis | | Non-inferiority Analysis | |
| Number of patients matched | 27,920 | Number of patients matched | 27,920 |
| Reference | 13,960 | Reference | 13,960 |
| Exposed | 13,960 | Exposed | 13,960 |
| Risk per 1,000 patients | 5.20 | Risk per 1,000 patients | 5.20 |
| Desired HR from RCT | 0.66 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.46 |
| Number of events expected | 145.184 | Number of events expected | 145.184 |
| Power | 0.70656205 | Power | 0.625504572 |

# o Medicare

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | 44,640 | Number of patients matched | 44,640 |
| Reference | 22,320 | Reference | 22,320 |
| Exposed | 22,320 | Exposed | 22,320 |
| Risk per 1,000 patients | 6.04 | Risk per 1,000 patients | 6.04 |
| Desired HR from RCT | 0.66 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.46 |
| Number of events expected | 269.6256 | Number of events expected | 269.6256 |
| Power | 0.926676361 | Power | 0.874319968 |

 Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 9/8/20 |
|-------------------------|------------------|----------------|---------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 9/29/20 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

#### 11. Study Confidence and Concerns

Deadline for voting on study confidence and listing concerns:

Date votes and concerns are summarized:

- If final feasibility and power analyses are reviewed and approved, proceed to the remaining protocol steps.
- All study team and advisory board members that review this protocol should at this stage provide their level of confidence for the
  success of the RWD study in the <u>Google Form</u>. This form also provides space for reviewers to list any concerns that they feel may
  contribute to a failure to replicate the findings of the RCT, including differences in study populations, poor measurement of study
  variables, or residual confounding. All responses will be kept confidential and individual-level results will only be shared with the
  individual respondent.
- After the deadline for voting has passed, provide the distribution of responses and summarize all concerns here.

### 12. Register study protocol on clinicalTrials.gov

#### Date conducted:

• Register the study on <u>clinicalTrials.gov</u> and upload this document.

#### 13. Comparative Analyses

Action report name:

Date conducted:

### 13.1 For primary analysis:

## 13.2 For sensitivity analyses:

### 14. Requested Results

### 14.1 <u>Table 1: Baseline characteristics before and after adjustment</u>

| | Before adjustment | | | After adjustment | | |
|---|---|---|---|---|---|---|
| Variable | Referent | Exposur | Std. diff. | Referent | Exposur | Std. diff. |
| | | e | | | e | |
| Number of | | | - | | | - |
| patients | | | | | | |
| Age categories | | | | | | |

### 14.2 <u>Table 2: Follow-up time</u>

| Patient Group | Median Follow-Up Time (Days) [IQR] |
|----------------------------|------------------------------------|
| Overall Patient Population | |
| Referent | |
| Exposure | |

## 14.3 <u>Table 3: Censoring events</u>

| Overall | Referent | Exposure |
|---------|----------|----------|

| Outcome |
|---------------------------------|
| Death |
| Start of an additional exposure |
| End of index exposure |
| Specified date reached |
| End of patient data |
| End of patient enrollment |

### 14.4 <u>Table 4: Results from primary analyses;</u>

| Analysis | No. exposed events | No. referent events | Exposed rate | Referent rate | HR (95% CI) |
|---|---|---|---|---|---|
| Crude | | | | | |
| Analysis 1 | | | | | |
| Analysis 2 | | | | | |

HR, Hazard Ratio; CI, Confidence Interval.

## 14.5 <u>Table 5: Results from secondary analyses;</u>

### 15. References

Chow S, Shao J, Wang H. 2008. *Sample Size Calculations in Clinical Research*. 2nd Ed. Chapman & Hall/CRC Biostatistics Series. **page 177** 

Connolly SJ, Ezekowitz MD, Yusuf S, et al. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med. 2009; 361:113951.

| | DE IV trial definitions | Implementation in venting care | References/Rationale | Color coding |
|---|---|---|---|---|
| # | RE-LY trial definitions | Implementation in routine care | | coror county |
| | | | Please see the following Google Drive for further details or any missing information: | |
| | | | https://drive.google.com/open?id=1WD618wrywYjEaXzfLTcuK-VCcnb6b- | Criteria |
| | Trial details- Primary approval; U | nintended S with label change | gV | |
| | | | ICD-10 codes are not listed in this document because of excel cell size | |
| | | | limitations and excessive number of ICD-10 codes. Full ICD-10 code lists will be available in the above Google Drive Folder (link above). ICD-9 to ICD | |
| | | | 10 code conversions were completed using a SAS macro that implements | Adequate mapping in claims |
| | | | forward/ backward mapping based on the CMS ICD-9 to ICD-10 mapping: | |
| 1 | EXPOSURE vs. C | OMPARICON | https://www.nber.org/data/icd9-icd-10-cm-and-pcs-crosswalk-general- | |
| - | Fixed doses of dabigatran (110 mg or 150 mg twice daily) vs. adjusted-dose warfarin | DAMPARISON Dabigatran (110mg or 150mg twice daily) vs adjusted-dose warfarin | сумняется парридании | Intermediate mapping in claims |
| $\vdash$ | The source of sourbarian (TTO IIIE of The IIIE raice daily) as adjusted dose Mariann | Para-Param (1770m) or 190m) raice nemy) as enforced-noise manifelm | | |
| | PRIMARY OF | JTCOME | | Poor mapping or cannot be measured in claim: |
| | | Measured 1 day after drug initiation in diagnosis position and care setting specified below. | | |
| | | | For stroke: | |
| | | For stroke: | PPV of 85% or higher for ischemic stroke | |
| | | Primary diagnosis position in inpatient care setting<br>430.xx Subarachnoid hemorrhage (SAH) | PPV ranging from 80% to 98% for hemorrhagic stroke | |
| | | 431.xx Intracerebral hemorrhage (ICH) | → [Andrade SE, Harrold LR, Tjia J, et al. A systematic review of validated methods for identifying cerebrovascular accident or transient ischemic | |
| | | 433.x1 Occlusion and stenosis of precerebral arteries with cerebral infarction | attack using administrative data. Pharmacoepidemiology and Drug Safety | Can't be measured in claims but not important |
| | The primary outcome is a composite of stroke (including hemorrhagic) and systemic embolism event | 434.xx (excluding 434.x0) Occlusion and stenosis of cerebral arteries with cerebral infarction | 2012;21 Suppl 1:100-28.] | for the analysis |
| | | 436.x Acute, but ill-defined cerebrovascular events | →[Tirschwell DL, Longstreth WT, Jr. Validating administrative data in stroke<br>research. Stroke; a journal of cerebral circulation 2002;33:2465-70.] | |
| | | Systemic embolism (Arterial embolism and thrombosis): | → [Roumie CL, Mitchel E, Gideon PS, Varas-Lorenzo C, Castellsague J, Griffin | |
| 1 | | Primary diagnosis position in inpatient care setting | MR. Validation of ICD-9 codes with a high positive predictive value for | |
| 1 | | ICD-9: 444.xx | incident strokes resulting in hospitalization using Medicaid health data. Pharmacoepidemiology and drug safety 2008;17:20-6.] | |
| 1 | | ICD-10: I74.x | r narmacoepiueiniology and drug salety 2008;17:20-6.] | |
| | INCLUSION ( AF documented as follows: (1a or 1b or 1c) | CRITERIA TOTAL CONTROLL CONTROL CONTR | | 4 |
| | An accumented as rollows. (18 or 10 or 10) | Measured 4 weeks prior to and including day of drug initiation in any diagnosis position and any care setting | | 1 |
| | | Intersured 4 weeks prior to and including day of drug initiation in any diagnosis position and any care setting | | |
| 1: | There is ECG documented AF on the day of screening or randomization | Atrial fibrillation | | |
| 10 | - There is Eco documented Ar on the day of screening of fandomization | ICD-9 diagnosis: 427.31 | | |
| | | ICD-10 diagnosis: I48.0x, I48.1x, I48.2x, I48.9x | 1 | ĺ |
| | | Measured 12 months prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient | <del> </del> | 1 |
| | | Measured 12 months prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting | 1 | ĺ |
| | The second secon | | | |
| 11 | The patient has had a symptomatic episode of paroxysmal or persistent AF documented by 12-lead ECG within 6 m before randomization | Atrial fibrillation | | |
| | TO TO THE PARTY OF | ICD-9 diagnosis: 427.31 | | |
| | | ICD-10 diagnosis: I48.0x, I48.1x, I48.2x, I48.9x | 1 | ĺ |
| | There is documentation of symptomatic or asymptomatic paroxysmal or persistent AF on 2 separate occasions, at least 1 day | >2 Diagnoses separated by 1 day to 30 days, measured 12 months prior to and including day of drug initiation in any | | 1 |
| | <ul> <li>There is documentation of symptomatic or asymptomatic paroxysmal or persistent AF on 2 separate occasions, at least 1 day apart, one of which is within 6 m before randomization.</li> </ul> | >2 Diagnoses separated by 1 day to 30 days, measured 12 months prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting | 1 | |
| 4. | In this case, AF may be documented by 12 lead ECG, rhythm strip, pacemaker/ICD electrogram, or Holter ECG. The duration of | | 1 | ĺ |
| 10 | AF should be at least 30 s. | <u>Atrial fibrillation</u> | | |
| | Electrograms (not marker channels or mode switch episodes) from pacemakers and defibrillators can be used to document | ICD-9 diagnosis: 427.31 | 1 | ĺ |
| | only 1 episode of paroxysmal or persistent AF<br>In addition to documented AF, patients must have one of the following: (2a or 2b or 2c or 2d or 2e) | ICD-10 diagnosis: I48.0x, I48.1x, I48.2x, I48.9x | | 4 |
| | in addition to documented Ar., patients must have <b>one</b> of the following: <b>(2a or 20 or 20 or 20 or 20 or 20</b> | | | 1 |
| | | Measured any time prior to and including day of drug initiation in any diagnosis position and inpatient care setting Any stroke | 1 | ĺ |
| | | Any stroke<br>ICD-9 diagnosis: 430.xx, 431.xx, 433.xx, 434.xx, 436.xx | | |
| | | the sugarest seems, seems, results, results, results | | |
| 20 | History of previous stroke, TIA, or systemic embolism | Systemic embolism | 1 | ĺ |
| 20 | instary or premous second, they of systemic embolism | ICD-9 diagnosis: 444.xx (arterial embolism) | | |
| | | ICD-10 diagnosis: I74.x arterial embolism and thrombosis | 1 | ĺ |
| | | TIA | | |
| | | ICD-9 diagnosis: 435.xx ( Transient cerebral ischemia) | 1 | ĺ |
| | | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient care setting | | 1 |
| | | ivieasureu 100 uays prior to and including day of drug initiation in any diagnosis position and inpatient care setting | 1 | ĺ |
| | Ejection fraction <40% documented by echocardiogram, radionuclide or contrast angiogram | Heart failure, systolic | 1 | ĺ |
| 21 | in the last 6 m | ICD-9 diagnosis: 428.2x, 428.4x | 1 | ĺ |
| | | ICD-10 diagnosis: I50.2x, I50.4x | | |
| | | | | 4 |
| | | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient care setting | | |
| 20 | Symptomatic heart failure, New York Heart Association class 2 or higher in the last 6 m | Congestive heart failure | | |
| 1 | The state of the s | ICD-9 diagnosis: 428.x, 398.91, 402.01, 402.11, 402.91, 404.01, 404.11, 404.91, 404.03, 404.13, 404.93 | 1 | ĺ |
| | | ICD-10 diagnosis: I50.1, I50.2x, I50.3x, I50.4x, I50.8x, I50.9, I09.81, I11.0, I13.0, I13.2 | | j |
| | | Measured on the day of drug initiation | | 1 |
| 20 | • Age ≥75 y | | | |
| | | Age ≥75 | | j |

| Note of the second process of the second pro | 2e | • Age ≥65 y <b>and</b> one of the following: | Measured on the day of drug initiation |
|---|---|---|---|
| Action Millinations are promitted: 10.70 degrons: 413.xx CP3 degro | - | – Diabetes mellitus on treatment | Measured any time prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting Diabetes mellitus. ICD-9 diagnosis: 250.x1, 250.x3, 250.x0, 250.x2 ICD-10 diagnosis: 250.x1, 250.x3, 250.x0, 250.x2 ICD-10 diagnosis: 210.x, E11.x AND At least one of the following drug prescriptions from 0 to 30 days after diagnosis*: Boolus Insulin insulin human regular, Insulin Aspart, Insulin Gilulisine, Insulin Ispro, Insulin Aspart/Insulin Aspart Protamine, Insulin Ispro/Insulin Lispro Protamine, insulin,pork purified Basal Insulin: Insulin human isophane (NPH), Insulin human regular/ Insulin human isophane (NPH), Insulin Debemir, Insulin Glargine, Insulin Degludec, Insulin zinc human rec, Insulin zinc extend human rec, Insulin nph human recom/insulin regular human rec, Insulin zinc human rec, Insulin pin human recom/insulin regular human rec Metformin DDP4 inhibitors: Alogliptin, Linagliptin, Saxagliptin, Sitagliptin Sulfonylureas Acetohexamide, Chlorpropamide, tolazamide, tolbutamide, Glipizide, Glyburide, Glimepiride Meglitinide derivatives Repaglinide, Nateglinide Alpha-glucosidase inhibitors Acarbose, Miglitol Thiazolidimediones (TZDs) Rossiglitazone, Pioglitazone Glucagonilke peptide—1 (G1P-1) agonists Exenatide, Liraglutide, Lixisenatide, Albiglutide, Dulaglutide, semaglutide SG121 hibibitors Canaglificior, Dapaglificor, Empaglificior, Erruglificior |
| Care setting Hypertension ICD 9 diagnosis: 401.x – 405.x AND Al least one drug prescriptions from 0 to 14 days after diagnosis*: ACE inhibitor Benazepril, captopril, enalapril, fosinopril, lisinopril, mexipril, perindopril, quinapril, ramipril, trandolapril ARB Azilsartan, candesartan, eprosartan, irbesartan, losartan, olmesartan, telmisartan, valsartan Beta blocker Acebutolol, atenolol, betavolol, bisoprolol, caredolo, caredolo, caredolo, enetoprolol succinate, propranolol, penbutolol, penbutolol, penbutolol, penbutolol, of periodiol, desidolol, timolol Calcium channel blocker Diltiazem, mibefradil, verapamil, amlodipine, clevidipine, bepridil, felodipine, isradipine, nicardipine, penbutolol, sold, aliskiren, apraclonidine Other hypertension drugs Doxazosin, eplerenone, prazosin, terazosin, clonidine, guanadrel, guanethidine, guanfacine, hydralazine, methyldopa, metyrosine, reserpine, minoxidil, aliskiren, apraclonidine Measured on the day of drug initiation Age >18 | | – Documented coronary artery disease (any of: prior myocardial infarction, positive stress test, positive nuclear perfusion study, prior CABG surgery or PCI, angiogram showing ≥75% stenosis in a major coronary artery | Acute MI (Inpatient, any position): ICD-9 diagnosis: 410.xx Old MI (Inpatient, any position): ICD-9 diagnosis: 412.xx Angina sectors (Inpatient, any position): ICD-9 diagnosis: 412.xx ICD-9 diagnosis: 412.xx ICD-9 diagnosis: 413.x ICD-9 diagnosis: 413.x ICD-9 diagnosis: 413.x ICD-9 diagnosis: 414.xx ICD-10 diagnosis: 141.xx ICD-10 procedure: 361.xx ICD-10 procedure: 361.xx ICD-10 procedure: 361.xx ICD-10 procedure: 00.66, 36.01, 36.02, 36.03, 36.03, 36.09 ICD-10 procedure: Coronary bypass in Coronary Revascularization sheet ICD-10 procedure: Coronary bypass in Coronary Revascularization sheet ICD-11 coronary Revascularization sheet ICD-12 procedure: 361.xx ICD-13 procedure: 361.xx ICD-10 procedure: Coronary Revascularization sheet ICD-12 procedure: Coronary Revascularization sheet ICD-13 procedure: 361.xx ICD-14 coronary Revascularization sheet ICD-15 procedure: 361.xx ICD-16 procedure: 361.xx ICD-17 coronary Revascularization sheet ICD-17 coronary Revascularization sheet ICD-17 coronary Revascularization sheet ICD-18 procedure: 361.xx ICD-19 procedure: 361.xx ICD-10 procedure: 3 |
| 3 Age >18 y at entry Age >18 | - | – Hypertension requiring medical treatment | care setting Hypertension ICD-9 diagnosis: 401.x – 405.x AND At least one drug prescriptions from 0 to 14 days after diagnosis*: ACE inhibitor Benazepri, captopri, enalapril, fosinopril, lisinopril, moexipril, perindopril, quinapril, ramipril, trandolapril ARB Azilsartan, candesartan, eprosartan, ibestartan, losartan, telmisartan, valsartan Beta blocker Acebutolol, atenolol, betavolol, bisoprolol, carteolol, carvedilol, esmolol, labetalol, metoprolol succinate, propranolol, penbutolol, polindolol, adolol), nebivolol, sotalol, timdol Calcium channel blocker Diltiazem, mibefradil, verapamil, amlodipine, clevidipine, bepridil, felodipine, isradipine, nicardipine, nimodipine, nisodipine Other hypertension drugs Doxaszoin, eplerenone, prazosin, terazosin, clonidine, guanabenz, guanabenz, guanatidine, |
| 4 Written, informed consent N/A | | | Age >18 |
| 4 Written, informed corsent IN/A EXCLUSION CRITERIA | 4 1 | | |

| | | Measured anytime prior to and including day of drug initiation in any diagnosis position and inpatient care setting 394 x (diseases of mitral valve), 395 x (diseases of a cortic valve), 395 x (diseases of mitral and a ortic valve) 397.x (diseases of other endocardial incructures), 398.9 x (other and unspecified rheumatic heart diseases) V42.2 (heart valve replaced by transplant), V43.3 (heart valve replaced by a mechanical device/prosthesis) |
|---|---|---|
| 1 | History of heart valve disorders (ie, prosthetic valve or hemodynamically relevant valve disease) | OR. ICD-9 procedure code 35.1x (open heart valvuloplasty without replacement), 35.2x (replacement of heart valve) OR- one of the following CPT codes: 33660-33665 (atrioventricular valve repair) 33400-33405 (artic valve valvuloplasty) 33400-33405 (artic valve valvuloplasty) 33405 (Replacement, aortic valve, with cardiopulmonary bypass; with prosthetic valve other than homograft or stentless valve) 33420-33430 (mitral valve repair/valvuloplasty/replacement) 33460-33463 (irticuspid valve repair/valvuloplasty/replacement) 33465-33466 (tricuspid valve repair/valvuloplasty/replacement) 33475 (replacement, pulmonary valve) 33496 (prosthetic valve dysfunction repair) 02577 (implantation of catheter-delivered prosthetic aortic heart valve; open thoracic approach) 02581 (transthoracic cardiac exposure for catheter-delivered aortic valve replacement; without cardiopulmonary bypass) 02627 (implantation of catheter-delivered prosthetic pulmonary valve, endovascular approach) |
| 2 | or<br>Any stroke within the previous 14 days | 1) Disabling stroke effects Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting ICD-9 diagnosis: 438.xx (Late effects of cerebrovascular disease) ICD-10 diagnosis: 169 (Sequelae of cerebrovascular disease) ICD-10 diagnosis: 169 (Sequelae of cerebrovascular disease) ICD-10 diagnosis: 273.6 (Limitation of activities due to disability) -OR- 2) Any stroke: Measured 14 days prior to and including day of drug initiation in primary diagnosis position and inpatient care setting ICD-9 diagnosis: 430.xx, 431.xx, 433.xx, 434.xx, 436.xx |
| 3 | Conditions associated with an increased risk of bleeding: | |
| 3a | Major surgery in the <b>previous month</b> | Measured 30 days prior to and including day of drug initiation in any procedure position and inpatient or outpatient care setting: 10-9 procedure codes: Major surgery selected from codes range 34.x-84.x 30-34 Operations On The Respiratory System 35-39 Operations On The Cardiovascular System 40-41 Operations On The Hemic And Lymphatic System 42-54 Operations On The Urinary System 55-59 Operations On The Urinary System 60-64 Operations On The Home Genital Organs 65-71 Operations On The Hemic And System 72-75 Obstetrical Procedures 72-75 Obstetrical Procedures 78-84 Operations On The Musculoskeletal System |
| 3b | Planned surgery or intervention in the next 3 m | N/A |
| 3с | History of intracranial, intraocular, spinal, retroperitoneal or atraumatic intra-articular bleeding | Measured anytime prior to and including day of drug initiation in any diagnosis position and inpatient care setting Intracranial hemorrhage: ICD-9: 430.x, 431.x, 432.x Intraocular hemorrhage: 379.23 vitreous hemorrhage, |
| | | 362.81 retinal hemorrhage<br>H35.6x |

| $\overline{}$ | | |
|---|---|---|
| | | Measured 365 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting: |
| | | ICD-9 diagnosis: 578.x Gastrointestinal hemorrhage |
| 3d | | ICD-10 diagnosis: K92.2: Gastrointestinal hemorrhage, unspecified acute hemorrhagic gastritis (K29.01) peptic ulcer with hemorrhage (K25.4 - excluding K25.9 - K26.x - excluding K26.9 - K27.x-K28.x) gastritis and duodenitis with hemorrhage (K29.x) diverticular disease with hemorrhage (K57.x) anglodysplasia of stomach with hemorrhage (K31.811) |
| | | CPT/HCPCS: OW3P8ZZ - (ICD10) Control Bleeding in Gastrointestinal Tract, Via Natural or Artificial Opening Endoscopic 43255 - (IHCPCS) Esophagogastroduodenoscopy, flexible, transoral; with control of bleeding, any method / Upper gastrointestinal endoscopy including esophagus, stomach, and either the duodenum and/or jejunum as appropriate; with control of bleeding, any method 44.43 - (ICD9) ENDOSCOPIC CONTROL OF GASTRIC OR DUODENAL BLEEDING |
| | | Measured 30 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting: |
| 3е | Symptomatic or endoscopically documented gastroduodenal ulcer disease in the previous 30 days | ICD-9 diagnosis: Disease of esophagus: 530.1x-530.4x, 530.8x, 530.9x Gastric ulcer: 531.x Duodenal ulcer: 532.x Peptic ulcer: 533.x Acute gastritis: 535.0x Other specified gastritis: 535.4x Unspecified gastritis: 535.6x Duodenitis: 535.6x |
| | | ICD-10 diagnosis: Peptic ulcer, site unspecified K27.x K25.9 - Gastric ulcer, unspecified as acute or chronic, without hemorrhage or perforation K26.9 Duodenal ulcer, unspecified as acute or chronic, without hemorrhage or perforation |
| | | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting |
| 3f | • Hemorrhagic disorder or bleeding diathesis | Bleeding diathesis: ICD-9 diagnosis: 287.x Purpura and other hemorrhagic conditions ICD-10 diagnosis: D65.x Disseminated intravascular coagulation [defibrination syndrome] D66.x Hereditary factor VIII deficiency D67.x Hereditary factor VX deficiency D68.x Other coagulation defects |
| | | D69.x Purpura and other hemorrhagic conditions |
| 3g | Need for anticoagulant treatment of disorders other than Atrial fibrillation | N/A We will censor the patients upon initiating these drugs after cohort entry: |
| 3h | • Fibrinolytic agents within 48 h of study entry | Fibrinolytic agent: Alteplase, reteplase, tenecteplase, streptokinase, urkinase |
| 3i | Uncontrolled hypertension (systolic blood pressure >180 mm Hg and/ or diastolic blood pressure >100 mm Hg) | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting Malignant hypertension: ICD-9 diagnosis: 401.0x (no ICD-10) Hypertensive urgency/ Hypertensive crisis: ICD-10 diagnosis: I16.x (no ICD-9) |
| | Recent malignancy or radiation therapy (≤6 m) <u>and</u> not expected to survive 3 y | N/A |
| | Contraindication to warfarin treatment Reversible causes of atrial fibrillation (eg, cardiac surgery, pulmonary embolism, | N/A |
| , | untreated hyperthyroidism). | N/A |
| 6 | Plan to perform a pulmonary vein ablation or surgery for cure of the AF | N/A Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting |
| 7 | Severe renal impairment (estimated creatinine clearance ≤30 mL/min) | <u>CKD stage 4/5/ESRD</u><br>ICD-9 diagnosis: 585.4x, 585.5x, 585.6x<br>ICD-10 diagnosis: N18.4x, N18.5x, N18.6x |
| 1 | | <u>Dialysis/ Renal transplant</u> Codes are in the sheet "Dialysis and Renal Transplant" |

| Active infective endocarditis | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting Infective endocarditis | |
|---|---|---|
| | ICD-9 diagnosis: 421.x ICD-10 diagnosis: l33.x | |
| Active liver disease, including but not limited to: | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting Acute Liver Disease: ICD-9 diagnosis: 070.xx, 570.xx, 576.xx, 782.4x, 789.5x ICD-10 diagnosis: 815.x, B16.x, B17.x, K76.x, R17.x, R18.x, K72.00, K76.2 | |
| Persistent ALT, AST, Alk Phos > 2x LILN | N/A | |
| Active nepatitis A | N/A | |
| Women who are pregnant or of childbearing potential who refuse to use a medically acceptable form of contraception throughout the study | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting | |
| | coues are in the sheet. Fregulaticy | |
| Anemia (hemoglobin level < $100 g/L$ ) or thrombocytopenia (platelet count < $100 \times 109/L$ ) | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting Anemia (non-deficiency/neoplastic/chemotherapy/hemorrhagic assoicated) ICD-9 diagnosis: 282.x, 283.x, 284.x, 285.x ICD-10 diagnosis: D62, D63.0 Thrombocytopenia: ICD-9 diagnosis: 287.3x, 287.4x, 287.5x ICD-10 diagnosis: D69.3x, D69.4x, D69.5x, D69.6x | |
| Patients who have developed transaminase elevations upon exposure to ximelagatran. | | |
| Patients who have received an investigational drug in the past 30 d | N/A | |
| Patients considered unreliable by the investigator or have a life expectancy less than the expected duration of the trial because of concomitant disease, or has any condition which in the opinion of the investigator, would not allow safe participation in the study (eg. drug addiction, alcohol abuse) | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting CCI >=10 (life expectancy less than the expected duration of the trial) -OR- Alcohol abuse or dependence ICD-9 diagnosis: 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x (CMS has not released mapping for new ICD10 for this code), V11.3x ICD-10 diagnosis: F10.x, K70x, G62.1, I42.6, 099.31x Drug abuse or dependence 292.xx, 304.xx, 305.2x-305.9x, 648.3x 965.0x, 967.xx, 969.4x-969.6x, 969.72-969.79, 970.81 ICD-10 diagnosis: F11.x, F12.x, F13.x, F14x, F15.x, F18.x, F19.x, G62.0, 099.32x | |
| Any known hypersensitivity to galactose if the warfarin used contains galactose. | N/A | |
| | Active liver disease, including but not limited to: Persistent ALT, AST, Alk Phos > 2× ULN Known active hepatitis C (positive HCV RNA) Active hepatitis B (HBS antigen +, anti HBc IgM+) Active hepatitis B (sas antigen +, anti HBc IgM+) Active hepatitis B (hBS antigen +, anti HBC IgM+) Active hepatitis B (hBS antigen +, anti HBC IgM+) Active hepatitis B ( | Active infective endocariditis Control disprace Control disprace |

| <u>Trial ID</u> | pNDA22 |
|---|---|
| Trial Name (with web links) | <u>RE-LY</u> |
| <u>NCT</u> | NCT00262600 |
| Therapeutic Area | Cardiology/Vascular Diseases |
| <b>Brand Name</b> | <u>Pradaxa</u> |
| <b>Generic Name</b> | dabigatran etexilate mesylate |
| Sponsor | Boehringer Ingelheim |
| <u>Year</u> | 2010 |
| pNDA Indication | For the risk reduction of stroke and embolism due to atrial fibrillation |
| Measurable endpoint | primary composite endpoint of stroke and systemic embolism |
| Trial finding | Rates of the primary outcome were 1.69% per year in the warfarin group, as compared with 1.53% per year in the group that received 110 mg of dabigatran (relative risk with dabigatran, 0.91; 95% confidence interval [CI], 0.74 to 1.11; P<0.001 for noninferiority) and 1.11% per year in the group that received 150 mg of dabigatran (relative risk, 0.66; 95% CI, 0.53 to 0.82; P<0.001 for superiority). |
| Blinding | fixed doses of dabigatran — 110 mg or 150 mg twice daily —each administered in a blinded manner, and adjusted-dose warfarin in an unblinded fashion |
| No. of Patients | 18,113 |
| Comparator | Active |

72.3 HIGH FORCEPS OPERATION

## **Pregnancy** Diagnosis codes 650 NORMAL DELIVERY 660 OBSTRUCTED LABOR 661 ABNORMALITY OF FORCES OF LABOR 662 LONG LABOR 663 UMBILICAL CORD COMPLICATIONS DURING LABOR AND DELIVERY 664 TRAUMA TO PERINEUM AND VULVA DURING DELIVERY 665 OTHER OBSTETRICAL TRAUMA 667 RETAINED PLACENTA OR MEMBRANES WITHOUT HEMORRHAGE 668 COMPLICATIONS OF THE ADMINISTRATION OF ANESTHETIC OR OTHER SEDATION IN LABOR AND DELIVERY 669.94 UNSPECIFIED COMPLICATION OF LABOR AND DELIVERY POSTPARTUM CONDITION OR COMPLICATION V24 POSTPARTUM CARE AND EXAMINATION V24.0 POSTPARTUM CARE AND EXAMINATION IMMEDIATELY AFTER DELIVERY V24.1 POSTPARTUM CARE AND EXAMINATION OF LACTATING MOTHER V24.2 ROUTINE POSTPARTUM FOLLOW V27 OUTCOME OF DELIVERY V27.0 MOTHER WITH SINGLE LIVEBORN V27.1 MOTHER WITH SINGLE STILLBORN+A2:J81 V27.2 MOTHER WITH TWINS BOTH LIVEBORN V27.3 MOTHER WITH TWINS ONE LIVEBORN AND ONE STILLBORN V27.4 MOTHER WITH TWINS BOTH STILLBORN V27.5 MOTHER WITH OTHER MULTIPLE BIRTH ALL LIVEBORN V27.6 MOTHER WITH OTHER MULTIPLE BIRTH SOME LIVEBORN V27.7 MOTHER WITH OTHER MULTIPLE BIRTH ALL STILLBORN V27.9 MOTHER WITH UNSPECIFIED OUTCOME OF DELIVERY Procedure codes 72.0 LOW FORCEPS OPERATION 72.1 LOW FORCEPS OPERATION WITH EPISIOTOMY 72.2 MID FORCEPS OPERATION 72.21 MID FORCEPS OPERATION WITH EPISIOTOMY 72.29 OTHER MID FORCEPS OPERATION

- 72.31 HIGH FORCEPS OPERATION WITH EPISIOTOMY
- 72.39 OTHER HIGH FORCEPS OPERATION
- 72.4 FORCEPS ROTATION OF FETAL HEAD
- 72.5 BREECH EXTRACTION
- 72.51 PARTIAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD
- 72.52 OTHER PARTIAL BREECH EXTRACTION
- 72.53 TOTAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD
- 72.54 OTHER TOTAL BREECH EXTRACTION
- 72.6 FORCEPS APPLICATION TO AFTERCOMING HEAD
- 72.7 VACUUM EXTRACTION
- 72.71 VACUUM EXTRACTION WITH EPISIOTOMY
- 72.79 OTHER VACUUM EXTRACTION
- 72.8 OTHER SPECIFIED INSTRUMENTAL DELIVERY
- 72.9 UNSPECIFIED INSTRUMENTAL DELIVERY
- 73.0 ARTIFICIAL RUPTURE OF MEMBRANES
- 73.01 INDUCTION OF LABOR BY ARTIFICIAL RUPTURE OF MEMBRANES
- 73.09 OTHER ARTIFICIAL RUPTURE OF MEMBRANES
- 73.1 OTHER SURGICAL INDUCTION OF LABOR
- 73.2 INTERNAL AND COMBINED VERSION AND EXTRACTION
- 73.21 INTERNAL AND COMBINED VERSION WITHOUT EXTRACTION
- 73.22 INTERNAL AND COMBINED VERSION WITH EXTRACTION
- 73.3 FAILED FORCEPS
- 73.4 MEDICAL INDUCTION OF LABOR
- 73.5 MANUALLY ASSISTED DELIVERY
- 73.51 MANUAL ROTATION OF FETAL HEAD
- 73.59 OTHER MANUALLY ASSISTED DELIVERY
- 73.6 EPISIOTOMY
- 73.8 OPERATIONS ON FETUS TO FACILITATE DELIVERY
- 73.9 OTHER OPERATIONS ASSISTING DELIVERY
- 73.91 EXTERNAL VERSION ASSISTING DELIVERY
- 73.92 REPLACEMENT OF PROLAPSED UMBILICAL CORD
- 73.93 INCISION OF CERVIX TO ASSIST DELIVERY
- 73.94 PUBIOTOMY TO ASSIST DELIVERY
- 73.99 OTHER OPERATIONS ASSISTING DELIVERY
- 74.0 CLASSICAL CESAREAN SECTION

- 74.1 LOW CERVICAL CESAREAN SECTION
- 74.2 EXTRAPERITONEAL CESAREAN SECTION
- 74.3 REMOVAL OF EXTRATUBAL ECTOPIC PREGNANCY
- 74.4 CESAREAN SECTION OF OTHER SPECIFIED TYPE
- 74.9 CESAREAN SECTION OF UNSPECIFIED TYPE
- 74.91 HYSTEROTOMY TO TERMINATE PREGNANCY
- 74.99 OTHER CESAREAN SECTION OF UNSPECIFIED TYPE
- 75.4 MANUAL REMOVAL OF RETAINED PLACENTA
- 75.5 REPAIR OF CURRENT OBSTETRIC LACERATION OF UTERUS
- 75.6 REPAIR OF OTHER CURRENT OBSTETRIC LACERATION
- 75.7 MANUAL EXPLORATION OF UTERINE CAVITY, POSTPARTUM
- 75.9 OTHER OBSTETRIC OPERATIONS

#### Dialysis codes

ESRD, defined as 2 codes (either inpatient or outpatient), separated by at least 30 days

Codes include:

- ICD9 prox codes:

39.95, Hemodialysis

54.98, Peritoneal dialysis

-ICD9 dx codes:

585.5x, Chronic kidney disease, Stage V (for ESRD with no mention of dialysis)

585.6x, End stage renal disease (for ESRD with dialysis)

V56.0x, encounter for dialysis NOS

V56.8x, encounter for peritoneal dialysis

V45.1x, renal dialysis status

- CPT4 codes:

90957, 90960, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 4 or more face-to-face physician visits per month

90958, 90961, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 2-3 face-to-face physician visits per month

90959, 90962, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 1 face-to-face physician visit per month

90920, 90921, ESRD related services per full month; for patients 12-19 and twenty years of age and over

90924, 90925, ESRD related services (less than full month), per day; for patients 12-19 and twenty years of age and over

90935, Hemodialysis procedure with single physician evaluation

90937, Hemodialysis procedure requiring repeated evaluation(s) with or without substantial revision of dialysis prescription

90945, Dialysis procedure other than hemodialysis (eg, peritoneal dialysis, hemofiltration, or other continuous renal replacement therapies), with single physician evaluation

90947, Dialysis procedure other than hemodialysis (eg, peritoneal dialysis, hemofiltration, or other continuous renal replacement therapies) requiring repeated physician evaluations, with or without substantial revision of dialysis prescription

90965, 90966, ESRD related services for home dialysis per full month, for patients 12-19 and 20 years of age and older

90969, 90970, ESRD related services for dialysis less than a full month of service, per day; for patients 12-19 and 20 years of age and older

90989 Dialysis training natient including helner where annlicable any mode completed course

ooooo, piaryois training, patient, meraanig nerper where appheasie, any mode, completed course

90993, Dialysis training, patient, including helper where applicable, any mode, course not completed, per training session

90999, Unlisted dialysis procedure, inpatient or outpatient

99512, Home visit for hemodialysis

- HCPCS codes:

G0257, Unscheduled or emergency dialysis treatment for ESRD patient in a hospital outpatient dept. that is not certified as an ESRD facility

G0314, G0317, ESRD related services during the course of treatment, for patients 12-19 and 20 yrs of age an over to include monitoring for the adequacy of nutrition, etc. w/4 or more physician visit per month

G0315, G0318, ESRD related services during the course of treatment, for patients 12-19 and 20yrs of age and over to include monitoring for the adequacy of nutrition, etc. w/2 or 3 physician visit per month

G0316, G0319, ESRD related services during the course of treatment, for patients 12-19 and 20 yrs of age and over to include monitoring for the adequacy of nutrition, etc. w/1 physician visit per month

G0322, G0323, ESRD related services for home dialysis patients per full month: for patients 12-19 and 20 yrs of age and over to include monitoring for adequacy of nutrition and etc.

G0326, G0327, ESRD related services for home dialysis (less than full month), per day; for patients 12-19 and 20 yrs of age and over

S9335, Home therapy, hemodialysis; administrative services, professional pharmacy services, care coordination, and all necessary supplies and equipment (drugs and nursing services coded separately), per diem

S9339, Home therapy, peritoneal dialysis, administrative services, care coordination and all necessary supplies and equipment, per diem

OR

Kidney transplant, defined as either 1 inpatient or 1 outpatient code

Codes include:

-ICD9 dx codes:

V42.0x, Kidney transplant status

996.81 Complications of transplanted kidney

-ICD9 prox codes:

55.6x, Transplant of kidney (Exclude 55.61)

- CPT4 codes:

50360, Renal allotransplantation, implantation, graft, w/o donor & recipient nephrectomy

50365, Renal allotransplantation, implantation, graft, w/donor & recipient nephrectomy

#### **Documented Coronary Artery Disease**

```
ICD10: Coronary Bypass -
```

```
02.10083, 02.1008x, 02.1009x, 02.100Ax, 02.100Jx, 02.100Kx, 02.100Zx, 02.10483, 02.10488, 02.10489,
02.1048x, 02.1049x, 02.1049x, 02.104Ax, 02.104Jx, 02.104Kx, 02.104Zx, 02.1108x, 02.1109x, 02.110Ax,
02.110Jx, 02.110Kx, 02.110Zx, 02.1148x, 02.1149x, 02.114Ax, 02.114Jx, 02.114Kx, 02.114Zx, 02.1208x,
02.1209x, 02.120Ax, 02.120Jx, 02.120Kx, 02.120Zx, 02.1248x, 02.1249x, 02.124Ax, 02.124Jx, 02.124Kx,
02.124Zx, 02.1308x, 02.1309x, 02.130Ax, 02.130Jx, 02.130Kx, 02.130Zx, 02.1348x, 02.1349x, 02.134Ax,
02.134x, 02.134Kx, 02.134Zx, 02.1K0Zx, 02.1K4Zx, 02.1L08X, 02.1L09x, 02.1L0Ax, 02.1L0Jx, 02.1L0Kx, 02.1l0Zx,
02.1L0Zx, 02.1L48X, 02.1L49x, 02.1L4xx, 02.7004x, 02.7006x, 02.7007x, 02.700Dx, 02.700Ex, 02.700Fx,
02.700Gx, 02.700Tx, 02.700Zx, 02.703xx, 02.704xx, 02.7104x, 02.7105x, 02.7106x, 02.7107x, 02.710Dx,
02.710Ex, 02.710Fx, 02.710Gx, 02.710Tx, 02.710Zx, 02.7134x, 02.7135x, 02.7136x, 02.7137x, 02.713Dx,
02.713Ex, 02.713Fx, 02.713Gx, 02.713Tx, 02.713Zx, 02.7144x, 02.7145x, 02.7146x, 02.7147x, 02.714Dx,
02.714Ex, 02.714Fx, 02.714Gx, 02.714Tx, 02.714Zx, 02.7204x, 02.72056, 02.72066, 02.7206Z, 02.72076,
02.7207Z, 02.720Dx, 02.720Ex, 02.720Fx, 02.720Tx, 02.720Zx, 02.7234x, 02.7235x, 02.7236x, 02.7237x,
02.7237x, 02.723Dx, 02.723Ex, 02.723Fx, 02.723Gx, 02.723Tx, 02.723Tx, 02.723Zx, 02.723Zx, 02.7244x,
02.7245x, 02.7246x, 02.7247x, 02.724Dx, 02.724Ex, 02.724Fx, 02.724Gx, 02.724Tx, 02.7304x, 02.7304x,
02.7305x, 02.7306x, 02.7307x, 02.730Dx, 02.730Ex, 02.730Fx, 02.730Gx, 02.730Tx, 02.730Zx, 02.7334x,
02.7335x, 02.7336x, 02.7337x, 02.733Dx, 02.733Ex, 02.733Fx, 02.733Gx, 02.733Tx, 02.733Zx, 02.7344x,
02.7345x, 02.7346x, 02.7347x, 02.734Dx, 02.734Ex, 02.734Fx, 02.734Gx, 02.734Tx, 02.734Zx, 02.C00Zx,
02.C03Zx, 02.C04Zx, 02.C10Zx, 02.C13Zx, 02.C14Zx, 02.C20Zx, 02.C23Zx, 02.C24Zx, 02.C30Zx, 02.C33Zx, 02.C34Zx
```

#### Stenting:

Inpatient CPT-4:

92980, 92981, 92928-92929, 92933-92934

OR-

Inpatient ICD-9 Procedure:

36.06

36.07

Inpatient ICD-10 Procedure:

02.7004x, 02.7005x, 02.7006x, 02.7007x, 02.700Dx, 02.700Ex, 02.700Fx, 02.700Gx, 02.700Tx, 02.700Zx, 02.7034x, 02.7035x, 02.7036x, 02.7037x, 02.703Dx, 02.703Ex, 02.703Fx, 02.703Gx, 02.703Tx, 02.703Zx, 02.7044x, 02.7045x, 02.7046x, 02.7047x, 02.704Dx, 02.704Ex, 02.704Fx, 02.704Gx, 02.704Tx, 02.704Zx, 02.7104x, 02.7105x, 02.7106x, 02.7107x, 02.710Dx, 02.710Ex, 02.710Fx, 02.710Gx, 02.710Tx, 02.710Zx,

02.71346. 02.7134Z, 02.71356, 02.7135Z, 02.71366, 02.7136Z, 02.71376, 02.7137Z, 02.713D6, 02.713DZ, 02.713E6, 02.713EZ, 02.713F6, 02.713F2, 02.713G6, 02.713G2, 02.713T6, 02.713T2, 02.713Z6, 02.713Z2, 02.71446, 02.71447, 02.71456, 02.71457, 02.71466, 02.71467, 02.71476, 02.71477, 02.71406, 02.71407, 02.714E6, 02.714EZ, 02.714F6, 02.714F2, 02.714G6, 02.714GZ, 02.714T6, 02.714TZ, 02.714ZZ, 02.72046, 02.7204z, 02.72056, 02.7205z, 02.72066, 02.7206z, 02.72076, 02.7207z, 02.720D6, 02.720Dz, 02.720E6, 02.720EZ, 02.720F6, 02.720FZ, 02.720G6, 02.720GZ, 02.720T6, 02.720TZ, 02.720Z6, 02.720ZZ, 02.72346, 02.7234Z, 02.72356, 02.7235Z, 02.72366, 02.7236Z, 02.7237G, 02.7237Z, 02.723DG, 02.723DZ, 02.723EG, 02.723EZ, 02.723F6, 02.723FZ, 02.723G6, 02.723GZ, 02.723T6, 02.723TZ, 02.723Z6, 02.723ZZ, 02.72446, 02.7244Z, 02.72456, 02.7245Z, 02.72466, 02.7246Z, 02.7247G, 02.7247Z, 02.724DG, 02.724DZ, 02.724EG, 02.724EZ, 02.724F6, 02.724FZ, 02.724G6, 02.724T6, 02.724TZ, 02.724Z6, 02.724ZZ, 02.73046, 02.7304Z, 02.73056, 02.7305Z, 02.73066, 02.7306Z, 02.73076, 02.7307Z, 02.730D6, 02.730DZ, 02.730E6, 02.730EZ, 02.730F6, 02.730FZ, 02.730G6, 02.730GZ, 02.730T6, 02.730TZ, 02.730TZ, 02.730Z6, 02.730ZZ, 02.73346, 02.7334Z, 02.73356, 02.7335Z, 02.73366, 02.7336Z, 02.73376, 02.73376, 02.7337Z, 02.733DG, 02.733DZ, 02.735DZ, 02.735DZ, 02.735DZ, 02.755DZ, 02.702.733E6, 02.733EZ, 02.733F6, 02.733FZ, 02.733G6, 02.733GZ, 02.733T6, 02.733TZ, 02.733Z6, 02.733ZZ, 02.733ZZ, 02.73446, 02.7344Z, 02.73456, 02.7345Z, 02.73466, 02.73476, 02.7347Z, 02.34D6, 02.734DZ, 02.734E6, 02.734EZ, 02.734F6, 02.734FZ, 02.734G6, 02.734GZ, 02.734T6, 02.734TZ, 02.734Z6, 02.734ZZ, 02.C00Z6, 02.C03Z6, 02.C03ZZ, 02.C04Z6, 02.C10Z6, 02.C13Z6, 02.C13ZZ, 02.C14Z6, 02.C20Z6, 02.C23Z6, 02.C23ZZ, 02.C24Z6, 02.C30Z6, 02.C33ZZ, 02.C34Z6



| | | | | | Unmatched | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Optur | n I | | Market | | | M | edicare | | | POOLED | |
| Variable | WARFARIN | Dabigatran 150mg | St. Diff. | Reference - warfarin | Forestone Debientone 150mm | St. Diff. | Reference - warfarin | Function Debies to 150mm | St. Diff. | Reference - warfarin | Exposure - Dabigatran<br>150mg | St. Diff. |
| Number of patients | 22.665 | 2.936 | St. Diff. | Keterence - wartarın<br>67,790 | Exposure - Dabigatran 150mg<br>14.929 | St. Diff. | 136,087 | Exposure - Dabigatran 150mg<br>25.230 | St. Diff. | Reference - warfarin<br>226.542 | 150mg<br>43.095 | St. Diff. |
| Age | 22,003 | 2,550 | | 07,750 | 14,323 | | 130,007 | 23,230 | | 220,542 | 43,033 | |
| mean (sd) | 77.97 (6.21) | 74.91 (7.65) | 0.44 | 78.02 (9.20) | 74.13 (9.67) | 0.41 | 79.43 (7.37) | 76.93 (6.88) | 0.35 | 78.86 (7.86) | 75.82 (8.01) | 0.38 |
| median [IOR] | 79.00 [76.00, 82.00] | 77.00 [70.00, 80.00] | 0.29 | 79.00 [74.00, 84.00] | 76.00 [68.00, 81.00] | 0.32 | 79.00 [75.00, 84.00] | 77.00 [73.00, 81.00] | 0.28 | 79.00 (7.86) | 76.65 (8.01) | 0.30 |
| Age categories without zero category | 75.00 [70.00, 82.00] | 77.00 [70.00, 80.00] | 0.25 | 75.00 [74.00, 84.00] | 70.00 [08.00, 81.00] | 0.32 | 75.00 [75.00, 84.00] | 77.00 [73.00, 81.00] | 0.28 | 75.00 (7.80) | 70.03 (8.01) | 0.30 |
| 18 - 54; n (%) | 128 (0.6%) | 54 (1.8%) | -0.11 | 1.319 (1.9%) | 586 (3.9%) | -0.12 | 586 (0.4%) | 123 (0.5%) | -0.01 | 2.033 (0.9%) | 763 (1.8%) | -0.08 |
| 55 - 64; n (%) | 573 (2.5%) | 198 (6.7%) | -0.20 | 4,878 (7.2%) | 1,917 (12.8%) | -0.12 | 1,594 (1.2%) | 351 (1.4%) | -0.02 | 7,045 (3.1%) | 2,466 (5.7%) | -0.13 |
| 65 - 74; n (%) | 3,335 (14.7%) | 705 (24.0%) | -0.24 | 11,624 (17.1%) | 3,645 (24.4%) | -0.18 | 26,002 (19.1%) | 7,382 (29.3%) | -0.24 | 40,961 (18.1%) | 11,732 (27.2%) | -0.22 |
| >= 75; n (%) | 18,629 (82.2%) | 1,979 (67.4%) | 0.35 | 49,969 (73.7%) | 8,781 (58.8%) | 0.32 | 107,905 (79.3%) | 17,374 (68.9%) | 0.24 | 176,503 (77.9%) | 28,134 (65.3%) | 0.28 |
| Gender without zero category- United | /(/ | _, | | , | 2,122 (2012). | | | | | | | |
| Males; n (%) | 12,791 (56.4%) | 1,776 (60.5%) | -0.08 | 36,708 (54.1%) | 8,819 (59.1%) | -0.10 | 72,765 (53.5%) | 14,393 (57.0%) | -0.07 | 122,264 (54.0%) | 24,988 (58.0%) | -0.08 |
| Females; n (%) | 9,874 (43.6%) | 1,160 (39.5%) | 0.08 | 31,082 (45.9%) | 6,110 (40.9%) | 0.10 | 63,322 (46.5%) | 10,837 (43.0%) | 0.07 | 104,278 (46.0%) | 18,107 (42.0%) | 0.08 |
| Race | | | | | | | | | | | | |
| White; n (%) | | | | | | | 127,987 (94.0%) | 23,447 (92.9%) | | 127,987 (94.0%) | 23,447 (92.9%) | 0.00 |
| Black; n (%) | | | | | | | 3,795 (2.8%) | 714 (2.8%) | | 3,795 (2.8%) | 714 (2.8%) | 0.00 |
| Asian; n (%) | | | | | | | 1,217 (0.9%) | 344 (1.4%) | | 1,217 (0.9%) | 344 (1.4%) | 0.00 |
| Hispanic; n (%) | | | | | | | 1,169 (0.9%) | 245 (1.0%) | | 1,169 (0.9%) | 245 (1.0%) | 0.00 |
| North American Native; n (%) | | | | | | | 428 (0.3%) | 70 (0.3%) | | 428 (0.3%) | 70 (0.3%) | 0.00 |
| Other/Unknown; n (%) | | | | | | | 1,491 (1.1%) | 410 (1.6%) | | 1,491 (1.1%) | 410 (1.6%) | 0.00 |
| Region without zero category- United v3 (lumping | | | | | | | | | | | | |
| missing&other category with West) | | | _ | | | | | | | | | |
| Northeast; n (%) | 2,860 (12.6%) | 428 (14.6%) | -0.06 | 15,592 (23.0%) | 3,464 (23.2%) | 0.00 | 27,525 (20.2%) | 4,871 (19.3%) | 0.02 | 45,977 (20.3%) | 8,763 (20.3%) | 0.00 |
| South; n (%) | 5,965 (26.3%) | 1,026 (34.9%) | -0.19 | 21,981 (32.4%) | 3,920 (26.3%) | 0.13 | 44,598 (32.8%) | 10,023 (39.7%) | -0.14 | 72,544 (32.0%) | 14,969 (34.7%) | -0.06 |
| Midwest; n (%) | 4,585 (20.2%) | 473 (16.1%) | 0.11 | 18,724 (27.6%) | 5,249 (35.2%) | -0.16 | 38,803 (28.5%) | 5,759 (22.8%) | 0.13 | 62,112 (27.4%) | 11,481 (26.6%) | 0.02 |
| West; n (%) | 9,255 (40.8%) | 1,009 (34.4%) | 0.13 | 11,263 (16.6%) | 2,233 (15.0%) | 0.04 | 25,161 (18.5%) | 4,577 (18.1%) | 0.01 | 45,679 (20.2%) | 7,819 (18.1%) | 0.05 |
| Unknown+missing; n (%) | N/A | N/A | #VALUE! | 230 (0.3%) | 63 (0.4%) | -0.02 | N/A | N/A | #VALUE! | 230 (0.3%) | 63 (0.4%) | -0.02 |
| CV Covariates | | | | | | | | | | | | |
| Ischemic heart disease; n (%) | 5,796 (25.6%) | 854 (29.1%) | -0.08 | 22,356 (33.0%) | 5,213 (34.9%) | -0.04 | 37,673 (27.7%) | 8,145 (32.3%) | -0.10 | 65,825 (29.1%) | 14,212 (33.0%) | -0.08 |
| Acute MI; n (%) | 192 (0.8%) | 19 (0.6%) | 0.02 | 1,721 (2.5%) | 411 (2.8%) | -0.02 | 1,928 (1.4%) | 380 (1.5%) | -0.01 | 3841 (1.7%) | 810 (1.9%) | -0.02 |
| ACS/unstable angina; n (%) | 196 (0.9%) | 30 (1.0%) | -0.01 | 1,436 (2.1%) | 412 (2.8%) | -0.05 | 1,896 (1.4%) | 456 (1.8%) | -0.03 | 3528 (1.6%) | 898 (2.1%) | -0.04 |
| Old MI; n (%) | 654 (2.9%) | 72 (2.5%) | 0.02 | 2,040 (3.0%) | 506 (3.4%) | -0.02 | 4,824 (3.5%) | 1,089 (4.3%) | -0.04 | 7518 (3.3%) | 1667 (3.9%) | -0.03 |
| Stable angina; n (%) | 557 (2.5%) | 99 (3.4%) | -0.05 | 2,157 (3.2%) | 612 (4.1%) | -0.05 | 3,376 (2.5%) | 966 (3.8%) | -0.07 | 6,090 (2.7%) | 1,677 (3.9%) | -0.07 |
| Coronary atherosclerosis and other forms of chronic | | | | | | | | | | | | |
| ischemic heart disease; n (%) | 5,348 (23.6%) | 808 (27.5%) | -0.09 | 20,511 (30.3%) | 4,710 (31.5%) | -0.03 | 34,808 (25.6%) | 7,439 (29.5%) | -0.09 | 60,667 (26.8%) | 12,957 (30.1%) | -0.07 |
| Other atherosclerosis with ICD10 v2 Copy; n (%) | 291 (1.3%) | 50 (1.7%) | -0.03 | 1,283 (1.9%) | 237 (1.6%) | 0.02 | 1,625 (1.2%) | 346 (1.4%) | -0.02 | 3199 (1.4%) | 633 (1.5%) | -0.01 |
| Previous cardiac procedure (CABG or PTCA or Stent) | | | | | | | | | | | | |
| v4; n (%) | 19 (0.1%) | 7 (0.2%) | -0.03 | 712 (1.1%) | 161 (1.1%) | 0.00 | 893 (0.7%) | 154 (0.6%) | 0.01 | 1624 (0.7%) | 322 (0.7%) | 0.00 |
| History of CABG or PTCA; n (%) | 1,022 (4.5%) | 146 (5.0%) | -0.02 | 2,582 (3.8%) | 672 (4.5%) | -0.04 | 8,074 (5.9%) | 2,028 (8.0%) | -0.08 | 11,678 (5.2%) | 2,846 (6.6%) | -0.06 |
| Any stroke; n (%) | 1,585 (7.0%) | 271 (9.2%) | -0.08 | 5,866 (8.7%) | 1,426 (9.6%) | -0.03 | 8,312 (6.1%) | 1,840 (7.3%) | -0.05 | 15,763 (7.0%) | 3,537 (8.2%) | -0.05 |
| Ischemic stroke (w and w/o mention of cerebral | 4.570 (7.00) | 270 (0.201) | | 5.042 (0.50() | 4 424 (0 50) | | 0.050 (5.40) | 4 000 (7 00) | | 45 500 (5 00) | 2 522 (0 201) | |
| infarction); n (%) | 1,579 (7.0%) | 270 (9.2%) | -0.08 | 5,843 (8.6%) | 1,421 (9.5%) | -0.03 | 8,268 (6.1%) | 1,832 (7.3%) | -0.05 | 15,690 (6.9%) | 3,523 (8.2%) | -0.05 |
| Hemorrhagic stroke; n (%) | 12 (0.1%)<br>627 (2.8%) | 3 (0.1%)<br>151 (5.1%) | 0.00<br>-0.12 | 41 (0.1%)<br>2.260 (3.3%) | 8 (0.1%)<br>759 (5.1%) | 0.00<br>-0.09 | 56 (0.0%)<br>3.166 (2.3%) | 9 (0.0%)<br>811 (3.2%) | #DIV/0!<br>-0.06 | 109 (0.0%)<br>6053 (2.7%) | 20 (0.0%)<br>1721 (4.0%) | #DIV/0!<br>-0.07 |
| TIA; n (%) | 627 (2.8%)<br>386 (1.7%) | 151 (5.1%)<br>54 (1.8%) | -0.12<br>-0.01 | , , | 759 (5.1%)<br>315 (2.1%) | 0.09 | 2,122 (1.6%) | 811 (3.2%)<br>433 (1.7%) | -0.06 | 3925 (1.7%) | 1721 (4.0%)<br>802 (1.9%) | -0.07 |
| Other cerebrovascular disease; n (%) | , | | | 1,417 (2.1%) | | | , , , , , , | | | | , | |
| Late effects of cerebrovascular disease; n (%) | 110 (0.5%) | 10 (0.3%) | 0.03<br>#DIV/01 | 77 (0.1%) | 19 (0.1%)<br>25 (0.2%) | 0.00 | 511 (0.4%) | 69 (0.3%) | 0.02 | 698 (0.3%)<br>166 (0.1%) | 98 (0.2%) | 0.02 |
| Cerebrovascular procedure; n (%) | 2 (0.0%) | - () | | 73 (0.1%) | () | | 91 (0.1%) | 21 (0.1%) | | () | 46 (0.1%) | |
| Heart failure (CHF); n (%) | 3,108 (13.7%) | 335 (11.4%) | 0.07 | 15,297 (22.6%) | 3,232 (21.6%) | 0.02 | 17,205 (12.6%) | 2,846 (11.3%) | 0.04 | 35,610 (15.7%) | 6,413 (14.9%) | 0.02 |
| Peripheral Vascular Disease (PVD) or PVD Surgery v2;<br>n (%) | 1,790 (7.9%) | 210 (7.2%) | 0.03 | 5,549 (8.2%) | 974 (6.5%) | 0.07 | 8,046 (5.9%) | 1,363 (5.4%) | 0.02 | 15,385 (6.8%) | 2,547 (5.9%) | 0.04 |
| * * | 21,440 (94.6%) | 2,786 (94.9%) | -0.01 | 61,508 (90.7%) | 14,189 (95.0%) | -0.17 | 121,089 (89.0%) | 21,872 (86.7%) | 0.02 | 204,037 (90.1%) | 38,847 (90.1%) | 0.00 |
| Atrial fibrillation; n (%) | 10,235 (45.2%) | 2,786 (94.9%)<br>1.233 (42.0%) | -0.01 | 18.823 (27.8%) | 14,189 (95.0%)<br>4,688 (31.4%) | -0.17 | 121,089 (89.0%)<br>47,883 (35.2%) | 21,872 (86.7%)<br>8,912 (35.3%) | 0.07 | 76,941 (34.0%) | 38,847 (90.1%)<br>14.833 (34.4%) | -0.01 |
| Other cardiac dysrhythmia; n (%) Cardiac conduction disorders; n (%) | 10,235 (45.2%) | 1,233 (42.0%) | -0.04 | 18,823 (27.8%) | 4,688 (31.4%)<br>953 (6.4%) | -0.08 | 47,883 (35.2%)<br>6.776 (5.0%) | 8,912 (35.3%)<br>1.425 (5.6%) | -0.03 | 76,941 (34.0%)<br>11903 (5.3%) | 14,833 (34.4%)<br>2561 (5.9%) | -0.01 |
| Other CVD; n (%) | 2,744 (12.1%) | 358 (12.2%) | 0.04 | 18,692 (27.6%) | 4,297 (28.8%) | -0.03 | 14,045 (10.3%) | 2,647 (10.5%) | -0.03 | 35,481 (15.7%) | 7,302 (16.9%) | -0.03 |
| Diabetes-related complications | 2,744 (12.1%) | 330 (12.2%) | 0.00 | 10,052 (27.0%) | 4,257 (20.6%) | -0.03 | 14,043 (10.5%) | 2,047 (10.3%) | -0.01 | 33,461 (13.7%) | 7,302 (10.5%) | -0.03 |
| Diabetic retinopathy; n (%) | 311 (1.4%) | 41 (1.4%) | 0.00 | 852 (1.3%) | 196 (1.3%) | 0.00 | 1,343 (1.0%) | 229 (0.9%) | 0.01 | 2,506 (1.1%) | 466 (1.1%) | 0.00 |
| | 511 (1.4%) | 41 (1.4%) | 0.00 | 852 (1.3%) | 190 (1.3%) | 0.00 | 1,343 (1.0%) | 229 (0.9%) | 0.01 | 2,500 (1.1%) | 400 (1.1%) | 0.00 |
| Diabetes with other ophthalmic manifestations; n (%) | 24 (0.1%) | 2 (0.1%) | 0.00 | 710 (1.0%) | 130 (0.9%) | 0.01 | 866 (0.6%) | 162 (0.6%) | 0.00 | 1600 (0.7%) | 294 (0.7%) | 0.00 |
| Retinal detachment, vitreous hemorrhage, | 24 (0.170) | 2 (0.1/0) | 5.00 | /10(1.0%) | 130 (0.3%) | 0.01 | 000 (0.0%) | 102 (0.0/0) | 0.00 | 1000 (0.7%) | 234 (0.770) | 0.00 |
| vitrectomy; n (%) | 41 (0.2%) | 7 (0.2%) | 0.00 | 157 (0.2%) | 35 (0.2%) | 0.00 | 214 (0.2%) | 40 (0.2%) | 0.00 | 412 (0.2%) | 82 (0.2%) | 0.00 |
| Retinal laser coagulation therapy; n (%) | 23 (0.1%) | 2 (0.1%) | 0.00 | 127 (0.2%) | 34 (0.2%) | 0.00 | 199 (0.1%) | 35 (0.1%) | 0.00 | 349 (0.2%) | 71 (0.2%) | 0.00 |
| Occurrence of Diabetic Neuropathy v2 Copy; n (%) | 1,095 (4.8%) | 116 (4.0%) | 0.04 | 2,494 (3.7%) | 485 (3.2%) | 0.00 | 3,720 (2.7%) | 626 (2.5%) | 0.01 | 7309 (3.2%) | 1227 (2.8%) | 0.00 |
| Occurrence of diabetic nephropathy V3 with ICD10 | 2,033 (4.070) | -10 (0/0) | 0- | 2,-3- (3.770) | 303 (3.270) | 0.03 | -,, 20 (2.770) | 020 (2.3.0) | 0.01 | . 303 (3.270) | | 0.02 |
| Copy; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | #VALUE! | 000 (0.0%) | #VALUE! |
| Hypoglycemia v2; n (%) | 148 (0.7%) | 19 (0.6%) | 0.01 | 780 (1.2%) | 138 (0.9%) | 0.03 | 1,333 (1.0%) | 221 (0.9%) | 0.01 | 2261 (1.0%) | 378 (0.9%) | 0.01 |
| Hyperglycemia: n (%) | 775 (3.4%) | 114 (3.9%) | -0.03 | 1.082 (1.6%) | 303 (2.0%) | -0.03 | 5,641 (4.1%) | 1.169 (4.6%) | -0.02 | 7498 (3.3%) | 1586 (3.7%) | -0.02 |
| Disorders of fluid electrolyte and acid-base balance; n | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | -17 (3.370) | 2.03 | 1,002 (1.070) | 353 (2.5%) | 0.03 | -,0-1 (170) | 1,100 (4.0.0) | 0.02 | . 430 (3.370) | _300 (3.770) | 0.02 |
| (%) | 797 (3.5%) | 111 (3.8%) | -0.02 | 4,181 (6.2%) | 939 (6.3%) | 0.00 | 5,781 (4.2%) | 1,199 (4.8%) | -0.03 | 10759 (4.7%) | 2249 (5.2%) | -0.02 |
| Diabetic ketoacidosis; n (%) | 12 (0.1%) | 2 (0.1%) | 0.00 | 65 (0.1%) | 9 (0.1%) | 0.00 | 107 (0.1%) | 23 (0.1%) | 0.00 | 184 (0.1%) | 34 (0.1%) | 0.00 |
| Hyperosmolar hyperglycemic nonketotic syndrome | 12 (0.170) | 2 (0.270) | 2.00 | 05 (0.170) | 3 (0.170) | 0.00 | 10, (0.170) | 25 (5.2,0) | 0.00 | 20- (0.270) | 5-1(0.270) | 0.50 |
| (HONK); n (%) | 17 (0.1%) | 1 (0.0%) | 0.04 | 49 (0.1%) | 7 (0.0%) | 0.04 | 91 (0.1%) | 24 (0.1%) | 0.00 | 157 (0.1%) | 32 (0.1%) | 0.00 |
| Diabetes with peripheral circulatory disorders with | (/9) | - \/ | | (/0) | . (2.374) | | ( 170) | () | | (/0) | () | 2.50 |
| | 554 (2.4%) | 48 (1.6%) | 0.06 | 1,275 (1.9%) | 239 (1.6%) | 0.02 | 2,694 (2.0%) | 433 (1.7%) | 0.02 | 4523 (2.0%) | 720 (1.7%) | 0.02 |
| ICD-10 v2 Copy: n (%) | JJ- (E70) | | | | | | | | 0.04 | | | |
| ICD-10 v2 Copy; n (%) Diabetic Foot: n (%) | 413 (1.8%) | 39 (1.3%) | 0.04 | 1.743 (2.6%) | 268 (1.8%) | 0.05 | 3.207 (2.4%) | 457 (1.8%) | | 5363 (2.4%) | 764 (1.8%) | 0.04 |
| Diabetic Foot; n (%) | 413 (1.8%)<br>19 (0.1%) | 39 (1.3%)<br>1 (0.0%) | 0.04 | 1,743 (2.6%)<br>103 (0.2%) | 268 (1.8%)<br>16 (0.1%) | 0.05<br>0.03 | 3,207 (2.4%)<br>108 (0.1%) | 457 (1.8%)<br>12 (0.0%) | 0.04 | 5363 (2.4%)<br>230 (0.1%) | 764 (1.8%)<br>29 (0.1%) | 0.04 |
| | 413 (1.8%)<br>19 (0.1%)<br>55 (0.2%) | | | | | | | 457 (1.8%)<br>12 (0.0%)<br>39 (0.2%) | | | | |

| Skin infections v2; n (%) | 1.050 (4.6%) | 137 (4.7%) | 0.00 | 4,516 (6.7%) | 784 (5.3%) | 0.06 | 7,183 (5.3%) | 1,151 (4.6%) | 0.03 | 12749 (5.6%) | 2072 (4.8%) | 0.04 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Erectile dysfunction; n (%) | 343 (1.5%) | 69 (2.4%) | -0.07 | 726 (1.1%) | 237 (1.6%) | -0.04 | 904 (0.7%) | 232 (0.9%) | -0.02 | 1973 (0.9%) | 538 (1.2%) | -0.03 |
| Diabetes with unspecified complication; n (%) | 187 (0.8%) | 20 (0.7%) | 0.01 | 519 (0.8%) | 101 (0.7%) | 0.01 | 764 (0.6%) | 139 (0.6%) | 0.00 | 1470 (0.6%) | 260 (0.6%) | 0.00 |
| Diabetes mellitus without mention of complications; | | | | | | | | | | | | |
| n (%) | 5,754 (25.4%) | 833 (28.4%) | -0.07 | 16,310 (24.1%) | 3,721 (24.9%) | -0.02 | 34,888 (25.6%) | 6,813 (27.0%) | -0.03 | 56,952 (25.1%) | 11,367 (26.4%) | -0.03 |
| Hypertension: 1 inpatient or 2 outpatient claims within 365 days; n (%) | 16.322 (72.0%) | 2.239 (76.3%) | -0.10 | 42,997 (63.4%) | 9.870 (66.1%) | -0.06 | 108.842 (80.0%) | 21.120 (83.7%) | -0.10 | 168.161 (74.2%) | 33.229 (77.1%) | -0.07 |
| Hyperlipidemia v2; n (%) | 11.780 (52.0%) | 1.804 (61.4%) | -0.19 | 25.573 (37.7%) | 6.296 (42.2%) | -0.09 | 59.674 (43.8%) | 12,723 (50.4%) | -0.13 | 97.027 (42.8%) | 20.823 (48.3%) | -0.11 |
| Edema; n (%) | 1,814 (8.0%) | 243 (8.3%) | -0.01 | 5,614 (8.3%) | 1.040 (7.0%) | 0.05 | 8.853 (6.5%) | 1,425 (5.6%) | 0.04 | 16281 (7.2%) | 2708 (6.3%) | 0.04 |
| Renal Dysfunction (non-diabetic) v2; n (%) | 7 (0.0%) | 1 (0.0%) | #DIV/0! | 50 (0.1%) | 6 (0.0%) | 0.04 | 33 (0.0%) | ** | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Occurrence of acute renal disease v2; n (%) | 2 (0.0%) | 1 (0.0%) | #DIV/0! | 46 (0.1%) | 6 (0.0%) | 0.04 | 23 (0.0%) | ** | #VALUE! | 71 (0.0%) | #VALUE! | #VALUE! |
| Occurrence of chronic renal insufficiency; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | ** | 0 (0.0%) | #VALUE! | #VALUE! | 000 (0.0%) | #VALUE! |
| Chronic kidney disease v2; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | #VALUE! | 000 (0.0%) | #VALUE! |
| CKD Stage 3-4; n (%) Occurrence of hypertensive nephropathy; n (%) | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%) | #DIV/0!<br>#DIV/0! | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%)<br>0 (0.0%) | #DIV/0!<br>#DIV/0! | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%)<br>0 (0.0%) | #DIV/0!<br>#DIV/0! | #VALUE!<br>#VALUE! | 000 (0.0%)<br>000 (0.0%) | #VALUE!<br>#VALUE! |
| Occurrence of miscellaneous renal insufficiency v2; n | 0 (0.0%) | 0 (0.0%) | #DIV/0: | 0 (0.0%) | 0 (0.0%) | #DIV/0: | 0 (0.0%) | 0 (0.0%) | #DIV/0: | #VALUE: | 000 (0.0%) | #VALUE: |
| (%) | 1 (0.0%) | 0 (0.0%) | #DIV/0! | 4 (0.0%) | 0 (0.0%) | #DIV/0! | ** | 0 (0.0%) | #VALUE! | #VALUE! | 000 (0.0%) | #VALUE! |
| Glaucoma or cataracts v2; n (%) | 5,118 (22.6%) | 675 (23.0%) | -0.01 | 15,190 (22.4%) | 3,243 (21.7%) | 0.02 | 1,139 (0.8%) | 160 (0.6%) | 0.02 | 21,447 (9.5%) | 4,078 (9.5%) | 0.00 |
| Cellulitis or abscess of toe; n (%) | 191 (0.8%) | 17 (0.6%) | 0.02 | 500 (0.7%) | 93 (0.6%) | 0.01 | 2,821 (2.1%) | 399 (1.6%) | 0.04 | 3512 (1.6%) | 509 (1.2%) | 0.03 |
| Foot ulcer; n (%) | 422 (1.9%) | 40 (1.4%) | 0.04 | 1,801 (2.7%) | 271 (1.8%) | 0.06 | 128 (0.1%) | 27 (0.1%) | 0.00 | 2351 (1.0%) | 338 (0.8%) | 0.02 |
| Bladder stones; n (%) | 26 (0.1%) | 5 (0.2%) | -0.03<br>-0.03 | 78 (0.1%) | 28 (0.2%) | -0.03<br>-0.03 | 1,422 (1.0%) | 293 (1.2%) | -0.02<br>0.04 | 1526 (0.7%) | 326 (0.8%) | -0.01<br>0.02 |
| Kidney stones; n (%)<br>Urinary tract infections (UTIs); n (%) | 171 (0.8%)<br>1.630 (7.2%) | 33 (1.1%)<br>185 (6.3%) | 0.03 | 813 (1.2%)<br>5.324 (7.9%) | 228 (1.5%)<br>927 (6.2%) | 0.03 | 12,492 (9.2%)<br>40,989 (30.1%) | 2,078 (8.2%)<br>8.320 (33.0%) | -0.06 | 13476 (5.9%)<br>47.943 (21.2%) | 2339 (5.4%)<br>9.432 (21.9%) | -0.02 |
| Dipstick urinalysis: n (%) | 5,873 (25.9%) | 901 (30.7%) | -0.11 | 13,373 (19.7%) | 3,156 (21.1%) | -0.03 | 14,042 (10.3%) | 2,978 (11.8%) | -0.05 | 33,288 (14.7%) | 7,035 (16.3%) | -0.02 |
| Non-dipstick urinalysis; n (%) | 2,541 (11.2%) | 355 (12.1%) | -0.03 | 3,103 (4.6%) | 801 (5.4%) | -0.04 | 5,152 (3.8%) | 1,026 (4.1%) | -0.02 | 10,796 (4.8%) | 2,182 (5.1%) | -0.01 |
| Urine function test; n (%) | 687 (3.0%) | 102 (3.5%) | -0.03 | 2,778 (4.1%) | 638 (4.3%) | -0.01 | 2,169 (1.6%) | 447 (1.8%) | -0.02 | 5634 (2.5%) | 1187 (2.8%) | -0.02 |
| Cytology; n (%) | 250 (1.1%) | 38 (1.3%) | -0.02 | 1,664 (2.5%) | 358 (2.4%) | 0.01 | 2,833 (2.1%) | 519 (2.1%) | 0.00 | 4747 (2.1%) | 915 (2.1%) | 0.00 |
| Cystoscopy; n (%) | 380 (1.7%) | 48 (1.6%) | 0.01 | 1,732 (2.6%) | 378 (2.5%) | 0.01 | #REF! | #REF! | #REF! | #REF! | #REF! | #REF! |
| Other Covariates | 84 (0.4%) | 14 (0.5%) | -0.01 | 343 (0.5%) | 98 (0.7%) | -0.03 | 443 (0.3%) | 100 (0.4%) | -0.02 | 870 (0.4%) | 212 (0.5%) | -0.01 |
| Liver disease; n (%) Osteoarthritis; n (%) | 84 (0.4%)<br>3,538 (15.6%) | 14 (0.5%)<br>497 (16.9%) | -0.01<br>-0.04 | 343 (0.5%)<br>10,558 (15.6%) | 98 (0.7%)<br>2,139 (14.3%) | -0.03<br>0.04 | 443 (0.3%)<br>21,641 (15.9%) | 100 (0.4%)<br>3,936 (15.6%) | -0.02<br>0.01 | 870 (0.4%)<br>35737 (15.8%) | 212 (0.5%)<br>6572 (15.3%) | -0.01<br>0.01 |
| Other arthritis, arthropathies and musculoskeletal | 3,336 (13.0%) | 457 (10.5%) | -0.04 | 10,536 (15.0%) | 2,135 (14.3%) | 0.04 | 21,041 (13.5%) | 3,530 (13.0%) | 0.01 | 33/3/ (13.6%) | 0372 (13.3%) | 0.01 |
| pain; n (%) | 7,087 (31.3%) | 897 (30.6%) | 0.02 | 23,692 (34.9%) | 4,746 (31.8%) | 0.07 | 41,341 (30.4%) | 7,342 (29.1%) | 0.03 | 72120 (31.8%) | 12985 (30.1%) | 0.04 |
| Dorsopathies; n (%) | 3,877 (17.1%) | 535 (18.2%) | -0.03 | 12,398 (18.3%) | 2,723 (18.2%) | 0.00 | 22,378 (16.4%) | 4,307 (17.1%) | -0.02 | 38653 (17.1%) | 7565 (17.6%) | -0.01 |
| Fractures; n (%) | 627 (2.8%) | 65 (2.2%) | 0.04 | 3,305 (4.9%) | 496 (3.3%) | 0.08 | 5,148 (3.8%) | 760 (3.0%) | 0.04 | 9080 (4.0%) | 1321 (3.1%) | 0.05 |
| Falls v2; n (%) | 688 (3.0%) | 67 (2.3%) | 0.04 | 1,133 (1.7%) | 149 (1.0%) | 0.06 | 2,111 (1.6%) | 262 (1.0%) | 0.05 | 3932 (1.7%) | 478 (1.1%) | 0.05 |
| Osteoporosis; n (%) | 1,758 (7.8%) | 188 (6.4%) | 0.05<br>-0.01 | 5,295 (7.8%) | 1,008 (6.8%) | 0.04 | 10,526 (7.7%) | 1,911 (7.6%) | 0.00<br>-0.03 | 17579 (7.8%) | 3107 (7.2%) | 0.02<br>-0.02 |
| Hyperthyroidism; n (%)<br>Hypothyroidism v2; n (%) | 163 (0.7%)<br>3,397 (15.0%) | 23 (0.8%)<br>425 (14.5%) | 0.01 | 494 (0.7%)<br>7.128 (10.5%) | 104 (0.7%)<br>1.551 (10.4%) | 0.00 | 1,000 (0.7%)<br>15.444 (11.3%) | 248 (1.0%)<br>3.025 (12.0%) | -0.03 | 1657 (0.7%)<br>25969 (11.5%) | 375 (0.9%)<br>5001 (11.6%) | 0.02 |
| Other disorders of thyroid gland V2; n (%) | 505 (2.2%) | 74 (2.5%) | -0.02 | 1.546 (2.3%) | 387 (2.6%) | -0.02 | 2.907 (2.1%) | 676 (2.7%) | -0.04 | 4958 (2.2%) | 1137 (2.6%) | -0.03 |
| Depression; n (%) | 1,103 (4.9%) | 144 (4.9%) | 0.00 | 3,463 (5.1%) | 728 (4.9%) | 0.01 | 6,172 (4.5%) | 1,217 (4.8%) | -0.01 | 10738 (4.7%) | 2089 (4.8%) | 0.00 |
| Anxiety; n (%) | 973 (4.3%) | 154 (5.2%) | -0.04 | 2,440 (3.6%) | 592 (4.0%) | -0.02 | 5,217 (3.8%) | 1,082 (4.3%) | -0.03 | 8630 (3.8%) | 1828 (4.2%) | -0.02 |
| Sleep_Disorder; n (%) | 1,509 (6.7%) | 291 (9.9%) | -0.12 | 6,461 (9.5%) | 1,761 (11.8%) | -0.07 | 7,241 (5.3%) | 1,661 (6.6%) | -0.05 | 15211 (6.7%) | 3713 (8.6%) | -0.07 |
| Dementia; n (%) | 1,070 (4.7%) | 113 (3.8%) | 0.04 | 3,564 (5.3%) | 483 (3.2%) | 0.10 | 6,660 (4.9%) | 919 (3.6%) | 0.06 | 11294 (5.0%) | 1515 (3.5%) | 0.07 |
| Delirium; n (%) | 85 (0.4%)<br>119 (0.5%) | 16 (0.5%)<br>13 (0.4%) | -0.01<br>0.01 | 960 (1.4%)<br>772 (1.1%) | 124 (0.8%)<br>104 (0.7%) | 0.06<br>0.04 | 1,006 (0.7%)<br>944 (0.7%) | 154 (0.6%)<br>177 (0.7%) | 0.01 | 2051 (0.9%)<br>1835 (0.8%) | 294 (0.7%)<br>294 (0.7%) | 0.02<br>0.01 |
| Psychosis; n (%) Obesity; n (%) | 1,627 (7.2%) | 283 (9.6%) | -0.09 | 3,572 (5.3%) | 1,075 (7.2%) | -0.08 | 9,935 (7.3%) | 2,313 (9.2%) | -0.07 | 15134 (6.7%) | 3671 (8.5%) | -0.07 |
| Overweight; n (%) | 619 (2.7%) | 83 (2.8%) | -0.01 | 498 (0.7%) | 96 (0.6%) | 0.01 | 2.324 (1.7%) | 441 (1.7%) | 0.00 | 3441 (1.5%) | 620 (1.4%) | 0.01 |
| Smoking; n (%) | 1,391 (6.1%) | 228 (7.8%) | -0.07 | 2,660 (3.9%) | 831 (5.6%) | -0.08 | 14,879 (10.9%) | 3,432 (13.6%) | -0.08 | 18930 (8.4%) | 4491 (10.4%) | -0.07 |
| Alcohol abuse or dependence; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Drug abuse or dependence; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| COPD; n (%) | 2,521 (11.1%) | 302 (10.3%) | 0.03 | 9,289 (13.7%) | 1,896 (12.7%) | 0.03 | 12,605 (9.3%) | 2,316 (9.2%) | 0.00 | 24415 (10.8%) | 4514 (10.5%) | 0.01 |
| Asthma; n (%) | 928 (4.1%)<br>1,465 (6.5%) | 134 (4.6%)<br>273 (9.3%) | -0.02<br>-0.10 | 3,235 (4.8%) | 799 (5.4%)<br>1,465 (9.8%) | -0.03<br>-0.07 | 4,679 (3.4%)<br>5,922 (4.4%) | 1,016 (4.0%) | -0.03<br>-0.06 | 8842 (3.9%)<br>12589 (5.6%) | 1949 (4.5%)<br>3158 (7.3%) | -0.03<br>-0.07 |
| Obstructive sleep apnea; n (%) Pneumonia: n (%) | 479 (2.1%) | 2/3 (9.3%)<br>46 (1.6%) | 0.04 | 5,202 (7.7%)<br>4,419 (6.5%) | 880 (5.9%) | 0.07 | 4.846 (3.6%) | 1,420 (5.6%)<br>865 (3.4%) | 0.01 | 9744 (4.3%) | 1791 (4.2%) | 0.00 |
| Imaging; n (%) | 3 (0.0%) | 1 (0.0%) | #DIV/0! | 115 (0.2%) | 18 (0.1%) | 0.03 | 2,821 (2.1%) | 399 (1.6%) | 0.04 | 2939 (1.3%) | 418 (1.0%) | 0.03 |
| Other Medications | | | | | | | | | | | | |
| Use of ACE inhibitors; n (%) | 7,637 (33.7%) | 997 (34.0%) | -0.01 | 23,436 (34.6%) | 5,249 (35.2%) | -0.01 | 47,332 (34.8%) | 8,768 (34.8%) | 0.00 | 78405 (34.6%) | 15014 (34.8%) | 0.00 |
| Use of ARBs; n (%) | 4,045 (17.8%) | 571 (19.4%) | -0.04 | 14,719 (21.7%) | 3,547 (23.8%) | -0.05 | 26,443 (19.4%) | 5,734 (22.7%) | -0.08 | 45207 (20.0%) | 9852 (22.9%) | -0.07 |
| Use of Loop Diuretics - United; n (%) | 4,781 (21.1%) | 482 (16.4%)<br>91 (3.1%) | 0.12 | 21,128 (31.2%) | 3,432 (23.0%) | 0.19 | 34,289 (25.2%) | 4,812 (19.1%) | 0.15 | 60198 (26.6%) | 8726 (20.2%)<br>1681 (3.9%) | 0.15 |
| Use of other diuretics- United; n (%) Use of nitrates-United; n (%) | 859 (3.8%)<br>1,267 (5.6%) | 91 (3.1%)<br>146 (5.0%) | 0.04 | 4,266 (6.3%)<br>6,398 (9.4%) | 730 (4.9%)<br>1,249 (8.4%) | 0.06<br>0.04 | 6,138 (4.5%)<br>10,986 (8.1%) | 860 (3.4%)<br>1,964 (7.8%) | 0.06<br>0.01 | 11263 (5.0%)<br>18651 (8.2%) | 3359 (7.8%) | 0.05<br>0.01 |
| Use of other hypertension drugs; n (%) | 1,739 (7.7%) | 228 (7.8%) | 0.00 | 5,200 (7.7%) | 1,037 (6.9%) | 0.03 | 9,777 (7.2%) | 1,817 (7.2%) | 0.00 | 16716 (7.4%) | 3082 (7.2%) | 0.01 |
| Use of digoxin- United; n (%) | 3,142 (13.9%) | 318 (10.8%) | 0.09 | 13,308 (19.6%) | 2,168 (14.5%) | 0.14 | 20,843 (15.3%) | 2,997 (11.9%) | 0.10 | 37293 (16.5%) | 5483 (12.7%) | 0.11 |
| Use of Anti-arrhythmics; n (%) | 2,154 (9.5%) | 459 (15.6%) | -0.18 | 9,822 (14.5%) | 3,029 (20.3%) | -0.15 | 15,578 (11.4%) | 4,366 (17.3%) | -0.17 | 27554 (12.2%) | 7854 (18.2%) | -0.17 |
| Use of COPD/asthma meds- United; n (%) | 3,022 (13.3%) | 435 (14.8%) | -0.04 | 12,353 (18.2%) | 2,900 (19.4%) | -0.03 | 20,518 (15.1%) | 4,170 (16.5%) | -0.04 | 35893 (15.8%) | 7505 (17.4%) | -0.04 |
| Use of statins; n (%) | 12,189 (53.8%) | 1,579 (53.8%) | 0.00 | 37,940 (56.0%) | 8,310 (55.7%) | 0.01 | 74,659 (54.9%) | 14,235 (56.4%) | -0.03 | 124788 (55.1%) | 24124 (56.0%) | -0.02 |
| Use of other lipid-lowering drugs; n (%) | 1,345 (5.9%) | 221 (7.5%) | -0.06<br>-0.11 | 6,440 (9.5%)<br>8,223 (12.1%) | 1,567 (10.5%) | -0.03<br>-0.13 | 9,683 (7.1%) | 2,038 (8.1%) | -0.04<br>-0.14 | 17468 (7.7%) | 3826 (8.9%) | -0.04<br>-0.14 |
| Use of antiplatelet agents; n (%) Use of heparin and other low-molecular weight | 1,466 (6.5%) | 282 (9.6%) | -0.11 | 8,223 (12.1%) | 2,505 (16.8%) | -0.13 | 12,346 (9.1%) | 3,435 (13.6%) | -0.14 | 22035 (9.7%) | 6222 (14.4%) | -0.14 |
| heparins; n (%) | 501 (2.2%) | 11 (0.4%) | 0.16 | 29 (0.0%) | 2 (0.0%) | #DIV/0! | 5,084 (3.7%) | 125 (0.5%) | 0.22 | 5614 (2.5%) | 138 (0.3%) | 0.19 |
| Use of NSAIDs; n (%) | 1,606 (7.1%) | 290 (9.9%) | -0.10 | 5,269 (7.8%) | 1,572 (10.5%) | -0.09 | 11,395 (8.4%) | 3,015 (12.0%) | -0.12 | 18270 (8.1%) | 4877 (11.3%) | -0.11 |
| Use of oral corticosteroids; n (%) | 3,335 (14.7%) | 475 (16.2%) | -0.04 | 12,514 (18.5%) | 2,819 (18.9%) | -0.01 | 23,765 (17.5%) | 4,688 (18.6%) | -0.03 | 39614 (17.5%) | 7982 (18.5%) | -0.03 |
| Use of bisphosphonate (United); n (%) | 961 (4.2%) | 109 (3.7%) | 0.03 | 3,457 (5.1%) | 681 (4.6%) | 0.02 | 5,374 (3.9%) | 1,024 (4.1%) | -0.01 | 9792 (4.3%) | 1814 (4.2%) | 0.00 |
| Use of opioids- United; n (%) | 4,335 (19.1%) | 569 (19.4%) | -0.01 | 16,765 (24.7%) | 3,550 (23.8%) | 0.02 | 30,560 (22.5%) | 5,619 (22.3%) | 0.00 | 51660 (22.8%) | 9738 (22.6%) | 0.00 |
| Use of antidepressants; n (%) Use of antipsychotics: n (%) | 3,538 (15.6%)<br>225 (1.0%) | 473 (16.1%)<br>25 (0.9%) | -0.01<br>0.01 | 12,223 (18.0%)<br>1,128 (1.7%) | 2,578 (17.3%)<br>168 (1.1%) | 0.02<br>0.05 | 24,350 (17.9%)<br>2.318 (1.7%) | 4,457 (17.7%)<br>392 (1.6%) | 0.01<br>0.01 | 40111 (17.7%)<br>3671 (1.6%) | 7508 (17.4%)<br>585 (1.4%) | 0.01<br>0.02 |
| Use of antipsychotics; n (%) Use of anticonvulsants: n (%) | 2.045 (9.0%) | 25 (0.9%) | 0.01 | 1,128 (1.7%) 6.508 (9.6%) | 1.262 (8.5%) | 0.05 | 2,318 (1.7%)<br>13.821 (10.2%) | 2.344 (9.3%) | 0.01 | 36/1 (1.6%)<br>22374 (9.9%) | 3854 (8.9%) | 0.02 |
| Use of lithium- United; n (%) | 16 (0.1%) | 3 (0.1%) | 0.00 | 46 (0.1%) | 14 (0.1%) | 0.00 | 57 (0.0%) | 23 (0.1%) | -0.04 | 119 (0.1%) | 40 (0.1%) | 0.00 |
| Use of Benzos- United; n (%) | 1,463 (6.5%) | 205 (7.0%) | -0.02 | 8,662 (12.8%) | 1,940 (13.0%) | -0.01 | 10,944 (8.0%) | 1,679 (6.7%) | 0.05 | 21069 (9.3%) | 3824 (8.9%) | 0.01 |

| Use of anxiolytics/hypnotics- United; n (%) | 937 (4.1%) | 184 (6.3%) | -0.10 | 4,377 (6.5%) | 1,073 (7.2%) | -0.03 | 7,226 (5.3%) | 1,699 (6.7%) | -0.06 | 12540 (5.5%) | 2956 (6.9%) | -0.06 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Use of dementia meds- United; n (%) | 840 (3.7%) | 98 (3.3%) | 0.02 | 3,200 (4.7%) | 474 (3.2%) | 0.08 | 6,279 (4.6%) | 927 (3.7%) | 0.05 | 10319 (4.6%) | 1499 (3.5%) | 0.06 |
| Use of antiparkinsonian meds- United; n (%) | 492 (2.2%) | 43 (1.5%) | 0.05 | 1,880 (2.8%) | 371 (2.5%) | 0.02 | 3,833 (2.8%) | 682 (2.7%) | 0.01 | 6205 (2.7%) | 1096 (2.5%) | 0.01 |
| Any use of pramlintide; n (%) | 2 (0.0%) | 0 (0.0%) | #DIV/0! | 19 (0.0%) | 8 (0.1%) | -0.04 | 11 (0.0%) | ** | #VALUE! | 32 (0.0%) | #VALUE! | #VALUE! |
| Any use of 1st generation sulfonylureas; n (%) | 1 (0.0%) | 0 (0.0%) | #DIV/0! | 19 (0.0%) | 5 (0.0%) | #DIV/0! | ** | ** | #VALUE! | #VALUE! | #VALUE! | 0.00 |
| Entresto (sacubitril/valsartan); n (%) | 21 (0.1%) | 3 (0.1%) | 0.00 | 18 (0.0%) | 2 (0.0%) | #DIV/0! | 30 (0.0%) | ** | #VALUE! | 69 (0.0%) | #VALUE! | 0.00 |
| Labs | 21 (0.170) | 3 (0.1%) | 0.00 | 10 (0.0%) | 2 (0.070) | | 50 (0.0%) | | WWW.COL. | 90.455 | 17,865 | 0.00 |
| Lab values- HbA1c (%) v3: n (%) | 2.340 (10.3%) | 328 (11.2%) | -0.03 | 682 (1.0%) | 109 (0.7%) | 0.03 | N/A | N/A | #VALUE! | 3,022 (3,3%) | 437 (2.4%) | 0.05 |
| Lab values- HbA1c (%) (within 3 months) v3; n (%) | 1,502 (6.6%) | 212 (7.2%) | -0.03 | 480 (0.7%) | 69 (0.5%) | 0.03 | N/A | N/A | #VALUE! | 1.982 (2.2%) | 281 (1.6%) | 0.03 |
| | | | | | , | | , | , | | , | | |
| Lab values- HbA1c (%) (within 6 months) v3; n (%) | 2,340 (10.3%) | 328 (11.2%) | -0.03 | 682 (1.0%) | 109 (0.7%) | 0.03 | N/A | N/A | #VALUE! | 3,022 (3.3%) | 437 (2.4%) | 0.05 |
| Lab values- BNP; n (%) | 227 (1.0%) | 28 (1.0%) | 0.00 | 45 (0.1%) | 17 (0.1%) | 0.00 | N/A | N/A | #VALUE! | 272 (0.3%) | 045 (0.3%) | 0.00 |
| Lab values- BNP (within 3 months); n (%) | 165 (0.7%) | 24 (0.8%) | -0.01 | 36 (0.1%) | 14 (0.1%) | 0.00 | N/A | N/A | #VALUE! | 201 (0.2%) | 038 (0.2%) | 0.00 |
| Lab values- BNP (within 6 months); n (%) | 227 (1.0%) | 28 (1.0%) | 0.00 | 45 (0.1%) | 17 (0.1%) | 0.00 | N/A | N/A | #VALUE! | 272 (0.3%) | 045 (0.3%) | 0.00 |
| Lab values- BUN (mg/dl); n (%) | 4,553 (20.1%) | 704 (24.0%) | -0.09 | 559 (0.8%) | 166 (1.1%) | -0.03 | N/A | N/A | #VALUE! | 5,112 (5.7%) | 870 (4.9%) | 0.04 |
| Lab values- BUN (mg/dl) (within 3 months); n (%) | 3,091 (13.6%) | 479 (16.3%) | -0.08 | 387 (0.6%) | 117 (0.8%) | -0.02 | N/A | N/A | #VALUE! | 3,478 (3.8%) | 596 (3.3%) | 0.03 |
| Lab values- BUN (mg/dl) (within 6 months); n (%) | 4,553 (20.1%) | 704 (24.0%) | -0.09 | 559 (0.8%) | 166 (1.1%) | -0.03 | N/A | N/A | #VALUE! | 5,112 (5.7%) | 870 (4.9%) | 0.04 |
| Lab values- Creatinine (mg/dl) v2; n (%) | 4,643 (20.5%) | 718 (24.5%) | -0.10 | 577 (0.9%) | 182 (1.2%) | -0.03 | N/A | N/A | #VALUE! | 5,220 (5.8%) | 900 (5.0%) | 0.04 |
| Lab values- Creatinine (mg/dl) (within 3 months) v2; | | | | , | | | • | , | | -, -, -, | | |
| n (%) | 3,146 (13.9%) | 489 (16.7%) | -0.08 | 402 (0.6%) | 125 (0.8%) | -0.02 | N/A | N/A | #VALUE! | 3,548 (3.9%) | 614 (3.4%) | 0.03 |
| Lab values- Creatinine (mg/dl) (within 6 months) v2; | | (2011) | | 102 (01011) | | | | | | 2,2 12 (2121-) | () | |
| n (%) | 4.643 (20.5%) | 718 (24.5%) | -0.10 | 577 (0.9%) | 182 (1.2%) | -0.03 | N/A | N/A | #VALUE! | 5,220 (5.8%) | 900 (5.0%) | 0.04 |
| Lab values- HDL level (mg/dl); n (%) | 3,264 (14.4%) | 532 (18.1%) | -0.10 | 539 (0.8%) | 125 (0.8%) | 0.00 | N/A | N/A | #VALUE! | 3,803 (4.2%) | 657 (3.7%) | 0.03 |
| Lab values- HDE level (Ilig/ul), Il (76) | 3,204 (14.4%) | 352 (18.1%) | -0.10 | 339 (0.8%) | 123 (0.8%) | 0.00 | N/A | IN/A | #VALUE: | 3,003 (4.270) | 037 (3.7%) | 0.03 |
| 1 - h d 11D1 d ( /d ) ( i + h i - 2 + h - ) (0) | 2 0 44 (0 00%) | 240 (11 69) | -0.09 | 367 (0.5%) | 77 (0.5%) | 0.00 | N/A | N/A | 40/01/151 | 2 400 (2 70/) | 447 (2.20() | 0.03 |
| Lab values- HDL level (mg/dl) (within 3 months); n (% | 5) 2,041 (9.0%) | 340 (11.6%) | -0.09 | 367 (0.5%) | //(0.5%) | 0.00 | N/A | N/A | #VALUE! | 2,408 (2.7%) | 417 (2.3%) | 0.03 |
| Laboration (ID) Invalent (ID) (ID) (ID) (ID) | 3.264 (14.4%) | E22 (40 40'' | -0.10 | E20 to 00** | 125 (0.8%) | 0.00 | N/A | N/A | #VALUE! | 2 002 (4 20) | CER (0. 20/) | 0.03 |
| Lab values- HDL level (mg/dl) (within 6 months); n (% | | 532 (18.1%) | | 539 (0.8%) | () | | | , | | 3,803 (4.2%) | 657 (3.7%) | |
| Lab values- LDL level (mg/dl) v2; n (%) | 3,488 (15.4%) | 561 (19.1%) | -0.10 | 689 (1.0%) | 134 (0.9%) | 0.01 | N/A | N/A | #VALUE! | 4,177 (4.6%) | 695 (3.9%) | 0.03 |
| Lab values- LDL level (mg/dl) (within 3 months) v2; n | | | | | | | | | | | | |
| (%) | 2,174 (9.6%) | 359 (12.2%) | -0.08 | 460 (0.7%) | 83 (0.6%) | 0.01 | N/A | N/A | #VALUE! | 2,634 (2.9%) | 442 (2.5%) | 0.02 |
| Lab values- LDL level (mg/dl) (within 6 months) v2; n | | | | | | | | | | | | |
| (%) | 3,488 (15.4%) | 561 (19.1%) | -0.10 | 689 (1.0%) | 134 (0.9%) | 0.01 | N/A | N/A | #VALUE! | 4,177 (4.6%) | 695 (3.9%) | 0.03 |
| Lab values- NT-proBNP; n (%) | 20 (0.1%) | 2 (0.1%) | 0.00 | 3 (0.0%) | 0 (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | 23 (0.0%) | 2 (0.0%) | #DIV/0! |
| Lab values- NT-proBNP (within 3 months); n (%) | 16 (0.1%) | 1 (0.0%) | 0.04 | 2 (0.0%) | 0 (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | 18 (0.0%) | 1 (0.0%) | - |
| Lab values- NT-proBNP (within 6 months); n (%) | 20 (0.1%) | 2 (0.1%) | 0.00 | 3 (0.0%) | 0 (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | 23 (0.0%) | 2 (0.0%) | - |
| Lab values-Total cholesterol (mg/dl) v2; n (%) | 3,311 (14.6%) | 542 (18.5%) | -0.11 | 560 (0.8%) | 136 (0.9%) | -0.01 | N/A | N/A | #VALUE! | 3,871 (4.3%) | 678 (3.8%) | 0.03 |
| Lab values-Total cholesterol (mg/dl) (within 3 | 5,511 (14.570) | 342 (20.3%) | 0.11 | 300 (0.0%) | 150 (0.570) | 0.01 | .,,,, | 14/1 | WWW.COL. | 3,072 (4.370) | 070 (3.070) | 0.03 |
| months) v2: n (%) | 2.069 (9.1%) | 346 (11.8%) | -0.09 | 377 (0.6%) | 82 (0.5%) | 0.01 | N/A | N/A | #VALUE! | 2.446 (2.7%) | 428 (2.4%) | 0.02 |
| | 2,005 (5.170) | 340 (11.070) | -0.03 | 377 (0.0%) | 82 (0.5%) | 0.01 | 14/0 | 11/15 | #VALUE: | 2,440 (2.770) | 420 (2.470) | 0.02 |
| Lab values-Total cholesterol (mg/dl) (within 6<br>months) v2: n (%) | 3.311 (14.6%) | 542 (18.5%) | -0.11 | 560 (0.8%) | 136 (0.9%) | -0.01 | N/A | N/A | #VALUE! | 3.871 (4.3%) | 678 (3.8%) | 0.03 |
| | -,- ( , | | -0.11 | | | 0.00 | N/A | N/A | #VALUE! | -,- , , | | 0.03 |
| Lab values- Triglyceride level (mg/dl); n (%) | 3,262 (14.4%) | 537 (18.3%) | -0.11 | 535 (0.8%) | 126 (0.8%) | 0.00 | N/A | N/A | #VALUE! | 3,797 (4.2%) | 663 (3.7%) | 0.03 |
| Lab values- Triglyceride level (mg/dl) (within 3 | | | | | | | | | | | | |
| months); n (%) | 2,035 (9.0%) | 343 (11.7%) | -0.09 | 358 (0.5%) | 77 (0.5%) | 0.00 | N/A | N/A | #VALUE! | 2,393 (2.6%) | 420 (2.4%) | 0.01 |
| Lab values-Triglyceride level (mg/dl) (within 6 | | | | | | | | | | | | |
| months); n (%) | 3,262 (14.4%) | 537 (18.3%) | -0.11 | 535 (0.8%) | 126 (0.8%) | 0.00 | N/A | N/A | #VALUE! | 3,797 (4.2%) | 663 (3.7%) | 0.03 |
| Lab result number- HbA1c (%) mean (only 2 to 20 | | | | | | | | | | | | |
| included) v4 | 2,323 | 326 | | 534 | 101 | | N/A | N/A | | 2,857 | 427 | |
| mean (sd) | 6.47 (1.11) | 6.53 (1.34) | -0.05 | 6.97 (1.28) | 6.79 (1.17) | 0.15 | N/A | N/A | #VALUE! | 6.56 (1.14) | 6.59 (1.30) | -0.02 |
| median [IQR] | 6.25 [5.80, 6.90] | 6.30 [5.80, 6.91] | -0.04 | 6.60 [6.15, 7.50] | 6.50 [5.95, 7.35] | 0.08 | N/A | N/A | #VALUE! | 6.32 (1.14) | 6.35 (1.30) | -0.02 |
| Missing; n (%) | 20,342 (89.8%) | 2,610 (88.9%) | 0.03 | 67,256 (99.2%) | 14,828 (99.3%) | -0.01 | N/A | N/A | #VALUE! | 87,598 (96.8%) | 17,438 (97.6%) | -0.05 |
| Lab result number- BNP mean v2 | 227 | 28 | | 45 | 17 | | N/A | N/A | | 272 | 45 | |
| mean (sd) | 261.46 (277.83) | 214.33 (164.51) | 0.21 | 247.18 (218.19) | 180.30 (209.53) | 0.31 | N/A | N/A | #VALUE! | 259.10 (269.51) | 201.47 (184.72) | 0.25 |
| median [IQR] | 198.60 [99.39, 339.40] | 170.15 [69.72, 343.75] | 0.12 | 174.00 [78.80, 330.50] | 121.00 [59.00, 245.00] | 0.25 | N/A | N/A | #VALUE! | 194.53 (269.51) | 151.58 (184.72) | 0.19 |
| Missing; n (%) | 22.438 (99.0%) | 2.908 (99.0%) | 0.00 | 67,745 (99.9%) | 14.912 (99.9%) | 0.00 | N/A | N/A | #VALUE! | 90.183 (99.7%) | 17,820 (99.7%) | 0.00 |
| Lab result number- BUN (mg/dl) mean v2 | 4,553 | 704 | 0.00 | 57,743 (33.370) | 166 | 0.00 | N/A | N/A | WYNEGE. | 5,112 | 870 | 0.00 |
| | 18.85 (6.58) | 17.70 (5.20) | 0.19 | 19.96 (8.62) | 18.29 (6.07) | 0.22 | N/A<br>N/A | N/A<br>N/A | #VALUE! | 18.97 (6.83) | 17.81 (5.38) | 0.19 |
| mean (sd)<br>median [IQR] | 18.85 (6.58)<br>18.00 [15.00, 22.00] | | 0.19 | 19.96 (8.62) | 18.29 (6.07) | 0.22 | N/A<br>N/A | N/A<br>N/A | #VALUE! | 18.97 (6.83) | 17.81 (5.38) | 0.19 |
| Missing; n (%) | 18,112 (79.9%) | 2,232 (76.0%) | 0.09 | 67,231 (99.2%) | 14,763 (98.9%) | 0.03 | N/A | N/A | #VALUE! | 85,343 (94.3%) | 16,995 (95.1%) | -0.04 |
| Lab result number- Creatinine (mg/dl) mean (only 0.: | | | | | | | 21/2 | | | | | |
| to 15 included) v3 | 4,611 | 714 | | 571 | 178 | | N/A | N/A | | 5,182 | 892 | |
| mean (sd) | 1.01 (0.25) | 0.98 (0.21) | 0.13 | 1.05 (0.30) | 0.98 (0.24) | 0.26 | N/A | N/A | #VALUE! | 1.01 (0.26) | 0.98 (0.22) | 0.12 |
| median [IQR] | 0.98 [0.84, 1.14] | 0.96 [0.83, 1.10] | 0.09 | 1.00 [0.85, 1.18] | 0.96 [0.80, 1.13] | 0.15 | N/A | N/A | #VALUE! | 0.98 (0.26) | 0.96 (0.22) | 0.08 |
| Missing; n (%) | 18,054 (79.7%) | 2,222 (75.7%) | 0.10 | 67,219 (99.2%) | 14,751 (98.8%) | 0.04 | N/A | N/A | #VALUE! | 85,273 (94.3%) | 16,973 (95.0%) | -0.03 |
| Lab result number- HDL level (mg/dl) mean (only | | | | | | | | | | | | |
| =<5000 included) v2 | 3,264 | 532 | | 539 | 125 | | N/A | N/A | | 3,803 | 657 | |
| mean (sd) | 51.06 (16.33) | 52.25 (17.04) | -0.07 | 45.82 (14.49) | 48.92 (17.38) | -0.19 | N/A | N/A | #VALUE! | 50.32 (16.08) | 51.62 (17.12) | -0.08 |
| median [IQR] | 48.00 [40.00, 60.00] | 49.00 [41.00, 61.00] | -0.06 | 44.00 [37.00, 53.00] | 48.00 [36.75, 60.00] | -0.25 | N/A | N/A | #VALUE! | 47.43 (16.08) | 48.81 (17.12) | -0.08 |
| Missing; n (%) | 19,401 (85.6%) | 2,404 (81.9%) | 0.10 | 67,251 (99.2%) | 14,804 (99.2%) | 0.00 | N/A | N/A | #VALUE! | 86,652 (95.8%) | 17,208 (96.3%) | -0.03 |
| Lab result number- LDL level (mg/dl) mean (only | | | | | | | | | | | | |
| =<5000 included) v2 | 3,405 | 545 | | 552 | 128 | | N/A | N/A | | 3,957 | 673 | |
| mean (sd) | 86.00 (31.67) | 87.70 (33.74) | -0.05 | 84.18 (33.47) | 82.01 (35.36) | 0.06 | N/A | N/A | #VALUE! | 85.75 (31.93) | 86.62 (34.08) | -0.03 |
| median [IQR] | 82.00 [65.00, 104.00] | 82.00 [66.00, 109.00] | 0.00 | 81.00 [62.25, 101.00] | 81.00 [59.00, 102.75] | 0.00 | N/A | N/A | #VALUE! | 81.86 (31.93) | 81.81 (34.08) | 0.00 |
| Missing; n (%) | 19,260 (85.0%) | 2,391 (81.4%) | 0.10 | 67,238 (99.2%) | 14,801 (99.1%) | 0.01 | N/A | N/A | #VALUE! | 86,498 (95.6%) | 17,192 (96.2%) | -0.03 |
| Lab result number-Total cholesterol (mg/dl) mean | 15,200 (05.070) | 2,332 (02.470) | 0.20 | 0.,230 (33.270) | 1-7,001 (33.170) | 0.01 | | /^ | | 00,430 (33.070) | 1,152 (50.270) | 0.03 |
| (only =<5000 included) v2 | 3.310 | 542 | | 560 | 136 | | N/A | N/A | | 3.870 | 678 | |
| mean (sd) | 163.13 (39.87) | 165.20 (40.26) | -0.05 | 157.07 (40.57) | 160.25 (40.19) | -0.08 | N/A | N/A | #VALUE! | 162.25 (39.98) | 164.21 (40.28) | -0.05 |
| | 159.00 [137.00, 186.00] | | -0.05 | 157.07 (40.57) | 160.50 [137.25, 183.38] | -0.08 | N/A<br>N/A | N/A<br>N/A | #VALUE! | 152.25 (39.98) | 159.70 (40.28) | -0.03 |
| median [IQR] | | | | | | | , | , | | | | |
| Missing; n (%) | 19,355 (85.4%) | 2,394 (81.5%) | 0.11 | 67,230 (99.2%) | 14,793 (99.1%) | 0.01 | N/A | N/A | #VALUE! | 86,585 (95.7%) | 17,187 (96.2%) | -0.03 |
| Lab result number-Triglyceride level (mg/dl) mean | | | | | | | 21/2 | | | | | |
| (only =<5000 included) v2 | 3,262 | 537 | | 535 | 126 | | N/A | N/A | | 3,797 | 663 | |
| mean (sd) | 129.05 (78.48) | 121.50 (66.86) | 0.10 | 139.12 (74.65) | 141.59 (94.40) | -0.03 | N/A | N/A | #VALUE! | 130.47 (77.96) | 125.32 (72.93) | 0.07 |
| median [IQR] | 111.00 [82.00, 156.00] | 107.00 [77.50, 145.00] | 0.05 | 122.00 [88.00, 175.00] | 125.50 [89.38, 157.38] | -0.04 | N/A | N/A | #VALUE! | 112.55 (77.96) | 110.52 (72.93) | 0.03 |

| Missing; n (%) | 19,403 (85.6%) | 2,399 (81.7%) | 0.11 | 67,255 (99.2%) | 14,803 (99.2%) | 0.00 | N/A | N/A | #VALUE! | 86,658 (95.8%) | 17,202 (96.3%) | -0.03 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Lab result number- Hemoglobin mean (only >0 | | | | | | | | | | | | |
| included) | 3,295 | 521 | | 359 | 114 | | N/A | N/A | | 3,654 | 635 | |
| mean (sd) | 13.87 (1.59) | 14.08 (1.40) | -0.14 | 13.42 (1.59) | 13.63 (2.34) | -0.10 | N/A | N/A | #VALUE! | 13.83 (1.59) | 14.00 (1.61) | -0.11 |
| median [IQR] | 13.90 [12.90, 14.90] | 14.00 [13.20, 15.00] | -0.07 | 13.50 [12.40, 14.40] | 13.95 [12.94, 15.00] | -0.22 | N/A | N/A | #VALUE! | 13.86 (1.59) | 13.99 (1.61) | -0.08 |
| Missing; n (%) | 19,370 (85.5%) | 2,415 (82.3%) | 0.09 | 67,431 (99.5%) | 14,815 (99.2%) | 0.04 | N/A | N/A | #VALUE! | 86,801 (96.0%) | 17,230 (96.4%) | -0.02 |
| Lab result number- Serum sodium mean (only > 90 | | | | | | | | | | | | |
| and < 190 included) | 4,380 | 685 | | 456 | 142 | | N/A | N/A | | 4,836 | 827 | |
| mean (sd) | 140.12 (2.88) | 140.14 (3.00) | -0.01 | 139.70 (2.75) | 139.32 (2.94) | 0.13 | N/A | N/A | #VALUE! | 140.08 (2.87) | 140.00 (2.99) | 0.03 |
| median [IQR] | 140.00 [139.00, 142.00] | | 0.00 | 140.00 [138.00, 141.00] | 139.33 [138.00, 141.00] | 0.24 | N/A | N/A | #VALUE! | 140.00 (2.87) | 139.88 (2.99) | 0.04 |
| Missing; n (%) | 18,285 (80.7%) | 2,251 (76.7%) | 0.10 | 67,334 (99.3%) | 14,787 (99.0%) | 0.03 | N/A | N/A | #VALUE! | 85,619 (94.7%) | 17,038 (95.4%) | -0.03 |
| Lab result number- Albumin mean (only >0 and <=10 | | | | | | | | | | | | |
| included) | 3,911 | 632 | | 366 | 120 | | N/A | N/A | | 4,277 | 752 | |
| mean (sd) | 4.14 (0.32) | 4.19 (0.31) | -0.16 | 4.05 (0.49) | 4.06 (0.47) | -0.02 | N/A | N/A | #VALUE! | 4.13 (0.34) | 4.17 (0.34) | -0.12 |
| median [IQR] | 4.15 [3.95, 4.35] | 4.20 [4.00, 4.40] | -0.16 | 4.10 [3.85, 4.30] | 4.10 [3.90, 4.30] | 0.00 | N/A | N/A | #VALUE! | 4.15 (0.34) | 4.18 (0.34) | -0.09 |
| Missing; n (%) | 18,754 (82.7%) | 2,304 (78.5%) | 0.11 | 67,424 (99.5%) | 14,809 (99.2%) | 0.04 | N/A | N/A | #VALUE! | 86,178 (95.3%) | 17,113 (95.8%) | -0.02 |
| Lab result number- Glucose (fasting or random) mean | | | | | | | | | | | | |
| (only 10-1000 included) | 4,320 | 676 | | 439 | 130 | | N/A | N/A | | 4,759 | 806 | |
| mean (sd) | 109.88 (33.22) | 111.68 (39.94) | -0.05 | 130.34 (49.02) | 127.55 (43.03) | 0.06 | N/A | N/A | #VALUE! | 111.77 (34.98) | 114.24 (40.48) | -0.07 |
| median [IQR] | 101.00 [91.00, 118.00] | 100.17 [91.00, 116.88] | 0.02 | 116.50 [98.00, 148.00] | 114.50 [101.81, 138.31] | 0.04 | N/A | N/A | #VALUE! | 102.43 (34.98) | 102.48 (40.48) | 0.00 |
| Missing; n (%) | 18,345 (80.9%) | 2,260 (77.0%) | 0.10 | 67,351 (99.4%) | 14,799 (99.1%) | 0.03 | N/A | N/A | #VALUE! | 85,696 (94.7%) | 17,059 (95.5%) | -0.04 |
| Lab result number- Potassium mean (only 1-7 | | | | | | | | | | | | |
| included) | 4,610 | 711 | | 552 | 164 | | N/A | N/A | | 5,162 | 875 | |
| mean (sd) | 4.35 (0.44) | 4.38 (0.44) | -0.07 | 4.33 (0.43) | 4.37 (0.38) | -0.10 | N/A | N/A | #VALUE! | 4.35 (0.44) | 4.38 (0.43) | -0.07 |
| median [IQR] | 4.30 [4.10, 4.60] | 4.40 [4.10, 4.60] | -0.23 | 4.30 [4.10, 4.60] | 4.40 [4.15, 4.60] | -0.25 | N/A | N/A | #VALUE! | 4.30 (0.44) | 4.40 (0.43) | -0.23 |
| Missing; n (%) | 18,055 (79.7%) | 2,225 (75.8%) | 0.09 | 67,238 (99.2%) | 14,765 (98.9%) | 0.03 | N/A | N/A | #VALUE! | 85,293 (94.3%) | 16,990 (95.1%) | -0.04 |
| Comorbidity Scores | | | | | | | | | | | | |
| CCI (180 days)- ICD9 and ICD10 v2 | | | | | | | | | | | | |
| mean (sd) | 2.62 (1.44) | 2.62 (1.34) | 0.00 | 2.78 (1.68) | 2.79 (1.56) | -0.01 | 1.42 (1.41) | 1.32 (1.38) | 0.07 | 1.95 (1.50) | 1.92 (1.44) | 0.02 |
| median [IQR] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 0.00 | 2.00 [2.00, 4.00] | 2.00 [2.00, 4.00] | 0.00 | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.00 | 1.40 (1.50) | 1.41 (1.44) | -0.01 |
| Non-Frailty; n (%) | 12,577 (55.5%) | 1,612 (54.9%) | 0.01 | 33,237 (49.0%) | 7,284 (48.8%) | 0.00 | 3,400 (2.5%) | 524 (2.1%) | 0.03 | 49,214 (21.7%) | 9,420 (21.9%) | 0.00 |
| Frailty Score (mean): Empirical Version 365 days, v2 | | | | | | | | | | | _ | |
| mean (sd) | 0.17 (0.04) | 0.17 (0.04) | 0.00 | 0.18 (0.05) | 0.17 (0.05) | 0.20 | 12.15 (9.76) | 10.54 (9.32) | 0.17 | 7.37 (7.56) | 6.24 (7.13) | 0.15 |
| median [IQR] | 0.16 [0.14, 0.19] | 0.16 [0.14, 0.19] | 0.00 | 0.17 [0.15, 0.21] | 0.16 [0.14, 0.19] | 0.20 | 10.13 [5.57, 16.45] | 8.75 [4.29, 14.71] | 0.14 | 6.15 (7.56) | 5.19 (7.13) | 0.13 |
| Healthcare Utilization | | | | | | | | | | | | |
| Any hospitalization; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 17,074 (25.2%) | 4,804 (32.2%) | -0.16 | 19,589 (14.4%) | 4,815 (19.1%) | -0.13 | 36,663 (16.2%) | 9,619 (22.3%) | -0.16 |
| Any hospitalization within prior 30 days; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 9,626 (14.2%) | 3,296 (22.1%) | -0.21 | 11,829 (8.7%) | 2,910 (11.5%) | -0.09 | 21455 (9.5%) | 6206 (14.4%) | -0.15 |
| Any hospitalization during prior 31-180 days; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 8,232 (12.1%) | 1,717 (11.5%) | 0.02 | 8,606 (6.3%) | 2,082 (8.3%) | -0.08 | 16838 (7.4%) | 3799 (8.8%) | -0.05 |
| Endocrinologist Visit; n (%) | 436 (1.9%) | 84 (2.9%) | -0.07 | 1,932 (2.8%) | 501 (3.4%) | -0.03 | 4,050 (3.0%) | 874 (3.5%) | -0.03 | 6418 (2.8%) | 1459 (3.4%) | -0.03 |
| Endocrinologist Visit (30 days prior); n (%) | 139 (0.6%) | 21 (0.7%) | -0.01 | 633 (0.9%) | 176 (1.2%) | -0.03 | 1,150 (0.8%) | 276 (1.1%) | -0.03 | 1922 (0.8%) | 473 (1.1%) | -0.03 |
| Endocrinologist Visit (31 to 180 days prior); n (%) | 381 (1.7%) | 72 (2.5%) | -0.06 | 1,650 (2.4%) | 413 (2.8%) | -0.03 | 3,536 (2.6%) | 755 (3.0%) | -0.02 | 5567 (2.5%) | 1240 (2.9%) | -0.02 |
| Internal medicine/family medicine visits; n (%) | 19,784 (87.3%) | 2,435 (82.9%) | 0.12 | 52,971 (78.1%) | 11,827 (79.2%) | -0.03 | 108,913 (80.0%) | 20,381 (80.8%) | -0.02 | 181668 (80.2%) | 34643 (80.4%) | -0.01 |
| Internal medicine/family medicine visits (30 days | | | | | | | | | | | | |
| prior) v2; n (%) | 13,564 (59.8%) | 1,529 (52.1%) | 0.16 | 33,572 (49.5%) | 7,777 (52.1%) | -0.05 | 68,566 (50.4%) | 12,510 (49.6%) | 0.02 | 115702 (51.1%) | 21816 (50.6%) | 0.01 |
| Internal medicine/family medicine visits (31 to 180 | | | | | | | | | | | | |
| days prior) v2; n (%) | 17,797 (78.5%) | 2,119 (72.2%) | 0.15 | 48,286 (71.2%) | 10,294 (69.0%) | 0.05 | 95,817 (70.4%) | 17,389 (68.9%) | 0.03 | 161900 (71.5%) | 29802 (69.2%) | 0.05 |
| Cardiologist visit; n (%) | 11,235 (49.6%) | 1,976 (67.3%) | -0.37 | 35,004 (51.6%) | 9,003 (60.3%) | -0.18 | 85,057 (62.5%) | 19,330 (76.6%) | -0.31 | 131296 (58.0%) | 30309 (70.3%) | -0.26 |
| Number of Cardiologist visits (30 days prior); n (%) | 6,801 (30.0%) | 1,379 (47.0%) | -0.35 | 20,128 (29.7%) | 6,908 (46.3%) | -0.35 | 53,448 (39.3%) | 14,249 (56.5%) | -0.35 | 80377 (35.5%) | 22536 (52.3%) | -0.34 |
| Number of Cardiologist visits (31 to 180 days prior); | | | | | | | | | | | | |
| n (%) | 8,195 (36.2%) | 1,255 (42.7%) | -0.13 | 27,617 (40.7%) | 5,842 (39.1%) | 0.03 | 61,773 (45.4%) | 12,141 (48.1%) | -0.05 | 97585 (43.1%) | 19238 (44.6%) | -0.03 |
| Electrocardiogram v2; n (%) | 11,225 (49.5%) | 2,064 (70.3%) | -0.43 | 39,015 (57.6%) | 11,173 (74.8%) | -0.37 | 77,673 (57.1%) | 19,434 (77.0%) | -0.43 | 127913 (56.5%) | 32671 (75.8%) | -0.42 |
| Use of glucose test strips; n (%) | 176 (0.8%) | 33 (1.1%) | -0.03 | 475 (0.7%) | 113 (0.8%) | -0.01 | 1,262 (0.9%) | 261 (1.0%) | -0.01 | 1913 (0.8%) | 407 (0.9%) | -0.01 |
| Dialysis; n (%) | 4 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | ** | 0 (0.0%) | #VALUE! | #VALUE! | 0 (0.0%) | #VALUE! |
| number of different/distinct medication | | | | | | | | | | | | |
| prescriptions | | | | | | | | | | | | |
| mean (sd) | 7.72 (3.82) | 8.13 (4.07) | -0.10 | 9.26 (4.52) | 9.27 (4.58) | 0.00 | 8.30 (3.85) | 8.59 (4.06) | -0.07 | 8.53 (4.06) | 8.79 (4.25) | 0.00 |
| median [IQR] | 7.00 [5.00, 10.00] | 8.00 [5.00, 10.00] | -0.25 | 9.00 [6.00, 12.00] | 9.00 [6.00, 12.00] | 0.00 | 8.00 [6.00, 10.00] | 8.00 [6.00, 11.00] | 0.00 | 5.79 (4.76) | 6.43 (4.80) | 0.00 |
| Number of Hospitalizations | | | | | | | | | | | | |
| mean (sd) | 0.00 (0.00) | 0.00 (0.00) | #DIV/0! | 0.28 (0.51) | 0.35 (0.55) | -0.13 | 0.16 (0.43) | 0.21 (0.47) | -0.11 | 0.18 (0.43) | 0.24 (0.48) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | #DIV/0! | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.52) | 0.00 (0.55) | 0.00 |
| Number of hospital days | | | | | | | | | | | | |
| mean (sd) | 0.00 (0.11) | 0.00 (0.00) | 0.00 | 1.61 (4.76) | 1.50 (3.28) | 0.03 | 0.80 (2.85) | 0.85 (2.46) | -0.02 | 0.96 (3.41) | 1.02 (2.70) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 2.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (4.30) | 0.00 (3.14) | 0.00 |
| Number of Emergency Department (ED) visits v3 | | | | | | | | | | | | |
| mean (sd) | 0.33 (0.88) | 0.42 (1.03) | -0.09 | 0.38 (1.65) | 0.45 (1.73) | -0.04 | 0.57 (1.27) | 0.63 (1.27) | -0.05 | 0.49 (1.36) | 0.55 (1.43) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (1.64) | 0.00 (1.66) | 0.00 |
| Number of Office visits | | | | | | | | | | | | |
| mean (sd) | 5.17 (4.16) | 5.24 (3.67) | -0.02 | 6.39 (5.10) | 5.79 (4.33) | 0.13 | 11.99 (11.24) | 11.79 (10.20) | 0.02 | 9.63 (9.24) | 9.27 (8.27) | 0.00 |
| median [IQR] | 4.00 [2.00, 7.00] | 4.00 [3.00, 7.00] | 0.00 | 5.00 [3.00, 9.00] | 5.00 [3.00, 8.00] | 0.00 | 9.00 [4.00, 16.00] | 9.00 [5.00, 16.00] | 0.00 | 4.59 (9.66) | 5.12 (8.53) | 0.00 |
| Number of Endocrinologist visits | | | | | | | | | | | | |
| mean (sd) | 0.07 (0.76) | 0.11 (1.08) | -0.04 | 0.11 (0.99) | 0.11 (0.87) | 0.00 | 0.13 (1.28) | 0.17 (1.51) | -0.03 | 0.12 (1.16) | 0.15 (1.29) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.28) | 0.00 (1.36) | 0.00 |
| Number of internal medicine/family medicine visits | | | | | | | | | | | | |
| mean (sd) | 10.57 (13.09) | 8.08 (12.69) | 0.19 | 7.44 (10.97) | 6.42 (9.19) | 0.10 | 7.40 (9.26) | 6.44 (7.85) | 0.11 | 7.73 (10.23) | 6.54 (8.74) | 0.00 |
| median [IQR] | 6.00 [2.00, 15.00] | 4.00 [1.00, 10.00] | 0.16 | 4.00 [1.00, 10.00] | 4.00 [1.00, 8.00] | 0.00 | 4.00 [1.00, 10.00] | 4.00 [1.00, 9.00] | 0.00 | 2.99 (11.87) | 3.04 (9.82) | 0.00 |
| Number of Cardiologist visits | | | | | | | | | | | | |
| mean (sd) | 2.53 (4.49) | 3.44 (4.50) | -0.20 | 3.04 (5.45) | 3.42 (5.10) | -0.07 | 3.93 (6.21) | 4.80 (5.92) | -0.14 | 3.52 (5.84) | 4.23 (5.56) | 0.00 |
| median [IQR] | 0.00 [0.00, 3.00] | 2.00 [0.00, 5.00] | -0.44 | 1.00 [0.00, 4.00] | 2.00 [0.00, 5.00] | -0.19 | 2.00 [0.00, 5.00] | 3.00 [1.00, 7.00] | -0.16 | 0.90 (6.56) | 1.87 (6.09) | 0.00 |
| Number electrocardiograms received v2 | | | | | | | | | | | | |
| mean (sd) | 0.96 (1.50) | 1.61 (1.87) | -0.38 | 1.26 (1.82) | 1.79 (1.99) | -0.28 | 1.24 (1.68) | 1.89 (1.96) | -0.36 | 1.22 (1.71) | 1.84 (1.96) | 0.00 |

| median [IQR] | 0.00 [0.00, 1.00] | 1.00 [0.00, 2.00] | -0.59 | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.00 | 1.00 [0.00, 2.00] | 1.00 [1.00, 3.00] | 0.00 | 0.60 (1.98) | 0.76 (2.19) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number of HbA1c tests ordered | | | | | | | | | | | | |
| mean (sd) | 0.36 (0.67) | 0.39 (0.70) | -0.04 | 0.14 (0.45) | 0.16 (0.48) | -0.04 | 0.37 (0.69) | 0.41 (0.72) | -0.06 | 0.30 (0.63) | 0.32 (0.65) | 0.00 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (0.67) | 0.00 (0.69) | 0.00 |
| Number of glucose tests ordered | | | | | | | | | | | | |
| mean (sd) | 0.11 (0.90) | 0.16 (0.94) | -0.05 | 0.10 (0.54) | 0.11 (0.58) | -0.02 | 0.11 (0.52) | 0.13 (0.49) | -0.04 | 0.11 (0.58) | 0.13 (0.56) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.65) | 0.00 (0.63) | 0.00 |
| Number of lipid tests ordered | | | | | | | | | | | | |
| mean (sd) | 0.59 (0.80) | 0.69 (0.85) | -0.12 | 0.22 (0.62) | 0.26 (0.68) | -0.06 | 0.59 (0.71) | 0.70 (0.75) | -0.15 | 0.48 (0.69) | 0.55 (0.73) | 0.00 |
| median [IQR] | 0.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | -1.21 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | -1.37 | 0.00 (0.77) | 0.41 (0.81) | -0.01 |
| Number of creatinine tests ordered | | | | | | | | | | | | |
| mean (sd) | 0.06 (0.32) | 0.07 (0.32) | -0.03 | 0.07 (0.41) | 0.05 (0.27) | 0.06 | 0.09 (0.38) | 0.09 (0.37) | 0.00 | 0.08 (0.38) | 0.07 (0.34) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.44) | 0.00 (0.36) | 0.00 |
| Number of BUN tests ordered | | | | | | | | | | | | |
| mean (sd) | 0.03 (0.24) | 0.05 (0.25) | -0.08 | 0.04 (0.31) | 0.03 (0.23) | 0.04 | 0.05 (0.29) | 0.06 (0.28) | -0.04 | 0.05 (0.29) | 0.05 (0.26) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.34) | 0.00 (0.28) | 0.00 |
| Number of tests for microal buminuria | | | | | | | | | | | | |
| mean (sd) | 0.18 (0.61) | 0.19 (0.64) | -0.02 | 0.06 (0.36) | 0.08 (0.39) | -0.05 | 0.10 (0.37) | 0.12 (0.39) | -0.05 | 0.10 (0.40) | 0.11 (0.41) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.44) | 0.00 (0.45) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at the 3rd | | | | | | | | | | | | |
| digit level Copy | | | | | | | | | | | | |
| mean (sd) | 3.20 (4.99) | 3.00 (5.09) | 0.04 | 2.23 (5.06) | 2.21 (4.86) | 0.00 | | 3.93 (6.39) | -0.01 | 3.32 (5.90) | 3.27 (5.82) | 0.00 |
| median [IQR] | 0.00 [0.00, 5.00] | 0.00 [0.00, 5.00] | 0.00 | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 | 0.00 [0.00, 6.00] | 0.00 [0.00, 6.00] | 0.00 | 0.00 (6.52) | 0.00 (6.28) | 0.00 |
| For PS | | | | | | | | | | | | |
| Hemorrhagic stroke+Other cerebrovascular | | | | , | | | | | | | | |
| disease+Cerebrovascular procedure (for PS); n (%) | 392 (1.7%) | 56 (1.9%) | -0.02 | 1,508 (2.2%) | 344 (2.3%) | -0.01 | 2,242 (1.6%) | 461 (1.8%) | -0.02 | 4142 (1.8%) | 861 (2.0%) | -0.01 |
| Occurrence of creatinine tests ordered (for PS); n (%) | 1,003 (4.4%) | 167 (5.7%) | -0.06 | 3,079 (4.5%) | 535 (3.6%) | 0.05 | 9,217 (6.8%) | 1,813 (7.2%) | -0.02 | 13299 (5.9%) | 2515 (5.8%) | 0.00 |
| Occurrence of creatinine tests ordered (for PS); n (%) Occurrence of BUN tests ordered (for PS); n (%) | | | | | | 0.05 | | | -0.02<br>-0.02 | | | -0.02 |
| Occurrence of BUN tests ordered (for PS); n (%) Occurrence of chronic renal insufficiency w/o CKD | 611 (2.7%) | 112 (3.8%) | -0.06 | 1,812 (2.7%) | 365 (2.4%) | 0.02 | 5,615 (4.1%) | 1,169 (4.6%) | -0.02 | 8038 (3.5%) | 1646 (3.8%) | -0.02 |
| (for PS) v2; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Chronic kidney disease Stage 1-2 (for PS); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Chronic kidney disease Stage 1-2 (for PS); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/01 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | • | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Bladder stones+Kidney stones (for PS): n (%) | 187 (0.8%) | 36 (1.2%) | -0.04 | 861 (1.3%) | 245 (1.6%) | -0.03 | 1,494 (1.1%) | 311 (1.2%) | -0.01 | 2542 (1.1%) | 592 (1.4%) | -0.03 |
| Diabetes with peripheral circulatory | 187 (0.878) | 30 (1.2%) | -0.04 | 801 (1.3%) | 245 (1.0%) | -0.03 | 1,454 (1.170) | 311 (1.270) | -0.01 | 2542 (1.170) | 332 (1.470) | -0.03 |
| disorders+Gangrene+Osteomyelitis(for PS) v3 with | | | | | | | | | | | | |
| ICD10 Copy; n (%) | 601 (2.7%) | 51 (1.7%) | 0.07 | 1,554 (2.3%) | 285 (1.9%) | 0.03 | 3,124 (2.3%) | 485 (1.9%) | 0.03 | 5279 (2.3%) | 821 (1.9%) | 0.03 |
| Alcohol abuse or dependence+Drug abuse or | 001 (2.770) | 31 (1.770) | 0.07 | 1,554 (2.576) | 203 (2:370) | 0.03 | 3,124 (2.370) | 403 (1.570) | 0.03 | 3273 (2.370) | 021 (1:570) | 0.05 |
| dependence (for PS); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Diabetes with other ophthalmic | , | , | | | , | | | | | , | , | |
| manifestations+Retinal detachment, vitreous | | | | | | | | | | | | |
| hemorrhage, vitrectomy+Retinal laser coagulation | | | | | | | | | | | | |
| therapy (for PS); n (%) | 86 (0.4%) | 11 (0.4%) | 0.00 | 937 (1.4%) | 183 (1.2%) | 0.02 | 1,247 (0.9%) | 226 (0.9%) | 0.00 | 2270 (1.0%) | 420 (1.0%) | 0.00 |
| Other atherosclerosis+Cardiac conduction | | | | | | | | | | | | |
| disorders+Other CVD (for PS) v2 Copy; n (%) | 3,880 (17.1%) | 540 (18.4%) | -0.03 | 21,635 (31.9%) | 4,994 (33.5%) | -0.03 | 20,779 (15.3%) | 4,065 (16.1%) | -0.02 | 46294 (20.4%) | 9599 (22.3%) | -0.05 |
| Previous cardiac procedure (CABG or PTCA or Stent) | | | | | | | | | | | | |
| History of CABG or PTCA (for PS) v3; n (%) | 1,033 (4.6%) | 148 (5.0%) | -0.02 | 3,026 (4.5%) | 771 (5.2%) | -0.03 | 8,489 (6.2%) | 2,092 (8.3%) | -0.08 | 12548 (5.5%) | 3011 (7.0%) | -0.06 |
| Hyperthyroidism + Hypothyroidism + Other disorder | | | | | | | | | | | | |
| of thyroid gland (for PS); n (%) | 3,831 (16.9%) | 479 (16.3%) | 0.02 | 8,436 (12.4%) | 1,861 (12.5%) | 0.00 | 17,662 (13.0%) | 3,549 (14.1%) | -0.03 | 29929 (13.2%) | 5889 (13.7%) | -0.01 |
| Delirium + Psychosis (for PS); n (%) | 198 (0.9%) | 29 (1.0%) | -0.01 | 1,554 (2.3%) | 211 (1.4%) | 0.07 | 1,839 (1.4%) | 311 (1.2%) | 0.02 | 3591 (1.6%) | 551 (1.3%) | 0.03 |
| Any use of Meglitinides (for PS); n (%) | 38 (0.2%) | 3 (0.1%) | 0.03 | 324 (0.5%) | 74 (0.5%) | 0.00 | 377 (0.3%) | 74 (0.3%) | 0.00 | 739 (0.3%) | 151 (0.4%) | -0.02 |
| Any use of AGIs (for PS); n (%) | 17 (0.1%) | 4 (0.1%) | 0.00 | 69 (0.1%) | 28 (0.2%) | -0.03 | 109 (0.1%) | 30 (0.1%) | 0.00 | 195 (0.1%) | 62 (0.1%) | 0.00 |
| CKD stage 3-6 + dialysis (for PS); n (%) | 4 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | | 0 (0.0%) | #VALUE! | #VALUE! | 0 (0.0%) | #VALUE! |
| Use of thiazide-United; n (%) | 2,786 (12.3%) | 342 (11.6%) | 0.02 | 7,453 (11.0%) | 1,623 (10.9%) | 0.00 | | 3,212 (12.7%) | -0.01 | 27210 (12.0%) | 5177 (12.0%) | 0.00 |
| Use of beta blockers; n (%) | 13,713 (60.5%) | 1,820 (62.0%) | -0.03 | 44,683 (65.9%) | 10,110 (67.7%) | -0.04 | 87,512 (64.3%) | 16,625 (65.9%) | -0.03 | 145908 (64.4%) | 28555 (66.3%) | -0.04 |
| Use of calcium channel blockers; n (%) | 7,737 (34.1%) | 1,075 (36.6%) | -0.05 | 24,743 (36.5%) | 5,699 (38.2%) | -0.04 | 48,655 (35.8%) | 9,878 (39.2%) | -0.07 | 81135 (35.8%) | 16652 (38.6%) | -0.06 |
| All antidiabetic medications except Insulin; n (%) | 4,109 (18.1%) | 615 (20.9%) | -0.07<br>-0.03 | 12,310 (18.2%) | 2,931 (19.6%) | -0.04<br>0.02 | | 5,082 (20.1%) | -0.04<br>0.01 | 41628 (18.4%) | 8628 (20.0%) | -0.04<br>0.00 |
| DM Medications - Insulin Copy; n (%) | 864 (3.8%)<br>8.138 (35.9%) | 128 (4.4%)<br>964 (32.8%) | -0.03<br>0.07 | 3,888 (5.7%)<br>23.820 (35.1%) | 795 (5.3%)<br>4.901 (32.8%) | 0.02 | 5,129 (3.8%)<br>48.921 (35.9%) | 926 (3.7%)<br>8.854 (35.1%) | 0.01 | 9881 (4.4%)<br>80879 (35.7%) | 1849 (4.3%)<br>14719 (34.2%) | 0.00 |
| Use of Low Intensity Statins; n (%) Use of High Intensity Statins; n (%) | 8,138 (35.9%)<br>4.085 (18.0%) | 964 (32.8%)<br>619 (21.1%) | -0.08 | 23,820 (35.1%)<br>13,552 (20.0%) | 4,901 (32.8%)<br>3,233 (21.7%) | -0.05 | | 8,854 (35.1%)<br>5,459 (21.6%) | -0.06 | 80879 (35.7%)<br>43735 (19.3%) | 14719 (34.2%)<br>9311 (21.6%) | -0.06 |
| | 4,085 (18.0%)<br>693 (3.1%) | 107 (3.6%) | -0.08 | 13,552 (20.0%)<br>27,053 (39.9%) | 3,233 (21.7%)<br>6,491 (43.5%) | -0.04 | | 5,459 (21.6%)<br>4,133 (16.4%) | -0.06 | 43735 (19.3%)<br>44503 (19.6%) | 10731 (24.9%) | -0.06 |
| Malignant hypertension; n (%)<br>Cardiovascular stress test; n (%) | 58 (0.3%) | 13 (0.4%) | -0.03 | 27,053 (39.9%)<br>449 (0.7%) | 6,491 (43.5%) | 0.07 | 579 (0.4%) | 4,133 (10.4%) | 0.12 | 1086 (0.5%) | 189 (0.4%) | 0.01 |
| Echocardiogram; n (%) | 3,464 (15.3%) | 835 (28.4%) | -0.32 | 23,390 (34.5%) | 7,438 (49.8%) | -0.31 | | 9,331 (37.0%) | -0.34 | 56652 (25.0%) | 17604 (40.8%) | -0.34 |
| Number of BNP tests | 3,404 (13.3%) | 833 (28.4%) | -0.32 | 23,390 (34.3%) | 7,438 (45.6%) | -0.51 | 25,750 (21.5%) | 3,331 (37.0%) | -0.54 | 30032 (23.0%) | 17004 (40.6%) | -0.54 |
| mean (sd) | 0.08 (0.35) | 0.09 (0.36) | -0.03 | 0.07 (0.40) | 0.08 (0.35) | -0.03 | 0.11 (0.41) | 0.13 (0.42) | -0.05 | 0.10 (0.40) | 0.11 (0.39) | -0.03 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.46) | 0.00 (0.43) | 0.03 |
| median [iQn] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.40) | 0.00 (0.43) | 0.00 |
| Number of Cardiac biomarkers tests (tropnin, CK-MB | Bs, Myoglobin, CPK) | | | | | | | | | | | |
| mean (sd) | 0.22 (0.91) | 0.37 (1.23) | -0.14 | 0.21 (0.98) | 0.32 (1.30) | -0.10 | 0.19 (0.49) | 0.25 (0.56) | -0.11 | 0.20 (0.72) | 0.28 (0.93) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.90) | 0.00 (1.13) | 0.00 |
| * ** | | | | | | | 1 | | | | | |
| Number of Ambulatory Blood pressure monitoring t | ests | | | | | | | | | | | |
| mean (sd) | 0.00 (0.03) | 0.00 (0.03) | 0.00 | 0.00 (0.04) | 0.00 (0.04) | 0.00 | 0.00 (0.02) | 0.00 (0.04) | 0.00 | 0.00 (0.03) | 0.00 (0.04) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.04) | 0.00 (0.04) | 0.00 |
| N of days on antihypertensive medications during ba | | | | | | | 0 | 0 | | | | |
| mean (sd) | 130.02 (68.95) | 129.85 (66.94) | 0.00 | 135.76 (65.79) | 131.96 (67.63) | 0.06 | 138.23 (64.13) | 137.11 (64.13) | 0.02 | 136.67 (65.13) | 134.83 (65.56) | 0.00 |
| median [IQR] | 171.00 [89.00, 181.00] | 168.00 [91.00, 181.00] | 0.04 | 174.00 [110.00, 181.00] | 171.00 [94.00, 181.00] | 0.04 | 174.00 [122.00, 181.00] | 173.00 [116.00, 181.00] | 0.02 | 121.24 (74.47) | 130.61 (73.42) | 0.00 |
| N of days in database anytime prior | | 1.753.82 (1.191.57) | 0.00 | 2,172.37 (1,246.30) | 2,083.21 (1,203.95) | 0.07 | 0<br>833.53 (537.51) | 0<br>873.46 (457.48) | -0.08 | 1325.93 (889.77) | 1352.52 (849.34) | |
| | | | | | | | | | | | | 0.00 |
| mean (sd) | 1,750.74 (1,238.00) | 1,733.82 (1,131.37) | 0.00 | 2,172.37 (1,240.30) | 2,003.21 (1,203.33) | 0.07 | 833.33 (337.31) | 073.40 (437.40) | -0.00 | 1323.53 (865.77) | 1332.32 (043.34) | 0.00 |

| andia (ION) | 1,541.00 [660.00,<br>2,568.00] | 1,604.00 [712.50,<br>2.511.00] | 0.05 | 2 222 00 (4 052 00 2 470 25) | 2 004 00 (007 50 2 005 00) | 0.10:0 | 20.00 (440.00 1.004.00) | 014 00 [520 00 4 005 00] | 0.35 | 1024.05 (1122.40) | 1116.67 (1033.38) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| median [IQR] | , | 2,511.00] | -0.05 | 2,222.00 [1,052.00, 3,178.25] | 2,094.00 [997.50, 3,086.00] | 0.10 % | 38.00 [448.00, 1,064.00] | 814.00 [530.00, 1,095.00] | -0.25 | 1024.96 (1122.48) | 1116.67 (1033.38) | 0.00 |
| Mean Copay for per prescription cost (charges in U.S. \$ | | | | | | | 0 | 0 | | | | |
| mean (sd) | 30.18 (42.11) | 31.24 (39.86) | -0.03 | 20.81 (20.98) | 22.85 (23.53) | -0.09 | 119.85 (114.12) | 114.07 (117.32) | 0.05 | 81.24 (90.18) | 76.83 (91.42) | 0.00 |
| median [IQR] | 18.00 [8.44, 36.45] | 20.77 [9.54, 39.82] | -0.07<br>0.11 | 16.05 [8.20, 27.50] | 17.50 [8.75, 30.19] | -0.07 | 95.08 [66.22, 140.00] | 90.00 [62.61, 132.00] | 0.04 | 35.06 (90.91) | 38.66 (92.15) | 0.00 |
| Missing; n (%) | 897 (4.0%)<br>527 (2.3%) | 62 (2.1%)<br>97 (3.3%) | -0.06 | 1,967 (2.9%)<br>1.843 (2.7%) | 447 (3.0%)<br>500 (3.3%) | -0.01<br>-0.04 | 3,658 (2.7%)<br>3.176 (2.3%) | 516 (2.0%)<br>762 (3.0%) | 0.05<br>-0.04 | 6522 (2.9%)<br>5546 (2.4%) | 1025 (2.4%)<br>1359 (3.2%) | 0.03<br>-0.05 |
| Colonoscopy; n (%) Fecal occult blood (FOB) test; n (%) | 738 (3.3%) | 119 (4.1%) | -0.06 | 1,273 (1.9%) | 340 (2.3%) | -0.04 | 2,831 (2.1%) | 762 (3.0%) | -0.04 | 4842 (2.1%) | 1201 (2.8%) | -0.05 |
| Flu vaccine; n (%) | 4,911 (21.7%) | 569 (19.4%) | 0.04 | 8,030 (11.8%) | 1,549 (10.4%) | 0.03 | 45,927 (33.7%) | 8,362 (33.1%) | 0.05 | 58868 (26.0%) | 10480 (24.3%) | 0.04 |
| Mammogram; n (%) | 1.643 (7.2%) | 230 (7.8%) | -0.02 | 3,465 (5.1%) | 794 (5.3%) | -0.01 | 9.038 (6.6%) | 1.984 (7.9%) | -0.05 | 14146 (6.2%) | 3008 (7.0%) | -0.03 |
| Pap smear; n (%) | 238 (1.1%) | 45 (1.5%) | -0.02 | 876 (1.3%) | 243 (1.6%) | -0.01 | 1,723 (1.3%) | 566 (2.2%) | -0.03 | 2837 (1.3%) | 854 (2.0%) | -0.05 |
| Pneumonia vaccine; n (%) | 2,371 (10.5%) | 268 (9.1%) | 0.05 | 2,176 (3.2%) | 469 (3.1%) | 0.01 | 16,663 (12.2%) | 2,980 (11.8%) | 0.01 | 21210 (9.4%) | 3717 (8.6%) | 0.03 |
| PSA test or Prostate exam for DRE; n (%) | 3,062 (13.5%) | 511 (17.4%) | -0.11 | 3,858 (5.7%) | 1.151 (7.7%) | -0.08 | 18,750 (13.8%) | 4,597 (18.2%) | -0.12 | 25670 (11.3%) | 6259 (14.5%) | -0.10 |
| Bone mineral density; n (%) | 705 (3.1%) | 107 (3.6%) | -0.03 | 1,213 (1.8%) | 266 (1.8%) | 0.00 | 3.836 (2.8%) | 858 (3.4%) | -0.03 | 5754 (2.5%) | 1231 (2.9%) | -0.02 |
| Use of Sympatomimetic agents; n (%) | 45 (0.2%) | 11 (0.4%) | -0.04 | 231 (0.3%) | 91 (0.6%) | -0.04 | 267 (0.2%) | 61 (0.2%) | 0.00 | 543 (0.2%) | 163 (0.4%) | -0.04 |
| Use of CNS stimulants; n (%) | 24 (0.1%) | 3 (0.1%) | 0.00 | 250 (0.4%) | 84 (0.6%) | -0.03 | 183 (0.1%) | 33 (0.1%) | 0.00 | 457 (0.2%) | 120 (0.3%) | -0.02 |
| Use of estrogens, progestins, androgens; n (%) | 465 (2.1%) | 88 (3.0%) | -0.06 | 2,275 (3.4%) | 696 (4.7%) | -0.07 | 3,175 (2.3%) | 880 (3.5%) | -0.07 | 5915 (2.6%) | 1664 (3.9%) | -0.07 |
| Use of Angiogenesis inhibitors; n (%) | 4 (0.0%) | 1 (0.0%) | #DIV/0! | 28 (0.0%) | 5 (0.0%) | #DIV/0! | 29 (0.0%) | 12 (0.0%) | #DIV/0! | 61 (0.0%) | 18 (0.0%) | #DIV/0! |
| Use of Oral Immunosuppressants; n (%) | 6 (0.0%) | 1 (0.0%) | #DIV/0! | 69 (0.1%) | 8 (0.1%) | 0.00 | 19 (0.0%) | ** | #VALUE! | 94 (0.0%) | #VALUE! | #VALUE! |
| Use of fondaparinux or Bivalirudin; n (%) | 3 (0.0%) | 1 (0.0%) | #DIV/0! | 61 (0.1%) | 11 (0.1%) | 0.00 | 61 (0.0%) | ** | #VALUE! | 125 (0.1%) | #VALUE! | #VALUE! |
| Use of other direct thrombin inhibitors (lepirudin, | | | | | | | | | | | | |
| desirudin, argatroban); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Use of Ticagrelor ON CED; n (%) | 2 (0.0%) | 2 (0.1%) | -0.04 | 43 (0.1%) | 12 (0.1%) | 0.00 | 26 (0.0%) | ** | #VALUE! | 71 (0.0%) | #VALUE! | #VALUE! |
| Use of Ticagrelor; n (%) | 6 (0.0%) | 3 (0.1%) | -0.04 | 62 (0.1%) | 19 (0.1%) | 0.00 | 165 (0.1%) | 37 (0.1%) | 0.00 | 233 (0.1%) | 59 (0.1%) | 0.00 |
| Number of D-dimer tests | 0.01 (0.12) | 0.02 (0.15) | -0.07 | 0.01 (0.12) | 0.02 (0.16) | -0.07 | 0.02 (0.16) | 0.03 (0.18) | -0.06 | 0.02 (0.15) | 0.03 (0.17) | 0.00 |
| mean (sd)<br>median (IQR) | 0.01 (0.12) | 0.02 (0.15) | -0.07 | 0.01 (0.12) | 0.02 (0.16) | -0.07 | 0.02 (0.16) | 0.03 (0.18) | -0.06<br>0.00 | 0.02 (0.15) | 0.03 (0.17) | 0.00 |
| median [IQK] Numbe of CRP, high-sensitivity CRP tests | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | U.UU (U.16) | U.UU (U.19) | 0.00 |
| mean (sd) | 0.04 (0.31) | 0.06 (0.32) | -0.06 | 0.03 (0.23) | 0.03 (0.20) | 0.00 | 0.06 (0.35) | 0.07 (0.36) | -0.03 | 0.05 (0.31) | 0.06 (0.31) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.34) | 0.00 (0.31) | 0.00 |
| Number of PT or aPTTt tests | (,) | (,, | | (,) | (,) | | () | (,) | | () | () | |
| mean (sd) | 3.36 (4.06) | 0.45 (1.50) | 0.95 | 1.97 (3.43) | 0.38 (1.42) | 0.61 | 3.73 (4.31) | 0.40 (1.30) | 1.05 | 3.17 (4.04) | 0.40 (1.36) | 0.01 |
| median [IQR] | 2.00 [0.00, 6.00] | 0.00 [0.00, 0.00] | 0.65 | 0.00 [0.00, 3.00] | 0.00 [0.00, 0.00] | 0.00 | 2.00 [0.00, 6.00] | 0.00 [0.00, 0.00] | 0.63 | 0.80 (4.46) | 0.00 (1.52) | 0.00 |
| Number of Bleeding time tests | | | | | | | | | | | | |
| mean (sd) | 0.00 (0.01) | 0.00 (0.00) | 0.00 | 0.00 (0.01) | 0.00 (0.01) | 0.00 | 0.00 (0.02) | 0.00 (0.02) | 0.00 | 0.00 (0.02) | 0.00 (0.02) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.02) | 0.00 (0.02) | 0.00 |
| HAS-BLED Score (ICD-9 and ICD-10), 180 days | | | | | | | | | | | | |
| mean (sd) | 3.18 (0.65) | 3.23 (0.68) | -0.08 | 3.23 (0.70) | 3.24 (0.75) | -0.01 | 3.23 (0.61) | 3.29 (0.62) | -0.10 | 3.22 (0.64) | 3.27 (0.67) | 0.00 |
| median [IQR] | 3.00 [3.00, 3.00] | 3.00 [3.00, 4.00] | 0.00 | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 2.10 (0.75) | 2.28 (0.77) | 0.00 |
| N of Generic name drugs | | | | | | | | | | | | |
| mean (sd) | 15.76 (13.47) | 14.43 (12.65) | 0.10 | 13.67 (9.58) | 12.24 (9.51) | 0.15 | 15.17 (11.23) | 14.50 (11.57) | 0.06 | 14.78 (11.02) | 13.71 (10.98) | 0.00 |
| median [IQR] | 12.00 [7.00, 20.00] | 11.00 [6.00, 19.00] | 0.08 | 12.00 [7.00, 18.00] | 10.00 [6.00, 16.00] | 0.21 | 13.00 [8.00, 19.00] | 12.00 [7.00, 19.00] | 0.09 | 8.68 (12.21) | 8.37 (11.93) | 0.00 |
| N of Brand name drugs | | | | () | | | | | | | / / | |
| mean (sd)<br>median (IOR) | 2.94 (4.50)<br>1.00 [0.00, 4.00] | 4.77 (5.14)<br>3.00 (1.00, 6.00) | -0.38<br>-0.41 | 4.27 (4.65)<br>3.00 [1.00, 6.00] | 5.81 (5.28)<br>4.00 [2.00, 8.00] | -0.31<br>-0.20 | 3.12 (4.33)<br>2.00 [0.00, 5.00] | 5.05 (5.37)<br>3.00 (1.00, 7.00) | -0.40<br>-0.21 | 3.45 (4.45)<br>1.60 (5.13) | 5.29 (5.32)<br>2.63 (5.92) | 0.00 |
| Use of clopidogrel ; n (%) | 1.00 (0.00, 4.00) | 190 (6.5%) | -0.41 | 5.477 (8.1%) | 1.823 (12.2%) | -0.20 | 8.774 (6.4%) | 2.571 (10.2%) | -0.21 | 15267 (6.7%) | 4584 (10.6%) | -0.14 |
| Systemic embolism; n (%) | 1,010 (4.5%) | 12 (0.4%) | 0.01 | 588 (0.9%) | 58 (0.4%) | 0.14 | 713 (0.5%) | 2,371 (10.2%)<br>87 (0.3%) | 0.03 | 1418 (0.6%) | 157 (0.4%) | 0.03 |
| DVT: n (%) | 887 (3.9%) | 33 (1.1%) | 0.01 | 3.510 (5.2%) | 214 (1.4%) | 0.00 | 6.763 (5.0%) | 280 (1.1%) | 0.03 | 11160 (4.9%) | 527 (1.2%) | 0.22 |
| PE; n (%) | 406 (1.8%) | 4 (0.1%) | 0.18 | 2,009 (3.0%) | 91 (0.6%) | 0.18 | 3,175 (2.3%) | 74 (0.3%) | 0.18 | 5590 (2.5%) | 169 (0.4%) | 0.18 |
| Diabetes: 1 inpatient or 2 outpatient claims within | 400 (1.070) | 4 (0.270) | 0.10 | 2,005 (5.0%) | 31 (0.0%) | 0.10 | 3,273 (2.370) | 74 (0.5%) | 0.20 | 3330 (E.370) | 103 (0.470) | 0.10 |
| 183 days ; n (%) | 5,727 (25.3%) | 791 (26.9%) | -0.04 | 16,089 (23.7%) | 3,565 (23.9%) | 0.00 | 33,792 (24.8%) | 6,369 (25.2%) | -0.01 | 55608 (24.5%) | 10725 (24.9%) | -0.01 |
| Intracranial or retroperitoneal hemorrhage: 1 | | | | | | | | | | | | |
| inpatient or 2 outpatient claims within 183 days; n | | | | | | | | | | | | |
| (%) | 27 (0.1%) | 1 (0.0%) | 0.04 | 89 (0.1%) | 8 (0.1%) | 0.00 | 90 (0.1%) | 18 (0.1%) | 0.00 | 206 (0.1%) | 27 (0.1%) | 0.00 |
| Peptic Ulcer Disease; n (%) | 1,599 (7.1%) | 222 (7.6%) | -0.02 | 3,997 (5.9%) | 908 (6.1%) | -0.01 | 8,879 (6.5%) | 1,855 (7.4%) | -0.04 | 14475 (6.4%) | 2985 (6.9%) | -0.02 |
| Upper GI bleed; n (%) | 2 (0.0%) | 0 (0.0%) | #DIV/0! | 17 (0.0%) | 4 (0.0%) | #DIV/0! | 18 (0.0%) | ** | #VALUE! | 37 (0.0%) | #VALUE! | #VALUE! |
| Lower/unspecified GI bleed; n (%) | 127 (0.6%) | 25 (0.9%) | -0.03 | 491 (0.7%) | 102 (0.7%) | 0.00 | 705 (0.5%) | 154 (0.6%) | -0.01 | 1323 (0.6%) | 281 (0.7%) | -0.01 |
| Urogenital bleed; n (%) | 686 (3.0%) | 91 (3.1%)<br>28 (1.0%) | -0.01 | 2,289 (3.4%) | 451 (3.0%)<br>163 (1.1%) | 0.02 | 4,121 (3.0%)<br>1,919 (1.4%) | 727 (2.9%)<br>259 (1.0%) | 0.01 | 7096 (3.1%) | 1269 (2.9%) | 0.01 |
| Other bleeds; n (%) | 297 (1.3%) | () | 0.03 | 1,189 (1.8%) | () | | -, (, | () | 0.04 | 3405 (1.5%) | 450 (1.0%) | |
| Prior cancer; n (%) Aspirin; n (%) | 2,605 (11.5%)<br>58 (0.3%) | 307 (10.5%)<br>13 (0.4%) | -0.02 | 6,550 (9.7%)<br>593 (0.9%) | 1,366 (9.1%)<br>180 (1.2%) | 0.02<br>-0.03 | 13,998 (10.3%)<br>348 (0.3%) | 2,691 (10.7%)<br>118 (0.5%) | -0.01<br>-0.03 | 23153 (10.2%)<br>999 (0.4%) | 4364 (10.1%)<br>311 (0.7%) | 0.00<br>-0.04 |
| Aspirin; n (%)<br>Aspirin/dipyridamole; n (%) | 36 (0.2%) | 11 (0.4%) | -0.02 | 243 (0.4%) | 83 (0.6%) | -0.03 | 295 (0.2%) | 103 (0.4%) | -0.03 | 574 (0.3%) | 197 (0.5%) | -0.04 |
| Other antiplatelet agents; n (%) | 108 (0.5%) | 13 (0.4%) | 0.04 | 407 (0.6%) | 83 (0.6%) | 0.00 | 604 (0.4%) | 148 (0.6%) | -0.04 | 1119 (0.5%) | 244 (0.6%) | -0.03 |
| PGP inhibitors; n (%) | 8,231 (36.3%) | 1,160 (39.5%) | -0.07 | 30,813 (45.5%) | 7,267 (48.7%) | -0.06 | 54,573 (40.1%) | 11,181 (44.3%) | -0.09 | 93617 (41.3%) | 19608 (45.5%) | -0.01 |
| Other gastroprotective agents; n (%) | 89 (0.4%) | 17 (0.6%) | -0.03 | 525 (0.8%) | 142 (1.0%) | -0.02 | 866 (0.6%) | 178 (0.7%) | -0.01 | 1480 (0.7%) | 337 (0.8%) | -0.01 |
| Number of lipid tests ordered | () | (/ | 2.23 | (0/4) | | | (/9) | () | | .== (=) | ·=· (=:=:d) | |
| mean (sd) | 0.59 (0.80) | 0.69 (0.85) | -0.12 | 0.22 (0.62) | 0.26 (0.68) | -0.06 | 0.62 (0.78) | 0.74 (0.83) | -0.15 | 0.50 (0.74) | 0.57 (0.78) | 0.00 |
| median [IQR] | 0.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | -1.21 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | -1.24 | 0.00 (0.81) | 0.41 (0.85) | 0.00 |
| Proton pump inhibitor; n (%) | 3,648 (16.1%) | 468 (15.9%) | 0.01 | 13,322 (19.7%) | 2,930 (19.6%) | 0.00 | 25,610 (18.8%) | 4,816 (19.1%) | -0.01 | 42580 (18.8%) | 8214 (19.1%) | -0.01 |
| H2 receptor antagonist; n (%) | 704 (3.1%) | 99 (3.4%) | -0.02 | 2,254 (3.3%) | 422 (2.8%) | 0.03 | 5,175 (3.8%) | 1,006 (4.0%) | -0.01 | 8133 (3.6%) | 1527 (3.5%) | 0.01 |
| Vitamin K therapy; n (%) | 18 (0.1%) | 0 (0.0%) | 0.04 | 180 (0.3%) | 8 (0.1%) | 0.04 | 101 (0.1%) | ** | #VALUE! | 299 (0.1%) | #VALUE! | #VALUE! |
| Number of neurologist visits | | | | | | | | | | | | |
| mean (sd) | 0.15 (0.97) | 0.17 (1.00) | -0.02 | 0.18 (1.18) | 0.21 (1.01) | -0.03 | 0.20 (1.29) | 0.24 (1.22) | -0.03 | 0.19 (1.23) | 0.22 (1.14) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.39) | 0.00 (1.24) | 0.00 |
| Number of INR (prothrombin) tests ordered | | | | | | | | | | | | |
| mean (sd) | 3.26 (3.99) | 0.35 (1.30) | 0.98 | 1.88 (3.34) | 0.29 (1.24) | 0.63 | 3.71 (4.27) | 0.37 (1.27) | 1.06 | 3.12 (3.99) | 0.34 (1.26) | 0.01 |
| median [IQR] | 1.00 [0.00, 6.00] | 0.00 [0.00, 0.00]<br>1.387 (47.2%) | 0.34<br>-0.35 | 0.00 [0.00, 2.00] | 0.00 [0.00, 0.00]<br>8.267 (55.4%) | 0.00<br>-0.42 | 2.00 [0.00, 6.00]<br>53,448 (39,3%) | 0.00 [0.00, 0.00] | 0.63<br>-0.35 | 0.70 (4.39)<br>84002 (37.1%) | 0.00 (1.40) | 0.00<br>-0.38 |
| Treating prescriber - Cardiologist; n (%) Treating prescriber - Primary Care Physician: n (%) | 6,838 (30.2%)<br>14,075 (62.1%) | 1,387 (47.2%)<br>1,646 (56.1%) | -0.35<br>0.12 | 23,716 (35.0%)<br>18,447 (27.2%) | 8,267 (55.4%)<br>4,421 (29.6%) | -0.42<br>-0.05 | 53,448 (39.3%)<br>32,984 (24.2%) | 14,249 (56.5%)<br>5,914 (23.4%) | -0.35<br>0.02 | 84002 (37.1%)<br>65506 (28.9%) | 23903 (55.5%)<br>11981 (27.8%) | -0.38 |
| reacing prescriber - rinnary care rnysiciali; ii (%) | 14,073 (02.1%) | 1,040 (30.1%) | 0.12 | 10,447 (27.2%) | 4,421 (29.0%) | -0.05 | 32,304 (24.2%) | 3,314 (23.4%) | 0.02 | 03300 (20.3%) | 11701 (27.8%) | 0.02 |

| Treating prescriber - Other; n (%) | 16,132 (71.2%) | 2,151 (73.3%) | -0.05 | 50,911 (75.1%) | 11,444 (76.7%) | -0.04 | 103,947 (76.4%) | 19,204 (76.1%) | 0.01 | 170990 (75.5%) | 32799 (76.1%) | -0.01 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Alpha blockers; n (%) | 3,017 (13.3%) | 415 (14.1%) | -0.02 | 9,114 (13.4%) | 1,933 (12.9%) | 0.01 | 18,132 (13.3%) | 3,523 (14.0%) | -0.02 | 30263 (13.4%) | 5871 (13.6%) | -0.01 |
| CHADS2 score, 180 days, V | | | | | | | | | | | | |
| mean (sd) | 1.86 (1.00) | 1.87 (1.01) | -0.01 | 1.97 (1.09) | 1.90 (1.08) | 0.06 | 3.02 (1.28) | 2.92 (1.27) | 0.08 | 2.59 (1.20) | 2.50 (1.19) | 0.00 |
| median [IQR] | 2.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 0.00 | 2.00 [1.00, 3.00] | 2.00 [1.00, 2.50] | 0.00 | 3.00 [2.00, 4.00] | 3.00 [2.00, 4.00] | 0.00 | 1.70 (1.34) | 1.87 (1.30) | 0.00 |
| Use of Prasugrel; n (%) | 14 (0.1%) | 7 (0.2%) | -0.03 | 138 (0.2%) | 72 (0.5%) | -0.05 | 11 (0.0%) | ** | #VALUE! | 163 (0.1%) | #VALUE! | #VALUE! |
| Use of Loop Diuretics+other diuretics+other | | | | | | | | | | | | |
| hypertension drugs; n (%) | 6,341 (28.0%) | 695 (23.7%) | 0.10 | 25,337 (37.4%) | 4,384 (29.4%) | 0.17 | 43,001 (31.6%) | 6,494 (25.7%) | 0.13 | 74679 (33.0%) | 11573 (26.9%) | 0.13 |
| Commercial vs Medicare Advantage- Business Type | | | | | | | | | | | | |
| Code - CORRECT ONE - OPTUM | | | | | | | | | | | | |
| Commercial; n (%) | 2,194 (9.7%) | 653 (22.2%) | -0.35 | 61,780 (91.1%) | 12,464 (83.5%) | 0.23 | | - | #VALUE! | 63,974 (70.7%) | 13,117 (73.4%) | -0.06 |
| Medicare Advantage; n (%) | 20,471 (90.3%) | 2283 (77.8%) | 0.35 | 6,010 (8.9%) | 2,465 (16.5%) | -0.23 | - | - | #VALUE! | 26,481 (29.3%) | 4,748 (26.6%) | 0.06 |
| Commercial vs Medicare Advantage- Business Type | | | | | | | | | | | | |
| Code | | | | | | | | | | | | |
| COM = COMMERCIAL; n (%) | 2,194 (9.7%) | 653 (22.2%) | -0.35 | - | - | | | - | #VALUE! | 2,194 (9.7%) | 653 (22.2%) | -0.35 |
| MCR = MEDICARE; n (%) | 20,471 (90.3%) | 2,283 (77.8%) | 0.35 | - | - | | - | - | #VALUE! | 20,471 (90.3%) | 2,283 (77.8%) | 0.35 |
| MCD = MEDICAID; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | | | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| NONE = NO BUSINESS LINE CODE (added in 2015); n | | | | | | | | | | | | |
| (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | | | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| UNK = UNKNOWN (added in 2015); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Commercial vs Medicare Advantage- Data Type | | | | | | | | | | | | |
| 1 - Fee For Service; n (%) | | | | 5,285 (7.8%) | 2,211 (14.8%) | -0.22 | - | - | | 5,285 (7.8%) | 2,211 (14.8%) | -0.22 |
| 2 - Encounter; n (%) | | | | 725 (1.1%) | 254 (1.7%) | -0.05 | | - | | 725 (1.1%) | 254 (1.7%) | -0.05 |
| 3 - Medicare; n (%) | | | | 54,723 (80.7%) | 11,573 (77.5%) | 0.08 | | - | | 54,723 (80.7%) | 11,573 (77.5%) | 0.08 |
| 4 - Medicare Encounter; n (%) | | | | 7,057 (10.4%) | 891 (6.0%) | 0.16 | - | - | | 7,057 (10.4%) | 891 (6.0%) | 0.16 |
| Metropolitan Statistical Area - Urban (any MSA) vs | | | | | | | | | | | | |
| Rural (non-MSA) | | | | | | | | | | 0 | 0 | 0.00 |
| Urban; n (%) | | | | 53,890 (79.5%) | 11,905 (79.7%) | 0.00 | | - | | 53,890 (79.5%) | 11,905 (79.7%) | 0.00 |
| Rural; n (%) | | | | 649 (1.0%) | 117 (0.8%) | 0.02 | | | | 649 (1.0%) | 117 (0.8%) | 0.02 |
| Unknown/Missing; n (%) | | | | 13,251 (19.5%) | 2,907 (19.5%) | 0.00 | | - | | 13,251 (19.5%) | 2,907 (19.5%) | 0.00 |

Due to CMS cell suppression policy, all values less

| | | | | | PS-matched | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Optun | 1 | I | Mai | ketScan | | Med | licare | | | POOLED | |
| Variable Number of patients | WARFARIN<br>2,790 | Dabigatran 150mg<br>2,790 | St. Diff. | Reference - warfarin<br>13,960 | Exposure - Dabigatran 150mg<br>13,960 | St. Diff. | Reference - warfarin<br>22,320 | Exposure - Dabigatran 150mg<br>22,320 | St. Diff. | Reference - warfarin<br>39,070 | Exposure - Dabigatran 150mg<br>39,070 | St. Diff |
| Age | | | | | | | | | | | | |
| mean (sd) | 75.41 (7.35) | 75.41 (7.13) | 0.00 | 74.41 (10.11) | 74.76 (9.22) | -0.04 | 77.04 (7.31) | 77.18 (6.88) | -0.02 | 75.98 (8.42) | 76.19 (7.81) | -0.03 |
| median [IQR] | 77.00 [71.00, 81.00] | 77.00 [71.00, 81.00] | 0.00 | 76.00 [69.00, 81.00] | 76.00 [69.00, 81.00] | 0.00 | 77.00 [73.00, 82.00] | 77.00 [73.00, 82.00] | 0.00 | 76.64 (8.42) | 76.64 (7.81) | 0.00 |
| Age categories without zero category | EO (1 89/) | 22 (1 19/) | 0.06 | 628 (4.5%) | 439 (3.19/) | 0.07 | 209 (0.9%) | 02 (0.49/) | 0.06 | 887 (2.3%) | EE2 (1 49/) | 0.07 |
| 18 - 54; n (%)<br>55 - 64; n (%) | 50 (1.8%)<br>145 (5.2%) | 32 (1.1%)<br>153 (5.5%) | -0.01 | 1.527 (10.9%) | 428 (3.1%)<br>1.634 (11.7%) | -0.03 | 414 (1.9%) | 92 (0.4%)<br>310 (1.4%) | 0.06 | 2.086 (5.3%) | 552 (1.4%)<br>2,097 (5.4%) | 0.07 |
| 65 - 74; n (%) | 661 (23.7%) | 665 (23.8%) | 0.00 | 3,394 (24.3%) | 3,359 (24.1%) | 0.00 | 6,138 (27.5%) | 6,223 (27.9%) | -0.01 | 10,193 (26.1%) | 10,247 (26.2%) | 0.00 |
| >= 75; n (%) | 1,934 (69.3%) | 1,940 (69.5%) | 0.00 | 8,411 (60.3%) | 8,539 (61.2%) | -0.02 | 15,559 (69.7%) | 15,695 (70.3%) | -0.01 | 25,904 (66.3%) | 26,174 (67.0%) | -0.01 |
| Gender without zero category- United | | | | | | | | | | | | |
| Males; n (%) | 1,675 (60.0%) | 1,675 (60.0%) | 0.00 | 8,106 (58.1%) | 8,134 (58.3%) | 0.00 | 12,689 (56.9%) | 12,580 (56.4%) | 0.01 | 22,470 (57.5%) | 22,389 (57.3%) | 0.00 |
| Females; n (%) | 1,115 (40.0%) | 1,115 (40.0%) | 0.00 | 5,854 (41.9%) | 5,826 (41.7%) | 0.00 | 9,631 (43.1%) | 9,740 (43.6%) | -0.01 | 16,600 (42.5%) | 16,681 (42.7%) | 0.00 |
| Race<br>White; n (%) | | | | | | | 20,699 (92.7%) | 20,744 (92.9%) | | 20,699 (92.7%) | 20,744 (92.9%) | 0.00 |
| Write; n (%)<br>Black; n (%) | | | | | | | 663 (3.0%) | 656 (2.9%) | | 663 (3.0%) | 656 (2.9%) | 0.00 |
| Asian; n (%) | | | | | | | 289 (1.3%) | 290 (1.3%) | | 289 (1.3%) | 290 (1.3%) | 0.00 |
| Hispanic; n (%) | | | | | | | 242 (1.1%) | 219 (1.0%) | | 242 (1.1%) | 219 (1.0%) | 0.00 |
| North American Native; n (%) | | | | | | | 73 (0.3%) | 67 (0.3%) | | 73 (0.3%) | 67 (0.3%) | 0.00 |
| Other/Unknown; n (%) | | | | | | | 354 (1.6%) | 344 (1.5%) | | 354 (1.6%) | 344 (1.5%) | 0.00 |
| Region without zero category- United v3 (lumping missing&other category with West) | | | | | | | | | | | | |
| Northeast; n (%) | 407 (14.6%) | 401 (14.4%) | 0.01 | 3,208 (23.0%) | 3,249 (23.3%) | -0.01 | 4,283 (19.2%) | 4,272 (19.1%) | 0.00 | 7,898 (20.2%) | 7,922 (20.3%) | 0.00 |
| South; n (%) | 945 (33.9%) | 945 (33.9%) | 0.00 | 3,797 (27.2%) | 3,765 (27.0%) | 0.00 | 8,706 (39.0%) | 8,595 (38.5%) | 0.01 | 13,448 (34.4%) | 13,305 (34.1%) | 0.01 |
| Midwest; n (%) | 453 (16.2%) | 456 (16.3%) | 0.00 | 4,767 (34.1%) | 4,766 (34.1%) | 0.00 | 5,278 (23.6%) | 5,344 (23.9%) | -0.01 | 10,498 (26.9%) | 10,566 (27.0%) | 0.00 |
| West; n (%) | 985 (35.3%) | 988 (35.4%) | 0.00 | 2,126 (15.2%) | 2,119 (15.2%) | 0.00 | 4,053 (18.2%) | 4,109 (18.4%) | -0.01 | 7,164 (18.3%) | 7,216 (18.5%) | -0.01 |
| Unknown+missing; n (%) | N/A | N/A | #VALUE! | 62 (0.4%) | 61 (0.4%) | 0.00 | N/A | N/A | #VALUE! | 62 (0.4%) | 61 (0.4%) | 0.00 |
| CV Covariates | 045 (00 00) | 000 (00 70) | | 4.070 (0.4.00) | 4.044 (0.4.704) | | 7 005 (04 50) | 5 000 (04 00) | | 40 740 (00 50) | 40.500.500.000 | 0.00 |
| Ischemic heart disease; n (%) Acute MI; n (%) | 815 (29.2%)<br>18 (0.6%) | 800 (28.7%)<br>19 (0.7%) | 0.01<br>-0.01 | 4,873 (34.9%)<br>394 (2.8%) | 4,841 (34.7%)<br>378 (2.7%) | 0.00<br>0.01 | 7,025 (31.5%)<br>320 (1.4%) | 6,988 (31.3%)<br>337 (1.5%) | 0.00<br>-0.01 | 12,713 (32.5%)<br>732 (1.9%) | 12,629 (32.3%)<br>734 (1.9%) | 0.00 |
| ACS/unstable angina; n (%) | 28 (1.0%) | 28 (1.0%) | 0.00 | 386 (2.8%) | 384 (2.8%) | 0.00 | 405 (1.8%) | 400 (1.8%) | 0.00 | 819 (2.1%) | 812 (2.1%) | 0.00 |
| Old MI: n (%) | 76 (2.7%) | 69 (2.5%) | 0.01 | 486 (3.5%) | 464 (3.3%) | 0.01 | 992 (4.4%) | 952 (4.3%) | 0.00 | 1554 (4.0%) | 1485 (3.8%) | 0.01 |
| Stable angina; n (%) | 100 (3.6%) | 94 (3.4%) | 0.01 | 556 (4.0%) | 549 (3.9%) | 0.01 | 864 (3.9%) | 822 (3.7%) | 0.01 | 1,520 (3.9%) | 1,465 (3.7%) | 0.01 |
| Coronary atherosclerosis and other forms of chronic | | | | | | | | | | | | |
| ischemic heart disease; n (%) | 759 (27.2%) | 754 (27.0%) | 0.00 | 4,442 (31.8%) | 4,376 (31.3%) | 0.01 | 6,399 (28.7%) | 6,373 (28.6%) | 0.00 | 11,600 (29.7%) | 11,503 (29.4%) | 0.01 |
| Other atherosclerosis with ICD10 v2 Copy; n (%) | 49 (1.8%) | 44 (1.6%) | 0.02 | 241 (1.7%) | 223 (1.6%) | 0.01 | 296 (1.3%) | 296 (1.3%) | 0.00 | 586 (1.5%) | 563 (1.4%) | 0.01 |
| Previous cardiac procedure (CABG or PTCA or Stent)<br>v4: n (%) | 3 (0.1%) | 7 (0.3%) | -0.04 | 221 (1.6%) | 142 (1.0%) | 0.05 | 222 (1.0%) | 125 (0.6%) | 0.04 | 446 (1.1%) | 274 (0.7%) | 0.04 |
| History of CABG or PTCA; n (%) | 152 (5.4%) | 139 (5.0%) | 0.02 | 585 (4.2%) | 611 (4.4%) | -0.01 | 1,677 (7.5%) | 1.720 (7.7%) | -0.01 | 2,414 (6.2%) | 2,470 (6.3%) | 0.04 |
| Any stroke: n (%) | 244 (8.7%) | 243 (8.7%) | 0.00 | 1,310 (9.4%) | 1,263 (9.0%) | 0.01 | 1,529 (6.9%) | 1,560 (7.0%) | 0.00 | 3,083 (7.9%) | 3,066 (7.8%) | 0.00 |
| Ischemic stroke (w and w/o mention of cerebral | , / | | | , , , , , , | ,, | | , | ,, | | | ,,,,,, | |
| infarction); n (%) | 243 (8.7%) | 243 (8.7%) | 0.00 | 1,307 (9.4%) | 1,258 (9.0%) | 0.01 | 1,521 (6.8%) | 1,552 (7.0%) | -0.01 | 3,071 (7.9%) | 3,053 (7.8%) | 0.00 |
| Hemorrhagic stroke; n (%) | 3 (0.1%) | 2 (0.1%) | 0.00 | 6 (0.0%) | 8 (0.1%) | -0.04 | ** | ** | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| TIA; n (%) | 132 (4.7%) | 137 (4.9%) | -0.01 | 655 (4.7%) | 636 (4.6%) | 0.00 | 690 (3.1%) | 663 (3.0%) | 0.01 | 1477 (3.8%) | 1436 (3.7%) | 0.01 |
| Other cerebrovascular disease; n (%) | 43 (1.5%) | 51 (1.8%) | -0.02<br>0.02 | 274 (2.0%) | 290 (2.1%) | -0.01<br>0.00 | 390 (1.7%) | 375 (1.7%) | 0.00 | 707 (1.8%) | 716 (1.8%) | 0.00 |
| Late effects of cerebrovascular disease; n (%) Cerebrovascular procedure; n (%) | 11 (0.4%)<br>0 (0.0%) | 9 (0.3%) 0 (0.0%) | #DIV/0! | 17 (0.1%)<br>21 (0.2%) | 19 (0.1%)<br>21 (0.2%) | 0.00 | 66 (0.3%)<br>19 (0.1%) | 68 (0.3%)<br>16 (0.1%) | 0.00 | 94 (0.2%)<br>040 (0.1%) | 96 (0.2%)<br>37 (0.1%) | 0.00 |
| Heart failure (CHF); n (%) | 325 (11.6%) | 326 (11.7%) | 0.00 | 3,066 (22.0%) | 3,013 (21.6%) | 0.01 | 2,500 (11.2%) | 2,580 (11.6%) | -0.01 | 5,891 (15.1%) | 5,919 (15.1%) | 0.00 |
| Peripheral Vascular Disease (PVD) or PVD Surgery v2; | () | ( | | 0,000 (==1011) | 0,000 (00.00,0 | | _,=== (=====, | -,, | | -, (, | 2,222 (22.2.2) | |
| n (%) | 209 (7.5%) | 203 (7.3%) | 0.01 | 898 (6.4%) | 922 (6.6%) | -0.01 | 1,212 (5.4%) | 1,199 (5.4%) | 0.00 | 2,319 (5.9%) | 2,324 (5.9%) | 0.00 |
| Atrial fibrillation; n (%) | 2,634 (94.4%) | 2,641 (94.7%) | -0.01 | 13,289 (95.2%) | 13,224 (94.7%) | 0.02 | 19,244 (86.2%) | 19,278 (86.4%) | -0.01 | 35,167 (90.0%) | 35,143 (89.9%) | 0.00 |
| Other cardiac dysrhythmia; n (%) | 1,200 (43.0%) | 1,187 (42.5%) | 0.01 | 4,384 (31.4%) | 4,311 (30.9%) | 0.01 | 8,194 (36.7%) | 8,120 (36.4%) | 0.01 | 13,778 (35.3%) | 13,618 (34.9%) | 0.01 |
| Cardiac conduction disorders; n (%) Other CVD; n (%) | 145 (5.2%)<br>363 (13.0%) | 174 (6.2%)<br>333 (11.9%) | -0.04<br>0.03 | 894 (6.4%)<br>4,082 (29.2%) | 888 (6.4%)<br>4,009 (28.7%) | 0.00<br>0.01 | 1,301 (5.8%)<br>2,342 (10.5%) | 1,265 (5.7%)<br>2,297 (10.3%) | 0.00<br>0.01 | 2340 (6.0%)<br>6,787 (17.4%) | 2327 (6.0%)<br>6,639 (17.0%) | 0.00<br>0.01 |
| Diabetes-related complications | 363 (13.0%) | 333 (11.9%) | 0.03 | 4,082 (29.2%) | 4,009 (28.7%) | 0.01 | 2,342 (10.5%) | 2,297 (10.3%) | 0.01 | 6,787 (17.4%) | 6,639 (17.0%) | 0.01 |
| Diabetic retinopathy; n (%) | 38 (1.4%) | 40 (1.4%) | 0.00 | 187 (1.3%) | 176 (1.3%) | 0.00 | 222 (1.0%) | 201 (0.9%) | 0.01 | #VALUE! | 417 (1.1%) | #VALUE! |
| Diabetes with other ophthalmic manifestations; n | () | (=) | | () | () | | (, | () | | | () | |
| (%) | 1 (0.0%) | 2 (0.1%) | -0.04 | 154 (1.1%) | 121 (0.9%) | 0.02 | 154 (0.7%) | 137 (0.6%) | 0.01 | 309 (0.8%) | 260 (0.7%) | 0.01 |
| Retinal detachment, vitreous hemorrhage, | | | | | | | | | | | | |
| vitrectomy; n (%) | 9 (0.3%) | 7 (0.3%) | 0.00 | 36 (0.3%) | 31 (0.2%) | 0.02 | 31 (0.1%) | 33 (0.1%) | 0.00 | 076 (0.2%) | 71 (0.2%) | 0.00 |
| Retinal laser coagulation therapy; n (%) | 1 (0.0%)<br>103 (3.7%) | 2 (0.1%) | -0.04 | 26 (0.2%) | 31 (0.2%) | 0.00 | 43 (0.2%) | 31 (0.1%)<br>569 (2.5%) | 0.03 | 70 (0.2%)<br>1109 (2.8%) | 64 (0.2%) | 0.00 |
| Occurrence of Diabetic Neuropathy v2 Copy; n (%) Occurrence of diabetic nephropathy V3 with ICD10 | 103 (3.7%) | 110 (3.9%) | -0.01 | 436 (3.1%) | 455 (3.3%) | -0.01 | 570 (2.6%) | 569 (2.5%) | 0.01 | 1109 (2.8%) | 1134 (2.9%) | -0.01 |
| Copy; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Hypoglycemia v2; n (%) | 15 (0.5%) | 18 (0.6%) | -0.01 | 151 (1.1%) | 128 (0.9%) | 0.02 | 244 (1.1%) | 190 (0.9%) | 0.02 | 410 (1.0%) | 336 (0.9%) | 0.01 |
| Hyperglycemia; n (%) | 117 (4.2%) | 105 (3.8%) | 0.02 | 255 (1.8%) | 282 (2.0%) | -0.01 | 1,028 (4.6%) | 1,049 (4.7%) | 0.00 | 1400 (3.6%) | 1436 (3.7%) | -0.01 |
| Disorders of fluid electrolyte and acid-base balance; n | | | | | | | | | | | | |
| (%) | 105 (3.8%) | 107 (3.8%) | 0.00 | 872 (6.2%) | 880 (6.3%) | 0.00 | 1,011 (4.5%) | 1,061 (4.8%) | -0.01 | 1988 (5.1%) | 2048 (5.2%) | 0.00 |
| Diabetic ketoacidosis; n (%) | 2 (0.1%) | 2 (0.1%) | 0.00 | 19 (0.1%) | 8 (0.1%) | 0.00 | 24 (0.1%) | 16 (0.1%) | 0.00 | 45 (0.1%) | 26 (0.1%) | 0.00 |
| Hyperosmolar hyperglycemic nonketotic syndrome<br>(HONK); n (%) | 2 (0.1%) | 1 (0.0%) | 0.04 | 12 (0.1%) | 5 (0.0%) | 0.04 | 17 (0.1%) | 21 (0.1%) | 0.00 | 31 (0.1%) | 27 (0.1%) | 0.00 |
| (HONK); n (%) Diabetes with peripheral circulatory disorders with | 2 (U.1%) | 1 (U.U%) | 0.04 | 12 (U.1%) | 5 (0.0%) | 0.04 | 1/(0.1%) | 21 (U.1%) | 0.00 | 31 (U.1%) | 27 (0.1%) | 0.00 |
| ICD-10 v2 Copy; n (%) | 68 (2.4%) | 46 (1.6%) | 0.06 | 242 (1.7%) | 225 (1.6%) | 0.01 | 361 (1.6%) | 384 (1.7%) | -0.01 | 671 (1.7%) | 655 (1.7%) | 0.00 |
| Diabetic Foot; n (%) | 46 (1.6%) | 38 (1.4%) | 0.02 | 243 (1.7%) | 261 (1.9%) | -0.02 | 358 (1.6%) | 423 (1.9%) | -0.02 | 647 (1.7%) | 722 (1.8%) | -0.01 |
| Gangrene v2; n (%) | 3 (0.1%) | 1 (0.0%) | 0.04 | 13 (0.1%) | 15 (0.1%) | 0.00 | 14 (0.1%) | 11 (0.0%) | 0.04 | 030 (0.1%) | 27 (0.1%) | 0.00 |
| Lower extremity amputation; n (%) | 2 (0.1%) | 8 (0.3%) | -0.04 | 15 (0.1%) | 27 (0.2%) | -0.03 | 33 (0.1%) | 38 (0.2%) | -0.03 | 050 (0.1%) | 073 (0.2%) | -0.03 |
| Osteomyelitis; n (%) | 5 (0.2%) | 4 (0.1%) | 0.03 | 40 (0.3%) | 48 (0.3%) | 0.00 | 43 (0.2%) | 47 (0.2%) | 0.00 | 88 (0.2%) | 99 (0.3%) | -0.02 |
| Skin infections v2; n (%) | 119 (4.3%) | 131 (4.7%) | -0.02 | 711 (5.1%) | 748 (5.4%) | -0.01 | 967 (4.3%) | 1,042 (4.7%) | -0.02 | 1797 (4.6%) | 1921 (4.9%) | -0.01 |
| Erectile dysfunction; n (%) | 58 (2.1%) | 63 (2.3%) | -0.01 | 215 (1.5%) | 215 (1.5%) | 0.00 | 223 (1.0%) | 192 (0.9%) | 0.01 | 496 (1.3%) | 470 (1.2%) | 0.01 |

| Diabetes with unspecified complication; n (%) | 19 (0.7%) | 19 (0.7%) | 0.00 | 115 (0.8%) | 92 (0.7%) | 0.01 | 150 (0.7%) | 125 (0.6%) | 0.01 | 284 (0.7%) | 236 (0.6%) | 0.01 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Diabetes mellitus without mention of complications; | | | | | | | | , | | | | |
| n (%)<br>Hypertension: 1 inpatient or 2 outpatient claims | 803 (28.8%) | 788 (28.2%) | 0.01 | 3,509 (25.1%) | 3,454 (24.7%) | 0.01 | 6,004 (26.9%) | 5,993 (26.9%) | 0.00 | 10,316 (26.4%) | 10,235 (26.2%) | 0.00 |
| within 365 days; n (%) | 2,143 (76.8%) | 2,129 (76.3%) | 0.01 | 9.249 (66.3%) | 9,189 (65.8%) | 0.01 | 18.608 (83.4%) | 18,599 (83,3%) | 0.00 | 30.000 (76.8%) | 29.917 (76.6%) | 0.00 |
| Hyperlipidemia v2; n (%) | 1,705 (61.1%) | 1,697 (60.8%) | 0.01 | 5,935 (42.5%) | 5,767 (41.3%) | 0.02 | 11,060 (49.6%) | 10,934 (49.0%) | 0.01 | 18,700 (47.9%) | 18,398 (47.1%) | 0.02 |
| Edema; n (%) | 233 (8.4%) | 230 (8.2%) | 0.01 | 1,038 (7.4%) | 981 (7.0%) | 0.02 | 1,262 (5.7%) | 1,296 (5.8%) | 0.00 | 2533 (6.5%) | 2507 (6.4%) | 0.00 |
| Renal Dysfunction (non-diabetic) v2; n (%) | 1 (0.0%) | 1 (0.0%) | #DIV/0! | 6 (0.0%) | 6 (0.0%) | #DIV/0! | ** | ** | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Occurrence of acute renal disease v2; n (%) | 0 (0.0%) | 1 (0.0%) | #DIV/0! | 6 (0.0%) | 6 (0.0%) | #DIV/0! | ** | ** | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Occurrence of chronic renal insufficiency; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0!<br>#DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Chronic kidney disease v2; n (%)<br>CKD Stage 3-4; n (%) | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%)<br>0 (0.0%) | #DIV/0!<br>#DIV/0! | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%)<br>0 (0.0%) | #DIV/0!<br>#DIV/0! | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%)<br>0 (0.0%) | #DIV/0!<br>#DIV/0! | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%)<br>0 (0.0%) | #DIV/0!<br>#DIV/0! |
| Occurrence of hypertensive nephropathy; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Occurrence of miscellaneous renal insufficiency v2; n | - () | - () | | - () | - () | | - () | - () | | - () | - () | |
| (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Glaucoma or cataracts v2; n (%) | 605 (21.7%) | 645 (23.1%) | -0.03 | 3,101 (22.2%) | 3,062 (21.9%) | 0.01 | 4,898 (21.9%) | 5,044 (22.6%) | -0.02 | 8,604 (22.0%) | 8,751 (22.4%) | -0.01 |
| Cellulitis or abscess of toe; n (%) Foot ulcer: n (%) | 15 (0.5%) | 16 (0.6%) | -0.01 | 68 (0.5%)<br>248 (1.8%) | 89 (0.6%) | -0.01 | 143 (0.6%) | 150 (0.7%) | -0.01 | 226 (0.6%) | 255 (0.7%) | -0.01 |
| Bladder stones; n (%) | 48 (1.7%)<br>8 (0.3%) | 39 (1.4%)<br>5 (0.2%) | 0.02 | 248 (1.8%)<br>15 (0.1%) | 264 (1.9%)<br>26 (0.2%) | -0.01<br>-0.03 | 310 (1.4%)<br>28 (0.1%) | 369 (1.7%)<br>23 (0.1%) | -0.02<br>0.00 | 606 (1.6%)<br>51 (0.1%) | 672 (1.7%)<br>54 (0.1%) | -0.01<br>0.00 |
| Kidney stones: n (%) | 29 (1.0%) | 32 (1.1%) | -0.01 | 181 (1.3%) | 213 (1.5%) | -0.02 | 270 (1.2%) | 257 (1.2%) | 0.00 | 480 (1.2%) | 502 (1.3%) | -0.01 |
| Urinary tract infections (UTIs); n (%) | 194 (7.0%) | 181 (6.5%) | 0.02 | 860 (6.2%) | 893 (6.4%) | -0.01 | 1,803 (8.1%) | 1,851 (8.3%) | -0.01 | 2,857 (7.3%) | 2,925 (7.5%) | -0.01 |
| Dipstick urinalysis; n (%) | 817 (29.3%) | 853 (30.6%) | -0.03 | 2,796 (20.0%) | 2,903 (20.8%) | -0.02 | 7,125 (31.9%) | 7,263 (32.5%) | -0.01 | 10,738 (27.5%) | 11,019 (28.2%) | -0.02 |
| Non-dipstick urinalysis; n (%) | 355 (12.7%) | 332 (11.9%) | 0.02 | 689 (4.9%) | 710 (5.1%) | -0.01 | 2,558 (11.5%) | 2,600 (11.6%) | 0.00 | 3,602 (9.2%) | 3,642 (9.3%) | 0.00 |
| Urine function test; n (%) | 106 (3.8%) | 93 (3.3%) | 0.03 | 623 (4.5%) | 599 (4.3%) | 0.01 | 888 (4.0%) | 889 (4.0%) | 0.00 | 1617 (4.1%) | 1581 (4.0%) | 0.01 |
| Cytology; n (%)<br>Cystoscopy; n (%) | 40 (1.4%)<br>50 (1.8%) | 37 (1.3%)<br>45 (1.6%) | 0.01 | 357 (2.6%)<br>342 (2.4%) | 338 (2.4%)<br>361 (2.6%) | 0.01<br>-0.01 | 365 (1.6%)<br>493 (2.2%) | 391 (1.8%)<br>456 (2.0%) | -0.02<br>0.01 | 762 (2.0%)<br>885 (2.3%) | 766 (2.0%)<br>862 (2.2%) | 0.00 |
| Other Covariates | 30 (1.6%) | 45 (1.0%) | 0.02 | 342 (2.470) | 301 (2.0%) | -0.01 | 453 (2.270) | 430 (2.0%) | 0.01 | 003 (2.3%) | 002 (2.2%) | 0.01 |
| Liver disease; n (%) | 12 (0.4%) | 13 (0.5%) | -0.01 | 85 (0.6%) | 84 (0.6%) | 0.00 | 93 (0.4%) | 90 (0.4%) | 0.00 | 190 (0.5%) | 187 (0.5%) | 0.00 |
| Osteoarthritis; n (%) | 488 (17.5%) | 471 (16.9%) | 0.02 | 2,145 (15.4%) | 2,035 (14.6%) | 0.02 | 3,559 (15.9%) | 3,519 (15.8%) | 0.00 | 6192 (15.8%) | 6025 (15.4%) | 0.01 |
| Other arthritis, arthropathies and musculoskeletal | | | | | | | | | | | | |
| pain; n (%) | 865 (31.0%) | 849 (30.4%) | 0.01 | 4,550 (32.6%) | 4,451 (31.9%) | 0.01 | 6,586 (29.5%) | 6,545 (29.3%) | 0.00 | 12001 (30.7%) | 11845 (30.3%) | 0.01 |
| Dorsopathies; n (%)<br>Fractures; n (%) | 503 (18.0%)<br>56 (2.0%) | 500 (17.9%)<br>62 (2.2%) | 0.00<br>-0.01 | 2,553 (18.3%)<br>474 (3.4%) | 2,541 (18.2%)<br>477 (3.4%) | 0.00 | 3,859 (17.3%)<br>701 (3.1%) | 3,772 (16.9%)<br>699 (3.1%) | 0.01 | 6915 (17.7%)<br>1231 (3.2%) | 6813 (17.4%)<br>1238 (3.2%) | 0.01 |
| Falls v2; n (%) | 74 (2.7%) | 67 (2.4%) | 0.01 | 124 (0.9%) | 135 (1.0%) | -0.01 | 260 (1.2%) | 252 (1.1%) | 0.00 | 458 (1.2%) | 454 (1.2%) | 0.00 |
| Osteoporosis: n (%) | 159 (5.7%) | 177 (6.3%) | -0.03 | 973 (7.0%) | 963 (6.9%) | 0.00 | 1,668 (7.5%) | 1,687 (7.6%) | 0.00 | 2800 (7.2%) | 2827 (7.2%) | 0.00 |
| Hyperthyroidism; n (%) | 23 (0.8%) | 23 (0.8%) | 0.00 | 122 (0.9%) | 92 (0.7%) | 0.02 | 187 (0.8%) | 207 (0.9%) | -0.01 | 332 (0.8%) | 322 (0.8%) | 0.00 |
| Hypothyroidism v2; n (%) | 381 (13.7%) | 405 (14.5%) | -0.02 | 1,399 (10.0%) | 1,455 (10.4%) | -0.01 | 2,639 (11.8%) | 2,604 (11.7%) | 0.00 | 4419 (11.3%) | 4464 (11.4%) | 0.00 |
| Other disorders of thyroid gland V2; n (%) | 56 (2.0%) | 68 (2.4%) | -0.03 | 344 (2.5%) | 361 (2.6%) | -0.01 | 593 (2.7%) | 567 (2.5%) | 0.01 | 993 (2.5%) | 996 (2.5%) | 0.00 |
| Depression; n (%) | 132 (4.7%) | 135 (4.8%) | 0.00 | 675 (4.8%) | 663 (4.7%) | 0.00 | 1,132 (5.1%) | 1,065 (4.8%) | 0.01 | 1939 (5.0%) | 1863 (4.8%) | 0.01 |
| Anxiety; n (%) Sleep_Disorder; n (%) | 144 (5.2%)<br>267 (9.6%) | 141 (5.1%)<br>255 (9.1%) | 0.00<br>0.02 | 545 (3.9%)<br>1,617 (11.6%) | 540 (3.9%)<br>1,579 (11.3%) | 0.00<br>0.01 | 1,013 (4.5%)<br>1,438 (6.4%) | 973 (4.4%)<br>1,405 (6.3%) | 0.00 | 1702 (4.4%)<br>3322 (8.5%) | 1654 (4.2%)<br>3239 (8.3%) | 0.01<br>0.01 |
| Dementia; n (%) | 117 (4.2%) | 106 (3.8%) | 0.02 | 466 (3.3%) | 469 (3.4%) | -0.01 | 822 (3.7%) | 843 (3.8%) | -0.01 | 1405 (3.6%) | 1418 (3.6%) | 0.00 |
| Delirium; n (%) | 21 (0.8%) | 15 (0.5%) | 0.04 | 110 (0.8%) | 121 (0.9%) | -0.01 | 135 (0.6%) | 133 (0.6%) | 0.00 | 266 (0.7%) | 269 (0.7%) | 0.00 |
| Psychosis; n (%) | 9 (0.3%) | 12 (0.4%) | -0.02 | 100 (0.7%) | 102 (0.7%) | 0.00 | 168 (0.8%) | 150 (0.7%) | 0.01 | 277 (0.7%) | 264 (0.7%) | 0.00 |
| Obesity; n (%) | 273 (9.8%) | 266 (9.5%) | 0.01 | 1,009 (7.2%) | 980 (7.0%) | 0.01 | 2,080 (9.3%) | 2,050 (9.2%) | 0.00 | 3362 (8.6%) | 3296 (8.4%) | 0.01 |
| Overweight; n (%) | 79 (2.8%) | 79 (2.8%) | 0.00 | 102 (0.7%) | 92 (0.7%) | 0.00 | 424 (1.9%) | 405 (1.8%) | 0.01 | 605 (1.5%) | 576 (1.5%) | 0.00 |
| Smoking; n (%) Alcohol abuse or dependence; n (%) | 230 (8.2%) | 213 (7.6%)<br>0 (0.0%) | 0.02<br>#DIV/0! | 743 (5.3%)<br>0 (0.0%) | 741 (5.3%)<br>0 (0.0%) | 0.00<br>#DIV/0! | 3,157 (14.1%)<br>0 (0.0%) | 3,046 (13.6%)<br>0 (0.0%) | 0.01<br>#DIV/0! | 4130 (10.6%)<br>0 (0.0%) | 4000 (10.2%)<br>0 (0.0%) | 0.01<br>#DIV/0! |
| Drug abuse or dependence; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| COPD; n (%) | 295 (10.6%) | 294 (10.5%) | 0.00 | 1.844 (13.2%) | 1.797 (12.9%) | 0.01 | 2.146 (9.6%) | 2.079 (9.3%) | 0.01 | 4285 (11.0%) | 4170 (10.7%) | 0.01 |
| Asthma; n (%) | 127 (4.6%) | 130 (4.7%) | 0.00 | 754 (5.4%) | 749 (5.4%) | 0.00 | 917 (4.1%) | 881 (3.9%) | 0.01 | 1798 (4.6%) | 1760 (4.5%) | 0.00 |
| Obstructive sleep apnea; n (%) | 270 (9.7%) | 242 (8.7%) | 0.03 | 1,345 (9.6%) | 1,319 (9.4%) | 0.01 | 1,262 (5.7%) | 1,225 (5.5%) | 0.01 | 2877 (7.4%) | 2786 (7.1%) | 0.01 |
| Pneumonia; n (%) | 33 (1.2%) | 45 (1.6%) | -0.03 | 833 (6.0%) | 848 (6.1%) | 0.00 | 772 (3.5%) | 783 (3.5%) | 0.00 | 1638 (4.2%) | 1676 (4.3%) | 0.00 |
| Imaging; n (%) Other Medications | 0 (0.0%) | 1 (0.0%) | #DIV/0! | 25 (0.2%) | 17 (0.1%) | 0.03 | 26 (0.1%) | 30 (0.1%) | 0.00 | 51 (0.1%) | 48 (0.1%) | 0.00 |
| Use of ACE inhibitors; n (%) | 961 (34.4%) | 951 (34.1%) | 0.01 | 4,940 (35.4%) | 4,936 (35.4%) | 0.00 | 7,744 (34.7%) | 7,830 (35.1%) | -0.01 | 13645 (34.9%) | 13717 (35.1%) | 0.00 |
| Use of ARBs; n (%) | 543 (19.5%) | 542 (19.4%) | 0.00 | 3,304 (23,7%) | 3,285 (23.5%) | 0.00 | 4,971 (22.3%) | 4,922 (22.1%) | 0.00 | 8818 (22.6%) | 8749 (22.4%) | 0.00 |
| Use of Loop Diuretics - United; n (%) | 467 (16.7%) | 464 (16.6%) | 0.00 | 3,441 (24.6%) | 3,280 (23.5%) | 0.03 | 4,396 (19.7%) | 4,390 (19.7%) | 0.00 | 8304 (21.3%) | 8134 (20.8%) | 0.01 |
| Use of other diuretics- United; n (%) | 80 (2.9%) | 84 (3.0%) | -0.01 | 716 (5.1%) | 693 (5.0%) | 0.00 | 727 (3.3%) | 771 (3.5%) | -0.01 | 1523 (3.9%) | 1548 (4.0%) | -0.01 |
| Use of nitrates-United; n (%) | 170 (6.1%) | 137 (4.9%) | 0.05 | 1,278 (9.2%) | 1,156 (8.3%) | 0.03 | 1,979 (8.9%) | 1,698 (7.6%) | 0.05 | 3427 (8.8%) | 2991 (7.7%) | 0.04 |
| Use of other hypertension drugs; n (%) | 225 (8.1%)<br>319 (11.4%) | 220 (7.9%)<br>302 (10.8%) | 0.01 | 904 (6.5%)<br>2,692 (19.3%) | 997 (7.1%)<br>2,018 (14.5%) | -0.02<br>0.13 | 1,616 (7.2%)<br>2,933 (13.1%) | 1,612 (7.2%)<br>2,579 (11.6%) | 0.00 | 2745 (7.0%)<br>5944 (15.2%) | 2829 (7.2%) | -0.01<br>0.08 |
| Use of digoxin- United; n (%) Use of Anti-arrhythmics; n (%) | 395 (14.2%) | 406 (14.6%) | -0.02 | 2,766 (19.8%) | 2,652 (19.0%) | 0.13 | 3,619 (16.2%) | 3,526 (15.8%) | 0.05 | 6780 (17.4%) | 4899 (12.5%)<br>6584 (16.9%) | 0.08 |
| Use of COPD/asthma meds- United; n (%) | 436 (15.6%) | 410 (14.7%) | 0.03 | 2,621 (18.8%) | 2,717 (19.5%) | -0.02 | 3,827 (17.1%) | 3,626 (16.2%) | 0.02 | 6884 (17.6%) | 6753 (17.3%) | 0.01 |
| Use of statins; n (%) | 1,516 (54.3%) | 1,505 (53.9%) | 0.01 | 7,744 (55.5%) | 7,735 (55.4%) | 0.00 | 12,406 (55.6%) | 12,391 (55.5%) | 0.00 | 21666 (55.5%) | 21631 (55.4%) | 0.00 |
| Use of other lipid-lowering drugs; n (%) | 228 (8.2%) | 203 (7.3%) | 0.03 | 1,425 (10.2%) | 1,428 (10.2%) | 0.00 | 1,695 (7.6%) | 1,671 (7.5%) | 0.00 | 3348 (8.6%) | 3302 (8.5%) | 0.00 |
| Use of antiplatelet agents; n (%) | 261 (9.4%) | 258 (9.2%) | 0.01 | 2,273 (16.3%) | 2,255 (16.2%) | 0.00 | 2,842 (12.7%) | 2,828 (12.7%) | 0.00 | 5376 (13.8%) | 5341 (13.7%) | 0.00 |
| Use of heparin and other low-molecular weight heparins: n (%) | 10 (0.4%) | 11 (0.4%) | 0.00 | 1 (0.0%) | 2 (0.0%) | #DIV/01 | 113 (0.5%) | 125 (0.6%) | -0.01 | 124 (0.3%) | 138 (0.4%) | -0.02 |
| Use of NSAIDs; n (%) | 284 (10.2%) | 269 (9.6%) | 0.00 | 1.482 (10.6%) | 1,438 (10.3%) | #DIV/0!<br>0.01 | 2,600 (11.6%) | 2,593 (11.6%) | 0.00 | 4366 (11.2%) | 4300 (11.0%) | 0.02 |
| Use of oral corticosteroids; n (%) | 443 (15.9%) | 443 (15.9%) | 0.00 | 2,669 (19.1%) | 2,624 (18.8%) | 0.01 | 4,130 (18.5%) | 4,126 (18.5%) | 0.00 | 7242 (18.5%) | 7193 (18.4%) | 0.00 |
| Use of bisphosphonate (United); n (%) | 85 (3.0%) | 102 (3.7%) | -0.04 | 671 (4.8%) | 644 (4.6%) | 0.01 | 894 (4.0%) | 892 (4.0%) | 0.00 | 1650 (4.2%) | 1638 (4.2%) | 0.00 |
| Use of opioids- United; n (%) | 534 (19.1%) | 536 (19.2%) | 0.00 | 3,392 (24.3%) | 3,321 (23.8%) | 0.01 | 5,044 (22.6%) | 4,995 (22.4%) | 0.00 | 8970 (23.0%) | 8852 (22.7%) | 0.01 |
| Use of antidepressants; n (%) | 452 (16.2%) | 448 (16.1%) | 0.00 | 2,414 (17.3%) | 2,392 (17.1%) | 0.01 | 4,003 (17.9%) | 3,947 (17.7%) | 0.01 | 6869 (17.6%) | 6787 (17.4%) | 0.01 |
| Use of antipsychotics; n (%) | 23 (0.8%) | 23 (0.8%) | 0.00 | 158 (1.1%) | 158 (1.1%) | 0.00 | 337 (1.5%) | 349 (1.6%) | -0.01 | 518 (1.3%) | 530 (1.4%) | -0.01 |
| Use of anticonvulsants; n (%) Use of lithium-United: n (%) | 262 (9.4%)<br>3 (0.1%) | 232 (8.3%)<br>3 (0.1%) | 0.04 | 1,177 (8.4%)<br>12 (0.1%) | 1,202 (8.6%)<br>13 (0.1%) | -0.01<br>0.00 | 2,161 (9.7%)<br>11 (0.0%) | 2,125 (9.5%)<br>19 (0.1%) | 0.01<br>-0.04 | 3600 (9.2%)<br>26 (0.1%) | 3559 (9.1%)<br>35 (0.1%) | 0.00 |
| Use of Benzos- United: n (%) | 177 (6.3%) | 186 (6.7%) | -0.02 | 1.811 (13.0%) | 1.800 (12.9%) | 0.00 | 1.595 (7.1%) | 1.599 (7.2%) | 0.00 | 3583 (9.2%) | 35 (0.1%) | 0.00 |
| Use of anxiolytics/hypnotics-United; n (%) | 167 (6.0%) | 165 (5.9%) | 0.00 | 1,000 (7.2%) | 984 (7.0%) | 0.01 | 1,478 (6.6%) | 1,447 (6.5%) | 0.00 | 2645 (6.8%) | 2596 (6.6%) | 0.01 |
| Use of dementia meds- United; n (%) | 103 (3.7%) | 94 (3.4%) | 0.02 | 447 (3.2%) | 458 (3.3%) | -0.01 | 856 (3.8%) | 821 (3.7%) | 0.01 | 1406 (3.6%) | 1373 (3.5%) | 0.01 |
| Use of antiparkinsonian meds- United; n (%) | 41 (1.5%) | 42 (1.5%) | 0.00 | 345 (2.5%) | 349 (2.5%) | 0.00 | 623 (2.8%) | 604 (2.7%) | 0.01 | 1009 (2.6%) | 995 (2.5%) | 0.01 |
| Any use of pramlintide; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 3 (0.0%) | 7 (0.1%) | -0.04 | ** | ** | #VALUE! | #VALUE! | #VALUE! | #VALUE! |

| Any use of 1st generation sulfonylureas; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 6 (0.0%) | 5 (0.0%) | #DIV/0! | ** | ** | #VALUE! | #VALUE! | #VALUE! | 0.00 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Entresto (sacubitril/valsartan); n (%) | 6 (0.2%) | 3 (0.1%) | 0.03 | 7 (0.1%) | 1 (0.0%) | 0.04 | ** | ** | #VALUE! | #VALUE! | #VALUE! | 0.00 |
| Labs | | | | | | | | | | 16,750 | 16,750 | |
| Lab values- HbA1c (%) v3: n (%) | 319 (11.4%) | 309 (11.1%) | 0.01 | 113 (0.8%) | 94 (0.7%) | 0.01 | N/A | N/A | #VALUE! | 432 (2.6%) | 403 (2.4%) | 0.01 |
| Lab values- HbA1c (%) (within 3 months) v3; n (%) | 205 (7.3%) | 202 (7.2%) | 0.00 | 87 (0.6%) | 61 (0.4%) | 0.03 | N/A | N/A | #VALUE! | 292 (1.7%) | 263 (1.6%) | 0.01 |
| Lab values- HbA1c (%) (within 6 months) v3; n (%) | 319 (11.4%) | 309 (11.1%) | 0.01 | 113 (0.8%) | 94 (0.7%) | 0.01 | N/A | N/A | #VALUE! | 432 (2.6%) | 403 (2.4%) | 0.01 |
| Lab values- BNP; n (%) | 27 (1.0%) | 28 (1.0%) | 0.00 | 10 (0.1%) | 17 (0.1%) | 0.00 | N/A | N/A | #VALUE! | 37 (0.2%) | 45 (0.3%) | -0.02 |
| Lab values- BNP (within 3 months); n (%) | 23 (0.8%) | | -0.01 | 8 (0.1%) | | 0.00 | N/A<br>N/A | N/A | #VALUE! | 31 (0.2%) | 38 (0.2%) | 0.02 |
| | | 24 (0.9%) | | | 14 (0.1%) | | | | | | | |
| Lab values- BNP (within 6 months); n (%) | 27 (1.0%) | 28 (1.0%) | 0.00 | 10 (0.1%) | 17 (0.1%) | 0.00 | N/A | N/A | #VALUE! | 37 (0.2%) | 45 (0.3%) | -0.02 |
| Lab values- BUN (mg/dl); n (%) | 604 (21.6%) | 673 (24.1%) | -0.06 | 111 (0.8%) | 144 (1.0%) | -0.02 | N/A | N/A | #VALUE! | 715 (4.3%) | 817 (4.9%) | -0.03 |
| Lab values- BUN (mg/dl) (within 3 months); n (%) | 421 (15.1%) | 456 (16.3%) | -0.03 | 83 (0.6%) | 105 (0.8%) | -0.02 | N/A | N/A | #VALUE! | 504 (3.0%) | 561 (3.3%) | -0.02 |
| Lab values- BUN (mg/dl) (within 6 months); n (%) | 604 (21.6%) | 673 (24.1%) | -0.06 | 111 (0.8%) | 144 (1.0%) | -0.02 | N/A | N/A | #VALUE! | 715 (4.3%) | 817 (4.9%) | -0.03 |
| Lab values- Creatinine (mg/dl) v2; n (%) | 614 (22.0%) | 686 (24.6%) | -0.06 | 111 (0.8%) | 159 (1.1%) | -0.03 | N/A | N/A | #VALUE! | 725 (4.3%) | 845 (5.0%) | -0.03 |
| Lab values- Creatinine (mg/dl) (within 3 months) v2; | | | | | | | | | | | | |
| n (%) | 427 (15.3%) | 465 (16.7%) | -0.04 | 82 (0.6%) | 112 (0.8%) | -0.02 | N/A | N/A | #VALUE! | 509 (3.0%) | 577 (3.4%) | -0.02 |
| Lab values- Creatinine (mg/dl) (within 6 months) v2; | | | | | ***** | | | | | | | |
| n (%) | 614 (22.0%) | 686 (24.6%) | -0.06 | 111 (0.8%) | 159 (1.1%) | -0.03 | N/A | N/A | #VALUE! | 725 (4.3%) | 845 (5.0%) | -0.03 |
| Lab values- HDL level (mg/dl); n (%) | 464 (16.6%) | 500 (17.9%) | -0.03 | 94 (0.7%) | 106 (0.8%) | -0.01 | N/A | N/A | #VALUE! | 558 (3.3%) | 606 (3.6%) | -0.02 |
| tab values institute (ing/ai/, ii (/a/ | 404 (10.0%) | 300 (17.370) | 0.03 | 34 (0.770) | 100 (0.0%) | 0.01 | 147. | 14,71 | WWW.COL. | 330 (3.3%) | 000 (5.0%) | 0.02 |
| Lab values- HDL level (mg/dl) (within 3 months); n (% | 6) 291 (10.4%) | 320 (11.5%) | -0.04 | 70 (0.5%) | 68 (0.5%) | 0.00 | N/A | N/A | #VALUE! | 361 (2.2%) | 388 (2.3%) | -0.01 |
| Lab values- HDL level (mg/di) (within 3 months); n (% | 6) 291 (10.4%) | 320 (11.5%) | -0.04 | 70 (0.5%) | 68 (0.5%) | 0.00 | N/A | N/A | #VALUE! | 301 (2.2%) | 388 (2.3%) | -0.01 |
| | | 500 (47 00) | | 0.4 (0.70) | 405 (0.00) | | *** | | | 550 (2.20) | 505 (2.50) | |
| Lab values- HDL level (mg/dl) (within 6 months); n (% | | 500 (17.9%) | -0.03 | 94 (0.7%) | 106 (0.8%) | -0.01 | N/A | N/A | #VALUE! | 558 (3.3%) | 606 (3.6%) | -0.02 |
| Lab values- LDL level (mg/dl) v2; n (%) | 487 (17.5%) | 527 (18.9%) | -0.04 | 117 (0.8%) | 115 (0.8%) | 0.00 | N/A | N/A | #VALUE! | 604 (3.6%) | 642 (3.8%) | -0.01 |
| Lab values- LDL level (mg/dl) (within 3 months) v2; n | | | | | | | | | | | | |
| (%) | 305 (10.9%) | 338 (12.1%) | -0.04 | 88 (0.6%) | 74 (0.5%) | 0.01 | N/A | N/A | #VALUE! | 393 (2.3%) | 412 (2.5%) | -0.01 |
| Lab values- LDL level (mg/dl) (within 6 months) v2; n | | | | | | | | | | | | |
| (%) | 487 (17.5%) | 527 (18.9%) | -0.04 | 117 (0.8%) | 115 (0.8%) | 0.00 | N/A | N/A | #VALUE! | 604 (3.6%) | 642 (3.8%) | -0.01 |
| Lab values- NT-proBNP; n (%) | 4 (0.1%) | 1 (0.0%) | 0.04 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | 04 (0.0%) | 1 (0.0%) | #DIV/0! |
| Lab values- NT-proBNP (within 3 months); n (%) | 3 (0.1%) | 0 (0.0%) | 0.04 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | 03 (0.0%) | 0 (0.0%) | - |
| Lab values- NT-proBNP (within 6 months); n (%) | 4 (0.1%) | 1 (0.0%) | 0.04 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | 04 (0.0%) | 1 (0.0%) | |
| Lab values- Total cholesterol (mg/dl) v2; n (%) | 467 (16.7%) | 508 (18.2%) | -0.04 | 95 (0.7%) | 117 (0.8%) | -0.01 | N/A | N/A | #VALUE! | 562 (3.4%) | 625 (3.7%) | -0.02 |
| Lab values- Total cholesterol (mg/dl) (within 3 | 407 (10.7%) | 500 (10.270) | -0.04 | 33 (0.7%) | 117 (0.070) | -0.01 | 19/6 | 14/15 | WALOE: | 302 (3.470) | 023 (3.7%) | -0.02 |
| months) v2; n (%) | 294 (10.5%) | 325 (11.6%) | -0.04 | 70 (0.5%) | 73 (0.5%) | 0.00 | N/A | N/A | #VALUE! | 364 (2.2%) | 398 (2.4%) | -0.01 |
| | 294 (10.5%) | 323 (11.0%) | -0.04 | 70 (0.5%) | 73 (0.5%) | 0.00 | N/A | N/A | #VALUE: | 304 (2.2%) | 350 (2.4%) | -0.01 |
| Lab values- Total cholesterol (mg/dl) (within 6 | 467.46.700 | 500 (40 00) | | 05 (0 70) | 117 (0.8%) | | *** | | | 552 (2.40) | 505 (0.70) | |
| months) v2; n (%) | 467 (16.7%) | 508 (18.2%) | -0.04 | 95 (0.7%) | () | -0.01 | N/A | N/A | #VALUE! | 562 (3.4%) | 625 (3.7%) | -0.02 |
| Lab values- Triglyceride level (mg/dl); n (%) | 464 (16.6%) | 503 (18.0%) | -0.04 | 94 (0.7%) | 107 (0.8%) | -0.01 | N/A | N/A | #VALUE! | 558 (3.3%) | 610 (3.6%) | -0.02 |
| Lab values- Triglyceride level (mg/dl) (within 3 | | | | | | | | | | | | |
| months); n (%) | 291 (10.4%) | 322 (11.5%) | -0.04 | 71 (0.5%) | 68 (0.5%) | 0.00 | N/A | N/A | #VALUE! | 362 (2.2%) | 390 (2.3%) | -0.01 |
| Lab values- Triglyceride level (mg/dl) (within 6 | | | | | | | | | | | | |
| months); n (%) | 464 (16.6%) | 503 (18.0%) | -0.04 | 94 (0.7%) | 107 (0.8%) | -0.01 | N/A | N/A | #VALUE! | 558 (3.3%) | 610 (3.6%) | -0.02 |
| Lab result number- HbA1c (%) mean (only 2 to 20 | | | | | | | | | | | | |
| included) v4 | 315 | 307 | | 100 | 87 | | N/A | N/A | | 415 | 394 | |
| mean (sd) | 6.57 (1.13) | 6.54 (1.37) | 0.02 | 7.01 (1.41) | 6.75 (1.08) | 0.21 | N/A | N/A | #VALUE! | 6.68 (1.20) | 6.59 (1.31) | 0.07 |
| median [IQR] | 6.20 [5.80, 7.00] | 6.30 [5.80, 7.00] | -0.08 | 6.60 [6.10, 7.77] | 6.50 [6.00, 7.25] | 0.08 | N/A | N/A | #VALUE! | 6.30 (1.20) | 6.34 (1.31) | -0.03 |
| Missing; n (%) | 2,475 (88.7%) | 2,483 (89.0%) | -0.01 | 13,860 (99.3%) | 13,873 (99.4%) | -0.01 | N/A | N/A | #VALUE! | 16,335 (97.5%) | 16,356 (97.6%) | -0.01 |
| Lab result number- BNP mean v2 | 2,473 (88.7%) | 2,463 (63.0%) | -0.01 | 10,000 (33.3%) | 13,873 (33.478) | -0.01 | N/A | N/A | WALOE: | 37 | 10,330 (37.0%) | -0.01 |
| | | 20 | | | | | , | | | | | 0.00 |
| mean (sd) | 358.65 (541.48) | 214.33 (164.51) | 0.36 | 217.51 (147.78) | 180.30 (209.53) | 0.21 | N/A | N/A | #VALUE! | 320.50 (479.58) | 201.47 (184.72) | 0.33 |
| median [IQR] | 216.30 [103.00, 361.00] | 170.15 [69.72, 343.75] | 0.12 | 233.50 [71.50, 328.00] | 121.00 [59.00, 245.00] | 0.62 | N/A | N/A | #VALUE! | 220.95 (479.58) | 151.58 (184.72) | 0.19 |
| Missing; n (%) | 2,763 (99.0%) | 2,762 (99.0%) | 0.00 | 13,950 (99.9%) | 13,943 (99.9%) | 0.00 | N/A | N/A | #VALUE! | 16,713 (99.8%) | 16,705 (99.7%) | 0.02 |
| Lab result number- BUN (mg/dl) mean v2 | 604 | 673 | | 111 | 144 | | N/A | N/A | | 715 | 817 | |
| mean (sd) | 17.89 (5.80) | 17.74 (5.21) | 0.03 | 17.65 (5.69) | 18.46 (5.89) | -0.14 | N/A | N/A | #VALUE! | 17.85 (5.79) | 17.87 (5.34) | 0.00 |
| median [IQR] | 17.50 [14.00, 21.00] | 17.00 [14.00, 21.00] | 0.09 | 17.00 [14.00, 21.00] | 18.00 [15.00, 22.00] | -0.17 | N/A | N/A | #VALUE! | 17.42 (5.79) | 17.18 (5.34) | 0.04 |
| Missing; n (%) | 2,186 (78.4%) | 2,117 (75.9%) | 0.06 | 13,849 (99.2%) | 13,816 (99.0%) | 0.02 | N/A | N/A | #VALUE! | 16,035 (95.7%) | 15,933 (95.1%) | 0.03 |
| Lab result number- Creatinine (mg/dl) mean (only 0. | 1 | | | | | | | | | | | |
| to 15 included) v3 | 607 | 682 | | 110 | 157 | | N/A | N/A | | 717 | 839 | |
| mean (sd) | 0.98 (0.25) | 0.98 (0.21) | 0.00 | 0.98 (0.22) | 0.98 (0.24) | 0.00 | N/A | N/A | #VALUE! | 0.98 (0.25) | 0.98 (0.22) | 0.00 |
| median [IQR] | 0.95 [0.82, 1.10] | 0.96 [0.83, 1.10] | -0.04 | 0.96 [0.81, 1.10] | 0.94 [0.80, 1.10] | 0.09 | N/A | N/A | #VALUE! | 0.95 (0.25) | 0.96 (0.22) | -0.04 |
| Missing; n (%) | 2,183 (78.2%) | 2,108 (75.6%) | 0.04 | 13,850 (99.2%) | 13,803 (98.9%) | 0.03 | N/A<br>N/A | N/A<br>N/A | #VALUE! | 16,033 (95.7%) | 15,911 (95.0%) | 0.04 |
| Missing; n (%)<br>Lab result number- HDL level (mg/dl) mean (only | 2,103 (/0.2%) | 2,100 (/3.0%) | 0.06 | 13,030 (33.270) | 13,003 (30.3%) | 0.05 | IN/M | N/A | #VALUE! | 10,033 (33.770) | 13,311 (33.070) | 0.05 |
| | 464 | 500 | | 94 | 106 | | 11/4 | N1/A | | 558 | 606 | |
| =<5000 included) v2 | | | | | | 0.10 | N/A | N/A | 40.44 | | | |
| mean (sd) | 51.27 (15.97) | 52.85 (17.18) | -0.10 | 45.87 (15.62) | 48.01 (17.14) | -0.13 | N/A | N/A | #VALUE! | 50.36 (15.93) | 52.00 (17.19) | -0.10 |
| median [IQR] | 48.25 [40.00, 60.00] | 50.00 [41.00, 62.00] | -0.11 | 45.50 [34.00, 54.12] | 47.50 [35.75, 59.25] | -0.12 | N/A | N/A | #VALUE! | 47.79 (15.93) | 49.56 (17.19) | -0.11 |
| Missing; n (%) | 2,326 (83.4%) | 2,290 (82.1%) | 0.03 | 13,866 (99.3%) | 13,854 (99.2%) | 0.01 | N/A | N/A | #VALUE! | 16,192 (96.7%) | 16,144 (96.4%) | 0.02 |
| Lab result number- LDL level (mg/dl) mean (only | | | | | | | | | | | | |
| =<5000 included) v2 | 472 | 512 | | 95 | 110 | | N/A | N/A | | 567 | 622 | |
| mean (sd) | 89.15 (32.99) | 87.59 (33.46) | 0.05 | 82.89 (29.91) | 79.99 (36.33) | 0.09 | N/A | N/A | #VALUE! | 88.10 (32.53) | 86.25 (34.01) | 0.06 |
| median [IQR] | 84.83 [68.50, 108.00] | 82.00 [66.00, 109.00] | 0.09 | 80.00 [64.50, 101.00] | 79.25 [57.38, 101.25] | 0.02 | N/A | N/A | #VALUE! | 84.02 (32.53) | 81.51 (34.01) | 0.08 |
| Missing; n (%) | 2,318 (83.1%) | 2,278 (81.6%) | 0.04 | 13,865 (99.3%) | 13,850 (99.2%) | 0.01 | N/A | N/A | #VALUE! | 16,183 (96.6%) | 16,128 (96.3%) | 0.02 |
| Lab result number- Total cholesterol (mg/dl) mean | , ()0/ | , () | | -,() | , (/0) | | *** | | | ., () | ., () | |
| (only =<5000 included) v2 | 467 | 508 | | 95 | 117 | | N/A | N/A | | 562 | 625 | |
| | 166.51 (40.78) | 165.12 (40.18) | 0.03 | 154.47 (33.16) | 157.68 (41.05) | -0.09 | N/A<br>N/A | N/A | #VALUE! | 164.47 (39.64) | 163.73 (40.38) | 0.02 |
| mean (cd) | 162.00 [139.00, 192.00] | | | 154.47 (33.16) | | -0.09 | N/A<br>N/A | N/A<br>N/A | #VALUE! | 164.47 (39.64) | 153.73 (40.38) | 0.02 |
| mean (sd) | | 159.00 [138.00, 192.00] | | | 159.00 [136.00, 181.75] | | | , | | | | |
| median [IQR] | | | 0.04 | 13,865 (99.3%) | 13,843 (99.2%) | 0.01 | N/A | N/A | #VALUE! | 16,188 (96.6%) | 16,125 (96.3%) | 0.02 |
| median [IQR]<br>Missing; n (%) | 2,323 (83.3%) | 2,282 (81.8%) | | | | | | | | | | |
| median [IQR]<br>Missing; n (%)<br>Lab result number-Triglyceride level (mg/dl) mean | 2,323 (83.3%) | , . , , | | _ | | | *** | | | | | |
| median [IQR]Missing; n (%) Lab result number-Triglyceride level (mg/dl) mean (only =<5000 included) v2 | 2,323 (83.3%)<br>464 | 503 | | 94 | 107 | | N/A | N/A | | 558 | 610 | |
| median [IQR]Missing; n (%) Lab result number-Triglyceride level (mg/dl) mean (only =<5000 included) v2mean (sd) | 2,323 (83.3%)<br>464<br>129.01 (76.77) | 503<br>119.47 (64.42) | 0.13 | 130.38 (67.84) | 144.37 (97.89) | -0.17 | N/A | N/A | #VALUE! | 129.24 (75.42) | 123.84 (71.45) | 0.07 |
| median [IQR]Missing; n (%) Lab result number-Triglyceride level (mg/dl) mean (only =<5000 included) v2 | 2,323 (83.3%)<br>464 | 503 | | | | -0.17<br>-0.14 | , | N/A<br>N/A | #VALUE! | | | 0.07<br>0.05 |
| median [IQR]Missing; n (%) Lab result number-Triglyceride level (mg/dl) mean (only =<5000 included) v2mean (sd) | 2,323 (83.3%) 464 129.01 (76.77) 112.00 [81.00, 151.38] | 503<br>119.47 (64.42) | 0.13 | 130.38 (67.84)<br>114.50 [81.38, 175.00] | 144.37 (97.89)<br>126.00 [91.00, 155.00] | | N/A | N/A | | 129.24 (75.42)<br>112.42 (75.42) | 123.84 (71.45)<br>108.68 (71.45) | |
| median [IQR]Missing; n (%) Lab result rumber-Triglyceride level (mg/dl) mean (only =<5000 included) v2mean (sd)median [IQR] | 2,323 (83.3%)<br>464<br>129.01 (76.77) | 503<br>119.47 (64.42)<br>105.00 [77.00, 144.00] | 0.13<br>0.10 | 130.38 (67.84) | 144.37 (97.89) | -0.14 | N/A<br>N/A | N/A<br>N/A | #VALUE! | 129.24 (75.42) | 123.84 (71.45) | 0.05 |
| median [IQR]Missing; n (%) Lab result number-Triglyceride level (mg/dl) mean (only ~5000 included) v2mean (sd)median [IQR]Missing; n (%) Lab result number-Hemoglobin mean (only >0 | 2,323 (83.3%) 464 129.01 (76.77) 112.00 [81.00, 151.38] | 503<br>119.47 (64.42)<br>105.00 [77.00, 144.00] | 0.13<br>0.10 | 130.38 (67.84)<br>114.50 [81.38, 175.00] | 144.37 (97.89)<br>126.00 [91.00, 155.00] | -0.14 | N/A<br>N/A | N/A<br>N/A | #VALUE! | 129.24 (75.42)<br>112.42 (75.42)<br>16,192 (96.7%) | 123.84 (71.45)<br>108.68 (71.45)<br>16,140 (96.4%) | 0.05 |
| median [IQR]Missing; n (%) Lab result number-Triglyceride level (mg/dl) mean (only =≤000 included) v2mean (sd)median [IQR]Missing; n (%) | 2,323 (83.3%) 464 129.01 (76.77) 112.00 [81.00, 151.38] 2,326 (83.4%) | 503<br>119.47 (64.42)<br>105.00 [77.00, 144.00]<br>2,287 (82.0%) | 0.13<br>0.10 | 130.38 (67.84)<br>114.50 [81.38, 175.00]<br>13,866 (99.3%) | 144.37 (97.89)<br>126.00 [91.00, 155.00]<br>13,853 (99.2%) | -0.14 | N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A | #VALUE! | 129.24 (75.42)<br>112.42 (75.42) | 123.84 (71.45)<br>108.68 (71.45) | 0.05 |
| median [IQR]Missing; n (%) Lab result number-Triglyceride level (mg/dl) mean (only <5000 included) v2mean (sd)median [IQR]Missing; n (%) Lab result number-Hemoglobin mean (only >0 included)mean (sd) | 2,323 (83.3%) 464 129.01 (76.77) 112.00 [81.00, 151.38] 2,326 (83.4%) 447 13.95 (1.46) | 503<br>119.47 (64.42)<br>105.00 [77.00, 144.00]<br>2,287 (82.0%)<br>494<br>14.06 (1.41) | 0.13<br>0.10<br>0.04 | 130.38 (67.84)<br>114.50 [81.38, 175.00]<br>13,866 (99.3%)<br>69<br>13.65 (1.51) | 144.37 (97.89)<br>126.00 [91.00, 155.00]<br>13,853 (99.2%)<br>99<br>13.64 (2.06) | -0.14<br>0.01 | N/A<br>N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A<br>N/A | #VALUE!<br>#VALUE! | 129.24 (75.42)<br>112.42 (75.42)<br>16,192 (96.7%)<br>516<br>13.91 (1.47) | 123.84 (71.45)<br>108.68 (71.45)<br>16,140 (96.4%)<br>593<br>13.99 (1.54) | 0.05<br>0.02 |
| median [IQR]Missing; n (%) Lab result number-Triglyceride level (mg/dl) mean (only <5000 included) v2mean (sd)median [IQR]Missing; n (%) Lab result number-Hemoglobin mean (only >0 included) | 2,323 (83.3%) 464 129.01 (76.77) 112.00 (81.00, 151.38) 2,326 (83.4%) | 503<br>119.47 (64.42)<br>105.00 [77.00, 144.00]<br>2,287 (82.0%) | 0.13<br>0.10<br>0.04 | 130.38 (67.84)<br>114.50 [81.38, 175.00]<br>13,866 (99.3%) | 144.37 (97.89)<br>126.00 [91.00, 155.00]<br>13,853 (99.2%) | -0.14<br>0.01 | N/A<br>N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A | #VALUE!<br>#VALUE! | 129.24 (75.42)<br>112.42 (75.42)<br>16,192 (96.7%) | 123.84 (71.45)<br>108.68 (71.45)<br>16,140 (96.4%) | 0.05<br>0.02 |

| Lab result number- Serum sodium mean (only > 90 | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| and < 190 included) | 579 | 654 | | 92 | 122 | | N/A | N/A | | 671 | 776 | |
| mean (sd) | 140.03 (2.74) | 140.11 (3.01) | -0.03 | 139.22 (2.71) | 139.28 (2.99) | -0.02 | N/A | N/A | #VALUE! | 139.92 (2.74) | 139.98 (3.01) | -0.02 |
| median [IQR] | 140.00 [138.50, 142.00] | 140.00 [139.00, 142.00] | | 139.80 [138.00, 141.00] | 139.83 [137.50, 141.00] | -0.01 | N/A | N/A | #VALUE! | 139.97 (2.74) | 139.97 (3.01) | 0.00 |
| Missing; n (%) | 2,211 (79.2%) | 2,136 (76.6%) | 0.06 | 13,868 (99.3%) | 13,838 (99.1%) | 0.02 | N/A | N/A | #VALUE! | 16,079 (96.0%) | 15,974 (95.4%) | 0.03 |
| Lab result number- Albumin mean (only >0 and <=10<br>included) | 530 | 601 | | 72 | 102 | | N/A | N/A | | 602 | 703 | |
| mean (sd) | 4.17 (0.31) | 4.19 (0.31) | -0.06 | 4.10 (0.58) | 4.03 (0.49) | 0.13 | N/A | N/A | #VALUE! | 4.16 (0.35) | 4.17 (0.34) | -0.03 |
| median [IQR] | 4.20 [4.00, 4.40] | 4.20 [4.00, 4.40] | 0.00 | 4.20 [3.90, 4.40] | 4.10 [3.89, 4.30] | 0.19 | N/A | N/A | #VALUE! | 4.20 (0.35) | 4.19 (0.34) | 0.03 |
| Missing; n (%) | 2,260 (81.0%) | 2,189 (78.5%) | 0.06 | 13,888 (99.5%) | 13,858 (99.3%) | 0.03 | N/A | N/A | #VALUE! | 16,148 (96.4%) | 16,047 (95.8%) | 0.03 |
| Lab result number- Glucose (fasting or random) mean | | | | | | | | | | | | |
| (only 10-1000 included) | 576 | 645 | | 91 | 111 | | N/A | N/A | | 667 | 756 | |
| mean (sd) | 110.45 (33.39) | 111.79 (39.37) | -0.04 | 139.94 (58.19) | 128.83 (44.07) | 0.22 | N/A | N/A | #VALUE! | 114.47 (37.74) | 114.29 (40.12) | 0.00 |
| median [IQR] | 101.00 [91.00, 118.88] | 100.50 [91.00, 117.00] | 0.01 | 122.00 [96.75, 162.50] | 117.00 [102.00, 140.00] | 0.10 | N/A | N/A | #VALUE! | 103.87 (37.74) | 102.92 (40.12) | 0.02 |
| Missing; n (%) | 2,214 (79.4%) | 2,145 (76.9%) | 0.06 | 13,869 (99.3%) | 13,849 (99.2%) | 0.01 | N/A | N/A | #VALUE! | 16,083 (96.0%) | 15,994 (95.5%) | 0.02 |
| Lab result number- Potassium mean (only 1-7<br>included) | 603 | 679 | | 108 | 143 | | N/A | N/A | | 711 | 822 | |
| mean (sd) | 4.35 (0.43) | 4.38 (0.44) | -0.07 | 4.35 (0.37) | 4.34 (0.38) | 0.03 | N/A | N/A | #VALUE! | 4.35 (0.42) | 4.37 (0.43) | -0.05 |
| median [IQR] | 4.30 [4.10, 4.60] | 4.40 [4.10, 4.65] | -0.23 | 4.30 [4.10, 4.60] | 4.36 [4.10, 4.60] | -0.16 | N/A | N/A | #VALUE! | 4.30 (0.42) | 4.39 (0.43) | -0.21 |
| Missing; n (%) | 2,187 (78.4%) | 2,111 (75.7%) | 0.06 | 13,852 (99.2%) | 13,817 (99.0%) | 0.02 | N/A | N/A | #VALUE! | 16,039 (95.8%) | 15,928 (95.1%) | 0.03 |
| Comorbidity Scores | | | | | | | | | | | | |
| CCI (180 days)-ICD9 and ICD10 v2 | | | | | | | | | | | | |
| mean (sd) | 2.63 (1.40) | 2.62 (1.35) | 0.01 | 2.81 (1.57) | 2.78 (1.56) | 0.02 | 1.33 (1.37) | 1.33 (1.39) | 0.00 | 1.95 (1.45) | 1.94 (1.45) | 0.01 |
| median [IQR] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 0.00 | 2.00 [2.00, 4.00] | 2.00 [2.00, 4.00] | 0.00 | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.00 | 1.43 (1.45) | 1.43 (1.45) | 0.00 |
| Non-Frailty; n (%) | 1,525 (54.7%) | 1,532 (54.9%) | 0.00 | 6,845 (49.0%) | 6,801 (48.7%) | 0.01 | 669 (3.0%) | 465 (2.1%) | 0.06 | 9,039 (23.1%) | 8,798 (22.5%) | 0.01 |
| Frailty Score (mean): Empirical Version 365 days, v2mean (sd) | 0.17 (0.04) | 0.17 (0.04) | 0.00 | 0.17 (0.05) | 0.17 (0.05) | 0.00 | 10.70 (9.15) | 10.66 (9.45) | 0.00 | 6.19 (6.92) | 6.16 (7.14) | 0.00 |
| median [IQR] | 0.16 [0.14, 0.19] | 0.16 [0.14, 0.19] | 0.00 | 0.17 [0.14, 0.20] | 0.17 [0.14, 0.20] | 0.00 | 8.94 [4.50, 14.92] | 8.82 [4.32, 14.85] | 0.01 | 5.18 (6.92) | 5.11 (7.14) | 0.01 |
| Healthcare Utilization | 0.10 (0.14, 0.15) | 0.10 [0.14, 0.15] | 0.00 | 0.17 [0.14, 0.20] | 0.17 [0.14, 0.10] | 0.00 | 0.54 [4.50, 14.52] | 0.02 [4.32, 14.03] | 0.01 | 3.10 (0.32) | 3.22(7.24) | 0.01 |
| Any hospitalization; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 4,495 (32.2%) | 4,381 (31.4%) | 0.02 | 4,193 (18.8%) | 4,147 (18.6%) | 0.01 | 8,688 (22.2%) | 8,528 (21.8%) | 0.01 |
| Any hospitalization within prior 30 days; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 3,098 (22.2%) | 2,998 (21.5%) | 0.02 | 2,640 (11.8%) | 2,607 (11.7%) | 0.00 | 5738 (14.7%) | 5605 (14.3%) | 0.01 |
| Any hospitalization during prior 31-180 days; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 1,606 (11.5%) | 1,567 (11.2%) | 0.01 | 1,741 (7.8%) | 1,691 (7.6%) | 0.01 | 3347 (8.6%) | 3258 (8.3%) | 0.01 |
| Endocrinologist Visit; n (%) | 67 (2.4%) | 77 (2.8%) | -0.03 | 474 (3.4%) | 451 (3.2%) | 0.01 | 783 (3.5%) | 731 (3.3%) | 0.01 | 1324 (3.4%) | 1259 (3.2%) | 0.01 |
| Endocrinologist Visit (30 days prior); n (%) | 24 (0.9%) | 19 (0.7%) | 0.02 | 165 (1.2%) | 156 (1.1%) | 0.01 | 233 (1.0%) | 222 (1.0%) | 0.00 | 422 (1.1%) | 397 (1.0%) | 0.01 |
| Endocrinologist Visit (31 to 180 days prior); n (%) | 56 (2.0%) | 66 (2.4%) | -0.03 | 395 (2.8%) | 374 (2.7%) | 0.01 | 669 (3.0%) | 636 (2.8%) | 0.01 | 1120 (2.9%) | 1076 (2.8%) | 0.01 |
| Internal medicine/family medicine visits; n (%)<br>Internal medicine/family medicine visits (30 days | 2,317 (83.0%) | 2,336 (83.7%) | -0.02 | 11,221 (80.4%) | 11,040 (79.1%) | 0.03 | 17,647 (79.1%) | 17,982 (80.6%) | -0.04 | 31185 (79.8%) | 31358 (80.3%) | -0.01 |
| prior) v2: n (%) | 1,469 (52.7%) | 1.468 (52.6%) | 0.00 | 7.381 (52.9%) | 7.282 (52.2%) | 0.01 | 11.348 (50.8%) | 11.109 (49.8%) | 0.02 | 20198 (51.7%) | 19859 (50.8%) | 0.02 |
| Internal medicine/family medicine visits (31 to 180 | 1,403 (32.770) | 1,400 (32.070) | 0.00 | 7,501 (52.570) | 7,202 (32.270) | 0.01 | 11,540 (50.070) | 11,105 (45.676) | 0.02 | 20130 (31.770) | 13033 (30.0%) | 0.02 |
| days prior) v2; n (%) | 2,048 (73.4%) | 2,033 (72.9%) | 0.01 | 9,897 (70.9%) | 9,621 (68.9%) | 0.04 | 14,888 (66.7%) | 15,277 (68.4%) | -0.04 | 26833 (68.7%) | 26931 (68.9%) | 0.00 |
| Cardiologist visit; n (%) | 1,715 (61.5%) | 1,844 (66.1%) | -0.10 | 8,643 (61.9%) | 8,241 (59.0%) | 0.06 | 15,939 (71.4%) | 16,749 (75.0%) | -0.08 | 26297 (67.3%) | 26834 (68.7%) | -0.03 |
| Number of Cardiologist visits (30 days prior); n (%) | 1,278 (45.8%) | 1,272 (45.6%) | 0.00 | 6,331 (45.4%) | 6,217 (44.5%) | 0.02 | 12,337 (55.3%) | 12,208 (54.7%) | 0.01 | 19946 (51.1%) | 19697 (50.4%) | 0.01 |
| Number of Cardiologist visits (31 to 180 days prior); | | | | | | | | | | | | |
| n (%) | 1,089 (39.0%) | 1,170 (41.9%) | -0.06 | 5,859 (42.0%) | 5,354 (38.4%) | 0.07 | 9,733 (43.6%) | 10,383 (46.5%) | -0.06 | 16681 (42.7%) | 16907 (43.3%) | -0.01 |
| Electrocardiogram v2; n (%) | 1,897 (68.0%)<br>26 (0.9%) | 1,931 (69.2%)<br>30 (1.1%) | -0.03<br>-0.02 | 9,862 (70.6%)<br>97 (0.7%) | 10,320 (73.9%)<br>101 (0.7%) | -0.07<br>0.00 | 16,644 (74.6%)<br>241 (1.1%) | 16,887 (75.7%)<br>229 (1.0%) | -0.03<br>0.01 | 28403 (72.7%)<br>364 (0.9%) | 29138 (74.6%) | -0.04<br>0.00 |
| Use of glucose test strips; n (%)<br>Dialysis; n (%) | 26 (0.9%) | 30 (1.1%)<br>0 (0.0%) | -0.02<br>#DIV/0! | 97 (0.7%) | 0 (0.0%) | 0.00<br>#DIV/01 | 241 (1.1%) | 229 (1.0%)<br>0 (0.0%) | #DIV/0! | 1 (0.0%) | 360 (0.9%)<br>0 (0.0%) | #DIV/0! |
| number of different/distinct medication | 1 (0.0%) | 0 (0.0%) | #514/0: | 0 (0.070) | 0 (0.0%) | #514/0: | 0 (0.070) | 0 (0.070) | #514/0: | 1 (0.070) | 0 (0.0%) | #D14/0: |
| prescriptions | | | | | | | | | | | | |
| mean (sd) | 8.18 (4.00) | 8.05 (4.00) | 0.03 | 9.29 (4.50) | 9.24 (4.56) | 0.01 | 8.57 (3.98) | 8.52 (4.04) | 0.01 | 8.80 (4.17) | 8.74 (4.23) | 0.01 |
| median [IQR] | 8.00 [5.00, 10.00] | 7.00 [5.00, 10.00] | 0.25 | 9.00 [6.00, 12.00] | 9.00 [6.00, 12.00] | 0.00 | 8.00 [6.00, 11.00] | 8.00 [6.00, 11.00] | 0.00 | 6.65 (4.66) | 6.57 (4.73) | 0.02 |
| Number of Hospitalizations | | | | | | | | | | | | |
| mean (sd) | 0.00 (0.00) | 0.00 (0.00) | #DIV/0! | 0.35 (0.55) | 0.34 (0.54) | 0.02 | 0.21 (0.47) | 0.21 (0.46) | 0.00 | 0.25 (0.48) | 0.24 (0.47) | 0.02 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | #DIV/0! | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.55) | 0.00 (0.54) | 0.00 |
| Number of hospital days | 0.00 (0.00) | 0.00 (0.00) | #DIV/0! | 1.59 (3.38) | 1.50 (3.34) | 0.03 | 0.88 (2.32) | 0.85 (2.52) | 0.01 | 1.07 (2.68) | 1.02 (2.76) | 0.02 |
| mean (sd)<br>median (IOR) | 0.00, 00.00 | 0.00 [0.00, 0.00] | #DIV/0! | 0.00 [0.00, 3.00] | 0.00 [0.00, 2.00] | 0.03 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.01 | 0.00 (3.10) | 0.00 (3.16) | 0.02 |
| Number of Emergency Department (ED) visits v3 | 0.00 (0.00, 0.00) | 0.00 (0.00, 0.00) | | 0.00 [0.00, 5.00] | 0.00 (0.00, 2.00) | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (3.10) | 0.00 (3.10) | 0.00 |
| mean (sd) | 0.40 (0.94) | 0.40 (0.99) | 0.00 | 0.44 (1.54) | 0.44 (1.72) | 0.00 | 0.64 (1.46) | 0.63 (1.26) | 0.01 | 0.55 (1.46) | 0.55 (1.43) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (1.62) | 0.00 (1.63) | 0.00 |
| Number of Office visits | | | | | | | | | | | | |
| mean (sd) | 5.25 (3.98) | 5.16 (3.64) | 0.02 | 5.89 (4.47) | 5.77 (4.32) | 0.03 | 11.61 (10.64) | 11.48 (9.99) | 0.01 | 9.11 (8.54) | 8.99 (8.04) | 0.01 |
| median [IQR] | 4.00 [3.00, 7.00] | 4.00 [3.00, 7.00] | 0.00 | 5.00 [3.00, 8.00] | 5.00 [3.00, 8.00] | 0.00 | 9.00 [5.00, 15.00] | 9.00 [5.00, 15.00] | 0.00 | 5.29 (8.79) | 5.29 (8.28) | 0.00 |
| Number of Endocrinologist visits | 0.00 (0.04) | 0.00 (0.05) | 0.00 | 0.13 (1.13) | 0.44 (0.07) | 0.02 | 0.17 (1.45) | 0.15 (1.39) | | 0.15 (1.31) | 0.13 (1.19) | 0.02 |
| mean (sd)<br>median [IQR] | 0.09 (0.81)<br>0.00 [0.00, 0.00] | 0.09 (0.86)<br>0.00 [0.00, 0.00] | 0.00 | | 0.11 (0.87)<br>0.00 [0.00, 0.00] | 0.02 | 0.00 [0.00, 0.00] | 0.15 (1.39) | 0.01<br>0.00 | 0.15 (1.31) | 0.13 (1.19) | 0.02 |
| median [IQK] Number of internal medicine/family medicine visits | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.41) | 0.00 (1.26) | 0.00 |
| mean (sd) | 8.11 (10.84) | 8.19 (12.81) | -0.01 | 6.56 (9.62) | 6.46 (9.25) | 0.01 | 6.41 (8.10) | 6.38 (7.75) | 0.00 | 6.58 (8.88) | 6.54 (8.75) | 0.00 |
| median [IOR] | 5.00 [2.00, 10.00] | 5.00 [1.00, 10.00] | 0.00 | 4.00 [1.00, 8.00] | 4.00 [1.00, 8.00] | 0.00 | 4.00 [1.00, 9.00] | 4.00 [1.00, 9.00] | 0.00 | 3.22 (9.94) | 3.22 (9.74) | 0.00 |
| Number of Cardiologist visits | | | | | | | | | | | , | |
| mean (sd) | 3.29 (4.91) | 3.30 (4.42) | 0.00 | 3.35 (4.99) | 3.29 (5.01) | 0.01 | 4.52 (6.31) | 4.46 (5.54) | 0.01 | 4.01 (5.78) | 3.96 (5.28) | 0.01 |
| median [IQR] | 2.00 [0.00, 5.00] | 2.00 [0.00, 5.00] | 0.00 | 2.00 [0.00, 5.00] | 1.50 [0.00, 5.00] | 0.10 | 2.00 [0.00, 6.00] | 3.00 [1.00, 6.00] | -0.17 | 1.57 (6.22) | 1.75 (5.77) | -0.03 |
| Number electrocardiograms received v2 | | | | | | | | | | | | |
| mean (sd) | 1.56 (2.08) | 1.54 (1.79) | 0.01 | 1.77 (2.23) | 1.72 (1.91) | 0.02 | 1.82 (2.02) | 1.80 (1.87) | 0.01 | 1.78 (2.10) | 1.75 (1.88) | 0.02 |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.00 | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.00 | 1.00 [0.00, 2.00] | 1.00 [1.00, 2.00] | 0.00 | 0.79 (2.34) | 0.79 (2.08) | 0.00 |
| Number of HbA1c tests ordered | 0.39 (0.69) | 0.39 (0.69) | 0.00 | 0.14 (0.45) | 0.15 (0.46) | -0.02 | 0.40 (0.71) | 0.40 (0.70) | 0.00 | 0.31 (0.63) | 0.31 (0.62) | 0.00 |
| mean (sd)<br>median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.02 | 0.40 (0.71) | 0.40 (0.70) | 0.00 | 0.31 (0.63) | 0.01 (0.62) | 0.00 |
| Number of glucose tests ordered | 2.22 [0.00, 2.00] | 2.25 [0.00, 2.00] | 0.00 | 2.22 [0.00, 0.00] | [0.00, 0.00] | 0.00 | [, 1] | 2.22 [0.00, 2.00] | 0.00 | 2.30 (0.00) | 0.00 (0.00) | 5.00 |
| mean (sd) | 0.13 (0.58) | 0.16 (0.96) | -0.04 | 0.10 (0.54) | 0.11 (0.58) | -0.02 | 0.13 (0.61) | 0.12 (0.48) | 0.02 | 0.12 (0.58) | 0.12 (0.56) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.63) | 0.00 (0.62) | 0.00 |
| Number of lipid tests ordered | | | | | | | | | | | | |

| mean (sd) | 0.67 (0.86) | 0.68 (0.84) | -0.01 | 0.25 (0.70) | 0.24 (0.63) | 0.02 | 0.68 (0.76) | 0.68 (0.74) | 0.00 | 0.53 (0.75) | 0.52 (0.71) | 0.01 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| median [IQR] | 0.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | -1.18 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 0.00 | 0.36 (0.81) | 0.43 (0.77) | -0.09 |
| Number of creatinine tests ordered | | | | | | | | | | | | |
| mean (sd) | 0.07 (0.33) | 0.07 (0.32) | 0.00 | 0.05 (0.28) | 0.05 (0.27) | 0.00 | 0.10 (0.39) | 0.09 (0.37) | 0.03 | 0.08 (0.35) | 0.07 (0.33) | 0.03 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.37) | 0.00 (0.36) | 0.00 |
| Number of BUN tests ordered | | | | | | | | | | | | |
| mean (sd) | 0.04 (0.23) | 0.05 (0.25) | -0.04 | 0.03 (0.22) | 0.03 (0.22) | 0.00 | 0.06 (0.30) | 0.05 (0.28) | 0.03 | 0.05 (0.27) | 0.04 (0.26) | 0.04 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.29) | 0.00 (0.28) | 0.00 |
| Number of tests for microal buminuria | | | | | | | | | | | | |
| mean (sd) | 0.21 (0.70) | 0.19 (0.64) | 0.03 | 0.07 (0.37) | 0.07 (0.37) | 0.00 | 0.12 (0.41) | 0.12 (0.39) | 0.00 | 0.11 (0.42) | 0.11 (0.41) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.46) | 0.00 (0.44) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at the 3rd | | | | | | | | | | | | |
| digit level Copy | 2.02 (4.05) | 2.04/5.12\ | 0.00 | 2 22 (4 07) | 2 24 (4 07) | 0.00 | 4.40 (6.63) | 4.00 (6.54) | 0.03 | 2.40 (5.04) | 2.24 (5.00) | 0.01 |
| mean (sd) | 3.02 (4.95) | 3.04 (5.12) | 0.00 | 2.23 (4.87) | 2.21 (4.87) | 0.00 | 4.18 (6.62) | 4.08 (6.51) | 0.02 | 3.40 (5.94) | 3.34 (5.88) | 0.01 |
| median [IQR]<br>For PS | 0.00 [0.00, 5.00] | 0.00 [0.00, 5.00] | 0.00 | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 | 0.00 [0.00, 6.00] | 0.00 [0.00, 6.00] | 0.00 | 0.00 (6.35) | 0.00 (6.30) | 0.00 |
| Hemorrhagic stroke+Other cerebrovascular<br>disease+Cerebrovascular procedure (for PS); n (%) | 45 (1.6%) | 52 (1.9%) | -0.02 | 297 (2.1%) | 316 (2.3%) | -0.01 | 416 (1.9%) | 398 (1.8%) | 0.01 | 758 (1.9%) | 766 (2.0%) | -0.01 |
| disease cerebrovascular procedure (101 + 5), 11 (70) | 45 (1.070) | 32 (1.370) | -0.02 | 237 (2.170) | 310 (2.3%) | -0.01 | 410 (1.570) | 330 (1.8%) | 0.01 | 730 (1.370) | 700 (2.0%) | -0.01 |
| Occurrence of creatinine tests ordered (for PS); n (%) | 148 (5.3%) | 154 (5.5%) | -0.01 | 495 (3.5%) | 495 (3.5%) | 0.00 | 1.648 (7.4%) | 1,562 (7.0%) | 0.02 | 2291 (5.9%) | 2211 (5.7%) | 0.01 |
| Occurrence of BUN tests ordered (for PS); n (%) | 95 (3.4%) | 103 (3.7%) | -0.02 | 311 (2.2%) | 333 (2.4%) | -0.01 | 1,063 (4.8%) | 1,001 (4.5%) | 0.01 | 1469 (3.8%) | 1437 (3.7%) | 0.01 |
| Occurrence of chronic renal insufficiency w/o CKD | | | | | | | ,, | , , | | , | | |
| (for PS) v2; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Chronic kidney disease Stage 1-2 (for PS); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 | 0 | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Chronic kidney disease Stage 3-6 (for PS); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Bladder stones+Kidney stones (for PS); n (%) | 35 (1.3%) | 35 (1.3%) | 0.00 | 191 (1.4%) | 229 (1.6%) | -0.02 | 283 (1.3%) | 274 (1.2%) | 0.01 | 509 (1.3%) | 538 (1.4%) | -0.01 |
| Diabetes with peripheral circulatory | | | | | | | | | | | | |
| disorders+Gangrene+Osteomyelitis(for PS) v3 with | | | | | | | | | | | | |
| ICD10 Copy; n (%) | 75 (2.7%) | 49 (1.8%) | 0.06 | 285 (2.0%) | 269 (1.9%) | 0.01 | 408 (1.8%) | 430 (1.9%) | -0.01 | 768 (2.0%) | 748 (1.9%) | 0.01 |
| Alcohol abuse or dependence+Drug abuse or | | | | | | | | | | | | |
| dependence (for PS); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Diabetes with other ophthalmic | | | | | | | | | | | | |
| manifestations+Retinal detachment, vitreous | | | | | | | | | | | | |
| hemorrhage, vitrectomy+Retinal laser coagulation<br>therapy (for PS); n (%) | 11 (0.4%) | 11 (0.4%) | 0.00 | 204 (1.5%) | 168 (1.2%) | 0.03 | 224 (1.0%) | 191 (0.9%) | 0.01 | 439 (1.1%) | 370 (0.9%) | 0.02 |
| Other atherosclerosis+Cardiac conduction | 11 (0.4%) | 11 (0.4%) | 0.00 | 204 (1.5%) | 168 (1.2%) | 0.03 | 224 (1.0%) | 191 (0.9%) | 0.01 | 439 (1.1%) | 370 (0.9%) | 0.02 |
| disorders+Other CVD (for PS) v2 Copy; n (%) | 515 (18.5%) | 505 (18.1%) | 0.01 | 4,706 (33.7%) | 4,661 (33.4%) | 0.01 | 3,619 (16.2%) | 3,549 (15.9%) | 0.01 | 8840 (22.6%) | 8715 (22.3%) | 0.01 |
| Previous cardiac procedure (CABG or PTCA or Stent) | | 303 (18.170) | 0.01 | 4,700 (33.770) | 4,001 (33.4%) | 0.01 | 3,013 (10.270) | 3,343 (13.5%) | 0.01 | 8040 (22.070) | 0713 (22.3%) | 0.01 |
| History of CABG or PTCA (for PS) v3; n (%) | 153 (5.5%) | 141 (5.1%) | 0.02 | 730 (5.2%) | 700 (5.0%) | 0.01 | 1,780 (8.0%) | 1,772 (7.9%) | 0.00 | 2663 (6.8%) | 2613 (6.7%) | 0.00 |
| Hyperthyroidism + Hypothyroidism + Other disorder | | (0.2, | | | ( , | | -, (, | _,(, | | | | |
| of thyroid gland (for PS); n (%) | 430 (15.4%) | 454 (16.3%) | -0.02 | 1,697 (12.2%) | 1,748 (12.5%) | -0.01 | 3,078 (13.8%) | 3,045 (13.6%) | 0.01 | 5205 (13.3%) | 5247 (13.4%) | 0.00 |
| Delirium + Psychosis (for PS); n (%) | 28 (1.0%) | 27 (1.0%) | 0.00 | 190 (1.4%) | 207 (1.5%) | -0.01 | 285 (1.3%) | 264 (1.2%) | 0.01 | 503 (1.3%) | 498 (1.3%) | 0.00 |
| Any use of Meglitinides (for PS); n (%) | 4 (0.1%) | 3 (0.1%) | 0.00 | 76 (0.5%) | 69 (0.5%) | 0.00 | 72 (0.3%) | 57 (0.3%) | 0.00 | 152 (0.4%) | 129 (0.3%) | 0.02 |
| Any use of AGIs (for PS); n (%) | 2 (0.1%) | 4 (0.1%) | 0.00 | 17 (0.1%) | 27 (0.2%) | -0.03 | 18 (0.1%) | 28 (0.1%) | 0.00 | 37 (0.1%) | 59 (0.2%) | -0.03 |
| CKD stage 3-6 + dialysis (for PS); n (%) | 1 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 1 (0.0%) | 0 (0.0%) | #DIV/0! |
| Use of thiazide; n (%) | 319 (11.4%) | 332 (11.9%) | -0.02 | 1,447 (10.4%) | 1,514 (10.8%) | -0.01 | 2,908 (13.0%) | 2,867 (12.8%) | 0.01 | 4674 (12.0%) | 4713 (12.1%) | 0.00 |
| Use of beta blockers; n (%) | 1,727 (61.9%) | 1,731 (62.0%) | 0.00 | 9,487 (68.0%) | 9,422 (67.5%) | 0.01 | 14,583 (65.3%) | 14,638 (65.6%) | -0.01 | 25797 (66.0%) | 25791 (66.0%) | 0.00 |
| Use of calcium channel blockers; n (%) | 1,068 (38.3%) | 1,010 (36.2%) | 0.04 | 5,367 (38.4%) | 5,347 (38.3%) | 0.00 | 8,746 (39.2%) | 8,649 (38.8%) | 0.01 | 15181 (38.9%) | 15006 (38.4%) | 0.01 |
| All antidiabetic medications except Insulin; n (%) | 603 (21.6%) | 585 (21.0%) | 0.01 | 2,704 (19.4%) | 2,727 (19.5%) | 0.00 | 4,497 (20.1%) | 4,460 (20.0%) | 0.00 | 7804 (20.0%) | 7772 (19.9%) | 0.00 |
| DM Medications - Insulin Copy; n (%) | 126 (4.5%) | 119 (4.3%) | 0.01 | 695 (5.0%) | 733 (5.3%) | -0.01 | 1,030 (4.6%) | 802 (3.6%) | 0.05 | 1851 (4.7%) | 1654 (4.2%) | 0.02 |
| Use of Low Intensity Statins; n (%) | 960 (34.4%) | 925 (33.2%) | 0.03 | 4,415 (31.6%) | 4,638 (33.2%) | -0.03 | 7,800 (34.9%) | 7,804 (35.0%) | 0.00 | 13175 (33.7%) | 13367 (34.2%) | -0.01 |
| Use of High Intensity Statins; n (%) | 553 (19.8%) | 586 (21.0%) | -0.03 | 3,170 (22.7%) | 2,952 (21.1%) | 0.04 | 4,696 (21.0%) | 4,665 (20.9%) | 0.00 | 8419 (21.5%) | 8203 (21.0%) | 0.01 |
| Malignant hypertension; n (%) | 108 (3.9%) | 103 (3.7%) | 0.01 | 6,144 (44.0%) | 5,989 (42.9%) | 0.02 | 3,405 (15.3%) | 3,554 (15.9%) | -0.02 | 9657 (24.7%) | 9646 (24.7%) | 0.00 |
| Cardiovascular stress test; n (%) | 6 (0.2%) | 13 (0.5%) | -0.05 | 96 (0.7%) | 63 (0.5%) | 0.03 | 105 (0.5%) | 85 (0.4%) | 0.01 | 207 (0.5%) | 161 (0.4%) | 0.01 |
| Echocardiogram; n (%) | 655 (23.5%) | 781 (28.0%) | -0.10 | 6,201 (44.4%) | 6,865 (49.2%) | -0.10 | 7,094 (31.8%) | 8,024 (35.9%) | -0.09 | 13950 (35.7%) | 15670 (40.1%) | -0.09 |
| Number of BNP tests | 0.00 | 0.00/5: | 0.6- | 0.07/5 | 0.07/5 | | 0.40.47 | 0.40.65 : | | 0.40/0.0-1 | 0.44/5 | |
| mean (sd) | 0.09 (0.43) | 0.09 (0.36) | 0.00 | 0.07 (0.32) | 0.07 (0.33) | 0.00 | 0.12 (0.40) | 0.13 (0.42) | -0.02 | 0.10 (0.38) | 0.11 (0.39) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.40) | 0.00 (0.42) | 0.00 |
| Number of Cardiac biomarkers tests (tropnin, CK-MB | s Munglohin CDK) | | | | | | | | | | | |
| mean (sd) | 0.31 (1.08) | 0.35 (1.15) | -0.04 | 0.27 (1.16) | 0.30 (1.23) | -0.03 | 0.24 (0.54) | 0.25 (0.55) | -0.02 | 0.26 (0.85) | 0.28 (0.90) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.01) | 0.00 (1.06) | 0.00 |
| realan (rept) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.01) | 0.00 (1.00) | 0.00 |
| Number of Ambulatory Blood pressure monitoring to | ests | | | | | | | | | | | |
| mean (sd) | 0.00 (0.02) | 0.00 (0.02) | 0.00 | 0.00 (0.03) | 0.00 (0.04) | 0.00 | 0.00 (0.02) | 0.00 (0.03) | 0.00 | 0.00 (0.02) | 0.00 (0.03) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.03) | 0.00 (0.04) | 0.00 |
| N of days on antihypertensive medications during ba | | | | | | | | | | | | |
| mean (sd) | 131.24 (67.61) | 130.11 (66.94) | 0.02 | 132.77 (67.41) | 132.32 (67.50) | 0.01 | 137.09 (64.11) | 136.78 (64.52) | 0.00 | 135.13 (65.56) | 134.71 (65.77) | 0.00 |
| median [IQR] | 170.00 [94.75, 181.00] | 169.00 [92.00, 181.00] | 0.01 | 172.00 [97.00, 181.00] | 171.00 [96.00, 181.00] | 0.01 | 173.00 [118.00, 181.00] | 173.00 [116.00, 181.00] | 0.00 | 135.41 (72.60) | 134.98 (72.81) | 0.00 |
| N of days in database anytime prior | | | | | | | | | | | | |
| mean (sd) | 1,737.28 (1,168.84) | 1,752.47 (1,196.68) | -0.01 | 2,106.30 (1,213.13) | 2,104.50 (1,207.54) | 0.00 | 860.39 (497.95) | 859.94 (468.49) | 0.00 | 1368.18 (874.66) | 1368.37 (865.24) | 0.00 |
| ii tool | 1,578.00 [699.75, | 4 500 00 (200 25 0 505) | | | | | == 00/400 00 4 0=:* | 775 00/544 00 4 005 | | | 4457 04/4005 | |
| median [IQR] | 2,481.50] | 1,600.00 [708.75, 2,508.25] | -0.02 )8 | 3.50 [1,036.00, 3,090.75] | 2,144.00 [1,017.00, 3,097.00] | -0.03 7 | 75.00 [499.00, 1,074.75] | 775.00 [511.00, 1,085.00] | 0.00 | 1142.98 (1039.21) | 1157.24 (1029.89) | 0.00 |
| Maan Consy for ner prescription sect (share | ¢\/190-1 day prior\ | | | | | | | | | | | |
| Mean Copay for per prescription cost (charges in U.Smean (sd) | . \$) (180-1 day prior)<br>32.13 (39.93) | 31.29 (40.47) | 0.02 | 22.72 (21.47) | 22.59 (23.48) | 0.01 | 113.35 (101.72) | 115.02 (120.71) | -0.01 | 75.17 (78.67) | 76.01 (92.94) | 0.00 |
| mean (sd)<br>median [IQR] | 32.13 (39.93)<br>19.94 [8.75, 41.24] | 20.38 [9.47, 39.44] | -0.02 | 18.19 [8.85, 30.64] | 22.59 (23.48)<br>17.21 [8.61, 29.98] | 0.01 | 90.00 [62.27, 132.46] | 90.94 [63.10, 132.85] | -0.01 | 75.17 (78.67)<br>40.08 (79.30) | 40.10 (93.57) | 0.00 |
| Missing; n (%) | 19.94 [8.75, 41.24]<br>56 (2.0%) | 20.38 [9.47, 39.44] | -0.01 | 420 (3.0%) | 422 (3.0%) | 0.04 | 482 (2.2%) | 502 (2.2%) | 0.00 | 958 (2.5%) | 985 (2.5%) | 0.00 |
| Colonoscopy; n (%) | 96 (3.4%) | 86 (3.1%) | 0.01 | 420 (3.0%) | 422 (3.0%) | 0.00 | 482 (2.2%)<br>621 (2.8%) | 639 (2.2%) | -0.01 | 1185 (3.0%) | 1184 (3.0%) | 0.00 |
| Fecal occult blood (FOB) test; n (%) | 112 (4.0%) | 111 (4.0%) | 0.02 | 316 (2.3%) | 303 (2.2%) | 0.01 | 621 (2.8%) | 603 (2.7%) | 0.01 | 1049 (2.7%) | 1017 (2.6%) | 0.00 |
| Flu vaccine; n (%) | 525 (18.8%) | 549 (19.7%) | -0.02 | 1.463 (10.5%) | 1.461 (10.5%) | 0.01 | 7.309 (32.7%) | 7.390 (33.1%) | -0.01 | 9297 (23.8%) | 9400 (24.1%) | -0.01 |
| Mammogram; n (%) | 227 (8.1%) | 220 (7.9%) | 0.01 | 782 (5.6%) | 732 (5.2%) | 0.02 | 1,723 (7.7%) | 1,707 (7.6%) | 0.00 | 2732 (7.0%) | 2659 (6.8%) | 0.01 |
| | 22, (0.1/0) | 220 (1.370) | 0.01 | , 02 (3.070) | , 32 (3.270) | 0.02 | -,, 25 (, ., 70) | 1,.0. (0/0) | 0.00 | 52 (1.070) | 2000 (0.070) | 0.01 |

| Pap smear; n (%) | 42 (1.5%) | 41 (1.5%) | 0.00 | 236 (1.7%) | 221 (1.6%) | 0.01 | 446 (2.0%) | 438 (2.0%) | 0.00 | 724 (1.9%) | 700 (1.8%) | 0.01 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Pneumonia vaccine; n (%) | 256 (9.2%) | 263 (9.4%) | -0.01 | 419 (3.0%) | 438 (3.1%) | -0.01 | 2,807 (12.6%) | 2,800 (12.5%) | 0.00 | 3482 (8.9%) | 3501 (9.0%) | 0.00 |
| PSA test or Prostate exam for DRE; n (%) | 483 (17.3%) | 471 (16.9%) | 0.01 | 1,011 (7.2%) | 980 (7.0%) | 0.01 | 3,880 (17.4%) | 3,854 (17.3%) | 0.00 | 5374 (13.8%) | 5305 (13.6%) | 0.01 |
| Bone mineral density; n (%) | 104 (3.7%) | 103 (3.7%) | 0.00 | 250 (1.8%) | 257 (1.8%) | 0.00 | 739 (3.3%) | 724 (3.2%) | 0.01 | 1093 (2.8%) | 1084 (2.8%) | 0.00 |
| Use of Sympatomimetic agents; n (%) | 10 (0.4%) | 8 (0.3%) | 0.02 | 70 (0.5%) | 79 (0.6%) | -0.01 | 48 (0.2%) | 53 (0.2%) | 0.00 | 128 (0.3%) | 140 (0.4%) | -0.02 |
| Use of CNS stimulants: n (%) | 4 (0.1%) | 3 (0.1%) | 0.00 | 78 (0.6%) | 73 (0.5%) | 0.01 | 28 (0.1%) | 30 (0.1%) | 0.00 | 110 (0.3%) | 106 (0.3%) | 0.00 |
| | 73 (2.6%) | 78 (2.8%) | -0.01 | 625 (4.5%) | 617 (4.4%) | 0.00 | | 703 (3.1%) | -0.01 | 1355 (3.5%) | 1398 (3.6%) | -0.01 |
| Use of estrogens, progestins, androgens; n (%) | , | - 1 | | , | | | 657 (2.9%) | /03 (3.1%) | | | , | |
| Use of Angiogenesis inhibitors; n (%) | 0 (0.0%) | 1 (0.0%) | #DIV/0! | 13 (0.1%) | 4 (0.0%) | 0.04 | ** | ** | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Use of Oral Immunosuppressants; n (%) | 2 (0.1%) | 1 (0.0%) | 0.04 | 14 (0.1%) | 7 (0.1%) | 0.00 | ** | ** | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Use of fondaparinux or Bivalirudin; n (%) | 0 (0.0%) | 1 (0.0%) | #DIV/0! | 12 (0.1%) | 10 (0.1%) | 0.00 | ** | ** | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| | 0 (0 00) | 0.40.0043 | | 0 (0 00) | 0.40.004 | up u 1/01 | 0 (0 00() | 0 (0 00) | up u //o1 | 0 (0 00() | 0 (0 00() | WP 11 / fo 1 |
| Use of other direct thrombin inhibitors (lepirudin, des | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Use of Ticagrelor ON CED; n (%) | 0 (0.0%) | 1 (0.0%) | #DIV/0! | 14 (0.1%) | 12 (0.1%) | 0.00 | 6 (0.0%) | 6 (0.0%) | #DIV/0! | 20 (0.1%) | 19 (0.0%) | 0.04 |
| Use of Ticagrelor; n (%) | 1 (0.0%) | 2 (0.1%) | -0.04 | 19 (0.1%) | 18 (0.1%) | 0.00 | 43 (0.2%) | 36 (0.2%) | 0.00 | 63 (0.2%) | 56 (0.1%) | 0.03 |
| Number of D-dimer tests | | | | | | | | | | | | |
| mean (sd) | 0.02 (0.14) | 0.02 (0.14) | 0.00 | 0.02 (0.15) | 0.02 (0.15) | 0.00 | 0.03 (0.18) | 0.03 (0.18) | 0.00 | 0.03 (0.17) | 0.03 (0.17) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.18) | 0.00 (0.18) | 0.00 |
| Numbe of CRP, high-sensitivity CRP tests | | | | | | | | | | | | |
| mean (sd) | 0.06 (0.33) | 0.06 (0.32) | 0.00 | 0.02 (0.20) | 0.02(0.19) | 0.00 | 0.07 (0.36) | 0.07 (0.34) | 0.00 | 0.05 (0.31) | 0.05 (0.29) | 0.00 |
| median (IOR) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.32) | 0.00 (0.23) | 0.00 |
| Number of PT or aPTTt tests | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.32) | 0.00 (0.31) | 0.00 |
| mean (sd) | 0.51 (1.32) | 0.46 (1.53) | 0.03 | 0.45 (1.36) | 0.38 (1.44) | 0.05 | 0.47 (1.25) | 0.43 (1.37) | 0.03 | 0.47 (1.30) | 0.41 (1.41) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.44) | 0.00 (1.56) | 0.00 |
| Number of Bleeding time tests | | | | | | | | | | | | |
| mean (sd) | 0.00 (0.00) | 0.00 (0.00) | #DIV/0! | 0.00 (0.02) | 0.00 (0.01) | 0.00 | 0.00 (0.01) | 0.00 (0.02) | 0.00 | 0.00 (0.01) | 0.00 (0.02) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | #DIV/0! | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.02) | 0.00 (0.02) | 0.00 |
| HAS-BLED Score (ICD-9 and ICD-10), 180 days | | | | | | | | | | | | |
| mean (sd) | 3.25 (0.70) | 3.23 (0.67) | 0.03 | 3.25 (0.74) | 3.25 (0.74) | 0.00 | 3.28 (0.63) | 3.28 (0.62) | 0.00 | 3.27 (0.68) | 3.27 (0.67) | 0.00 |
| median [IQR] | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 2.36 (0.76) | 2.36 (0.75) | 0.00 |
| N of Generic name drugs | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 2.50 (0.70) | 2.50 (0.75) | 0.00 |
| | 14.73 (11.91) | 14.51 (12.77) | 0.02 | 12.44 (8.50) | 12.33 (9.55) | 0.01 | 14.78 (10.66) | 14.67 (11.77) | 0.01 | 13.94 (10.04) | 13.82 (11.11) | 0.00 |
| mean (sd) | | | | | | | | | | | | |
| median [IQR] | 12.00 [7.00, 19.00] | 11.00 [6.00, 19.00] | 0.08 | 11.00 [7.00, 16.00] | 10.00 [6.00, 16.00] | 0.11 | 12.00 [8.00, 19.00] | 12.00 [7.00, 19.00] | 0.00 | 9.07 (10.79) | 8.65 (11.95) | 0.00 |
| N of Brand name drugs | | | | | | | | | | | | |
| mean (sd) | 4.80 (6.60) | 4.49 (4.60) | 0.05 | 5.59 (5.92) | 5.53 (4.85) | 0.01 | 4.64 (5.86) | 4.56 (4.70) | 0.02 | 4.99 (5.94) | 4.90 (4.75) | 0.00 |
| median [IQR] | 3.00 [0.00, 6.00] | 3.00 [1.00, 6.00] | 0.00 | 4.00 [2.00, 8.00] | 4.00 [2.00, 7.00] | 0.00 | 3.00 [1.00, 6.00] | 3.00 [1.00, 6.00] | 0.00 | 2.72 (6.54) | 2.72 (5.25) | 0.00 |
| Use of clopidogrel ; n (%) | 180 (6.5%) | 177 (6.3%) | 0.01 | 1,663 (11.9%) | 1,623 (11.6%) | 0.01 | 2,096 (9.4%) | 2,122 (9.5%) | 0.00 | 3939 (10.1%) | 3922 (10.0%) | 0.00 |
| Systemic embolism; n (%) | 13 (0.5%) | 11 (0.4%) | 0.01 | 50 (0.4%) | 58 (0.4%) | 0.00 | 77 (0.3%) | 80 (0.4%) | -0.02 | 140 (0.4%) | 149 (0.4%) | 0.00 |
| DVT; n (%) | 35 (1.3%) | 32 (1.1%) | 0.02 | 207 (1.5%) | 213 (1.5%) | 0.00 | 245 (1.1%) | 272 (1.2%) | -0.01 | 487 (1.2%) | 517 (1.3%) | -0.01 |
| PE; n (%) | 5 (0.2%) | 4 (0.1%) | 0.03 | 92 (0.7%) | 91 (0.7%) | 0.00 | 84 (0.4%) | 73 (0.3%) | 0.02 | 181 (0.5%) | 168 (0.4%) | 0.01 |
| r L, 11 (70) | 3 (0.270) | 4 (0.170) | 0.03 | 32 (0.770) | 51 (0.7%) | 0.00 | 84 (0.470) | 75 (0.5%) | 0.02 | 101 (0.570) | 100 (0.470) | 0.01 |
| Diabetes: 1 inpatient or 2 outpatient claims within 18 | 780 (28.0%) | 749 (26.8%) | 0.03 | 3,371 (24.1%) | 3,331 (23.9%) | 0.00 | 5,636 (25.3%) | 5,630 (25.2%) | 0.00 | 9787 (25.0%) | 9710 (24.9%) | 0.00 |
| Intracranial or retroperitoneal hemorrhage: 1 inpatier | 0 (0.0%) | 1 (0.0%) | #DIV/01 | 9 (0.1%) | 8 (0.1%) | 0.00 | 20 (0.1%) | 17 (0.1%) | 0.00 | 29 (0.1%) | 26 (0.1%) | 0.00 |
| Intracranial or retroperitoneal hemorrhage: 1 inpatier | - () | - () | #DIV/0! | - () | - (,-) | | () | () | | () | () | |
| Peptic Ulcer Disease; n (%) | 203 (7.3%) | 208 (7.5%) | -0.01 | 901 (6.5%) | 844 (6.0%) | 0.02 | 1,652 (7.4%) | 1,633 (7.3%) | 0.00 | 2756 (7.1%) | 2685 (6.9%) | 0.01 |
| Peptic Ulcer Disease; n (%)<br>Upper GI bleed; n (%) | 203 (7.3%) | 208 (7.5%) | -0.01<br>#DIV/0! | 901 (6.5%)<br>5 (0.0%) | 844 (6.0%)<br>4 (0.0%) | 0.02<br>#DIV/0! | 1,652 (7.4%)<br>0 (0.0%) | 1,633 (7.3%) | 0.00<br>#VALUE! | 2756 (7.1%)<br>5 (0.0%) | 2685 (6.9%)<br>#VALUE! | 0.01<br>#VALUE! |
| Peptic Ulcer Disease; n (%)<br>Upper Gi bleed; n (%)<br>Lower/ unspecified Gi bleed; n (%) | 203 (7.3%)<br>0 (0.0%)<br>21 (0.8%) | 208 (7.5%)<br>0 (0.0%)<br>24 (0.9%) | -0.01<br>#DIV/0!<br>-0.01 | 901 (6.5%)<br>5 (0.0%)<br>104 (0.7%) | 844 (6.0%)<br>4 (0.0%)<br>98 (0.7%) | 0.02<br>#DIV/0!<br>0.00 | 1,652 (7.4%)<br>0 (0.0%)<br>116 (0.5%) | 1,633 (7.3%)<br>**<br>132 (0.6%) | 0.00<br>#VALUE!<br>-0.01 | 2756 (7.1%)<br>5 (0.0%)<br>241 (0.6%) | 2685 (6.9%)<br>#VALUE!<br>254 (0.7%) | 0.01<br>#VALUE!<br>-0.01 |
| Peptic Ulcer Disease; n (%)<br>Upper Gl bleed; n (%)<br>Lower/ unspecified Gl bleed; n (%)<br>Urogenital bleed; n (%) | 203 (7.3%)<br>0 (0.0%)<br>21 (0.8%)<br>91 (3.3%) | 208 (7.5%)<br>0 (0.0%)<br>24 (0.9%)<br>85 (3.0%) | -0.01<br>#DIV/0!<br>-0.01<br>0.02 | 901 (6.5%)<br>5 (0.0%)<br>104 (0.7%)<br>441 (3.2%) | 844 (6.0%)<br>4 (0.0%)<br>98 (0.7%)<br>429 (3.1%) | 0.02<br>#DIV/0!<br>0.00<br>0.01 | 1,652 (7.4%)<br>0 (0.0%)<br>116 (0.5%)<br>671 (3.0%) | 1,633 (7.3%) ** 132 (0.6%) 628 (2.8%) | 0.00<br>#VALUE!<br>-0.01<br>0.01 | 2756 (7.1%)<br>5 (0.0%)<br>241 (0.6%)<br>1203 (3.1%) | 2685 (6.9%)<br>#VALUE!<br>254 (0.7%)<br>1142 (2.9%) | 0.01<br>#VALUE!<br>-0.01<br>0.01 |
| Peptic Ulcer Disease; n (%) Upper Gi bleed; n (%) Lower/ unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) | 203 (7.3%)<br>0 (0.0%)<br>21 (0.8%)<br>91 (3.3%)<br>29 (1.0%) | 208 (7.5%)<br>0 (0.0%)<br>24 (0.9%)<br>85 (3.0%)<br>27 (1.0%) | -0.01<br>#DIV/0!<br>-0.01<br>0.02<br>0.00 | 901 (6.5%)<br>5 (0.0%)<br>104 (0.7%)<br>441 (3.2%)<br>167 (1.2%) | 844 (6.0%)<br>4 (0.0%)<br>98 (0.7%)<br>429 (3.1%)<br>157 (1.1%) | 0.02<br>#DIV/0!<br>0.00<br>0.01<br>0.01 | 1,652 (7.4%)<br>0 (0.0%)<br>116 (0.5%)<br>671 (3.0%)<br>229 (1.0%) | 1,633 (7.3%) ** 132 (0.6%) 628 (2.8%) 243 (1.1%) | 0.00<br>#VALUE!<br>-0.01<br>0.01<br>-0.01 | 2756 (7.1%)<br>5 (0.0%)<br>241 (0.6%)<br>1203 (3.1%)<br>425 (1.1%) | 2685 (6.9%)<br>#VALUE!<br>254 (0.7%)<br>1142 (2.9%)<br>427 (1.1%) | 0.01<br>#VALUE!<br>-0.01<br>0.01<br>0.00 |
| Peptic Ulcer Disease; n (%) Upper Gi bleed; n (%) Lower (unspecified Gi bleed; n (%) Urogenital bleed; n (%) Urogenital bleed; n (%) Prior cancer; n (%) | 203 (7.3%)<br>0 (0.0%)<br>21 (0.8%)<br>91 (3.3%)<br>29 (1.0%)<br>285 (10.2%) | 208 (7.5%)<br>0 (0.0%)<br>24 (0.9%)<br>85 (3.0%)<br>27 (1.0%)<br>289 (10.4%) | -0.01<br>#DIV/0!<br>-0.01<br>0.02<br>0.00<br>-0.01 | 901 (6.5%)<br>5 (0.0%)<br>104 (0.7%)<br>441 (3.2%)<br>167 (1.2%)<br>1,288 (9.2%) | 844 (6.0%)<br>4 (0.0%)<br>98 (0.7%)<br>429 (3.1%)<br>157 (1.1%)<br>1,288 (9.2%) | 0.02<br>#DIV/0!<br>0.00<br>0.01<br>0.01 | 1,652 (7.4%)<br>0 (0.0%)<br>116 (0.5%)<br>671 (3.0%)<br>229 (1.0%)<br>2,427 (10.9%) | 1,633 (7.3%) ** 132 (0.6%) 628 (2.8%) 243 (1.1%) 2,334 (10.5%) | 0.00<br>#VALUE!<br>-0.01<br>0.01<br>-0.01 | 2756 (7.1%)<br>5 (0.0%)<br>241 (0.6%)<br>1203 (3.1%)<br>425 (1.1%)<br>4000 (10.2%) | 2685 (6.9%)<br>#VALUE!<br>254 (0.7%)<br>1142 (2.9%)<br>427 (1.1%)<br>3911 (10.0%) | 0.01<br>#VALUE!<br>-0.01<br>0.01<br>0.00 |
| Peptic Ulcer Disease; n (%) Upper Gi bleed; n (%) Lower/ unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) | 203 (7.3%)<br>0 (0.0%)<br>21 (0.8%)<br>91 (3.3%)<br>29 (1.0%) | 208 (7.5%)<br>0 (0.0%)<br>24 (0.9%)<br>85 (3.0%)<br>27 (1.0%) | -0.01<br>#DIV/0!<br>-0.01<br>0.02<br>0.00 | 901 (6.5%)<br>5 (0.0%)<br>104 (0.7%)<br>441 (3.2%)<br>167 (1.2%) | 844 (6.0%)<br>4 (0.0%)<br>98 (0.7%)<br>429 (3.1%)<br>157 (1.1%) | 0.02<br>#DIV/0!<br>0.00<br>0.01<br>0.01 | 1,652 (7.4%)<br>0 (0.0%)<br>116 (0.5%)<br>671 (3.0%)<br>229 (1.0%) | 1,633 (7.3%) ** 132 (0.6%) 628 (2.8%) 243 (1.1%) | 0.00<br>#VALUE!<br>-0.01<br>0.01<br>-0.01 | 2756 (7.1%)<br>5 (0.0%)<br>241 (0.6%)<br>1203 (3.1%)<br>425 (1.1%) | 2685 (6.9%)<br>#VALUE!<br>254 (0.7%)<br>1142 (2.9%)<br>427 (1.1%) | 0.01<br>#VALUE!<br>-0.01<br>0.01<br>0.00 |
| Peptic Ulcer Disease; n (%) Upper Gi bleed; n (%) Lower (unspecified Gi bleed; n (%) Urogenital bleed; n (%) Urogenital bleed; n (%) Prior cancer; n (%) | 203 (7.3%)<br>0 (0.0%)<br>21 (0.8%)<br>91 (3.3%)<br>29 (1.0%)<br>285 (10.2%) | 208 (7.5%)<br>0 (0.0%)<br>24 (0.9%)<br>85 (3.0%)<br>27 (1.0%)<br>289 (10.4%) | -0.01<br>#DIV/0!<br>-0.01<br>0.02<br>0.00<br>-0.01 | 901 (6.5%)<br>5 (0.0%)<br>104 (0.7%)<br>441 (3.2%)<br>167 (1.2%)<br>1,288 (9.2%) | 844 (6.0%)<br>4 (0.0%)<br>98 (0.7%)<br>429 (3.1%)<br>157 (1.1%)<br>1,288 (9.2%) | 0.02<br>#DIV/0!<br>0.00<br>0.01<br>0.01 | 1,652 (7.4%)<br>0 (0.0%)<br>116 (0.5%)<br>671 (3.0%)<br>229 (1.0%)<br>2,427 (10.9%) | 1,633 (7.3%) ** 132 (0.6%) 628 (2.8%) 243 (1.1%) 2,334 (10.5%) | 0.00<br>#VALUE!<br>-0.01<br>0.01<br>-0.01 | 2756 (7.1%)<br>5 (0.0%)<br>241 (0.6%)<br>1203 (3.1%)<br>425 (1.1%)<br>4000 (10.2%) | 2685 (6.9%)<br>#VALUE!<br>254 (0.7%)<br>1142 (2.9%)<br>427 (1.1%)<br>3911 (10.0%) | 0.01<br>#VALUE!<br>-0.01<br>0.01<br>0.00 |
| Peptic Ulcer Disease; n (%) Upper Gi bleed; n (%) Lower / unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) | 203 (7.3%)<br>0 (0.0%)<br>21 (0.8%)<br>91 (3.3%)<br>29 (1.0%)<br>285 (10.2%)<br>13 (0.5%) | 208 (7.5%)<br>0 (0.0%)<br>24 (0.9%)<br>85 (3.0%)<br>27 (1.0%)<br>289 (10.4%)<br>11 (0.4%) | -0.01<br>#DIV/0!<br>-0.01<br>0.02<br>0.00<br>-0.01 | 901 (6.5%)<br>5 (0.0%)<br>104 (0.7%)<br>441 (3.2%)<br>167 (1.2%)<br>1,288 (9.2%)<br>164 (1.2%) | 844 (6.0%)<br>4 (0.0%)<br>98 (0.7%)<br>429 (3.1%)<br>157 (1.1%)<br>1,288 (9.2%)<br>161 (1.2%) | 0.02<br>#DIV/0!<br>0.00<br>0.01<br>0.01<br>0.00<br>0.00 | 1,652 (7.4%)<br>0 (0.0%)<br>116 (0.5%)<br>671 (3.0%)<br>229 (1.0%)<br>2,427 (10.9%)<br>105 (0.5%) | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 2,334 (10.5%) 97 (0.4%) | 0.00<br>#VALUE!<br>-0.01<br>0.01<br>-0.01<br>0.01 | 2756 (7.1%)<br>5 (0.0%)<br>241 (0.6%)<br>1203 (3.1%)<br>425 (1.1%)<br>4000 (10.2%)<br>282 (0.7%) | 2685 (6.9%) #VALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) | 0.01<br>#VALUE!<br>-0.01<br>0.01<br>0.00<br>0.01 |
| Peptic Ulcer Disease; n (%) Upper Gl bleed; n (%) Lower / unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) | 203 (7.3%)<br>0 (0.0%)<br>21 (0.8%)<br>91 (3.3%)<br>29 (1.0%)<br>285 (10.2%)<br>13 (0.5%)<br>9 (0.3%) | 208 (7.5%)<br>0 (0.0%)<br>24 (0.9%)<br>85 (3.0%)<br>27 (1.0%)<br>289 (10.4%)<br>11 (0.4%)<br>9 (0.3%) | -0.01<br>#DIV/0!<br>-0.01<br>0.02<br>0.00<br>-0.01<br>0.01 | 901 (6.5%)<br>5 (0.0%)<br>104 (0.7%)<br>441 (3.2%)<br>167 (1.2%)<br>1,288 (9.2%)<br>164 (1.2%)<br>79 (0.6%) | 844 (6.0%)<br>4 (0.0%)<br>98 (0.7%)<br>429 (3.1%)<br>157 (1.1%)<br>1,288 (9.2%)<br>161 (1.2%)<br>71 (0.5%) | 0.02<br>#DIV/0!<br>0.00<br>0.01<br>0.01<br>0.00<br>0.00<br>0.00 | 1,652 (7.4%)<br>0 (0.0%)<br>116 (0.5%)<br>671 (3.0%)<br>229 (1.0%)<br>2,427 (10.9%)<br>105 (0.5%)<br>90 (0.4%) | 1,633 (7.3%) ** 132 (0.6%) 628 (2.8%) 243 (1.1%) 2,334 (10.5%) 97 (0.4%) 84 (0.4%) | 0.00<br>#VALUE!<br>-0.01<br>0.01<br>-0.01<br>0.01<br>0.01 | 2756 (7.1%)<br>5 (0.0%)<br>241 (0.6%)<br>1203 (3.1%)<br>425 (1.1%)<br>4000 (10.2%)<br>282 (0.7%)<br>178 (0.5%) | 2685 (6.9%) #WALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) | 0.01<br>#VALUE!<br>-0.01<br>0.01<br>0.00<br>0.01<br>0.00<br>0.01 |
| Peptic Ulcer Disease; n (%) Upper Gi bleed; n (%) Lower / unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin, n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGF inhibitors; n (%) | 203 (7.3%)<br>0 (0.0%)<br>21 (0.8%)<br>91 (3.3%)<br>92 (1.0%)<br>285 (10.2%)<br>13 (0.5%)<br>9 (0.3%)<br>17 (0.6%)<br>1,098 (39.4%) | 208 (7.5%)<br>0 (0.0%)<br>24 (0.9%)<br>85 (3.0%)<br>27 (1.0%)<br>289 (10.4%)<br>9 (0.3%)<br>13 (0.5%)<br>1,087 (39.0%) | -0.01<br>#DIV/0!<br>-0.01<br>0.02<br>0.00<br>-0.01<br>0.01<br>0.00<br>0.01 | 901 (6.5%)<br>5 (0.0%)<br>104 (0.7%)<br>441 (3.2%)<br>167 (1.2%)<br>1,288 (9.2%)<br>164 (1.2%)<br>79 (0.6%)<br>68 (0.5%)<br>6,825 (48.5%) | 844 (6.0%)<br>4 (0.0%)<br>98 (0.7%)<br>429 (3.1%)<br>157 (1.1%)<br>1,288 (9.2%)<br>161 (1.2%)<br>71 (0.5%)<br>77 (0.6%)<br>6,727 (48.2%) | 0.02<br>#DIV/0!<br>0.00<br>0.01<br>0.01<br>0.00<br>0.00<br>0.01<br>-0.01 | 1,652 (7.4%)<br>0 (0.0%)<br>116 (0.5%)<br>671 (3.0%)<br>229 (1.0%)<br>2,427 (10.9%)<br>105 (0.5%)<br>90 (0.4%)<br>134 (0.6%)<br>9,742 (43.6%) | 1,633 (7.3%) ** 132 (0.6%) 628 (2.8%) 243 (1.1%) 2,334 (10.5%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) | 0.00<br>#VALUE!<br>-0.01<br>0.01<br>-0.01<br>0.01<br>0.01<br>0.00<br>0.00 | 2756 (7.1%)<br>5 (0.0%)<br>241 (0.5%)<br>1203 (3.1%)<br>425 (1.1%)<br>4000 (10.2%)<br>282 (0.7%)<br>178 (0.5%)<br>219 (0.6%)<br>17655 (45.2%) | 2685 (6.9%) #WALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) | 0.01<br>#VALUE!<br>-0.01<br>0.01<br>0.00<br>0.01<br>0.00<br>0.01<br>0.00 |
| Peptic Ulcer Disease; n (%) Upper Gl bleed; n (%) Lower/ unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin/qibyridamole; n (%) Other antiplatelet agents; n (%) PGP Inhibitors, n (%) Other gastroprotective agents; n (%) Other gastroprotective agents; n (%) | 203 (7.3%)<br>0 (0.0%)<br>21 (0.8%)<br>91 (3.3%)<br>29 (1.0%)<br>285 (10.2%)<br>13 (0.5%)<br>9 (0.3%)<br>17 (0.6%) | 208 (7.5%)<br>0 (0.0%)<br>24 (0.9%)<br>85 (3.0%)<br>27 (1.0%)<br>289 (10.4%)<br>11 (0.4%)<br>9 (0.3%)<br>13 (0.5%) | -0.01<br>#DIV/0!<br>-0.01<br>0.02<br>0.00<br>-0.01<br>0.01<br>0.00<br>0.01 | 901 (6.5%)<br>5 (0.0%)<br>104 (0.7%)<br>441 (3.2%)<br>167 (1.2%)<br>1,288 (9.2%)<br>164 (1.2%)<br>79 (0.6%)<br>68 (0.5%) | 844 (6.0%)<br>4 (0.0%)<br>98 (0.7%)<br>429 (3.1%)<br>157 (1.1%)<br>1,288 (9.2%)<br>161 (1.2%)<br>71 (0.5%)<br>77 (0.5%) | 0.02<br>#DIV/0!<br>0.00<br>0.01<br>0.01<br>0.00<br>0.00<br>0.01 | 1,652 (7.4%)<br>0 (0.0%)<br>116 (0.5%)<br>671 (3.0%)<br>229 (1.0%)<br>2,427 (10.9%)<br>105 (0.5%)<br>90 (0.4%)<br>134 (0.6%) | 1,633 (7.3%) 132 (0.5%) 628 (2.8%) 243 (1.1%) 2,334 (10.5%) 84 (0.4%) 125 (0.6%) | 0.00<br>#VALUE!<br>-0.01<br>0.01<br>-0.01<br>0.01<br>0.01<br>0.00 | 2756 (7.1%)<br>5 (0.0%)<br>241 (0.6%)<br>1203 (3.1%)<br>425 (1.1%)<br>4000 (10.2%)<br>282 (0.7%)<br>178 (0.5%)<br>219 (0.6%) | 2685 (6.9%) #WALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) | 0.01<br>#VALUE!<br>-0.01<br>0.01<br>0.00<br>0.01<br>0.00<br>0.01<br>0.00 |
| Peptic Ulcer Disease; n (%) Upper Gl bleed; n (%) Lower/ unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number Of lipid tests ordered | 203 (7.3%)<br>0 (0.0%)<br>21 (0.8%)<br>91 (3.3%)<br>92 (1.0%)<br>285 (10.2%)<br>13 (0.5%)<br>9 (0.3%)<br>17 (0.6%)<br>1,098 (39.4%)<br>19 (0.7%) | 208 (7.5%)<br>0 (0.0%)<br>24 (0.9%)<br>85 (3.0%)<br>27 (1.0%)<br>289 (10.4%)<br>9 (0.3%)<br>13 (0.5%)<br>1,087 (39.0%) | -0.01<br>#DIV/0!<br>-0.01<br>0.02<br>0.00<br>-0.01<br>0.00<br>0.01<br>0.01<br>0.01 | 901 (6.5%)<br>5 (0.0%)<br>104 (0.7%)<br>441 (3.2%)<br>167 (1.2%)<br>1,288 (9.2%)<br>164 (1.2%)<br>79 (0.6%)<br>68 (0.5%)<br>6.825 (48.9%)<br>131 (0.9%) | 844 (6.0%)<br>4 (0.0%)<br>98 (0.7%)<br>429 (3.1%)<br>157 (1.1%)<br>1,288 (9.2%)<br>161 (1.2%)<br>77 (0.5%)<br>77 (0.5%)<br>6,727 (48.2%)<br>125 (0.9%) | 0.02<br>#DIV/0!<br>0.00<br>0.01<br>0.01<br>0.00<br>0.00<br>0.01<br>-0.01<br>0.01 | 1,652 (7.4%)<br>0 (0.0%)<br>116 (0.5%)<br>671 (3.0%)<br>229 (1.0%)<br>2,427 (10.9%)<br>105 (0.5%)<br>90 (0.4%)<br>134 (0.6%)<br>9,742 (43.6%)<br>165 (0.7%) | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 2,334 (10.5%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) | 0.00<br>#VALUE!<br>-0.01<br>0.01<br>-0.01<br>0.01<br>0.00<br>0.00<br>0.00 | 2756 (7.1%)<br>5 (0.0%)<br>241 (0.6%)<br>1203 (3.1%)<br>425 (1.1%)<br>4000 (10.2%)<br>282 (0.7%)<br>178 (0.5%)<br>219 (0.6%)<br>17665 (45.2%)<br>315 (0.8%) | 2685 (6.9%) #VALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 297 (0.8%) | 0.01<br>#VALUE!<br>-0.01<br>0.01<br>0.00<br>0.01<br>0.00<br>0.01<br>0.00<br>0.01 |
| Peptic Ulcer Disease; n (%) Upper Gl bleed; n (%) Lower (unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (6d) | 203 (7.3%)<br>0 (0.0%)<br>21 (0.8%)<br>91 (3.3%)<br>29 (1.0%)<br>285 (10.2%)<br>13 (0.5%)<br>9 (0.3%)<br>17 (0.6%)<br>1,098 (39.4%)<br>19 (0.7%) | 208 (7.5%)<br>0 (0.0%)<br>24 (0.9%)<br>85 (3.0%)<br>27 (1.0%)<br>289 (10.4%)<br>11 (0.4%)<br>9 (0.3%)<br>13 (0.5%)<br>1,087 (39.0%)<br>0.68 (0.84) | -0.01<br>#DIV/0!<br>-0.01<br>0.02<br>0.00<br>-0.01<br>0.00<br>0.01<br>0.01 | 901 (6.5%)<br>5 (0.0%)<br>104 (0.7%)<br>441 (3.2%)<br>167 (1.2%)<br>1,288 (9.2%)<br>164 (1.2%)<br>79 (0.6%)<br>68 (0.5%)<br>6.825 (48.9%)<br>131 (0.9%) | 844 (6.0%)<br>4 (0.0%)<br>98 (0.7%)<br>429 (3.3%)<br>157 (1.1%)<br>1,288 (9.2%)<br>161 (1.2%)<br>77 (0.5%)<br>6,727 (48.2%)<br>125 (0.9%) | 0.02<br>#DIV/01<br>0.00<br>0.01<br>0.01<br>0.00<br>0.00<br>0.01<br>-0.01<br>0.01 | 1,652 (7.4%)<br>0 (0.0%)<br>116 (0.5%)<br>671 (3.0%)<br>229 (1.0%)<br>105 (0.5%)<br>90 (0.4%)<br>134 (0.6%)<br>9,742 (43.6%)<br>165 (0.7%) | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 156 (0.7%) | 0.00<br>#VALUE!<br>-0.01<br>-0.01<br>-0.01<br>-0.01<br>-0.01<br>-0.00<br>-0.00<br>-0.00<br>-0.00 | 2756 (7.1%)<br>5 (0.0%)<br>241 (0.6%)<br>1203 (3.1%)<br>425 (1.1%)<br>4000 (10.2%)<br>282 (0.7%)<br>178 (0.5%)<br>219 (0.6%)<br>17665 (45.2%)<br>315 (0.8%)<br>0.54 (0.81) | 2685 (6.9%) #VALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17442 (44.6%) 297 (0.8%) 0.54 (0.75) | 0.01<br>#VALUE!<br>-0.01<br>0.00<br>0.01<br>0.00<br>0.01<br>0.00<br>0.01<br>0.00 |
| Peptic Ulcer Disease; n (%) Upper Gl bleed; n (%) Lower (unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) OG hinbitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd)median [loß] | 203 (7.3%) 0 (0.0%) 21 (0.8%) 21 (0.8%) 91 (3.3%) 29 (1.0%) 285 (10.2%) 9 (0.3%) 17 (0.6%) 1,098 (39.4%) 19 (0.7%) 0.67 (0.86) 0.00 (0.00, 1.00) | 208 (7.5%)<br>0 (0.0%)<br>24 (0.9%)<br>85 (3.0%)<br>27 (1.0%)<br>289 (10.4%)<br>9 (0.3%)<br>13 (0.5%)<br>1,087 (39.0%)<br>16 (0.6%) | -0.01<br>#DIV/0!<br>-0.01<br>0.02<br>0.00<br>-0.01<br>0.01<br>0.01<br>0.01<br>0.01 | 901 (6.5%) 5 (0.0%) 104 (0.7%) 441 (3.2%) 167 (1.2%) 1,288 (9.2%) 164 (1.2%) 79 (0.6%) 68 (0.5%) 6,825 (48.9%) 131 (0.9%) 0.25 (0.70) | 844 (6.0%)<br>4 (0.0%)<br>98 (0.7%)<br>429 (3.1%)<br>157 (1.1%)<br>1,288 (9.2%)<br>161 (1.2%)<br>71 (0.5%)<br>6,727 (48.2%)<br>125 (0.9%)<br>0.24 (0.63)<br>0.00 (0.00, 0.00) | 0.02<br>#DIV/01<br>0.00<br>0.01<br>0.01<br>0.00<br>0.00<br>0.01<br>-0.01<br>0.00 | 1,652 (7.4%)<br>0 (0.0%)<br>116 (0.5%)<br>671 (3.0%)<br>229 (1.0%)<br>2,427 (10.9%)<br>105 (0.5%)<br>90 (0.4%)<br>134 (0.6%)<br>9,742 (43.6%)<br>165 (0.7%)<br>0.71 (0.86) | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 2,334 (10.5%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 156 (0.7%) 0.71 (0.81) 1.00 (0.00, 1.00) | 0.00 #VALUE! -0.01 -0.01 -0.01 -0.01 -0.01 -0.01 -0.00 -0.00 -0.00 -0.00 -0.00 -0.00 -0.00 | 2756 (7.1%)<br>5 (0.0%)<br>241 (0.6%)<br>1203 (3.1%)<br>425 (1.1%)<br>4000 (10.2%)<br>282 (0.7%)<br>178 (0.5%)<br>219 (0.6%)<br>17665 (45.2%)<br>315 (0.8%)<br>0.54 (0.81)<br>0.36 (0.87) | 2685 (6.9%) #VALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 297 (0.8%) 0.54 (0.75) 0.43 (0.81) | 0.01<br>#VALUE!<br>-0.01<br>0.00<br>0.01<br>0.00<br>0.01<br>0.00<br>0.01<br>0.00 |
| Peptic Uter Disease; n (%) Upper Gi bleed; n (%) Lower/ unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin; n (%) Aspirinj dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd)median [LQR] Proton pump inhibitor; n (%) | 203 (7.3%)<br>0 (0.0%)<br>21 (0.8%)<br>91 (3.3%)<br>92 (1.0%)<br>285 (10.2%)<br>13 (0.5%)<br>9 (0.3%)<br>17 (0.6%)<br>1,098 (39.4%)<br>19 (0.7%)<br>0.67 (0.86)<br>0.00 [0.00, 1.00] | 208 (7.5%)<br>0 (0.0%)<br>24 (0.9%)<br>85 (3.0%)<br>27 (1.0%)<br>289 (10.4%)<br>9 (0.3%)<br>13 (0.5%)<br>1,087 (39.0%)<br>16 (0.6%)<br>0.68 (0.84)<br>1.00 (0.00, 1.00)<br>440 (15.8%) | -0.01 #DIV/0! -0.01 -0.02 -0.00 -0.01 -0.01 -0.00 -0.01 -0.01 -0.01 -0.01 -1.18 -0.03 | 901 (6.5%) 5 (0.0%) 104 (0.7%) 441 (3.2%) 167 (1.2%) 1,288 (9.2%) 164 (1.2%) 79 (0.6%) 68 (0.5%) 6.825 (48.9%) 131 (0.9%) 0.25 (0.70) 0.00 (0.00, 0.00) 2,736 (19.6%) | 844 (6.0%)<br>4 (0.0%)<br>98 (0.7%)<br>429 (3.1%)<br>157 (1.1%)<br>1,288 (9.2%)<br>161 (1.2%)<br>77 (0.6%)<br>6,727 (48.2%)<br>125 (0.9%)<br>0.24 (0.63)<br>0.00 (0.00, 0.00)<br>2,724 (19.5%) | 0.02<br>#DIV/01<br>0.00<br>0.01<br>0.01<br>0.00<br>0.00<br>0.01<br>-0.01<br>0.01 | 1,652 (7.4%)<br>0 (0.0%)<br>116 (0.5%)<br>671 (3.0%)<br>229 (1.0%)<br>2,427 (10.9%)<br>105 (0.5%)<br>90 (0.4%)<br>134 (0.6%)<br>9,742 (43.6%)<br>165 (0.7%)<br>0.71 (0.86)<br>1.00 (0.00, 1.00)<br>4,221 (18.9%) | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 2,334 (10.5%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 156 (0.7%) 0.71 (0.81) 1.00 (0.00) 1.00] 4,253 (19.1%) | 0.00 #VALUEI -0.01 -0.01 -0.01 -0.01 -0.01 -0.01 -0.00 -0.00 -0.00 -0.00 -0.00 -0.00 -0.00 | 2756 (7.1%)<br>5 (0.0%)<br>241 (0.6%)<br>1203 (3.1%)<br>425 (1.1%)<br>4000 (10.2%)<br>282 (0.7%)<br>178 (0.5%)<br>219 (0.6%)<br>17665 (45.2%)<br>315 (0.8%)<br>0.54 (0.81)<br>0.36 (0.87)<br>7427 (19.0%) | 2685 (6.9%) #VALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 297 (0.8%) 0.54 (0.75) 0.43 (0.81) 7417 (19.0%) | 0.01 #VALUE! -0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.00 |
| Peptic Ulcer Disease; n (%) Upper Gl bleed; n (%) Lower/ unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleed; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP Inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (6d)median [IQR] Proton pump Inhibitor; n (%) H2 receptor antagonist; n (%) | 203 (7.3%) 0 (0.0%) 21 (0.8%) 91 (3.3%) 29 (1.0%) 285 (10.2%) 13 (0.5%) 9 (0.3%) 17 (0.6%) 1,098 (39.4%) 19 (0.7%) 0.67 (0.86) 0.00 (0.00,1.00) 470 (16.8%) 91 (3.3%) | 208 (7.5%)<br>0 (0.0%)<br>24 (0.9%)<br>85 (3.0%)<br>27 (1.0%)<br>11 (0.4%)<br>9 (0.3%)<br>13 (0.5%)<br>1,087 (39.0%)<br>16 (0.6%)<br>0.68 (0.84)<br>1.00 (0.00, 1.00)<br>440 (15.8%)<br>93 (3.3%) | -0.01 #DIV/0! -0.01 -0.02 -0.00 -0.01 -0.00 | 901 (6.5%) 5 (0.0%) 104 (0.7%) 441 (3.2%) 167 (1.2%) 1,288 (9.2%) 164 (1.2%) 79 (0.6%) 68 (0.5%) 6,825 (48.9%) 131 (0.9%) 0.25 (0.70) 0.00 (0.00, 0.00) 2,736 (19.6%) 384 (2.8%) | 844 (6.0%)<br>4 (0.0%)<br>98 (0.7%)<br>429 (3.3%)<br>157 (1.1%)<br>1,288 (9.2%)<br>161 (1.2%)<br>71 (0.5%)<br>6,727 (48.2%)<br>125 (0.9%)<br>0.24 (0.63)<br>0.00 (0.00, 0.00)<br>2,724 (19.5%)<br>399 (2.9%) | 0.02<br>#DIV/01<br>0.00<br>0.01<br>0.01<br>0.00<br>0.00<br>0.01<br>-0.01<br>0.00<br>0.00 | 1,652 (7.4%) 0 (0.0%) 116 (0.5%) 671 (3.0%) 229 (1.0%) 105 (0.5%) 90 (0.4%) 134 (0.6%) 9,742 (43.6%) 105 (0.7%) 0.71 (0.86) 1.00 (0.00, 1.00) 4,221 (18.9%) 917 (4.1%) | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 624 (3.11%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 156 (0.7%) 0.71 (0.81) 1.00 (0.00, 1.00) 4,253 (19.1%) 890 (4.0%) | 0.00 #WALUEI -0.01 0.01 -0.01 0.01 0.01 0.00 0.00 0. | 2756 (7.1%)<br>5 (0.0%)<br>241 (0.6%)<br>1203 (3.1%)<br>425 (1.1%)<br>4000 (10.2%)<br>282 (0.7%)<br>178 (0.5%)<br>219 (0.6%)<br>17665 (45.2%)<br>315 (0.8%)<br>0.54 (0.81)<br>0.36 (0.87)<br>7427 (19.0%)<br>1392 (3.6%) | 2685 (6.9%) #VALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 297 (0.8%) 0.54 (0.75) 0.43 (0.81) 7417 (19.0%) 1382 (3.5%) | #VALUE! -0.01 0.01 0.01 0.00 |
| Peptic Ulcer Disease; n (%) Upper Gi bleed; n (%) Lower (unspecified Gi bleed; n (%) Urogenital bleed; n (%) Urogenital bleed; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGF inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd)median [loR] Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) | 203 (7.3%)<br>0 (0.0%)<br>21 (0.8%)<br>91 (3.3%)<br>92 (1.0%)<br>285 (10.2%)<br>13 (0.5%)<br>9 (0.3%)<br>17 (0.6%)<br>1,098 (39.4%)<br>19 (0.7%)<br>0.67 (0.86)<br>0.00 [0.00, 1.00] | 208 (7.5%)<br>0 (0.0%)<br>24 (0.9%)<br>85 (3.0%)<br>27 (1.0%)<br>289 (10.4%)<br>9 (0.3%)<br>13 (0.5%)<br>1,087 (39.0%)<br>16 (0.6%)<br>0.68 (0.84)<br>1.00 (0.00, 1.00)<br>440 (15.8%) | -0.01 #DIV/0! -0.01 -0.02 -0.00 -0.01 -0.01 -0.00 -0.01 -0.01 -0.01 -0.01 -1.18 -0.03 | 901 (6.5%) 5 (0.0%) 104 (0.7%) 441 (3.2%) 167 (1.2%) 1,288 (9.2%) 164 (1.2%) 79 (0.6%) 68 (0.5%) 6.825 (48.9%) 131 (0.9%) 0.25 (0.70) 0.00 (0.00, 0.00) 2,736 (19.6%) | 844 (6.0%)<br>4 (0.0%)<br>98 (0.7%)<br>429 (3.1%)<br>157 (1.1%)<br>1,288 (9.2%)<br>161 (1.2%)<br>77 (0.6%)<br>6,727 (48.2%)<br>125 (0.9%)<br>0.24 (0.63)<br>0.00 (0.00, 0.00)<br>2,724 (19.5%) | 0.02<br>#DIV/01<br>0.00<br>0.01<br>0.01<br>0.00<br>0.00<br>0.01<br>-0.01<br>0.01 | 1,652 (7.4%)<br>0 (0.0%)<br>116 (0.5%)<br>671 (3.0%)<br>229 (1.0%)<br>2,427 (10.9%)<br>105 (0.5%)<br>90 (0.4%)<br>134 (0.6%)<br>9,742 (43.6%)<br>165 (0.7%)<br>0.71 (0.86)<br>1.00 (0.00, 1.00)<br>4,221 (18.9%) | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 2,334 (10.5%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 156 (0.7%) 0.71 (0.81) 1.00 (0.00) 1.00] 4,253 (19.1%) | 0.00 #VALUEI -0.01 -0.01 -0.01 -0.01 -0.01 -0.01 -0.00 -0.00 -0.00 -0.00 -0.00 -0.00 -0.00 | 2756 (7.1%)<br>5 (0.0%)<br>241 (0.6%)<br>1203 (3.1%)<br>425 (1.1%)<br>4000 (10.2%)<br>282 (0.7%)<br>178 (0.5%)<br>219 (0.6%)<br>17665 (45.2%)<br>315 (0.8%)<br>0.54 (0.81)<br>0.36 (0.87)<br>7427 (19.0%) | 2685 (6.9%) #VALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 297 (0.8%) 0.54 (0.75) 0.43 (0.81) 7417 (19.0%) | 0.01 #VALUE! -0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.00 |
| Peptic Ulcer Disease; n (%) Upper Gl bleed; n (%) Lower (unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (6d)median [IGR] Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) | 203 (7.3%) 0 (0.0%) 21 (0.8%) 91 (3.3%) 29 (1.0%) 285 (10.2%) 13 (0.5%) 9 (0.3%) 17 (0.6%) 1,098 (39.4%) 0.67 (0.86) 0.00 (0.00, 1.00) 470 (16.8%) 91 (3.3%) 0 (0.0%) | 208 (7.5%) 0 (0.0%) 24 (0.9%) 85 (3.0%) 27 (1.0%) 289 (10.4%) 11 (0.4%) 9 (0.3%) 13 (0.5%) 1,087 (39.0%) 0.68 (0.84) 1.00 (0.00, 1.00) 440 (15.8%) 93 (3.3%) 0 (0.0%) | -0.01 #DIV/0! -0.01 -0.02 -0.00 -0.01 -0.01 -0.01 -0.01 -0.01 -0.01 -0.01 -1.18 -0.03 -0.00 #DIV/0! | 901 (6.5%) 5 (0.0%) 104 (0.7%) 441 (3.2%) 167 (1.2%) 167 (1.2%) 1,288 (9.2%) 164 (1.2%) 79 (0.6%) 68 (0.5%) 6.825 (48.9%) 131 (0.9%) 0.25 (0.70) 0.00 (0.00, 0.00) 2,73 6 (19.6%) 384 (2.8%) 11 (0.1%) | 844 (6.0%) 4 (0.0%) 98 (0.7%) 429 (3.1%) 157 (1.1%) 1,288 (9.2%) 161 (1.2%) 77 (0.5%) 77 (0.5%) 6,727 (48.2%) 125 (0.9%) 0.24 (0.63) 0.00 (0.00, 0.00) 2,724 (19.5%) 399 (2.9%) 8 (0.1%) | 0.02<br>#DIV/01<br>0.00<br>0.01<br>0.01<br>0.00<br>0.00<br>0.01<br>0.01<br>0 | 1,652 (7.4%) 0 (0.0%) 116 (0.5%) 671 (3.0%) 229 (1.0%) 105 (0.5%) 90 (0.4%) 134 (0.6%) 9,742 (43.6%) 1,742 (43.6%) 0.71 (0.86) 1.00 (0.00,1.00) 4,221 (18.9%) 917 (4.1%) 4 (0.0%) | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 0.71 (0.81) 1.00 (0.00, 1.00) 4,253 (19.1%) 890 (4.0%) 4 (0.0%) | 0.00 #WALUEI -0.01 0.01 -0.01 0.01 0.01 0.00 0.00 0. | 2756 (7.1%) 5 (0.0%) 241 (0.6%) 1203 (3.1%) 425 (1.1%) 4000 (10.2%) 282 (0.7%) 178 (0.5%) 219 (0.6%) 17665 (45.2%) 315 (0.8%) 0.54 (0.81) 0.36 (0.87) 7427 (19.0%) 1392 (3.6%) | 2685 (6.9%) #VALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 297 (0.8%) 0.54 (0.75) 0.43 (0.81) 7417 (19.0%) 1382 (3.5%) 12 (0.0%) | #VALUE! -0.01 0.01 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 |
| Peptic Ulcer Disease; n (%) Upper Gi bleed; n (%) Lower (unspecified Gi bleed; n (%) Urogenital bleed; n (%) Urogenital bleed; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGF inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd)median [loR] Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) | 203 (7.3%) 0 (0.0%) 21 (0.8%) 21 (0.8%) 91 (3.3%) 29 (1.0%) 13 (0.5%) 9 (0.3%) 17 (0.6%) 1,098 (39.4%) 19 (0.7%) 0.67 (0.86) 0.00 (0.00, 1.00) 470 (16.8%) 91 (3.3%) 0 (0.0%) | 208 (7.5%) 0 (0.0%) 24 (0.9%) 85 (3.0%) 27 (1.0%) 289 (10.4%) 9 (0.3%) 13 (0.5%) 1,087 (39.0%) 16 (0.6%) 0.68 (0.84) 1.00 (0.00, 1.00) 440 (15.8%) 93 (3.3%) 0 (0.0%) | -0.01 #DIV/0! -0.01 0.02 0.00 -0.01 0.01 0.01 0.01 0.01 -1.18 0.03 0.00 #DIV/0! | 901 (6.5%) 5 (0.0%) 104 (0.7%) 441 (3.2%) 167 (1.2%) 168 (9.2%) 164 (1.2%) 79 (0.6%) 68 (0.5%) 6.825 (48.3%) 131 (0.9%) 0.25 (0.70) 0.00 (0.00, 0.00) 2,736 (19.6%) 384 (2.8%) 11 (0.1%) 0.20 (1.18) | 844 (6.0%) 4 (0.0%) 98 (0.7%) 429 (3.1%) 157 (1.1%) 1,288 (9.2%) 161 (1.2%) 71 (0.5%) 77 (0.6%) 6,727 (48.2%) 125 (0.9%) 0.24 (0.63) 0.00 (0.00, 0.00) 2,724 (19.5%) 399 (2.9%) 8 (0.1%) 0.20 (1.00) | 0.02<br>#DIV/01<br>0.00<br>0.01<br>0.01<br>0.00<br>0.00<br>0.01<br>-0.01<br>0.00<br>0.00 | 1,652 (7.4%)<br>0 (0.0%)<br>116 (0.5%)<br>671 (3.0%)<br>229 (1.0%)<br>2,427 (10.9%)<br>105 (0.5%)<br>90 (0.4%)<br>134 (0.6%)<br>9,742 (43.6%)<br>165 (0.7%)<br>0.71 (0.86)<br>1.00 (0.00, 1.00)<br>4,221 (18.9%)<br>917 (4.1%)<br>4 (0.0%) | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 2,334 (10.5%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 156 (0.7%) 0.71 (0.81) 1.00 (0.00, 1.00) 4,253 (19.1%) 890 (4.0%) 4 (0.0%) | 0.00 #WALUEI -0.01 0.01 -0.01 0.01 0.01 0.00 0.00 0. | 2756 (7.1%)<br>5 (0.0%)<br>241 (0.6%)<br>1203 (3.1%)<br>425 (1.1%)<br>4000 (10.2%)<br>282 (0.7%)<br>178 (0.5%)<br>219 (0.6%)<br>17665 (45.2%)<br>315 (0.8%)<br>0.54 (0.81)<br>0.36 (0.87)<br>7427 (19.0%)<br>1392 (3.6%)<br>15 (0.0%) | 2685 (6.9%) #VALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 297 (0.8%) 0.54 (0.75) 0.43 (0.81) 7417 (19.0%) 1382 (3.5%) | 0.01 #VALUE! -0.01 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 |
| Peptic Ulcer Disease; n (%) Upper Gl bleed; n (%) Lower (unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (6d)median [IGR] Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) | 203 (7.3%) 0 (0.0%) 21 (0.8%) 91 (3.3%) 29 (1.0%) 285 (10.2%) 13 (0.5%) 9 (0.3%) 17 (0.6%) 1,098 (39.4%) 0.67 (0.86) 0.00 (0.00, 1.00) 470 (16.8%) 91 (3.3%) 0 (0.0%) | 208 (7.5%) 0 (0.0%) 24 (0.9%) 85 (3.0%) 27 (1.0%) 289 (10.4%) 11 (0.4%) 9 (0.3%) 13 (0.5%) 1,087 (39.0%) 0.68 (0.84) 1.00 (0.00, 1.00) 440 (15.8%) 93 (3.3%) 0 (0.0%) | -0.01 #DIV/0! -0.01 -0.02 -0.00 -0.01 -0.01 -0.01 -0.01 -0.01 -0.01 -0.01 -1.18 -0.03 -0.00 #DIV/0! | 901 (6.5%) 5 (0.0%) 104 (0.7%) 441 (3.2%) 167 (1.2%) 167 (1.2%) 1,288 (9.2%) 164 (1.2%) 79 (0.6%) 68 (0.5%) 6.825 (48.9%) 131 (0.9%) 0.25 (0.70) 0.00 (0.00, 0.00) 2,73 6 (19.6%) 384 (2.8%) 11 (0.1%) | 844 (6.0%) 4 (0.0%) 98 (0.7%) 429 (3.1%) 157 (1.1%) 1,288 (9.2%) 161 (1.2%) 77 (0.5%) 77 (0.5%) 6,727 (48.2%) 125 (0.9%) 0.24 (0.63) 0.00 (0.00, 0.00) 2,724 (19.5%) 399 (2.9%) 8 (0.1%) | 0.02<br>#DIV/01<br>0.00<br>0.01<br>0.01<br>0.00<br>0.00<br>0.01<br>0.01<br>0 | 1,652 (7.4%) 0 (0.0%) 116 (0.5%) 671 (3.0%) 229 (1.0%) 105 (0.5%) 90 (0.4%) 134 (0.6%) 9,742 (43.6%) 1,742 (43.6%) 0.71 (0.86) 1.00 (0.00,1.00) 4,221 (18.9%) 917 (4.1%) 4 (0.0%) | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 0.71 (0.81) 1.00 (0.00, 1.00) 4,253 (19.1%) 890 (4.0%) 4 (0.0%) | 0.00 #WALUEI -0.01 0.01 -0.01 0.01 0.01 0.00 0.00 0. | 2756 (7.1%) 5 (0.0%) 241 (0.6%) 1203 (3.1%) 425 (1.1%) 4000 (10.2%) 282 (0.7%) 178 (0.5%) 219 (0.6%) 17665 (45.2%) 315 (0.8%) 0.54 (0.81) 0.36 (0.87) 7427 (19.0%) 1392 (3.6%) | 2685 (6.9%) #VALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 297 (0.8%) 0.54 (0.75) 0.43 (0.81) 7417 (19.0%) 1382 (3.5%) 12 (0.0%) | #VALUE! -0.01 0.01 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 |
| Peptic Ulcer Disease; n (%) Upper Gl bleed; n (%) Lower Unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP Inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd)median [IQR] Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of neurologist visitsmean (sd) | 203 (7.3%) 0 (0.0%) 21 (0.8%) 21 (0.8%) 91 (3.3%) 29 (1.0%) 13 (0.5%) 9 (0.3%) 17 (0.6%) 1,098 (39.4%) 19 (0.7%) 0.67 (0.86) 0.00 (0.00, 1.00) 470 (16.8%) 91 (3.3%) 0 (0.0%) | 208 (7.5%) 0 (0.0%) 24 (0.9%) 85 (3.0%) 27 (1.0%) 289 (10.4%) 9 (0.3%) 13 (0.5%) 1,087 (39.0%) 16 (0.6%) 0.68 (0.84) 1.00 (0.00, 1.00) 440 (15.8%) 93 (3.3%) 0 (0.0%) | -0.01 #DIV/0! -0.01 0.02 0.00 -0.01 0.01 0.01 0.01 0.01 -1.18 0.03 0.00 #DIV/0! | 901 (6.5%) 5 (0.0%) 104 (0.7%) 441 (3.2%) 167 (1.2%) 168 (9.2%) 164 (1.2%) 79 (0.6%) 68 (0.5%) 6.825 (48.3%) 131 (0.9%) 0.25 (0.70) 0.00 (0.00, 0.00) 2,736 (19.6%) 384 (2.8%) 11 (0.1%) 0.20 (1.18) | 844 (6.0%) 4 (0.0%) 98 (0.7%) 429 (3.1%) 157 (1.1%) 1,288 (9.2%) 161 (1.2%) 71 (0.5%) 77 (0.6%) 6,727 (48.2%) 125 (0.9%) 0.24 (0.63) 0.00 (0.00, 0.00) 2,724 (19.5%) 399 (2.9%) 8 (0.1%) 0.20 (1.00) | 0.02<br>#DIV/01<br>0.00<br>0.01<br>0.01<br>0.00<br>0.00<br>0.01<br>-0.01<br>0.00<br>0.00 | 1,652 (7.4%)<br>0 (0.0%)<br>116 (0.5%)<br>671 (3.0%)<br>229 (1.0%)<br>2,427 (10.9%)<br>105 (0.5%)<br>90 (0.4%)<br>134 (0.6%)<br>9,742 (43.6%)<br>165 (0.7%)<br>0.71 (0.86)<br>1.00 (0.00, 1.00)<br>4,221 (18.9%)<br>917 (4.1%)<br>4 (0.0%) | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 2,334 (10.5%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 156 (0.7%) 0.71 (0.81) 1.00 (0.00, 1.00) 4,253 (19.1%) 890 (4.0%) 4 (0.0%) | 0.00 #WALUEI -0.01 0.01 0.01 0.01 0.01 0.00 0.00 0.0 | 2756 (7.1%)<br>5 (0.0%)<br>241 (0.6%)<br>1203 (3.1%)<br>425 (1.1%)<br>4000 (10.2%)<br>282 (0.7%)<br>178 (0.5%)<br>219 (0.6%)<br>17665 (45.2%)<br>315 (0.8%)<br>0.54 (0.81)<br>0.36 (0.87)<br>7427 (19.0%)<br>1392 (3.6%)<br>15 (0.0%) | 2685 (6.9%) #VALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 297 (0.8%) 0.54 (0.75) 0.43 (0.81) 7417 (19.0%) 1382 (3.5%) 12 (0.0%) | 0.01 #VALUE! -0.01 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 |
| Peptic Ulcer Disease; n (%) Upper Gi bleed; n (%) Lower/ unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin; n (%) Aspirinj dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd)median [loR] Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin Ktherapy; n (%) Number of neurologist visitsmean (sd)mean (sd)mean (sd)mean (sd)mean (sd)mean (sd)mean (sd)median [loR] | 203 (7.3%) 0 (0.0%) 21 (0.8%) 21 (0.8%) 91 (3.3%) 29 (1.0%) 13 (0.5%) 9 (0.3%) 17 (0.6%) 1,098 (39.4%) 19 (0.7%) 0.67 (0.86) 0.00 (0.00, 1.00) 470 (16.8%) 91 (3.3%) 0 (0.0%) | 208 (7.5%) 0 (0.0%) 24 (0.9%) 85 (3.0%) 27 (1.0%) 289 (10.4%) 9 (0.3%) 13 (0.5%) 1,087 (39.0%) 16 (0.6%) 0.68 (0.84) 1.00 (0.00, 1.00) 440 (15.8%) 93 (3.3%) 0 (0.0%) | -0.01 #DIV/0! -0.01 0.02 0.00 -0.01 0.01 0.01 0.01 0.01 -1.18 0.03 0.00 #DIV/0! | 901 (6.5%) 5 (0.0%) 104 (0.7%) 441 (3.2%) 167 (1.2%) 168 (9.2%) 164 (1.2%) 79 (0.6%) 68 (0.5%) 6.825 (48.3%) 131 (0.9%) 0.25 (0.70) 0.00 (0.00, 0.00) 2,736 (19.6%) 384 (2.8%) 11 (0.1%) 0.20 (1.18) | 844 (6.0%) 4 (0.0%) 98 (0.7%) 429 (3.1%) 157 (1.1%) 1,288 (9.2%) 161 (1.2%) 71 (0.5%) 77 (0.6%) 6,727 (48.2%) 125 (0.9%) 0.24 (0.63) 0.00 (0.00, 0.00) 2,724 (19.5%) 399 (2.9%) 8 (0.1%) 0.20 (1.00) | 0.02<br>#DIV/01<br>0.00<br>0.01<br>0.01<br>0.00<br>0.00<br>0.01<br>-0.01<br>0.00<br>0.00 | 1,652 (7.4%)<br>0 (0.0%)<br>116 (0.5%)<br>671 (3.0%)<br>229 (1.0%)<br>2,427 (10.9%)<br>105 (0.5%)<br>90 (0.4%)<br>134 (0.6%)<br>9,742 (43.6%)<br>165 (0.7%)<br>0.71 (0.86)<br>1.00 (0.00, 1.00)<br>4,221 (18.9%)<br>917 (4.1%)<br>4 (0.0%) | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 2,334 (10.5%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 156 (0.7%) 0.71 (0.81) 1.00 (0.00, 1.00) 4,253 (19.1%) 890 (4.0%) 4 (0.0%) | 0.00 #WALUEI -0.01 0.01 0.01 0.01 0.01 0.00 0.00 0.0 | 2756 (7.1%)<br>5 (0.0%)<br>241 (0.6%)<br>1203 (3.1%)<br>425 (1.1%)<br>4000 (10.2%)<br>282 (0.7%)<br>178 (0.5%)<br>219 (0.6%)<br>17665 (45.2%)<br>315 (0.8%)<br>0.54 (0.81)<br>0.36 (0.87)<br>7427 (19.0%)<br>1392 (3.6%)<br>15 (0.0%) | 2685 (6.9%) #VALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 297 (0.8%) 0.54 (0.75) 0.43 (0.81) 7417 (19.0%) 1382 (3.5%) 12 (0.0%) | 0.01 #VALUE! -0.01 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 |
| Peptic Ulcer Disease; n (%) Upper Gl bleed; n (%) Lower Unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (6d)median [IQR] Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of neurologist visitsmean (6d)median [IQR] Number of INR (prothrombin) tests ordered | 203 (7.3%) 0 (0.0%) 21 (0.8%) 21 (0.8%) 91 (3.3%) 29 (1.0%) 13 (0.5%) 9 (0.3%) 17 (0.6%) 1,098 (39.4%) 19 (0.7%) 0.67 (0.86) 0.00 (0.00,1.00) 470 (16.8%) 91 (3.3%) 0 (0.0%) 0.16 (0.98) | 208 (7.5%) 0 (0.0%) 24 (0.9%) 85 (3.0%) 27 (1.0%) 11 (0.4%) 9 (0.3%) 13 (0.5%) 1,087 (39.0%) 16 (0.6%) 0.68 (0.84) 1.00 (0.00, 1.00) 440 (15.8%) 93 (3.3%) 0 (0.0%) 0.16 (0.97) 0.00 [0.00, 0.00] | -0.01<br>#DIV/0!<br>-0.01<br>0.02<br>0.00<br>-0.01<br>0.01<br>0.01<br>0.01<br>-1.18<br>0.03<br>0.00<br>#DIV/0! | 901 (6.5%) 5 (0.0%) 104 (0.7%) 441 (3.2%) 167 (1.2%) 168 (9.2%) 164 (1.2%) 79 (0.6%) 68 (0.5%) 6,825 (48.9%) 131 (0.9%) 0.25 (0.70) 0.00 (0.00, 0.00) 2,736 (19.6%) 384 (2.8%) 11 (0.1%) 0.20 (1.18) 0.00 (0.00, 0.00) | 844 (6.0%) 4 (0.0%) 98 (0.7%) 429 (3.1%) 157 (1.1%) 1,288 (9.2%) 161 (1.2%) 71 (0.5%) 77 (0.5%) 6,727 (48.2%) 125 (0.5%) 0.24 (0.63) 0.00 (0.00, 0.00) 2,724 (19.5%) 399 (2.5%) 8 (0.1%) 0.20 (1.00) 0.00 (0.00, 0.00) | 0.02<br>#DIV/01<br>0.00<br>0.01<br>0.01<br>0.00<br>0.01<br>-0.01<br>0.01<br>0 | 1,652 (7.4%) 0 (0.0%) 116 (0.5%) 671 (3.0%) 229 (1.0%) 105 (0.5%) 90 (0.4%) 134 (0.6%) 9,742 (43.6%) 1.00 (0.0,0.1.00) 4,221 (18.9%) 917 (4.1%) 4 (0.0%) 0.24 (1.44) | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 156 (0.7%) 0.71 (0.81) 1.00 (0.00, 1.00) 4,253 (19.1%) 890 (4.0%) 4 (0.0%) 0.23 (1.23) 0.00 [0.00, 0.00] | 0.00 #WALUEI -0.01 0.01 0.01 0.01 0.01 0.00 0.00 0.0 | 2756 (7.1%) 5 (0.0%) 241 (0.6%) 1203 (3.1%) 425 (1.1%) 4800 (10.2%) 282 (0.7%) 178 (0.5%) 219 (0.6%) 17665 (45.2%) 315 (0.8%) 0.54 (0.81) 0.36 (0.87) 7427 (19.0%) 1392 (3.6%) 15 (0.0%) 0.22 (1.32) 0.00 (1.43) | 2685 (6.9%) #VALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 297 (0.8%) 0.54 (0.75) 0.43 (0.81) 7417 (19.0%) 1382 (3.5%) 12 (0.0%) 0.21 (1.14) 0.00 (1.23) | 0.01 #/ALUE! -0.01 0.01 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 #/BUV/01 |
| Peptic Ulcer Disease; n (%) Upper Gl bleed; n (%) Lower Junspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Other plate of the company of the com | 203 (7.3%) 0 (0.0%) 21 (0.8%) 91 (3.3%) 29 (1.0%) 13 (0.5%) 9 (0.3%) 17 (0.6%) 1,098 (39.4%) 0.67 (0.86) 0.00 (0.00, 1.00) 470 (16.8%) 9 (3.3%) 0 (0.0%) 0.16 (0.98) 0.00 (0.00, 0.00) | 208 (7.5%) 0 (0.0%) 24 (0.9%) 85 (3.0%) 27 (1.0%) 289 (10.4%) 11 (0.4%) 9 (0.3%) 13 (0.5%) 1,087 (39.0%) 0.68 (0.84) 1.00 (0.00, 1.00) 440 (15.8%) 93 (3.3%) 0 (0.0%) 0.16 (0.97) 0.00 (0.00, 0.00) 0.36 (1.33) 0.00 (0.00, 0.00) | -0.01 #DIV/0! -0.01 0.02 0.00 -0.01 0.01 0.01 0.01 0.01 -0.01 -1.18 0.03 0.00 #DIV/0! | 901 (6.5%) 5 (0.0%) 104 (0.7%) 441 (3.2%) 167 (1.2%) 167 (1.2%) 1,288 (9.2%) 164 (1.2%) 79 (0.6%) 68 (0.5%) 6.825 (48.9%) 131 (0.9%) 0.25 (0.70) 0.00 (0.00, 0.00) 2,736 (19.5%) 384 (2.8%) 11 (0.1%) 0.20 (1.18) 0.00 (0.00, 0.00) | 844 (6.0%) 4 (0.0%) 98 (0.7%) 429 (3.1%) 157 (1.1%) 1,288 (9.2%) 161 (1.2%) 77 (0.5%) 77 (0.5%) 6,727 (48.2%) 125 (0.9%) 0.24 (0.63) 0.00 (0.00, 0.00) 2,724 (19.5%) 399 (2.9%) 8 (0.1%) 0.20 (1.00) 0.00 (0.00, 0.00) | 0.02<br>#DIV/01<br>0.00<br>0.01<br>0.01<br>0.01<br>0.01<br>0.01<br>0.01<br>0 | 1,652 (7.4%) 0 (0.0%) 116 (0.5%) 671 (3.0%) 229 (1.0%) 105 (0.5%) 90 (0.4%) 134 (0.6%) 9,742 (43.6%) 0.71 (0.86) 1.00 [0.00, 1.00] 4,221 (18.9%) 917 (4.1%) 4 (0.0%) 0.24 (1.44) 0.00 [0.00, 0.00] | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 156 (0.7%) 0.71 (0.81) 1.00 (0.00, 1.00) 4,253 (19.1%) 890 (4.0%) 4 (0.0%) 0.23 (1.23) 0.00 (0.00, 0.00) 0.41 (1.34) 0.00 (0.00, 0.00) | 0.00 #WALUEI -0.01 0.01 0.01 0.01 0.01 0.00 0.00 0.0 | 2756 (7.1%) 5 (0.0%) 241 (0.6%) 1203 (3.1%) 425 (1.1%) 4000 (10.2%) 282 (0.7%) 178 (0.5%) 219 (0.6%) 17665 (45.2%) 315 (0.8%) 0.54 (0.81) 0.36 (0.87) 7427 (19.0%) 1392 (3.6%) 15 (0.0%) 0.22 (1.32) 0.00 (1.43) 0.41 (1.19) | 2685 (6.9%) #VALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 297 (0.8%) 0.54 (0.75) 0.43 (0.81) 7417 (19.0%) 1382 (3.5%) 12 (0.0%) 0.21 (1.14) 0.00 (1.23) 0.37 (1.32) | 0.01 #/ALUE! -0.01 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 |
| Peptic Ulcer Disease; n (%) Upper Gl bleed; n (%) Lower Unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP Inhibitors; n (%) OCHER gastroprotective agents; n (%) Number of lipid tests orderedmean (sd)median [lQR] Proton pump inhibitor; n (%) Vitamin K therapy; n (%) Number of neurologist visitsmean (sd)median [lQR] Number of INR (prothrombin) tests orderedmean (sd)median [lQR] Treating prescriber - Cardiologist; n (%) | 203 (7.3%) 0 (0.0%) 21 (0.8%) 91 (3.3%) 29 (1.0%) 13 (0.5%) 9 (0.3%) 17 (0.6%) 1,098 (39.4%) 19 (0.7%) 0.67 (0.86) 0.00 [0.00, 1.00] 470 (16.8%) 91 (3.3%) 0 (0.0%) 0.16 (0.98) 0.00 [0.00, 0.00] 0.41 (1.13) 0.00 [0.00, 0.00] 1,281 (45.9%) | 208 (7.5%) 0 (0.0%) 24 (0.9%) 85 (3.0%) 27 (1.0%) 289 (10.4%) 9 (0.3%) 13 (0.5%) 1,087 (39.0%) 16 (0.6%) 0.68 (0.84) 1.00 (0.00, 1.00) 440 (15.8%) 93 (3.3%) 0 (0.0%) 0.16 (0.97) 0.00 [0.00, 0.00] 0.36 (1.33) 0.00 (0.00, 0.00] 1,280 (45.9%) | -0.01 -0.01 0.02 0.00 -0.01 0.01 0.01 0.01 0.01 0.01 -1.18 0.03 0.00 #DIV/0! | 901 (6.5%) 5 (0.0%) 104 (0.7%) 441 (3.2%) 167 (1.2%) 167 (1.2%) 168 (9.2%) 164 (1.2%) 79 (0.6%) 68 (0.5%) 6,825 (48.9%) 131 (0.9%) 0.25 (0.70) 0.00 (0.00, 0.00) 2,736 (19.6%) 384 (2.8%) 11 (0.1%) 0.20 (1.18) 0.00 (0.00, 0.00) 0.36 (1.18) 0.00 (0.00, 0.00) 7,610 (54.5%) | 844 (6.0%) 4 (0.0%) 98 (0.7%) 98 (0.7%) 429 (3.1%) 1.57 (1.1%) 1,288 (9.2%) 161 (1.2%) 71 (0.5%) 6,727 (48.2%) 125 (0.9%) 0.24 (0.63) 0.00 (0.00, 0.00) 2,724 (19.5%) 399 (2.9%) 8 (0.1%) 0.20 (1.00) 0.00 (0.00, 0.00) 0.30 (1.28) 0.00 (0.00, 0.00) 7,447 (53.3%) | 0.02<br>#DIV/01<br>0.00<br>0.01<br>0.01<br>0.00<br>0.00<br>0.01<br>0.01<br>0 | 1,652 (7.4%) 0 (0.0%) 116 (0.5%) 671 (3.0%) 229 (1.0%) 105 (0.5%) 90 (0.4%) 134 (0.6%) 9,742 (43.6%) 165 (0.7%) 0.71 (0.86) 1.00 [0.00, 1.00] 4,221 (18.9%) 917 (4.1%) 0.24 (1.44) 0.00 [0.00, 0.00] 0.45 (1.21) 0.00 [0.00, 1.00] 12,337 (55.3%) | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 624 (2.8%) 2431 (1.5%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 156 (0.7%) 0.71 (0.81) 1.00 [0.00, 1.00] 4,253 (19.1%) 890 (4.0%) 4 (0.0%) 0.23 (1.23) 0.00 [0.00, 0.00] 0.41 (1.34) 0.00 [0.00, 0.00] 12,208 (54.7%) | 0.00 #WALUEI -0.01 0.01 0.01 0.01 0.01 0.00 0.00 0.0 | 2756 (7.1%) 5 (0.0%) 241 (0.6%) 1203 (3.1%) 425 (1.1%) 4000 (10.2%) 282 (0.7%) 178 (0.5%) 219 (0.6%) 17665 (45.2%) 315 (0.8%) 0.54 (0.81) 0.36 (0.87) 7427 (19.0%) 1392 (3.6%) 15 (0.0%) 0.22 (1.32) 0.00 (1.43) 0.41 (1.19) 0.00 (1.31) 21228 (54.3%) | 2685 (6.9%) #VALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 297 (0.8%) 0.54 (0.75) 0.43 (0.81) 7417 (19.0%) 1382 (3.5%) 12 (0.0%) 0.21 (1.14) 0.00 (1.23) 0.37 (1.32) 0.01 (1.45) 29935 (53.6%) | 0.01 #/ALUE! -0.01 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.00 0.01 #/DIV/01 |
| Peptic Ulcer Disease; n (%) Upper Gi bleed, n (%) Lower/ unspecified Gi bleed; n (%) Urogenital bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin, n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd)median [lQR] Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of INR (prothrombin) tests orderedmean (sd)median [lQR] Number of INR (prothrombin) tests orderedmean (sd)median [lQR] Treating prescriber - Primary Care Physician; n (%) Treating prescriber - Primary Care Physician; n (%) | 203 (7.3%) 0 (0.0%) 21 (0.8%) 91 (3.3%) 29 (1.0%) 285 (10.2%) 13 (0.5%) 9 (0.3%) 17 (0.6%) 1,098 (93.4%) 0.00 (0.00, 1.00) 470 (16.8%) 9 (0.3%) 0 (0.0%) 0.16 (9.98) 0.00 (0.00, 0.00) 0.41 (1.13) 0.00 (0.00, 0.00) 1,281 (45.9%) 1,757 (56.5%) | 208 (7.5%) 0 (0.0%) 24 (0.9%) 85 (3.0%) 27 (1.0%) 289 (10.4%) 11 (0.4%) 9 (0.3%) 13 (0.5%) 1,087 (39.0%) 0.68 (0.84) 1.00 (0.00, 1.00) 440 (15.8%) 0 (0.0%) 0.16 (0.97) 0.00 (0.00, 0.00) 1,280 (4.3%) 1,274 (5.4%) | -0.01 #DIV/01 -0.01 0.02 0.00 -0.01 0.01 0.01 0.01 0.01 -1.18 0.03 0.00 #DIV/01 0.00 0.00 0.00 0.00 0.00 0.00 0.00 | 901 (6.5%) 5 (0.0%) 104 (0.7%) 441 (3.2%) 167 (1.2%) 167 (1.2%) 168 (9.2%) 164 (1.2%) 79 (0.6%) 68 (0.5%) 6.825 (48.9%) 131 (0.9%) 0.25 (0.70) 0.00 (0.00, 0.00) 2,736 (19.6%) 384 (2.8%) 11 (0.1%) 0.20 (1.18) 0.00 (0.00, 0.00) 0.36 (1.18) 0.00 (0.00, 0.00) 7,610 (54.5%) 4,213 (30.2%) | 844 (6.0%) 4 (0.0%) 98 (0.7%) 429 (3.1%) 157 (1.1%) 1,288 (9.2%) 161 (1.2%) 77 (0.5%) 6,727 (48.2%) 0.24 (0.63) 0.00 (0.00, 0.00) 2,724 (19.5%) 8 (0.1%) 0.20 (1.00) 0.00 (0.00, 0.00) 1,744 (9.5%) 0.30 (1.28) 0.00 (0.00, 0.00) 7,447 (5.3.3%) 4,147 (29.3%) | 0.02<br>#DIV/01<br>0.00<br>0.01<br>0.01<br>0.01<br>0.01<br>0.01<br>0.01<br>0 | 1,652 (7.4%) 0 (0.0%) 116 (0.5%) 671 (3.0%) 229 (1.0%) 2,427 (10.9%) 134 (0.5%) 90 (0.4%) 134 (0.6%) 9,742 (43.6%) 165 (0.7%) 0.71 (0.86) 1.00 (0.00,1.00] 4,221 (18.9%) 917 (4.1%) 4 (0.0%) 0.24 (1.44) 0.00 (0.00,0.00] 0.45 (1.21) 0.00 (0.00,1.00] 12,337 (5.3.3%) 5,306 (23.8%) | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 100 (0.00, 1.00) 4,253 (19.1%) 890 (4.0%) 4 (0.0%) 0.23 (1.23) 0.00 (0.00, 0.00) 0.41 (1.34) 0.00 (0.00, 0.00) 12,208 (54.7%) 5,332 (23.9%) | 0.00 #WALUEI -0.01 0.01 -0.01 0.01 0.01 0.00 0.00 0. | 2756 (7.1%) 5 (0.0%) 241 (0.6%) 1203 (3.1%) 425 (1.1%) 4000 (10.2%) 282 (0.7%) 178 (0.5%) 219 (0.6%) 17655 (45.2%) 315 (0.8%) 0.54 (0.81) 0.36 (0.87) 7427 (19.0%) 15 (0.0%) 0.22 (1.32) 0.00 (1.43) 0.41 (1.19) 0.00 (1.31) 21228 (54.3%) | 2685 (6.9%) #VALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 0.54 (0.75) 0.43 (0.81) 7417 (19.0%) 1382 (3.5%) 12 (0.0%) 0.21 (1.14) 0.00 (1.23) 0.37 (1.32) 0.00 (1.45) 20935 (3.5%) 11053 (28.3%) | 0.01 #ALUEI -0.01 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 |
| Peptic Ulcer Disease; n (%) Upper Gl bleed; n (%) Lower Unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin (dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (6d)median [IQR] Proton pump inhibitor; n (%) Vitamin K therapy; n (%) Number of neurologist visitsmean (6d)median [IQR] Number of INR (prothrombin) tests orderedmean (6d)median [IQR] Number of INR (prothrombin) tests orderedmean (6d)median [IQR] Treating prescriber - Cardiologist; n (%) Treating prescriber - Cardiologist; n (%) Treating prescriber - Trimary Care Physician; n (%) Treating prescriber - Other; n (%) | 203 (7.3%) 0 (0.0%) 21 (0.8%) 91 (3.3%) 29 (1.0%) 13 (0.5%) 9 (0.3%) 17 (0.6%) 1,098 (39.4%) 19 (0.7%) 0.67 (0.86) 0.00 (0.00,1.00) 470 (16.8%) 91 (3.3%) 0 (0.0%) 0.16 (0.98) 0.00 (0.00,0.00) 0.41 (1.13) 0.00 (0.00,0.00) 1,281 (45.9%) 1,575 (56.5%) 1,997 (71.6%) | 208 (7.5%) 0 (0.0%) 24 (0.9%) 85 (3.0%) 27 (1.0%) 10 (0.4%) 9 (0.3%) 13 (0.5%) 1,087 (39.0%) 16 (0.6%) 0.68 (0.84) 1.00 (0.00, 1.00) 440 (15.8%) 93 (3.3%) 0 (0.0%) 0.16 (0.97) 0.00 (0.00, 0.00) 0.36 (1.33) 0.00 (0.00, 0.00) 1,280 (45.9%) 1,574 (56.4%) 2,025 (72.6%) | -0.01 #DIV/0! -0.01 0.02 0.00 -0.01 0.01 0.01 0.01 -0.01 -1.18 0.03 0.00 #DIV/0! 0.00 0.00 0.04 0.00 0.00 0.00 | 901 (6.5%) 5 (0.0%) 104 (0.7%) 441 (3.2%) 167 (1.2%) 167 (1.2%) 168 (9.2%) 164 (1.2%) 79 (0.6%) 68 (0.5%) 6.825 (48.9%) 131 (0.9%) 0.25 (0.70) 0.00 (0.00, 0.00) 2,736 (19.6%) 384 (2.8%) 11 (0.1%) 0.20 (1.18) 0.00 (0.00, 0.00) 0.36 (1.18) 0.00 (0.00, 0.00) 7,610 (54.5%) 4,213 (30.2%) 10,745 (77.0%) | 844 (6.0%) 4 (0.0%) 98 (0.7%) 429 (3.1%) 157 (1.1%) 1,288 (9.2%) 161 (1.2%) 71 (0.5%) 6,727 (48.2%) 125 (0.5%) 0.24 (0.63) 0.00 (0.00, 0.00) 2,724 (19.5%) 399 (2.5%) 8 (0.1%) 0.20 (1.00) 0.00 (0.00, 0.00) 1,744 (19.5%) 0.20 (1.00) 0.00 (0.00, 0.00) 7,447 (53.3%) 4,147 (29.7%) 10,635 (76.2%) | 0.02<br>#DIV/01<br>0.00<br>0.01<br>0.01<br>0.00<br>0.01<br>-0.01<br>0.01<br>0 | 1,652 (7.4%) 0 (0.0%) 116 (0.5%) 671 (3.0%) 229 (1.0%) 105 (0.5%) 90 (0.4%) 134 (0.6%) 9,742 (43.6%) 1.00 (0.0,0.1.00) 4,221 (18.9%) 917 (4.1%) 4 (0.0%) 0.24 (1.44) 0.00 (0.00,0.00) 0.45 (1.21) 0.00 (0.00,1.00) 12,337 (55.3%) 5,306 (23.8%) 17,177 (77.0%) | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 156 (0.7%) 0.71 (0.81) 1.00 (0.00, 1.00) 4,253 (19.1%) 890 (4.0%) 4 (0.0%) 0.23 (1.23) 0.00 (0.00, 0.00) 12,208 (54.7%) 5,332 (23.9%) 17,046 (76.4%) | 0.00 #WALUEI -0.01 0.01 0.01 0.01 0.01 0.00 0.00 0.0 | 2756 (7.1%) 5 (0.0%) 241 (0.6%) 1203 (3.1%) 425 (1.1%) 4000 (10.2%) 282 (0.7%) 178 (0.5%) 219 (0.6%) 17665 (45.2%) 315 (0.8%) 0.54 (0.81) 0.36 (0.87) 7427 (19.0%) 1392 (3.6%) 15 (0.0%) 0.22 (1.32) 0.00 (1.43) 0.41 (1.19) 0.00 (1.31) 21228 (54.3%) 11094 (28.4%) 29919 (76.6%) | 2685 (6.9%) #VALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 297 (0.8%) 0.54 (0.75) 0.43 (0.81) 7417 (19.0%) 1382 (3.5%) 12 (0.0%) 0.21 (1.14) 0.00 (1.23) 0.37 (1.32) 0.00 (1.45) 20935 (53.6%) 11053 (28.3%) 29706 (76.0%) | 0.01 #/ALUE! -0.01 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 #/DIV/01 0.00 0.00 0.01 #/DIV/01 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0 |
| Peptic Utcer Disease; n (%) Upper Gi bleed; n (%) Upper Gi bleed; n (%) Urogenital bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd)median [IQR] Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of fin8t (prothrombin) tests orderedmean (sd)median [IQR] Number of INR (prothrombin) tests orderedmean (sd)median [IQR] Treating prescriber - Primary Care Physician; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) | 203 (7.3%) 0 (0.0%) 21 (0.8%) 91 (3.3%) 29 (1.0%) 285 (10.2%) 13 (0.5%) 9 (0.3%) 17 (0.6%) 1,098 (93.4%) 0.00 (0.00, 1.00) 470 (16.8%) 9 (0.3%) 0 (0.0%) 0.16 (9.98) 0.00 (0.00, 0.00) 0.41 (1.13) 0.00 (0.00, 0.00) 1,281 (45.9%) 1,757 (56.5%) | 208 (7.5%) 0 (0.0%) 24 (0.9%) 85 (3.0%) 27 (1.0%) 289 (10.4%) 11 (0.4%) 9 (0.3%) 13 (0.5%) 1,087 (39.0%) 0.68 (0.84) 1.00 (0.00, 1.00) 440 (15.8%) 0 (0.0%) 0.16 (0.97) 0.00 (0.00, 0.00) 1,280 (4.3%) 1,274 (5.4%) | -0.01 #DIV/01 -0.01 0.02 0.00 -0.01 0.01 0.01 0.01 0.01 -1.18 0.03 0.00 #DIV/01 0.00 0.00 0.00 0.00 0.00 0.00 0.00 | 901 (6.5%) 5 (0.0%) 104 (0.7%) 441 (3.2%) 167 (1.2%) 167 (1.2%) 168 (9.2%) 164 (1.2%) 79 (0.6%) 68 (0.5%) 6.825 (48.9%) 131 (0.9%) 0.25 (0.70) 0.00 (0.00, 0.00) 2,736 (19.6%) 384 (2.8%) 11 (0.1%) 0.20 (1.18) 0.00 (0.00, 0.00) 0.36 (1.18) 0.00 (0.00, 0.00) 7,610 (54.5%) 4,213 (30.2%) | 844 (6.0%) 4 (0.0%) 98 (0.7%) 429 (3.1%) 157 (1.1%) 1,288 (9.2%) 161 (1.2%) 77 (0.5%) 6,727 (48.2%) 0.24 (0.63) 0.00 (0.00, 0.00) 2,724 (19.5%) 8 (0.1%) 0.20 (1.00) 0.00 (0.00, 0.00) 1,744 (9.5%) 0.30 (1.28) 0.00 (0.00, 0.00) | 0.02<br>#DIV/01<br>0.00<br>0.01<br>0.01<br>0.01<br>0.01<br>0.01<br>0.01<br>0 | 1,652 (7.4%) 0 (0.0%) 116 (0.5%) 671 (3.0%) 229 (1.0%) 2,427 (10.9%) 134 (0.5%) 90 (0.4%) 134 (0.6%) 9,742 (43.6%) 165 (0.7%) 0.71 (0.86) 1.00 (0.00,1.00] 4,221 (18.9%) 917 (4.1%) 4 (0.0%) 0.24 (1.44) 0.00 (0.00,0.00] 0.45 (1.21) 0.00 (0.00,1.00] 12,337 (5.3.3%) 5,306 (23.8%) | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 100 (0.00, 1.00) 4,253 (19.1%) 890 (4.0%) 4 (0.0%) 0.23 (1.23) 0.00 (0.00, 0.00) 0.41 (1.34) 0.00 (0.00, 0.00) 12,208 (54.7%) 5,332 (23.9%) | 0.00 #WALUEI -0.01 0.01 -0.01 0.01 0.01 0.00 0.00 0. | 2756 (7.1%) 5 (0.0%) 241 (0.6%) 1203 (3.1%) 425 (1.1%) 4000 (10.2%) 282 (0.7%) 178 (0.5%) 219 (0.6%) 17655 (45.2%) 315 (0.8%) 0.54 (0.81) 0.36 (0.87) 7427 (19.0%) 15 (0.0%) 0.22 (1.32) 0.00 (1.43) 0.41 (1.19) 0.00 (1.31) 21228 (54.3%) | 2685 (6.9%) #VALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 0.54 (0.75) 0.43 (0.81) 7417 (19.0%) 1382 (3.5%) 12 (0.0%) 0.21 (1.14) 0.00 (1.23) 0.37 (1.32) 0.00 (1.45) 20935 (3.5%) 11053 (28.3%) | 0.01 #ALUEI -0.01 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 |
| Peptic Ulcer Disease; n (%) Upper Gi bleed; n (%) Lower/ unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (6d)median [IQR] Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of neurologist visitsmean (6d)mean (6d)median [IQR] Number of INR (prothrombin) tests orderedmean (6d)median [IQR] Number of INR (prothrombin) tests orderedmean (6d)median [IQR] Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) Alpha blockers, n (%) CHADS2 socre, 180 days, V | 203 (7.3%) 0 (0.0%) 21 (0.8%) 91 (3.3%) 29 (1.0%) 285 (10.2%) 13 (0.5%) 9 (0.3%) 17 (0.6%) 1,098 (39.4%) 0.67 (0.86) 0.00 (0.00, 1.00) 470 (16.8%) 91 (3.3%) 0 (0.0%) 0.16 (0.98) 0.00 (0.00, 0.00) 0.15 (0.98) 0.00 (0.00, 0.00) 1,281 (45.9%) 1,575 (56.5%) 1,997 (71.6%) 400 (14.3%) | 208 (7.5%) 0 (0.0%) 24 (0.9%) 85 (3.0%) 27 (1.0%) 289 (10.4%) 11 (0.4%) 9 (0.3%) 13 (0.5%) 1,087 (39.0%) 0.68 (0.84) 1.00 (0.00, 1.00) 440 (15.8%) 93 (3.3%) 0 (0.0%) 0.16 (0.97) 0.00 (0.00, 0.00) 0.36 (1.33) 0.00 (0.00, 0.00) 1,280 (45.9%) 1,574 (56.4%) 2,025 (72.6%) 399 (14.3%) | -0.01 #DIV/01 #DIV/01 -0.01 0.02 0.00 -0.01 0.01 0.01 0.01 -0.01 -1.18 0.03 0.00 #DIV/01 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0 | 901 (6.5%) 5 (0.0%) 104 (0.7%) 441 (3.2%) 167 (1.2%) 167 (1.2%) 1,288 (9.2%) 164 (1.2%) 79 (0.6%) 68 (0.5%) 6.825 (48.9%) 131 (0.9%) 0.25 (0.70) 0.00 (0.00, 0.00) 2,736 (1.9.6%) 384 (2.8%) 11 (0.1%) 0.20 (1.18) 0.00 (0.00, 0.00) 0.36 (1.18) 0.00 (0.00, 0.00) 7,610 (54.5%) 4,213 (30.2%) 10,745 (77.0%) 1,835 (13.1%) | 844 (6.0%) 4 (0.0%) 98 (0.7%) 149 (3.1%) 157 (1.1%) 1,288 (9.2%) 161 (1.2%) 77 (0.5%) 77 (0.5%) 6,727 (48.2%) 125 (0.9%) 0.24 (0.63) 0.00 (0.00, 0.00) 2,724 (19.5%) 399 (2.9%) 8 (0.1%) 0.20 (1.00) 0.00 (0.00, 0.00) 7,447 (53.3%) 4,147 (29.7%) 10,635 (76.2%) 1,839 (13.2%) | 0.02<br>#DIV/01<br>0.00<br>0.01<br>0.01<br>0.01<br>0.01<br>0.01<br>0.01<br>0 | 1,652 (7.4%) 0 (0.0%) 116 (0.5%) 671 (3.0%) 229 (1.0%) 105 (0.5%) 90 (0.4%) 134 (0.6%) 9,742 (43.6%) 1,742 (43.6%) 0.71 (0.86) 1.00 [0.00,1.00] 4,221 (18.9%) 917 (4.1%) 4 (0.0%) 0.24 (1.44) 0.00 [0.00,0.00] 1.237 (55.3%) 5,306 (23.8%) 17,177 (77.0%) 3,188 (14.3%) | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 2,334 (10.5%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 156 (0.7%) 0.71 (0.81) 1.00 (0.00, 1.00) 4,253 (19.1%) 890 (4.0%) 4 (0.0%) 0.23 (1.23) 0.00 (0.00, 0.00) 12,208 (54.7%) 5,32 (23.9%) 17,046 (76.4%) 3,078 (13.8%) | 0.00 #WALUEI -0.01 0.01 0.01 0.01 0.01 0.00 0.00 0.0 | 2756 (7.1%) 5 (0.0%) 241 (0.6%) 1203 (3.1%) 425 (1.1%) 4000 (10.2%) 282 (0.7%) 178 (0.5%) 219 (0.6%) 17665 (45.2%) 315 (0.8%) 0.54 (0.81) 0.36 (0.87) 7427 (19.0%) 15 (0.0%) 0.22 (1.32) 0.00 (1.43) 0.41 (1.19) 0.00 (1.31) 21228 (54.3%) 11094 (28.4%) 29919 (76.6%) 5423 (13.9%) | 2685 (6.9%) #WALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 297 (0.8%) 0.54 (0.75) 0.43 (0.81) 7417 (19.0%) 1382 (3.5%) 12 (0.0%) 0.21 (1.14) 0.00 (1.23) 0.37 (1.32) 0.00 (1.45) 20935 (53.6%) 11053 (28.3%) 29706 (76.0%) 5316 (13.6%) | 0.01 #/ALUE! -0.01 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 #/DIV/OI 0.00 0.00 0.01 0.00 0.00 0.01 0.00 0.0 |
| Peptic Ulcer Disease; n (%) Upper Gl bleed; n (%) Lower Unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Prior cancer; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP Inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd)median [IQR] Proton pump inhibitor; n (%) Vitamin k therapy; n (%) Number of neurologist visitsmean (sd)median [IQR] Number of INR (prothrombin) tests orderedmean (sd)median [IQR] Treating prescriber - Cardiologist; n (%) Treating prescriber - Primary Care Physician; n (%) Alpha blockers; n (%) Alpha blockers; n (%) Alpha blockers; n (%)mean (sd)medidd)mediddiddiddiddiddiddiddiddiddiddiddiddid | 203 (7.3%) 0 (0.0%) 21 (0.8%) 91 (3.3%) 29 (1.0%) 13 (0.5%) 9 (0.3%) 17 (0.6%) 1,098 (39.4%) 19 (0.7%) 0.67 (0.86) 0.00 [0.00, 1.00] 470 (16.8%) 91 (3.3%) 0 (0.0%) 0.16 (0.98) 0.00 [0.00, 0.00] 0.41 (1.13) 0.00 [0.00, 0.00] 1,281 (45.9%) 1,597 (56.5%) 1,997 (71.6%) 400 (14.3%) | 208 (7.5%) 0 (0.0%) 24 (0.9%) 85 (3.0%) 27 (1.0%) 11 (0.4%) 9 (0.3%) 13 (0.5%) 1,087 (39.0%) 16 (0.6%) 0.68 (0.84) 1.00 (0.00, 1.00) 440 (15.5%) 93 (3.3%) 0 (0.0%) 0.16 (0.97) 0.00 [0.00, 0.00] 1,280 (45.9%) 1,574 (56.4%) 2,025 (72.6%) 399 (14.3%) | -0.01 -1.18 -0.03 -0.00 | 901 (6.5%) 5 (0.0%) 104 (0.7%) 441 (3.2%) 167 (1.2%) 167 (1.2%) 164 (1.2%) 79 (0.6%) 68 (0.5%) 6,825 (48.9%) 131 (0.9%) 0.25 (0.70) 0.00 (0.00, 0.00] 2,736 (19.6%) 384 (2.8%) 11 (0.1%) 0.20 (1.18) 0.00 (0.00, 0.00] 0.36 (1.18) 0.00 (0.00, 0.00] 7,510 (54.5%) 4,213 (30.2%) 10,745 (77.0%) 1,835 (13.1%) | 844 (6.0%) 4 (0.0%) 98 (0.7%) 98 (0.7%) 429 (3.1%) 157 (1.1%) 1,288 (9.2%) 161 (1.2%) 71 (0.5%) 77 (0.6%) 6,727 (48.2%) 125 (0.9%) 0.24 (0.63) 0.00 (0.00, 0.00) 2,724 (19.5%) 399 (2.9%) 8 (0.1%) 0.20 (1.00) 0.00 (0.00, 0.00) 0.30 (1.28) 0.00 (0.00, 0.00) 7,447 (53.3%) 4,147 (29.7%) 10,635 (76.2%) 11,839 (13.2%) | 0.02 #DIV/01 0.00 0.01 0.01 0.00 0.01 0.01 0.01 0 | 1,652 (7.4%) 0 (0.0%) 116 (0.5%) 671 (3.0%) 229 (1.0%) 105 (0.5%) 90 (0.4%) 134 (0.6%) 9,742 (43.6%) 105 (0.5%) 0.71 (0.86) 1.00 [0.00, 1.00] 4,221 (18.9%) 917 (4.1%) 0.02 (1.0%) 0.24 (1.44) 0.00 [0.00, 1.00] 0.45 (1.21) 0.00 [0.00, 1.00] 12,337 (55.3%) 5,306 (23.8%) 17,177 (77.0%) 3,188 (14.3%) | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 156 (0.7%) 0.71 (0.81) 1.00 [0.00, 1.00] 4,253 (19.1%) 890 (4.0%) 4 (0.0%) 0.23 (1.23) 0.00 [0.00, 0.00] 0.41 (1.34) 0.00 [0.00, 0.00] 12,208 (54.7%) 5,332 (23.9%) 17,046 (76.4%) 3,078 (13.8%) | 0.00 #WALUEI -0.01 -0.01 -0.01 -0.01 -0.01 -0.00 -0.00 -0.00 -0.01 -0.01 #DIV/0! | 2756 (7.1%) 5 (0.0%) 241 (0.6%) 1203 (3.1%) 425 (1.1%) 4000 (10.2%) 282 (0.7%) 178 (0.5%) 219 (0.6%) 17665 (45.2%) 315 (0.8%) 0.54 (0.81) 0.36 (0.87) 7427 (19.0%) 1392 (3.6%) 15 (0.0%) 0.22 (1.32) 0.00 (1.43) 0.41 (1.19) 0.00 (1.31) 21228 (54.3%) 11094 (28.4%) 2919 (76.6%) 5423 (13.9%) | 2685 (6.9%) #VALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 297 (0.8%) 0.54 (0.75) 0.43 (0.81) 7417 (19.0%) 1382 (3.5%) 12 (0.0%) 0.21 (1.14) 0.00 (1.23) 0.37 (1.32) 0.00 (1.45) 29706 (76.0%) 5316 (13.6%) | 0.01 #/ALUE! -0.01 -0.01 -0.00 -0.01 -0.00 -0.01 -0.00 -0.01 -0.00 -0.01 -0.00 -0.01 #/DIV/01 -0.00 -0 |
| Peptic Ulcer Disease; n (%) Upper Gi bleed, n (%) Lower/ unspecified Gi bleed; n (%) Urogenital bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin; n (%) Aspirinj dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (bd)median [lQR] Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin (k therapy; n (%) Number of lipid tests orderedmean (bd)median [lQR] Number of link (prothrombin) tests orderedmean (bd)median [lQR] Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHADS2 score, 180 days, Vmean (bd)mean (bd)mean (bd)mean (bd)mean (bd) | 203 (7.3%) 0 (0.0%) 21 (0.8%) 91 (3.3%) 29 (1.0%) 28 5 (10.2%) 13 (0.5%) 9 (0.3%) 17 (0.6%) 1,098 (93.4%) 1,098 (93.4%) 0.00 (0.00,1.00) 470 (16.8%) 9 (0.0%) 0.16 (0.98) 0.00 (0.00,0.00) 0.11,281 (45.9%) 1,282 (45.9%) 1,285 (65.5%) 1,997 (71.6%) 400 (14.3%) 1.88 (1.05) 2.00 (1.00),2.00] | 208 (7.5%) 0 (0.0%) 24 (0.9%) 85 (3.0%) 27 (1.0%) 8 (3.0%) 27 (1.0%) 9 (0.3%) 13 (0.5%) 1,087 (39.0%) 16 (0.6%) 0.68 (0.84) 1.00 (0.00, 1.00) 440 (15.8%) 93 (3.3%) 0 (0.0%) 0.16 (0.97) 0.00 [0.00, 0.00] 1,280 (45.9%) 1,574 (56.4%) 2,025 (72.6%) 399 (14.3%) 1,57 (1.00) 2.00 [1.00, 2.00] | -0.01 #DIV/01 -0.01 0.02 0.00 -0.01 0.01 0.01 0.01 0.01 -1.18 0.03 0.00 #DIV/01 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0 | 901 (6.5%) 5 (0.0%) 104 (0.7%) 441 (3.2%) 167 (1.2%) 167 (1.2%) 168 (9.2%) 164 (1.2%) 79 (0.6%) 68 (0.5%) 6.825 (48.9%) 131 (0.9%) 0.25 (0.70) 0.00 (0.00, 0.00) 2,736 (19.6%) 384 (2.8%) 11 (0.1%) 0.20 (1.18) 0.00 (0.00, 0.00) 0.36 (1.18) 0.00 (0.00, 0.00) 7,610 (54.5%) 4,213 (30.2%) 1,745 (77.0%) 1,835 (13.1%) 1,91 (1.09) | 844 (6.0%) 4 (0.0%) 98 (0.7%) 149 (3.1%) 157 (1.1%) 1,288 (9.2%) 161 (1.2%) 77 (0.5%) 6,727 (48.2%) 125 (0.9%) 0.24 (0.63) 0.00 (0.00, 0.00) 2,724 (19.5%) 399 (2.9%) 8 (0.1%) 0.20 (1.00) 0.00 (0.00, 0.00) 7,447 (53.3%) 4,147 (29.7%) 10,635 (76.2%) 1,839 (13.2%) 1,90 (1.07) 2,00 (1.07) | 0.02<br>#DIV/01<br>0.00<br>0.01<br>0.01<br>0.01<br>0.01<br>0.01<br>0.01<br>0 | 1,652 (7.4%) 0 (0.0%) 116 (0.5%) 671 (3.0%) 229 (1.0%) 2,427 (10.9%) 105 (0.5%) 90 (0.4%) 134 (0.6%) 9,742 (43.6%) 1,742 (43.6%) 0.71 (0.86) 1.00 [0.00,1.00] 4,221 (18.9%) 917 (4.1%) 4 (0.0%) 0.24 (1.44) 0.00 [0.00,0.00] 0.45 (1.21) 0.00 [0.00,1.00] 12,337 (55.3%) 5,306 (23.8%) 17,177 (77.0%) 3,188 (14.3%) 2.90 (1.27) 3.00 (2.00,4.00] | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 1.00 (0.00, 1.00) 4,253 (19.1%) 890 (4.0%) 4 (0.0%) 0.23 (1.23) 0.00 [0.00, 0.00] 12,208 (54.7%) 5,332 (23.9%) 17,046 (76.4%) 3,078 (13.8%) 2.92 (1.26) 3.00 [2.00, 4.00] | 0.00 #WALUEI -0.01 0.01 0.01 0.01 0.01 0.00 0.00 0.0 | 2756 (7.1%) 5 (0.0%) 241 (0.6%) 1203 (3.1%) 425 (1.1%) 4000 (10.2%) 282 (0.7%) 178 (0.5%) 219 (0.6%) 17655 (45.2%) 315 (0.8%) 0.54 (0.81) 0.36 (0.87) 7427 (19.0%) 1392 (3.6%) 15 (0.0%) 0.22 (1.32) 0.00 (1.43) 0.41 (1.19) 0.00 (1.31) 21228 (54.3%) 11994 (28.4%) 29919 (76.6%) 5423 (13.9%) 2.47 (1.19) 1.93 (1.30) | 2685 (6.9%) #VALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 0.54 (0.75) 0.43 (0.81) 7417 (19.0%) 1382 (3.5%) 12 (0.0%) 0.21 (1.14) 0.00 (1.23) 0.37 (1.32) 0.00 (1.45) 20935 (53.6%) 11053 (28.3%) 29706 (76.0%) 5316 (13.6%) 12.48 (1.18) 1.93 (1.28) | 0.01 #ALUE! -0.01 0.01 0.00 0.01 #DIV/0! |
| Peptic Ulcer Disease; n (%) Upper Gl bleed; n (%) Lower Unspecified Gl bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Prior cancer; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP Inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd)median [IQR] Proton pump inhibitor; n (%) Vitamin k therapy; n (%) Number of neurologist visitsmean (sd)median [IQR] Number of INR (prothrombin) tests orderedmean (sd)median [IQR] Treating prescriber - Cardiologist; n (%) Treating prescriber - Primary Care Physician; n (%) Alpha blockers; n (%) Alpha blockers; n (%) Alpha blockers; n (%)mean (sd)medidd)mediddiddiddiddiddiddiddiddiddiddiddiddid | 203 (7.3%) 0 (0.0%) 21 (0.8%) 91 (3.3%) 29 (1.0%) 13 (0.5%) 9 (0.3%) 17 (0.6%) 1,098 (39.4%) 19 (0.7%) 0.67 (0.86) 0.00 [0.00, 1.00] 470 (16.8%) 91 (3.3%) 0 (0.0%) 0.16 (0.98) 0.00 [0.00, 0.00] 0.41 (1.13) 0.00 [0.00, 0.00] 1,281 (45.9%) 1,597 (56.5%) 1,997 (71.6%) 400 (14.3%) | 208 (7.5%) 0 (0.0%) 24 (0.9%) 85 (3.0%) 27 (1.0%) 11 (0.4%) 9 (0.3%) 13 (0.5%) 1,087 (39.0%) 16 (0.6%) 0.68 (0.84) 1.00 (0.00, 1.00) 440 (15.5%) 93 (3.3%) 0 (0.0%) 0.16 (0.97) 0.00 [0.00, 0.00] 1,280 (45.9%) 1,574 (56.4%) 2,025 (72.6%) 399 (14.3%) | -0.01 -1.18 -0.03 -0.00 | 901 (6.5%) 5 (0.0%) 104 (0.7%) 441 (3.2%) 167 (1.2%) 167 (1.2%) 164 (1.2%) 79 (0.6%) 68 (0.5%) 6,825 (48.9%) 131 (0.9%) 0.25 (0.70) 0.00 (0.00, 0.00] 2,736 (19.6%) 384 (2.8%) 11 (0.1%) 0.20 (1.18) 0.00 (0.00, 0.00] 0.36 (1.18) 0.00 (0.00, 0.00] 7,510 (54.5%) 4,213 (30.2%) 10,745 (77.0%) 1,835 (13.1%) | 844 (6.0%) 4 (0.0%) 98 (0.7%) 98 (0.7%) 429 (3.1%) 157 (1.1%) 1,288 (9.2%) 161 (1.2%) 71 (0.5%) 77 (0.6%) 6,727 (48.2%) 125 (0.9%) 0.24 (0.63) 0.00 (0.00, 0.00) 2,724 (19.5%) 399 (2.9%) 8 (0.1%) 0.20 (1.00) 0.00 (0.00, 0.00) 0.30 (1.28) 0.00 (0.00, 0.00) 7,447 (53.3%) 4,147 (29.7%) 10,635 (76.2%) 11,839 (13.2%) | 0.02 #DIV/01 0.00 0.01 0.01 0.00 0.01 0.01 0.01 0 | 1,652 (7.4%) 0 (0.0%) 116 (0.5%) 671 (3.0%) 229 (1.0%) 105 (0.5%) 90 (0.4%) 134 (0.6%) 9,742 (43.6%) 105 (0.5%) 0.71 (0.86) 1.00 [0.00, 1.00] 4,221 (18.9%) 917 (4.1%) 0.02 (1.0%) 0.24 (1.44) 0.00 [0.00, 1.00] 0.45 (1.21) 0.00 [0.00, 1.00] 12,337 (55.3%) 5,306 (23.8%) 17,177 (77.0%) 3,188 (14.3%) | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 156 (0.7%) 0.71 (0.81) 1.00 [0.00, 1.00] 4,253 (19.1%) 890 (4.0%) 4 (0.0%) 0.23 (1.23) 0.00 [0.00, 0.00] 0.41 (1.34) 0.00 [0.00, 0.00] 12,208 (54.7%) 5,332 (23.9%) 17,046 (76.4%) 3,078 (13.8%) | 0.00 #WALUEI -0.01 -0.01 -0.01 -0.01 -0.01 -0.00 -0.00 -0.00 -0.01 -0.01 #DIV/0! | 2756 (7.1%) 5 (0.0%) 241 (0.6%) 1203 (3.1%) 425 (1.1%) 4000 (10.2%) 282 (0.7%) 178 (0.5%) 219 (0.6%) 17665 (45.2%) 315 (0.8%) 0.54 (0.81) 0.36 (0.87) 7427 (19.0%) 1392 (3.6%) 15 (0.0%) 0.22 (1.32) 0.00 (1.43) 0.41 (1.19) 0.00 (1.31) 21228 (54.3%) 11094 (28.4%) 2919 (76.6%) 5423 (13.9%) | 2685 (6.9%) #VALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 297 (0.8%) 0.54 (0.75) 0.43 (0.81) 7417 (19.0%) 1382 (3.5%) 12 (0.0%) 0.21 (1.14) 0.00 (1.23) 0.37 (1.32) 0.00 (1.45) 29706 (76.0%) 5316 (13.6%) | 0.01 #/ALUE! -0.01 -0.01 -0.00 -0.01 -0.00 -0.01 -0.00 -0.01 -0.00 -0.01 -0.00 -0.01 #/DIV/01 -0.00 -0 |
| Peptic Ulcer Disease; n (%) Upper Gi bleed; n (%) Lower/ unspecified Gi bleed; n (%) Urogenital bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin; n (%) Aspirinj (dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd)median [loR] Proton pump inhibitor; n (%) Number of neurologist visitsmean (sd)median [loR] Number of INR (prothrombin) tests orderedmean (sd)median [loR] Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) | 203 (7.3%) 0 (0.0%) 21 (0.8%) 91 (3.3%) 29 (1.0%) 285 (10.2%) 13 (0.5%) 9 (0.3%) 1,098 (93.4%) 1,098 (93.4%) 0.00 (0.00,1.00) 470 (16.8%) 9 (0.0%) 0.16 (0.98) 0.00 (0.00,0.00) 0.41 (1.13) 0.00 (0.00,0.00) 1,281 (45.9%) 1,575 (56.5%) 1,997 (71.6%) 400 (14.3%) 0.18 (1.05) 2.00 [1.00,2.00] 5 (0.2%) | 208 (7.5%) 0 (0.0%) 24 (0.9%) 85 (3.0%) 27 (1.0%) 85 (3.0%) 27 (1.0%) 10 (0.4%) 11 (0.4%) 9 (0.3%) 13 (0.5%) 1,087 (39.0%) 0.68 (0.84) 1.00 (0.00, 1.00) 440 (15.8%) 93 (3.3%) 0 (0.0%) 0.16 (0.97) 0.00 (0.00, 0.00) 1,280 (45.9%) 1,574 (56.4%) 2,025 (72.6%) 399 (14.3%) 1.87 (1.00) 2.00 [1.00, 2.00] 4 (0.1%) | -0.01 #DIV/01 #DIV/01 -0.01 0.02 0.00 -0.01 0.01 0.01 -0.01 -1.18 0.03 0.00 #DIV/0! 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0 | 901 (6.5%) 5 (0.0%) 104 (0.7%) 441 (3.2%) 167 (1.2%) 167 (1.2%) 1,288 (9.2%) 164 (1.2%) 79 (0.6%) 68 (0.5%) 6.825 (48.9%) 131 (0.9%) 0.25 (0.70) 0.00 (0.00, 0.00) 2,736 (19.6%) 384 (2.8%) 11 (0.1%) 0.20 (1.18) 0.00 (0.00, 0.00) 7,510 (54.5%) 4,213 (30.2%) 1,835 (13.1%) 1,931 (1.09) | 844 (6.0%) 4 (0.0%) 98 (0.7%) 429 (3.1%) 157 (1.1%) 1,288 (9.2%) 161 (1.2%) 77 (0.5%) 6,727 (48.2%) 0.24 (0.63) 0.00 (0.00, 0.00) 2,724 (19.5%) 8 (0.1%) 0.20 (1.00) 0.00 (0.00, 0.00) 7,447 (19.5%) 0.20 (1.00) 0.30 (1.28) 0.00 (0.00, 0.00) 7,447 (53.3%) 4,147 (29.7%) 1,635 (76.2%) 1,839 (13.2%) 1,90 (1.07) 2.00 [1.00, 2.00] | 0.02<br>#DIV/01<br>0.00<br>0.01<br>0.01<br>0.01<br>0.01<br>0.01<br>0.01<br>0 | 1,652 (7.4%) 0 (0.0%) 116 (0.5%) 671 (3.0%) 229 (1.0%) 2,427 (10.9%) 134 (0.6%) 97 (2.43.6%) 134 (0.6%) 9,742 (43.6%) 165 (0.7%) 0.71 (0.86) 1.00 (0.00,1.00) 4,221 (18.9%) 917 (4.1%) 4 (0.0%) 0.24 (1.44) 0.00 (0.00,0.00) 0.45 (1.21) 0.00 (0.00,0.00) 12,337 (55.3%) 5,306 (23.8%) 17,177 (77.0%) 3,188 (14.3%) 2.90 (1.27) 3.00 (2.00, 4.00) | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 100 (0.00, 1.00) 4,253 (19.1%) 890 (4.0%) 4 (0.0%) 0.23 (1.23) 0.00 (0.00, 0.00) 12,208 (54.7%) 5,332 (23.9%) 17,046 (76.4%) 3,078 (13.8%) 2.92 (1.26) 3.00 [2.00, 4.00] | 0.00 #WALUEI -0.01 -0.01 -0.01 -0.01 -0.01 -0.00 -0.00 -0.00 -0.00 -0.01 -0.02 -0.00 #WALUEI | 2756 (7.1%) 5 (0.0%) 241 (0.6%) 1203 (3.1%) 425 (1.1%) 4000 (10.2%) 282 (0.7%) 178 (0.5%) 219 (0.6%) 17655 (45.2%) 315 (0.8%) 0.54 (0.81) 0.36 (0.87) 7427 (19.0%) 1392 (3.6%) 15 (0.0%) 0.22 (1.32) 0.00 (1.43) 0.41 (1.19) 0.00 (1.31) 21228 (54.3%) 11094 (28.4%) 29919 (76.6%) 5423 (13.9%) 2.47 (1.19) 1.93 (1.30) #VALUE! | 2685 (6.9%) #VALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 0.54 (0.75) 0.43 (0.81) 7417 (19.0%) 1382 (3.5%) 12 (0.0%) 0.21 (1.14) 0.00 (1.23) 0.37 (1.32) 0.00 (1.45) 29936 (53.6%) 11053 (28.3%) 29706 (76.0%) 5316 (13.6%) 2.48 (1.18) 1.93 (1.28) #VALUE! | |
| Peptic Ulcer Disease; n (%) Upper Gi bleed, n (%) Lower/ unspecified Gi bleed; n (%) Urogenital bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin; n (%) Aspirinj dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (bd)median [lQR] Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin (k therapy; n (%) Number of lipid tests orderedmean (bd)median [lQR] Number of link (prothrombin) tests orderedmean (bd)median [lQR] Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHADS2 score, 180 days, Vmean (bd)mean (bd)mean (bd)mean (bd)mean (bd) | 203 (7.3%) 0 (0.0%) 21 (0.8%) 91 (3.3%) 29 (1.0%) 28 5 (10.2%) 13 (0.5%) 9 (0.3%) 17 (0.6%) 1,098 (93.4%) 1,098 (93.4%) 0.00 (0.00,1.00) 470 (16.8%) 9 (0.0%) 0.16 (0.98) 0.00 (0.00,0.00) 0.11,281 (45.9%) 1,282 (45.9%) 1,285 (65.5%) 1,997 (71.6%) 400 (14.3%) 1.88 (1.05) 2.00 (1.00),2.00] | 208 (7.5%) 0 (0.0%) 24 (0.9%) 85 (3.0%) 27 (1.0%) 8 (3.0%) 27 (1.0%) 9 (0.3%) 13 (0.5%) 1,087 (39.0%) 16 (0.6%) 0.68 (0.84) 1.00 (0.00, 1.00) 440 (15.8%) 93 (3.3%) 0 (0.0%) 0.16 (0.97) 0.00 [0.00, 0.00] 1,280 (45.9%) 1,574 (56.4%) 2,025 (72.6%) 399 (14.3%) 1,57 (1.00) 2.00 [1.00, 2.00] | -0.01 #DIV/01 -0.01 0.02 0.00 -0.01 0.01 0.01 0.01 0.01 -1.18 0.03 0.00 #DIV/01 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0 | 901 (6.5%) 5 (0.0%) 104 (0.7%) 441 (3.2%) 167 (1.2%) 167 (1.2%) 168 (9.2%) 164 (1.2%) 79 (0.6%) 68 (0.5%) 6.825 (48.9%) 131 (0.9%) 0.25 (0.70) 0.00 (0.00, 0.00) 2,736 (19.6%) 384 (2.8%) 11 (0.1%) 0.20 (1.18) 0.00 (0.00, 0.00) 0.36 (1.18) 0.00 (0.00, 0.00) 7,610 (54.5%) 4,213 (30.2%) 1,745 (77.0%) 1,835 (13.1%) 1,91 (1.09) | 844 (6.0%) 4 (0.0%) 98 (0.7%) 149 (3.1%) 157 (1.1%) 1,288 (9.2%) 161 (1.2%) 77 (0.5%) 6,727 (48.2%) 125 (0.9%) 0.24 (0.63) 0.00 (0.00, 0.00) 2,724 (19.5%) 399 (2.9%) 8 (0.1%) 0.20 (1.00) 0.00 (0.00, 0.00) 7,447 (53.3%) 4,147 (29.7%) 10,635 (76.2%) 1,839 (13.2%) 1,90 (1.07) 2,00 (1.07) | 0.02<br>#DIV/01<br>0.00<br>0.01<br>0.01<br>0.01<br>0.01<br>0.01<br>0.01<br>0 | 1,652 (7.4%) 0 (0.0%) 116 (0.5%) 671 (3.0%) 229 (1.0%) 2,427 (10.9%) 105 (0.5%) 90 (0.4%) 134 (0.6%) 9,742 (43.6%) 1,742 (43.6%) 0.71 (0.86) 1.00 [0.00,1.00] 4,221 (18.9%) 917 (4.1%) 4 (0.0%) 0.24 (1.44) 0.00 [0.00,0.00] 0.45 (1.21) 0.00 [0.00,1.00] 12,337 (55.3%) 5,306 (23.8%) 17,177 (77.0%) 3,188 (14.3%) 2.90 (1.27) 3.00 (2.00,4.00] | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 1.00 (0.00, 1.00) 4,253 (19.1%) 890 (4.0%) 4 (0.0%) 0.23 (1.23) 0.00 [0.00, 0.00] 12,208 (54.7%) 5,332 (23.9%) 17,046 (76.4%) 3,078 (13.8%) 2.92 (1.26) 3.00 [2.00, 4.00] | 0.00 #WALUEI -0.01 0.01 0.01 0.01 0.01 0.00 0.00 0.0 | 2756 (7.1%) 5 (0.0%) 241 (0.6%) 1203 (3.1%) 425 (1.1%) 4000 (10.2%) 282 (0.7%) 178 (0.5%) 219 (0.6%) 17655 (45.2%) 315 (0.8%) 0.54 (0.81) 0.36 (0.87) 7427 (19.0%) 1392 (3.6%) 15 (0.0%) 0.22 (1.32) 0.00 (1.43) 0.41 (1.19) 0.00 (1.31) 21228 (54.3%) 11994 (28.4%) 29919 (76.6%) 5423 (13.9%) 2.47 (1.19) 1.93 (1.30) | 2685 (6.9%) #VALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 0.54 (0.75) 0.43 (0.81) 7417 (19.0%) 1382 (3.5%) 12 (0.0%) 0.21 (1.14) 0.00 (1.23) 0.37 (1.32) 0.00 (1.45) 20935 (53.6%) 11053 (28.3%) 29706 (76.0%) 5316 (13.6%) 12.48 (1.18) 1.93 (1.28) | 0.01 #ALUE! -0.01 0.01 0.00 0.01 #DIV/0! |
| Peptic Utcer Disease; n (%) Upper Gi bleed; n (%) Lower/ unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGF inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd)median [LQR] Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of fin8 (prothrombin) tests orderedmean (sd)median [LQR] Number of INR (prothrombin) tests orderedmean (sd)median [LQR] Treating prescriber - Cardiologist; n (%) Treating prescriber - Primary Care Physician; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHADS2 score, 180 days, Vmean (sd)median [LQR] Use of Prasugre; n (%) | 203 (7.3%) 0 (0.0%) 21 (0.8%) 91 (3.3%) 29 (1.0%) 13 (0.5%) 9 (0.3%) 17 (0.6%) 1,098 (39.4%) 19 (0.7%) 0.67 (0.86) 0.00 [0.00, 1.00] 470 (16.8%) 91 (3.3%) 0 (0.0%) 0.16 (0.98) 0.00 [0.00, 0.00] 0.41 (1.13) 0.00 [0.00, 0.00] 1,281 (45.9%) 1,597 (56.5%) 1,997 (71.6%) 400 (14.3%) 1.88 (1.05) 2.00 [1.00, 2.00] 5 (0.2%) | 208 (7.5%) 0 (0.0%) 24 (0.9%) 85 (3.0%) 27 (1.0%) 85 (3.0%) 27 (1.0%) 10 (0.4%) 11 (0.4%) 9 (0.3%) 13 (0.5%) 1,087 (39.0%) 0.68 (0.84) 1.00 (0.00, 1.00) 440 (15.8%) 93 (3.3%) 0 (0.0%) 0.16 (0.97) 0.00 (0.00, 0.00) 1,280 (45.9%) 1,574 (56.4%) 2,025 (72.6%) 399 (14.3%) 1.87 (1.00) 2.00 [1.00, 2.00] 4 (0.1%) | -0.01 #DIV/01 #DIV/01 -0.01 0.02 0.00 -0.01 0.01 0.01 -0.01 -1.18 0.03 0.00 #DIV/0! 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0 | 901 (6.5%) 5 (0.0%) 104 (0.7%) 441 (3.2%) 167 (1.2%) 167 (1.2%) 1,288 (9.2%) 164 (1.2%) 79 (0.6%) 68 (0.5%) 6.825 (48.9%) 131 (0.9%) 0.25 (0.70) 0.00 (0.00, 0.00) 2,736 (19.6%) 384 (2.8%) 11 (0.1%) 0.20 (1.18) 0.00 (0.00, 0.00) 7,510 (54.5%) 4,213 (30.2%) 1,835 (13.1%) 1,931 (1.09) | 844 (6.0%) 4 (0.0%) 98 (0.7%) 429 (3.1%) 157 (1.1%) 1,288 (9.2%) 161 (1.2%) 77 (0.5%) 6,727 (48.2%) 0.24 (0.63) 0.00 (0.00, 0.00) 2,724 (19.5%) 8 (0.1%) 0.20 (1.00) 0.00 (0.00, 0.00) 7,447 (19.5%) 0.20 (1.00) 0.30 (1.28) 0.00 (0.00, 0.00) 7,447 (53.3%) 4,147 (29.7%) 1,635 (76.2%) 1,839 (13.2%) 1,90 (1.07) 2.00 [1.00, 2.00] | 0.02<br>#DIV/01<br>0.00<br>0.01<br>0.01<br>0.01<br>0.01<br>0.01<br>0.01<br>0 | 1,652 (7.4%) 0 (0.0%) 116 (0.5%) 671 (3.0%) 229 (1.0%) 2,427 (10.9%) 134 (0.6%) 97 (2.43.6%) 134 (0.6%) 9,742 (43.6%) 165 (0.7%) 0.71 (0.86) 1.00 (0.00,1.00) 4,221 (18.9%) 917 (4.1%) 4 (0.0%) 0.24 (1.44) 0.00 (0.00,0.00) 0.45 (1.21) 0.00 (0.00,0.00) 12,337 (55.3%) 5,306 (23.8%) 17,177 (77.0%) 3,188 (14.3%) 2.90 (1.27) 3.00 (2.00, 4.00) | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 100 (0.00, 1.00) 4,253 (19.1%) 890 (4.0%) 4 (0.0%) 0.23 (1.23) 0.00 (0.00, 0.00) 12,208 (54.7%) 5,332 (23.9%) 17,046 (76.4%) 3,078 (13.8%) 2.92 (1.26) 3.00 [2.00, 4.00] | 0.00 #WALUEI -0.01 -0.01 -0.01 -0.01 -0.01 -0.00 -0.00 -0.00 -0.00 -0.01 -0.02 -0.00 #WALUEI | 2756 (7.1%) 5 (0.0%) 241 (0.6%) 1203 (3.1%) 425 (1.1%) 4000 (10.2%) 282 (0.7%) 178 (0.5%) 219 (0.6%) 17655 (45.2%) 315 (0.8%) 0.54 (0.81) 0.36 (0.87) 7427 (19.0%) 1392 (3.6%) 15 (0.0%) 0.22 (1.32) 0.00 (1.43) 0.41 (1.19) 0.00 (1.31) 21228 (54.3%) 11094 (28.4%) 29919 (76.6%) 5423 (13.9%) 2.47 (1.19) 1.93 (1.30) #VALUE! | 2685 (6.9%) #VALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 0.54 (0.75) 0.43 (0.81) 7417 (19.0%) 1382 (3.5%) 12 (0.0%) 0.21 (1.14) 0.00 (1.23) 0.37 (1.32) 0.00 (1.45) 29936 (53.6%) 11053 (28.3%) 29706 (76.0%) 5316 (13.6%) 2.48 (1.18) 1.93 (1.28) #VALUE! | |
| Peptic Ulcer Disease; n (%) Upper Gi bleed; n (%) Lower/ unspecified Gi bleed; n (%) Urogenital bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin; n (%) Aspirinj (dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd)median [loR] Proton pump inhibitor; n (%) Number of neurologist visitsmean (sd)median [loR] Number of INR (prothrombin) tests orderedmean (sd)median [loR] Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) | 203 (7.3%) 0 (0.0%) 21 (0.8%) 91 (3.3%) 29 (1.0%) 13 (0.5%) 9 (0.3%) 17 (0.6%) 1,098 (39.4%) 19 (0.7%) 0.67 (0.86) 0.00 [0.00, 1.00] 470 (16.8%) 91 (3.3%) 0 (0.0%) 0.16 (0.98) 0.00 [0.00, 0.00] 0.41 (1.13) 0.00 [0.00, 0.00] 1,281 (45.9%) 1,597 (56.5%) 1,997 (71.6%) 400 (14.3%) 1.88 (1.05) 2.00 [1.00, 2.00] 5 (0.2%) | 208 (7.5%) 0 (0.0%) 24 (0.9%) 85 (3.0%) 27 (1.0%) 85 (3.0%) 27 (1.0%) 10 (0.4%) 9 (0.3%) 13 (0.5%) 1,087 (39.0%) 0.68 (0.84) 1.00 (0.00, 1.00] 440 (15.8%) 93 (3.3%) 0 (0.0%) 0.16 (0.97) 0.00 (0.00, 0.00) 1,280 (45.5%) 1,574 (56.4%) 2,025 (72.6%) 399 (14.3%) 1.87 (1.00) 2.00 [1.00, 2.00] 4 (0.1%) 668 (23.9%) | -0.01 #DIV/01 -0.01 0.02 0.00 -0.01 0.01 0.01 0.01 0.01 -0.01 -1.18 0.03 0.00 #DIV/01 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0 | 901 (6.5%) 5 (0.0%) 104 (0.7%) 441 (3.2%) 167 (1.2%) 167 (1.2%) 168 (9.2%) 164 (1.2%) 79 (0.6%) 68 (0.5%) 6.825 (48.9%) 131 (0.9%) 0.25 (0.70) 0.00 (0.00, 0.00) 2,736 (19.6%) 334 (2.8%) 11 (0.1%) 0.20 (1.18) 0.00 (0.00, 0.00) 0.36 (1.18) 0.00 (0.00, 0.00) 7,610 (54.5%) 4,213 (30.2%) 10,745 (77.0%) 1,835 (13.1%) 1.91 (1.09) 2.00 [1.00, 3.00] 56 (0.4%) 4,208 (30.1%) | 844 (6.0%) 4 (0.0%) 98 (0.7%) 198 (0.7%) 429 (3.1%) 157 (1.1%) 71 (0.5%) 77 (0.5%) 6,727 (48.2%) 125 (0.9%) 0.24 (0.63) 0.00 (0.00, 0.00) 2,724 (19.5%) 399 (2.9%) 8 (0.1%) 0.20 (1.00) 0.00 (0.00, 0.00) 7,447 (53.3%) 4,147 (29.7%) 10,635 (76.2%) 1,839 (13.2%) 1.90 (1.07) 2.00 (1.00) 2.01 (1.07) 2.00 (1.00) 2.01 (1.07) 2.00 (1.00) 2.01 (1.07) 2.00 (1.00) 2.01 (1.07) 2.00 (1.00) 3.01 (1.28) 3.06 (1.28) 3.07 (1.28) 3.08 (1.28) 3.09 (1.28) 3.09 (1.00) 3.00 (1.00) | 0.02 #DIV/01 0.00 0.01 0.01 0.01 0.01 0.01 0.01 0 | 1,652 (7.4%) 0 (0.0%) 116 (0.5%) 671 (3.0%) 229 (1.0%) 2,427 (10.9%) 134 (0.6%) 97 (2.43.6%) 134 (0.6%) 9,742 (43.6%) 165 (0.7%) 0.71 (0.86) 1.00 (0.00,1.00) 4,221 (18.9%) 917 (4.1%) 4 (0.0%) 0.24 (1.44) 0.00 (0.00,0.00) 0.45 (1.21) 0.00 (0.00,0.00) 12,337 (55.3%) 5,306 (23.8%) 17,177 (77.0%) 3,188 (14.3%) 2.90 (1.27) 3.00 (2.00, 4.00) | 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 100 (0.00, 1.00) 4,253 (19.1%) 890 (4.0%) 4 (0.0%) 0.23 (1.23) 0.00 (0.00, 0.00) 12,208 (54.7%) 5,332 (23.9%) 17,046 (76.4%) 3,078 (13.8%) 2.92 (1.26) 3.00 [2.00, 4.00] | 0.00 #WALUEI -0.01 -0.01 -0.01 -0.01 -0.01 -0.00 -0.00 -0.00 -0.01 -0.00 -0.01 -0.01 -0.00 -0.00 | 2756 (7.1%) 5 (0.0%) 241 (0.6%) 1203 (3.1%) 425 (1.1%) 4000 (10.2%) 282 (0.7%) 178 (0.5%) 219 (0.6%) 17655 (45.2%) 315 (0.8%) 0.54 (0.81) 0.36 (0.87) 7427 (19.0%) 15 (0.0%) 0.22 (1.32) 0.00 (1.43) 0.41 (1.19) 0.00 (1.31) 21228 (54.3%) 11094 (28.4%) 29919 (76.6%) 5423 (13.9%) 2.47 (1.19) 1.93 (1.30) #VALUE! | 2685 (6.9%) #WALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 297 (0.8%) 0.54 (0.75) 0.43 (0.81) 7417 (19.0%) 1382 (3.5%) 12 (0.0%) 0.21 (1.14) 0.00 (1.23) 0.37 (1.32) 0.00 (1.45) 20935 (53.6%) 11053 (28.3%) 29706 (76.0%) 5316 (13.6%) 2.48 (1.18) 1.93 (1.28) #WALUE! | 0.01 #/ALUE! -0.01 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 #/DIV/OI 0.00 0.00 0.01 #/DIV/OI 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0. |
| Peptic Utcer Disease; n (%) Upper Gi bleed; n (%) Lower/ unspecified Gi bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGF inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd)median [LQR] Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of fin8 (prothrombin) tests orderedmean (sd)median [LQR] Number of INR (prothrombin) tests orderedmean (sd)median [LQR] Treating prescriber - Cardiologist; n (%) Treating prescriber - Primary Care Physician; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHADS2 score, 180 days, Vmean (sd)median [LQR] Use of Prasugre; n (%) | 203 (7.3%) 0 (0.0%) 21 (0.8%) 91 (3.3%) 29 (1.0%) 13 (0.5%) 9 (0.3%) 17 (0.6%) 1,098 (39.4%) 19 (0.7%) 0.67 (0.86) 0.00 [0.00, 1.00] 470 (16.8%) 91 (3.3%) 0 (0.0%) 0.16 (0.98) 0.00 [0.00, 0.00] 0.41 (1.13) 0.00 [0.00, 0.00] 1,281 (45.9%) 1,597 (56.5%) 1,997 (71.6%) 400 (14.3%) 1.88 (1.05) 2.00 [1.00, 2.00] 5 (0.2%) | 208 (7.5%) 0 (0.0%) 24 (0.9%) 85 (3.0%) 27 (1.0%) 85 (3.0%) 27 (1.0%) 10 (0.4%) 11 (0.4%) 9 (0.3%) 13 (0.5%) 1,087 (39.0%) 0.68 (0.84) 1.00 (0.00, 1.00) 440 (15.8%) 93 (3.3%) 0 (0.0%) 0.16 (0.97) 0.00 (0.00, 0.00) 1,280 (45.9%) 1,574 (56.4%) 2,025 (72.6%) 399 (14.3%) 1.87 (1.00) 2.00 [1.00, 2.00] 4 (0.1%) | -0.01 #DIV/01 #DIV/01 -0.01 0.02 0.00 -0.01 0.01 0.01 -0.01 -1.18 0.03 0.00 #DIV/0! 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0 | 901 (6.5%) 5 (0.0%) 104 (0.7%) 441 (3.2%) 167 (1.2%) 167 (1.2%) 1,288 (9.2%) 164 (1.2%) 79 (0.6%) 68 (0.5%) 6.825 (48.9%) 131 (0.9%) 0.25 (0.70) 0.00 (0.00, 0.00) 2,736 (19.6%) 384 (2.8%) 11 (0.1%) 0.20 (1.18) 0.00 (0.00, 0.00) 7,510 (54.5%) 4,213 (30.2%) 1,835 (13.1%) 1,931 (1.09) | 844 (6.0%) 4 (0.0%) 98 (0.7%) 429 (3.1%) 157 (1.1%) 1,288 (9.2%) 161 (1.2%) 77 (0.5%) 6,727 (48.2%) 0.24 (0.63) 0.00 (0.00, 0.00) 2,724 (19.5%) 8 (0.1%) 0.20 (1.00) 0.00 (0.00, 0.00) 7,447 (19.5%) 0.20 (1.00) 0.30 (1.28) 0.00 (0.00, 0.00) 7,447 (53.3%) 4,147 (29.7%) 1,635 (76.2%) 1,839 (13.2%) 1,90 (1.07) 2.00 [1.00, 2.00] | 0.02<br>#DIV/01<br>0.00<br>0.01<br>0.01<br>0.01<br>0.01<br>0.01<br>0.01<br>0 | 1,652 (7.4%) 0 (0.0%) 116 (0.5%) 671 (3.0%) 229 (1.0%) 105 (0.5%) 90 (0.4%) 134 (0.6%) 9,742 (43.6%) 105 (0.5%) 0.71 (0.86) 1.00 [0.00, 1.00] 4,221 (18.9%) 917 (4.1%) 4 (0.0%) 0.24 (1.44) 0.00 [0.00, 1.00] 0.45 (1.21) 0.00 [0.00, 1.00] 12,337 (55.3%) 5,306 (23.8%) 17,177 (77.0%) 3,188 (14.3%) 2.90 (1.27) 3.00 [2.00, 4.00] | 1,633 (7.3%) 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 156 (0.7%) 0.71 (0.81) 1.00 [0.00, 1.00] 4,253 (19.1%) 890 (4.0%) 4 (0.0%) 0.23 (1.23) 0.00 [0.00, 0.00] 0.41 (1.34) 0.00 [0.00, 0.00] 12,208 (54.7%) 5,332 (23.9%) 17,046 (76.4%) 3,078 (13.8%) 2.92 (1.26) 3.00 [2.00, 4.00] ** 5,880 (26.3%) | 0.00 #WALUEI -0.01 -0.01 -0.01 -0.01 -0.01 -0.00 -0.00 -0.00 -0.00 -0.01 -0.02 -0.00 #WALUEI | 2756 (7.1%) 5 (0.0%) 241 (0.6%) 1203 (3.1%) 425 (1.1%) 4000 (10.2%) 282 (0.7%) 178 (0.5%) 219 (0.6%) 17655 (45.2%) 315 (0.8%) 0.54 (0.81) 0.36 (0.87) 7427 (19.0%) 1392 (3.6%) 15 (0.0%) 0.22 (1.32) 0.00 (1.43) 0.41 (1.19) 0.00 (1.31) 21228 (54.3%) 11094 (28.4%) 29919 (76.6%) 5423 (13.9%) 2.47 (1.19) 1.93 (1.30) #VALUE! | 2685 (6.9%) #VALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 0.54 (0.75) 0.43 (0.81) 7417 (19.0%) 1382 (3.5%) 12 (0.0%) 0.21 (1.14) 0.00 (1.23) 0.37 (1.32) 0.00 (1.45) 29936 (53.6%) 11053 (28.3%) 29706 (76.0%) 5316 (13.6%) 2.48 (1.18) 1.93 (1.28) #VALUE! | |
| Peptic Ulcer Disease; n (%) Upper Gi bled; n (%) Lower/ unspecified Gi bled; n (%) Lrogenital bleed; n (%) Urogenital bleed; n (%) Other bleeds; n (%) Prior cancer; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd)median [IQR] Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of Invital (%) Vitamin K therapy; n (%) Number of neurologist visitsmean (sd)median [IQR] Number of INR (prothrombin) tests orderedmean (sd)median [IQR] Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHADS2 score, 180 days, Vmean (sd)mean (sd)mean (sd)mean (sd) Use of Prasugrel; n (%) Use of Loop Diuretics+other diuretics+other hyperten: Commercial vs Medicare Advantage-Business Type Code | 203 (7.3%) 0 (0.0%) 21 (0.8%) 21 (0.8%) 91 (3.3%) 29 (1.0%) 13 (0.5%) 9 (0.3%) 17 (0.6%) 1,098 (93.4%) 1,098 (93.4%) 0.00 (0.00, 1.00) 470 (16.8%) 91 (3.3%) 0 (0.0%) 0.16 (0.98) 0.01 (0.00, 0.00) 0.41 (1.13) 0.00 (0.00, 0.00) 1,281 (45.9%) 1,575 (66.5%) 1,997 (71.6%) 400 (14.3%) 1.88 (1.05) 2.00 [1.00, 2.00] 5 (0.2%) | 208 (7.5%) 0 (0.0%) 24 (0.9%) 85 (3.0%) 27 (1.0%) 85 (3.0%) 27 (1.0%) 10 (0.4%) 9 (0.3%) 13 (0.5%) 1,087 (39.0%) 0.68 (0.84) 1.00 (0.00, 1.00] 440 (15.8%) 93 (3.3%) 0 (0.0%) 0.16 (0.97) 0.00 (0.00, 0.00) 1,280 (45.5%) 1,574 (56.4%) 2,025 (72.6%) 399 (14.3%) 1.87 (1.00) 2.00 [1.00, 2.00] 4 (0.1%) 668 (23.9%) | -0.01 #DIV/01 -0.01 0.02 0.00 -0.01 0.01 0.01 0.01 0.01 -0.01 -1.18 0.03 0.00 #DIV/01 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0 | 901 (6.5%) 5 (0.0%) 104 (0.7%) 441 (3.2%) 167 (1.2%) 167 (1.2%) 168 (9.2%) 164 (1.2%) 79 (0.6%) 68 (0.5%) 6.825 (48.9%) 131 (0.9%) 0.25 (0.70) 0.00 (0.00, 0.00) 2,736 (19.6%) 334 (2.8%) 11 (0.1%) 0.20 (1.18) 0.00 (0.00, 0.00) 0.36 (1.18) 0.00 (0.00, 0.00) 7,610 (54.5%) 4,213 (30.2%) 10,745 (77.0%) 1,835 (13.1%) 1.91 (1.09) 2.00 [1.00, 3.00] 56 (0.4%) 4,208 (30.1%) | 844 (6.0%) 4 (0.0%) 98 (0.7%) 198 (0.7%) 429 (3.1%) 157 (1.1%) 71 (0.5%) 77 (0.5%) 6,727 (48.2%) 125 (0.9%) 0.24 (0.63) 0.00 (0.00, 0.00) 2,724 (19.5%) 399 (2.9%) 8 (0.1%) 0.20 (1.00) 0.00 (0.00, 0.00) 7,447 (53.3%) 4,147 (29.7%) 10,635 (76.2%) 1,839 (13.2%) 1.90 (1.07) 2.00 (1.00) 2.01 (1.07) 2.00 (1.00) 2.01 (1.07) 2.00 (1.00) 2.01 (1.07) 2.00 (1.00) 2.01 (1.07) 2.00 (1.00) 3.01 (1.28) 3.06 (1.28) 3.07 (1.28) 3.08 (1.28) 3.09 (1.28) 3.09 (1.00) 3.00 (1.00) | 0.02 #DIV/01 0.00 0.01 0.01 0.01 0.01 0.01 0.01 0 | 1,652 (7.4%) 0 (0.0%) 116 (0.5%) 671 (3.0%) 229 (1.0%) 105 (0.5%) 90 (0.4%) 134 (0.6%) 9,742 (43.6%) 105 (0.5%) 0.71 (0.86) 1.00 [0.00, 1.00] 4,221 (18.9%) 917 (4.1%) 4 (0.0%) 0.24 (1.44) 0.00 [0.00, 1.00] 0.45 (1.21) 0.00 [0.00, 1.00] 12,337 (55.3%) 5,306 (23.8%) 17,177 (77.0%) 3,188 (14.3%) 2.90 (1.27) 3.00 [2.00, 4.00] | 1,633 (7.3%) 1,633 (7.3%) 132 (0.6%) 628 (2.8%) 243 (1.1%) 97 (0.4%) 84 (0.4%) 125 (0.6%) 9,629 (43.1%) 156 (0.7%) 0.71 (0.81) 1.00 [0.00, 1.00] 4,253 (19.1%) 890 (4.0%) 4 (0.0%) 0.23 (1.23) 0.00 [0.00, 0.00] 0.41 (1.34) 0.00 [0.00, 0.00] 12,208 (54.7%) 5,332 (23.9%) 17,046 (76.4%) 3,078 (13.8%) 2.92 (1.26) 3.00 [2.00, 4.00] ** 5,880 (26.3%) | 0.00 #WALUEI -0.01 -0.01 -0.01 -0.01 -0.01 -0.00 -0.00 -0.00 -0.01 -0.00 -0.01 -0.01 -0.00 -0.00 | 2756 (7.1%) 5 (0.0%) 241 (0.6%) 1203 (3.1%) 425 (1.1%) 4000 (10.2%) 282 (0.7%) 178 (0.5%) 219 (0.6%) 17655 (45.2%) 315 (0.8%) 0.54 (0.81) 0.36 (0.87) 7427 (19.0%) 15 (0.0%) 0.22 (1.32) 0.00 (1.43) 0.41 (1.19) 0.00 (1.31) 21228 (54.3%) 11094 (28.4%) 29919 (76.6%) 5423 (13.9%) 2.47 (1.19) 1.93 (1.30) #VALUE! | 2685 (6.9%) #WALUE! 254 (0.7%) 1142 (2.9%) 427 (1.1%) 3911 (10.0%) 269 (0.7%) 164 (0.4%) 215 (0.6%) 17443 (44.6%) 297 (0.8%) 0.54 (0.75) 0.43 (0.81) 7417 (19.0%) 1382 (3.5%) 12 (0.0%) 0.21 (1.14) 0.00 (1.23) 0.37 (1.32) 0.00 (1.45) 20935 (53.6%) 11053 (28.3%) 29706 (76.0%) 5316 (13.6%) 2.48 (1.18) 1.93 (1.28) #WALUE! | 0.01 #/ALUE! -0.01 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 0.00 0.01 #/DIV/OI 0.00 0.00 0.01 #/DIV/OI 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0. |

| Commercial vs Medicare Advantage-Business Type CodeCOM = COMMERCIAL; n (%)MCR = MEDICARE; n (%)MCD = MEDICAID; n (%) | 543 (19.5%)<br>2,247 (80.5%)<br>0 (0.0%) | 550 (19.7%)<br>2,240 (80.3%)<br>0 (0.0%) | -0.01<br>0.01<br>#DIV/0! | : | : | #VALUE!<br>#VALUE!<br>#VALUE! | : | | #VALUE!<br>#VALUE!<br>#VALUE! | 543 (19.5%)<br>2,247 (80.5%)<br>0 (0.0%) | 550 (19.7%)<br>2,240 (80.3%)<br>0 (0.0%) | -0.01<br>0.01<br>#DIV/0! |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| NONE = NO BUSINESS LINE CODE (added in 2015); n ( | 0 (0.0%) | 0 (0.0%) | #DIV/0! | | | #VALUE! | | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| UNK = UNKNOWN (added in 2015); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | | #VALUE! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Commercial vs Medicare Advantage- Data Type | - | | | 0 | 0 | | - | - | | | | |
| 1 - Fee For Service; n (%) | - | | | 1,842 (13.2%) | 1,816 (13.0%) | | - | - | | 1,842 (13.2%) | 1,816 (13.0%) | 0.00 |
| 2 - Encounter; n (%) | - | | | 228 (1.6%) | 210 (1.5%) | | - | - | | 228 (1.6%) | 210 (1.5%) | 0.00 |
| 3 - Medicare; n (%) | - | | | 11,016 (78.9%) | 11,069 (79.3%) | | - | - | | 11,016 (78.9%) | 11,069 (79.3%) | 0.00 |
| 4 - Medicare Encounter; n (%) | • | | | 874 (6.3%) | 865 (6.2%) | | • | - | | 874 (6.3%) | 865 (6.2%) | 0.00 |
| Metropolitan Statistical Area - Urban (any MSA) vs Rural (ı | non-MSA) | | | | | | | | | 0 | 0 | 0.00 |
| Urban; n (%) | - | | | 11,038 (79.1%) | 11,101 (79.5%) | | - | - | | 11,038 (79.1%) | 11,101 (79.5%) | 0.00 |
| Rural; n (%) | - | | | 101 (0.7%) | 111 (0.8%) | | - | - | | 101 (0.7%) | 111 (0.8%) | 0.00 |
| Unknown/Missing; n (%) | - | | | 2,821 (20.2%) | 2,748 (19.7%) | | - | | | 2,821 (20.2%) | 2,748 (19.7%) | 0.00 |

Due to CMS cell suppression policy, all values less than 11 are denoted with \*\*